- **Protocol number:** 156-08-276.
- **Document title:** A Phase 3b, Multicenter, Open-label, Randomized Withdrawal Trial of the Effects of Titrated Oral SAMSCA® (Tolvaptan) on Serum Sodium, Pharmacokinetics, and Safety in Children and Adolescent Subjects Hospitalized With Euvolemic or Hypervolemic Hyponatremia
- **Version number:** Amendment 5.
- Date of the document: 17 Nov 2015.
- EudraCT number: 2013-002005-59.

# Otsuka Pharmaceutical Development & Commercialization, Inc.

**Investigational Medicinal Product** 

SAMSCA<sup>®</sup>, Tolvaptan (OPC-41061)

#### REVISED CLINICAL PROTOCOL

A Phase 3b, Multicenter, Open-label, Randomized Withdrawal Trial of the Effects of Titrated Oral SAMSCA® (Tolvaptan) on Serum Sodium, Pharmacokinetics, and Safety in Children and Adolescent Subjects Hospitalized With Euvolemic or Hypervolemic Hyponatremia

Protocol No. 156-08-276 IND No. 54,200 NDA No. 22-275 EudraCT No. 2013-002005-59

#### CONFIDENTIAL – PROPRIETARY INFORMATION

Drug Development Phase: 3b

Sponsor: Otsuka Pharmaceutical Development &

Commercialization, Inc. 2440 Research Boulevard

Rockville, Maryland 20850, United States

Sponsor Representatives:

Phone ; Fax
E-mail:
Phone ; Fax

Immediately Reportable Event: INC Research (see Appendix 1)

E-mail:

Issue Date:

Date of Amendment 1:

Date of Amendment 2:

Date of Amendment 3:

Date of Amendment 4:

Date of Amendment 5:

O3 Jul 2013

04 Nov 2013

19 May 2014

26 February 2015

07 May 2015

17 Nov 2015

# **Protocol Synopsis**

| Name of Company: | Otsuka Pharmaceutical | Protocol No. 156-08-276 |
|---|---|---|
| Development & Com | | Protocol No. 156-08-2/6<br>IND No. 54,200 |
| Name of Product: SA | | NDA No. 22-275 |
| (OPC-41061) | AWISCA, Tolvapian | EudraCT No. 2013-002005-59 |
| Protocol Title: | A Phase 3h Multicenter Open | -label, Randomized Withdrawal |
| Trotocor ritic. | | |
| Trial of the Effects of Titrated Oral SAMSCA <sup>®</sup> (Tolvaptar<br>Serum Sodium, Pharmacokinetics, and Safety in Children<br>Adolescent Subjects Hospitalized With Euvolemic or<br>Hypervolemic Hyponatremia | | |
| Clinical Phase/Trial Type: | Phase 3b, therapeutic confirma | tory |
| Treatment | Euvolemic or hypervolemic hy | ponatremia |
| Indication: | | - |
| Objectives: | Primary Objective: | |
| | To demonstrate that tolvaptan effectively and safely increases and maintains serum sodium concentrations in children and adolescent subjects with euvolemic or hypervolemic hyponatremia. | |
| | Secondary Objective: | |
| | · · | 's pharmacokinetics (PK) and its effect on |
| fluid balance in children and adolescent subjects with | | |
| | euvolemic or hypervolemic hyp | ponatremia. |
| Trial Design: | This is an open-label, multicenter, multiple-dose, randomized withdrawal, parallel-group trial of tolvaptan in children and adolescent subjects hospitalized with euvolemic or hypervolemic hyponatremia. | |
| | to be screened for participation<br>demonstrate prior resistance to<br>will be excluded. All potential | ponatremia (serum sodium ersists despite initial standard ling fluid restriction) are eligible |
| | Since hyponatremia in this patient population can often be transient and/or may be secondary to hypovolemic states, potential subjects will be screened for hyponatremic histories well as clinically evaluated to rule out such cases. For the purpose of this protocol, persistent hyponatremia will be defined as serum sodium assessments < 130 mEq/L (mmol/L) | |

documented as present for at least 48 hours. Specifically, subjects must have at least 2 documented serum sodium assessments < 130 mEq/L (mmol/L) drawn at least 12 hours apart. These values can be documented using historical values previously obtained as per standard of care. A third (immediate [STAT]) serum sodium assessment < 130 mEq/L (mmol/L), which will serve as the baseline value for final trial qualification and clinical management strategy, is to be obtained within 2-4 hours prior to the first dose of tolvaptan. Additional qualification assessments will be performed as per etiology of hyponatremia. The first dose of tolvaptan will be administered upon successful completion of all screening procedures.

Subjects will be required to be in a hospital setting during initiation and titration of tolvaptan.

Overall, in this trial, subjects will undergo treatment (2 to 5 days of tolvaptan among 2 treatment phases) and a post-last dose follow-up phase of 14 days.

#### **Treatment Phase A**

After screening, all subjects will initially receive tolvaptan once daily for 2 days. If the desired serum sodium level target improvement is not reached after Day 2 of tolvaptan administration (post 2 doses), a third day (Day 2a) of treatment is required. At the end of Day 2 (or 2a), subjects will be assessed for a serum sodium level change of  $\geq 4$  mEq/L (mmol/L). At that time, subjects who are responders will enter Treatment Phase B, and be randomized to either the Early Withdrawal group or Late Withdrawal group. Responders are defined as those subjects who achieve an increase in serum sodium concentrations of  $\geq 4$  mEq/L (mmol/L); nonresponders are defined as subjects who do not achieve an increase in serum sodium concentration of  $\geq 4$  mEq/L (mmol/L).

#### **Treatment Phase B**

#### Responders

Responders from Treatment Phase A will be randomized to either the:

- Late Withdrawal group subjects continue tolvaptan treatment on Days 3 and 4
- Early Withdrawal group subjects do not receive additional tolvaptan treatment on Days 3 and 4.

Randomization will include stratification by age , serum sodium response

, and underlying etiology of

hyponatremia.

Subjects who are randomized to the Early Withdrawal group will initially be observed to determine whether additional intervention is required to maintain appropriate serum sodium levels. Those subjects whose serum sodium level declines by ≥ 4 mEq/L (mmol/L), or whose overall clinical condition requires further treatment to increase serum sodium level, will be treated per the investigator's preferred standard of care. Any intervention intended to raise serum sodium level during the first 48 hours of the Early Withdrawal phase (including fluid restriction) will be defined as rescue therapy. Subjects who receive rescue therapy will be considered to have reached their clinical endpoint, and their data will be censored from that time forward.

#### <u>Nonresponders</u>

If the subject remains a nonresponder at the end of Day 2a, the investigator decides to either (a) continue tolvaptan for 2 additional days, or (b) discontinue tolvaptan and treat the subject per the investigator's preferred standard of care during Days 3 and 4. Subjects will continue to follow scheduled assessments regardless of treatment.

#### All Subjects

All subjects will have serum sodium levels measured at 8, 12, and 24 hours post-first dose and thereafter every 12 ( $\pm$  4) hours through completion of Treatment Phase B. In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment will be obtained on Day 1 at 4 to 6 (-1 to  $\pm$  0.25) hours postdose and at 18 ( $\pm$  1) hours postdose. This sodium safety assessment will be repeated at 6 (-1 to  $\pm$  0.25) and 18 ( $\pm$  1) hours postdose each day for the remainder of titration.

#### Follow-up Phase C

All subjects will have an additional serum sodium assessment at 72 ( $\pm$  4) hours post-last dose and 7 ( $\pm$  1) days post-last dose. A final safety follow-up telephone contact/visit will be performed 14 ( $\pm$  2) days post-last dose.

### Pharmacokinetic Sampling

Blood samples for PK analysis will be obtained at 2 and 8 hours post-first dose, and at trough  $(24 [\pm 4] \text{ hours post-previous})$ 

dose) on Days 1, 2, 3, and 4 for all subjects dosed with tolvaptan on Days 1, 2, 3, and 4, respectively, regardless of responder status. Pharmacokinetic profiles will be evaluated on an ongoing basis to determine variability among subjects. Based on the findings, PK sampling will continue for as long as necessary to establish suitable estimates of clearance with a 90% confidence interval (CI), similar to that observed in adult subject populations. Once these estimates are achieved, sampling will be discontinued in subsequent subjects in order to minimize blood draws in this pediatric population.

## Subject Population:

This trial will enroll approximately 100 male and female subjects to get approximately 70 randomized subjects aged  $\geq 4$  weeks (or  $\geq 44$  weeks adjusted gestational age) to < 18 years who have been diagnosed with euvolemic or hypervolemic hyponatremia (< 130 mEq/L [mmol/L]) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). Age groups will be enrolled such that at least 50% of these subjects will be < 10 years old and at least 25% of subjects < 6 years old

Subjects with acute hyponatremia or hyponatremia expected to resolve spontaneously will be excluded from the trial. Children with an impaired ability to sense or communicate their thirst will either be required per protocol to undergo closer in-hospital observation, laboratory and urine output monitoring, or will be excluded from the trial if this is not possible.

The protocol entry criteria have been designed to ensure careful selection of subjects with chronic (≥ 48 hours) dilutional hyponatremia (euvolemic or hypervolemic) associated with heart failure, hepatocellular disease (including cirrhosis), or syndrome of inappropriate secretion of antidiuretic hormone/other, who may benefit from treatment with tolvaptan, while excluding those who have acute or transient hyponatremia, have overt symptoms of hyponatremia requiring immediate intervention, or who are at increased risk for developing hyponatremic encephalopathy or osmotic demyelination.

# Inclusion/Exclusion Criteria:

#### Key inclusion criteria:

- Male and female subjects  $\geq$  4 weeks (or  $\geq$  44 weeks adjusted gestational age) to  $\leq$  18 years old
- Subjects hospitalized with euvolemic or hypervolemic hyponatremia resistant to initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist) and who are deemed by the

- investigator as likely to benefit from a therapy that raises serum sodium levels
- Persistent euvolemic or hypervolemic hyponatremia defined as being documented as present for at least 48 hours, evidenced by at least 2 serum sodium assessments
   130 mEq/L (mmol/L) drawn at least 12 hours apart (these values can be documented using historical values previously obtained per standard of care); a third (STAT) serum sodium assessment < 130 mEq/L (mmol/L), which will serve as the baseline value for final trial qualification and clinical management strategy, is to be obtained within 2-4 hours prior to the first dose of tolvaptan</li>

#### Key exclusion criteria:

- Has evidence of hypovolemia or intravascular volume depletion (eg, hypotension, clinical evidence of volume depletion, response to saline challenge); if the subject has systolic blood pressure or heart rate outside of the normal range for that age, then volume status should be specifically clinically assessed to rule out volume depletion
- Has serum sodium level < 120 mEq/L (mmol/L), with or without associated neurologic impairment (ie, symptoms such as apathy, confusion, or seizures)
- Current use or expected use during the trial of potent cytochrome P450 (CYP) 3A4 inhibitors in subjects < 12 kg or moderate CYP3A4 inhibitors in subjects < 6 kg
- Has estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m<sup>2</sup>
- Has acute kidney injury defined as:
  - Increase in serum creatinine by  $\geq 0.3 \text{ mg/dL}$ ( $\geq 26.5 \text{ } \mu\text{mol/L}$ ) within 48 hours; or
  - Increase in serum creatinine to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or
  - Urine volume < 0.5 mL/kg/h for 6 hours
- Has had treatment for hyponatremia with:
  - Hypertonic saline (including normal saline challenge) within 8 hours of qualifying serum sodium assessments
  - Urea, lithium, demeclocycline, conivaptan, or tolvaptan within 4 days of qualifying serum sodium assessments
  - Other treatment for the purpose of increasing serum sodium concurrent with dosing of trial medication
- Has uncontrolled diabetes mellitus defined as fasting

glucose > 300 mg/dL (16.7 mEg/L [mmol/L])Has screening liver function values  $> 3 \times$  the upper limit of normal (ULN) Subjects who have cirrhosis and meet any of the following conditions: a major gastrointestinal (GI) bleed within the past 6 months, evidence of active bleeding (eg, epistaxis, petechiae/purpura, hematuria, or hematochezia), platelet count  $< 50,000/\mu L$ , or use of concomitant medications known to increase bleeding risk Trial Sites: The trial will be conducted at approximately 60 centers globally. Investigational Tolvaptan will be supplied as 3.75-, 7.5-, 15-, and 30-mg Medicinal Product, spray-dried tablets and, where approved, as a 1 mg/mL Dose, Formulation, (0.1% w/v) suspension. Mode of Administration: Tolvaptan tablets will be administered once daily, orally with a dose proportional amount of water. Doses of  $\geq 15$  mg tolvaptan will be given with 240 mL of water, 7.5 mg tolvaptan will be given with 120 mL of water, and 3.75 mg of tolvaptan will be given with 60 mL of water. The treatment duration will be up to 5 days. Tolvaptan suspension will be administered once daily, orally using the provided, appropriately-sized syringe (3 mL or 10 mL) to measure the volume. The lowest volume that can be administered is 0.3 mL (0.3 mg). Any initiation or titration of tolvaptan must occur in a hospital setting. The investigator has the option of performing a swallow test and providing coaching on swallowing techniques using placebo tablets if it is unknown if the subject is able to swallow tablets. Placebo tablets will be provided for use in performing this test at screening. Subjects will be administered tolvaptan on an age- and weight-based scale. Up-titration of tolvaptan doses will be based on serum sodium levels at > 20 hours following initiation of therapy and at > 20 hours following each additional dose; a change in serum sodium  $\leq 4 \text{ mEq/L (mmol/L)}$  from baseline should warrant up-titration, which is limited to no more than twice the previous dose. Subjects  $\geq$  4 weeks (or  $\geq$  44 weeks adjusted gestational age)

- to < 2 years of age and weighing  $\ge 3$  kg to < 6 kg will receive 0.1 mg/kg of the suspension on Day 1 with possible up-titration to 0.2 mg/kg and 0.4 mg/kg doses.
- Subjects  $\geq$  4 weeks (or  $\geq$  44 weeks adjusted gestational age) to < 2 years of age and weighing  $\geq$  6 kg to < 12 kg will receive 0.1 mg/kg of the suspension on Day 1 with possible up-titration to 0.2 mg/kg and 0.4 mg/kg doses.
- Subjects  $\geq 2$  to  $\leq 6$  years of age, weighing  $\leq 30$  kg will receive a 0.15 mg/kg dose of the suspension on Day 1 with possible up-titration to 0.3 mg/kg and 0.6 mg/kg doses.
- Subjects > 6 years of age, weighing ≤ 30 kg and who cannot safely swallow a tablet, will receive a 0.15 mg/kg dose of the suspension on Day 1 with possible up-titration to 0.3 mg/kg and 0.6 mg/kg doses.
- Subjects > 6 years of age and weighing 20 to 50 kg, inclusive, will receive a 7.5 mg tablet on Day 1 with possible up-titration to 15-mg and 30-mg doses.
- Subjects > 6 years of age and weighing > 50 kg, will receive a 15 mg tablet on Day 1 with possible up-titration to 30-mg and 60-mg doses.

The subjects will continue dosing according to a titration scheme targeting a final serum sodium concentration between 135 and 140 mEq/L (mmol/L). Titration will ideally achieve a change in serum sodium concentration of at least 4 to 8 mEq/L (mmol/L)/24 hours but not exceeding

#### Trial Assessments:

#### Efficacy:

• Serum sodium concentrations

#### Pharmacokinetic/pharmacodynamic:

- Blood sampling for tolvaptan and metabolite plasma concentrations
- Fluid intake
- Urine output
- Urine chemistry

#### Safety:

- Adverse event (AE) reporting
- Vital signs
- Clinical laboratory tests (hematology, coagulation, chemistry, urinalysis)
- Physical examinations, including body weight and neurological examinations

# Criteria for Evaluation:

#### **Primary Efficacy Endpoint**

• For subjects with serum sodium level increases of ≥ 4 mEq/L (mmol/L) (ie, responders), change in serum sodium concentration from Day 2 (or 2a) at the end of Treatment Phase A to the end of Treatment Phase B for Early compared to Late Withdrawal groups.

#### **Key Secondary Efficacy Endpoint**

• For all subjects, the key secondary endpoint is the change in serum sodium concentration at the end of Day 2 (or 2a) in Treatment Phase A from baseline.

# **Other Secondary Endpoints**

#### Safety:

- Percentage of subjects with overly rapid increase in serum sodium level
- Change in serum sodium level from 24 hours post-last dose to 7 days post-last dose
- Percentage of subjects requiring rescue therapy (other than fluid restriction) during Treatment Phase A and Treatment Phase B
- Percentage of subjects requiring fluid restriction during Treatment Phase A and Treatment Phase B
- Vital signs, blood pressure, clinical laboratory tests,

| | body weight, and neurological examinations |
|---|---|
| | Pharmacokinetic: |
| | • On Day 1 in Treatment Phase A, tolvaptan maximum |
| | (peak) plasma concentration ( $C_{max}$ ), time to maximum |
| | (peak) plasma concentration ( $t_{max}$ ), and area under the concentration-time curve from time zero to 24 hours (AUC <sub>0-24h</sub> ) |
| | Pharmacodynamic: |
| | Fluid intake, urine output, and fluid balance |
| | (intake minus output) every 6 hours on Days 1 and 2 in Treatment Phase A |
| | Exploratory Endpoints |
| | • Efficacy will be assessed in nonresponders continuing on tolvaptan therapy by change from baseline in serum sodium concentration at the end of Treatment Phase B compared to the end of Treatment Phase A. |
| | • In all subjects, 24-hour excretion of sodium, creatinine, and osmolality on Days 1 and 2 |
| | • 24-hour sodium clearance on Day 1 |
| | <ul> <li>Quality of life (QoL) assessments</li> </ul> |
| Statistical Methods: | The primary analysis will use a mixed-model repeated measures analysis based on the observed cases dataset. The key secondary analysis will be analyzed using a paired Student's t-test. Other secondary analyses will use a paired Student's t-test, descriptive statistics, and/or 2-sided 95% CIs. |
| Trial Duration: | Overall trial duration of enrollment is expected to be |
| | approximately 3 years with an enrollment rate of approximately |
| | 33 subjects per year. Nominal trial duration for each subject is up to 21 days. Treatment duration is up to 5 days with ongoing |
| | monitoring of serum sodium levels. A serum sodium |
| | assessment and AE follow-up visit will be performed 7 (+ 1) |
| | days post-last dose. A final safety follow-up telephone contact |
| | or visit will be performed 14 (+ 2) days post-last dose. |

# **Table of Contents**

| Otsu | ıka Pharmaceutical Development & Commercialization, Inc | 1 |
|-------|---------------------------------------------------------|---|
| Prot | ocol Synopsis | 2 |
| Tabl | le of Contents | 2 |
| | of In-text Tables | |
| List | of In-text Figures | 2 |
| List | of Appendices | 2 |
| List | of Abbreviations and Definitions of Terms | 2 |
| 1 | Introduction | 2 |
| 1.1 | Nonclinical Data | |
| 1.1.1 | Juvenile Animal Toxicity Data | 2 |
| 1.2 | Clinical Data | 2 |
| 1.2.1 | Pharmacokinetics | 2 |
| 1.2.2 | Pharmacodynamics | 2 |
| 1.2.3 | Clinical Efficacy | 2 |
| 1.3 | Known and Potential Risks and Benefits | 2 |
| 2 | Trial Rationale and Objectives | 2 |
| 2.1 | Trial Rationale | 2 |
| 2.1.1 | Dosing Rationale | 2 |
| 2.2 | Trial Objectives | 2 |
| 2.2.1 | Primary Objective | 2 |
| 2.2.2 | Secondary Objectives | 2 |
| 3 | Trial Design | 2 |
| 3.1 | Type/Design of Trial | 2 |
| 3.1.1 | Trial Phases. | 2 |
| 3.2 | Trial Treatments | 2 |
| 3.2.1 | Tablet Formulation | 2 |
| 3.2.2 | Suspension Formulation | 2 |
| 3.2.3 | Dosing Guidelines | 2 |
| 3.2.4 | Titration Guidelines and Rescue Therapy | 2 |
| 3.3 | Trial Population | 2 |

| 5.1 | Definitions | 2 |
|---|---|---|
| 5 | Reporting of Adverse Events | 2 |
| 4.2 | Other Restrictions | 2 |
| 4.1 | Prohibited Medications. | 2 |
| 4 | Restrictions | 2 |
| 3.13 | Protocol Deviations | 2 |
| 3.12 | Subject Compliance | 2 |
| 3.11 | Definition of Lost to Follow-up | 2 |
| 3.10 | Definition of Completed Subjects | 2 |
| 3.9 | Screen Failures | 2 |
| 3.8.3 | Individual Subject Discontinuation | 2 |
| 3.8.2 | Individual Site | 2 |
| 3.8.1 | Entire Trial or Treatment Arm(s) | 2 |
| 3.8 | Stopping Rules, Withdrawal Criteria and Procedures | 2 |
| 3.7.6 | Independent Data Monitoring Committee | |
| 3.7.5 | End of Trial | |
| 3.7.4 | Safety Assessments | |
| 3.7.3 | Pharmacokinetic/Pharmacodynamic Assessments | |
| 3.7.2 | Efficacy Assessments | |
| 3.7.1 | Schedule of Assessments | |
| 3.7 | Trial Procedures | |
| 3.6 | Measures to Minimize/Avoid Bias | |
| 3.5.4 | Exploratory Variables | |
| 3.5.3 | Other Secondary Outcome Variables | |
| 3.5.2 | Key Secondary Efficacy Outcome Variable | |
| 3.5.1 | Primary Efficacy Outcome Variable | |
| 3.4.3 | Outcome Variables | |
| 3.4.2 | Inclusion Criteria Exclusion Criteria | |
| 3.4.1 | Informed Consent/Assent | |
| 3.4<br>3.4.1 | Eligibility Criteria | |
| 3.3.1 | Subject Eligibility by Hyponatremia Etiology | |
| 2 2 1 | Code in at Edit il ilitar for Ideas on attraction Edit along | 2 |

| 5.2 | Eliciting and Reporting Adverse Events |
|---|---|
| 5.3 | Immediately Reportable Events |
| 5.3.1 | Hyponatremia-related Adverse Events |
| 5.4 | Potential Drug-induced Liver Injury |
| 5.4.1 | Liver Transaminase Elevations. |
| 5.5 | Pregnancy |
| 5.6 | Procedure for Breaking the Blind. |
| 5.7 | Follow-up of Adverse Events |
| 5.7.1 | Follow-up of Nonserious Adverse Events |
| 5.7.2 | Follow-up of Serious Adverse Events |
| 5.7.3 | Follow-up and Reporting of Serious Adverse Events Occurring After Last Scheduled Contact |
| 6 | Pharmacokinetic/Pharmacodynamic Analyses |
| 6.1 | Pharmacokinetic Analysis |
| 6.2 | Pharmacodynamic Analysis |
| 7 | Statistical Analysis |
| 7.1 | Sample Size |
| 7.1.1 | Sample Size for Efficacy |
| 7.1.2 | Sample Size for Pharmacokinetic Parameters |
| 7.2 | Datasets for Analysis |
| 7.3 | Handling of Missing Data |
| 7.4 | Primary and Secondary Outcome Analysis |
| 7.4.1 | Primary Outcome Analysis |
| 7.4.2 | Secondary Outcome Analyses |
| 7.4.3 | Exploratory Outcome Analyses |
| 7.4.4 | Interim Analysis |
| 7.5 | Analysis of Demographic and Baseline Characteristics |
| 7.6 | Safety Analysis |
| 7.6.1 | Adverse Events |
| 7.6.2 | Clinical Laboratory Assessment Data |
| 7.6.3 | Physical Examination and Vital Signs Data |
| 8 | Management of Investigational Medicinal Product |

| 8.1 | Packaging and Labeling | 2 |
|-----------|----------------------------------------------------|---|
| 8.2 | Storage | 2 |
| 8.3 | Accountability | 2 |
| 8.4 | Returns and Destruction | 2 |
| 8.5 | Reporting of Product Quality Complaints | 2 |
| 8.5.1 | Eliciting and Reporting Product Quality Complaints | 2 |
| 8.5.2 | Information Required for Reporting Purposes | 2 |
| 8.5.3 | Return Process | 2 |
| 8.5.4 | Assessment/Evaluation | 2 |
| 9 | Records Management | 2 |
| 9.1 | Source Documents | 2 |
| 9.2 | Data Collection | 2 |
| 9.3 | File Management at the Trial Site | 2 |
| 9.4 | Records Retention at the Trial Site | 2 |
| 10 | Quality Control and Quality Assurance | 2 |
| 10.1 | Monitoring | 2 |
| 10.2 | Auditing | 2 |
| 11 | Ethics and Responsibility | 2 |
| 12 | Confidentiality | |
| 13 | Amendment Policy | |
| 14 | Publication Authorship Requirements | |
| <b>15</b> | References | 2 |

# **List of In-text Tables**

| Table 2.1.1-1 | Starting Tolvaptan Tablet Doses as mg/kg of Body Weight | 2 |
|---|---|---|
| Table 3.2.3-1 | Starting Tolvaptan Doses With or Without Potent or Moderate CYP3A Inhibitors | 2 |
| Table 3.3.1.2-1 | Screening Algorithms by Hyponatremia Etiology | 2 |
| Table 3.4.2-1 | Inclusion Criteria | 2 |
| Table 3.4.3-1 | Exclusion Criteria | 2 |
| Table 3.7-1 | Schedule of Assessments | 2 |
| Table 3.7.2.1-1 | Serum Sodium Assessments | 2 |
| Table 3.7.4.2.3-1 | Clinical Laboratory Tests to be Performed Locally | 2 |
| Table 4.1-1 | List of Cytochrome P450 3A4 Inhibitors (Partial List) | 2 |
| Table 7.4.4-1 | Sample Size Re-estimation | 2 |

# **List of In-text Figures**

| Figure 1.2.3-1 | Mean (Standard Error) Changes From Baseline in Serum Sodium Concentration Following Tolvaptan or Placebo Treatment for 30 Days and at 7 Days Following Withdrawal of Therapy (Trials 156-02-235 and 156-03-238 [SALT 1 and 2] Combined) | 2 |
|---|---|---|
| Figure 1.2.3-2 | Mean (Standard Error) Serum Sodium Concentration Over<br>Time From the Parent Trials (156-02-235 and 156-03-238<br>[SALT 1 and 2]) to the Open-label Extension Trial (156-03-<br>244 [SALTWATER]); All Subjects (Observed Case) | 2 |
| Figure 3.1-1 | Trial Design Schematic | 2 |
| Figure 3.2.4-1 | Titration and Rescue Therapy Scheme | 2 |

# **List of Appendices**

| Appendix 1 | Names of Sponsor Personnel | 2 |
|------------|------------------------------------------------|---|
| Appendix 2 | Institutions Concerned With the Trial | 2 |
| Appendix 3 | Handling and Shipment of Bioanalytical Samples | 2 |
| Appendix 4 | Tanner Staging | 2 |
| Appendix 5 | Protocol Amendments | 2 |

# **List of Abbreviations and Definitions of Terms**

| TOPTU 7-day follow-up ADPKD Autosomal dominant polycystic kidney disease AE Adverse event AKI Acute kidney injury ALT Alanine transaminase AST Aspartate transaminase AUC Area under the concentration-time curve from time zero to 24 hours AUC <sub>0-24h</sub> Area under the concentration-time curve calculated to the last observable concentration at time t AUC <sub>τ</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CVV Coefficient of variation CVP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of sodium FE urea Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | A 1-1 | D. C |
|---|---|---|
| ADPKD AL Autosomal dominant polycystic kidney disease AE Adverse event AKI Acute kidney injury ALT Alanine transaminase AST Aspartate transaminase AST Aspartate transaminase AUC Area under the concentration-time curve AUC0-24h Area under the concentration-time curve from time zero to 24 hours AUCt Area under the concentration-time curve calculated to the last observable concentration at time t AUCt Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED3 Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of or uea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH Internsive care unit IDMC Independent data monitoring committee | Abbreviation | Definition 7 day fallow up |
| AE Adverse event AKI Acute kidney injury ALT Alanine transaminase AST Aspartate transaminase AUC Area under the concentration-time curve AUC <sub>0-24h</sub> Area under the concentration-time curve from time zero to 24 hours AUC <sub>t</sub> Area under the concentration-time curve calculated to the last observable concentration at time t AUC <sub>t</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CVP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DIL1 Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FENa Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | J 1 |
| AKI Acute kidney injury ALT Alanine transaminase AST Aspartate transaminase AUC Area under the concentration-time curve AUC <sub>0-24h</sub> Area under the concentration-time curve from time zero to 24 hours AUC <sub>1</sub> Area under the concentration-time curve calculated to the last observable concentration at time t AUC <sub>1</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CI/F Apparent clearance of drug from plasma after extravascular administration C <sub>max</sub> Maximum (peak) plasma concentration CV Coefficient of variation CVP Cytochrome P450 DDAVP I-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | |
| ALT Aspartate transaminase AST Aspartate transaminase AUC Area under the concentration-time curve AUC <sub>0-24h</sub> Area under the concentration-time curve from time zero to 24 hours AUC <sub>1</sub> Area under the concentration-time curve calculated to the last observable concentration at time t AUC <sub>1</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP I-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electroic ase report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | |
| AST Apartate transaminase AUC Area under the concentration-time curve AUC <sub>0-24h</sub> Area under the concentration-time curve from time zero to 24 hours AUC <sub>t</sub> Area under the concentration-time curve calculated to the last observable concentration at time t AUC <sub>t</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP I-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENA Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFF Heart failure HFF Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | 2 3 2 |
| AUC AUC <sub>0-24h</sub> Area under the concentration-time curve AUC <sub>1</sub> Area under the concentration-time curve from time zero to 24 hours AUC <sub>1</sub> Area under the concentration-time curve calculated to the last observable concentration at time t AUC <sub>1</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration CV CV Coefficient of variation CYP Cytochrome P450 DDAVP I-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | |
| AUC <sub>0-24h</sub> Area under the concentration-time curve from time zero to 24 hours AUC <sub>t</sub> Area under the concentration-time curve calculated to the last observable concentration at time t AUC <sub>t</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED3 Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | |
| AUC <sub>t</sub> Area under the concentration-time curve calculated to the last observable concentration at time t AUC <sub>t</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | |
| observable concentration at time t AUC <sub>T</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP I-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | V = | |
| AUC <sub>T</sub> Area under the concentration-time curve during the dosing interval at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DIL1 Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED3 Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | $AUC_t$ | |
| at steady state AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED3 Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | ATTG | |
| AVP Arginine vasopressin BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED3 Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | $AUC_{\tau}$ | |
| BUN Blood urea nitrogen BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED3 Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | ΛVD | • |
| BW Body weight CHF Congestive heart failure CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED3 Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | <del>-</del> |
| CHF CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED3 Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | <u>e</u> |
| CI Confidence interval CL/F Apparent clearance of drug from plasma after extravascular administration Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED3 Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | · · · |
| CL/F Apparent clearance of drug from plasma after extravascular administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | C |
| administration Cmax Maximum (peak) plasma concentration CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | | |
| CV Coefficient of variation CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | CL/I | |
| CYP Cytochrome P450 DDAVP 1-deamino-8-D-arginine vasopressin DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | $C_{max}$ | Maximum (peak) plasma concentration |
| DDAVP DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | CV | Coefficient of variation |
| DILI Drug-induced liver injury ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | CYP | Cytochrome P450 |
| ECG Electrocardiogram eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | DDAVP | 1-deamino-8-D-arginine vasopressin |
| eCRF Electronic case report form ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | DILI | Drug-induced liver injury |
| ED <sub>3</sub> Dose required to triple the urine output eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | ECG | Electrocardiogram |
| eGFR Estimated glomerular filtration rate EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | eCRF | Electronic case report form |
| EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Independent data monitoring committee | $ED_3$ | Dose required to triple the urine output |
| EMA European Medicines Agency ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Independent data monitoring committee | eGFR | Estimated glomerular filtration rate |
| ET Early termination FDA Food and Drug Administration FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Independent data monitoring committee | EMA | |
| FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Independent data monitoring committee | ET | <u> </u> |
| FENa Fractional excretion of sodium FE urea Fractional excretion of urea GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Independent data monitoring committee | FDA | Food and Drug Administration |
| GCP Good Clinical Practice GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | FENa | |
| GI Gastrointestinal HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | FE urea | Fractional excretion of urea |
| HF Heart failure HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | GCP | Good Clinical Practice |
| HFI Hereditary fructose intolerance IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | GI | Gastrointestinal |
| IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | HF | Heart failure |
| IB Investigator's Brochure ICF Informed consent form ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | HFI | Hereditary fructose intolerance |
| ICH International Conference on Harmonisation ICU Intensive care unit IDMC Independent data monitoring committee | IB | |
| ICU Intensive care unit IDMC Independent data monitoring committee | ICF | Informed consent form |
| IDMC Independent data monitoring committee | ICH | International Conference on Harmonisation |
| | ICU | Intensive care unit |
| IEC Independent ethics committee | | Independent data monitoring committee |
| | IEC | Independent ethics committee |

IMP Investigational medicinal product

IND Investigational new drug
INR International normalized ratio
IRB Institutional review board
IRE Immediately reportable event

ITT Intent-to-treat IV Intravenous

IWRS Interactive web response system

K<sub>i</sub> Inhibition constant

LOCF Last observation carried forward

LS Least squares

MHRA Medicines and Healthcare Products Regulatory

MMRM Mixed-model repeated measures

OAPI-EQC Otsuka America Pharmaceutical, Inc.-Ethics, Quality and

Compliance

OC Observed cases

OPDC Otsuka Pharmaceutical Development & Commercialization, Inc.

PD Pharmacodynamic(s)
PDCO Paediatric Committee
PI Principal investigator
PK Pharmacokinetic(s)

PO By mouth

PQC Product quality complaint
PREA Pediatric Research Equity Act

QoL Quality of life RBC Red blood cell

SAE Serious adverse event

SALT Study of Ascending Levels of Tolvaptan in Hyponatremia
SALTWATER Safety and sodium Assessment of Long-term Tolvaptan With

hyponatremia: A year-long, open-label Trial to gain Experience

under Real-world conditions

SAP Statistical analysis plan SD Standard deviation

SIADH Syndrome of inappropriate secretion of antidiuretic hormone

STAT Immediate

 $t_{1/2,z}$  Terminal-phase elimination half-life TEAE Treatment-emergent adverse event

t<sub>max</sub> Time to maximum (peak) plasma concentration

TSH Thyroid-stimulating hormone

ULN Upper limit of normal

US United States
WBC White blood cell

WOCBP Women of childbearing potential

#### 1 Introduction

Sodium is the major extracellular electrolyte and is a key factor in maintaining extracellular osmolality and transmembrane electrical and chemical potentials. Serum sodium concentration is maintained within a narrow range (normally 135 to 145 mEq/L [mmol/L]) to facilitate optimal cellular hydration and neuromuscular function. Sodium concentration is normally balanced through integrated actions of the cardiovascular, renal, endocrine, gastrointestinal (GI), and nervous systems.

Hyponatremia is a disease seen in all age groups, including pediatrics, and across a wide range of patients "from asymptomatic to the critically ill." It is characterized by a subnormal concentration of sodium in the blood (serum sodium < 135 mEq/L [mmol/L]) and is manifest by a range of neurological symptoms which, left untreated, can lead to seizure, obtundation, hypoxia, and death. Hyponatremia is rarely seen in isolation and typically is found in association with disorders, behaviors, or circumstances which promote an imbalance of fluid/sodium homeostasis. Children, in particular those hospitalized and receiving parenteral fluids (eg, post-operative maintenance and hydration with hypotonic fluid), are at risk for developing hyponatremia. <sup>2,3</sup>

Both forms of hyponatremia, dilutional and depletional, impair normal neurological function and therefore represent a disease state. Furthermore, there is evidence suggesting that, in both children and adults, hyponatremia has more serious consequences than previously believed. 4 Various clinical and nonclinical experiments and case studies have documented the role of sodium in maintaining extracellular osmolality and transmembrane electrical and chemical potentials. Sudden decreases in the concentration of extracellular sodium lead to influx of water into cells, often resulting in cerebral edema, irreversible neurological damage, respiratory arrest, brainstem herniation, and death if not treated quickly and appropriately. When hyponatremia persists, osmotic adjustments can occur over hours to days through metabolic elimination of electrolytes and then osmotically-active organic compounds from the cells. While these compensatory mechanisms can prevent acute brain herniation, chronic symptoms of hyponatremia may arise from electrochemical imbalances in cations that are important for nerve conduction and/or imbalances in amino acids and neurotransmitters dependent on sodium for transport. Disturbances in these physiological processes lead to symptoms and outcomes which depend on a number of factors, including rapidity of onset, severity of hyponatremia, persistence of underlying disease, and clinical context (age, gender, baseline neurological function). In many cases, morbidity and mortality associated with

hyponatremia can be shown to be prevented or reversed with appropriate and timely correction of serum sodium concentration.

In the adult population, hyponatremia occurs in 7% to 8% of elderly, ambulatory patients and 15% to 20% of hospitalized patients making it the most common serum electrolyte abnormality that physicians encounter, and a prevalent problem for those hospitalized for a wide variety of critical illnesses. A similar situation exists for children in which approximately 25% of hospitalized children were found to have mild hyponatremia (serum sodium < 135 mEq/L [mmol/L]) and approximately 1% were found to have moderate hyponatremia (serum sodium < 130 mEq/L [mmol/L]). Hyponatremia is associated with significant additional hospital morbidity and cost. 10

Children, especially infants, are particularly vulnerable to sodium and other electrolyte imbalances due to their relatively immature renal function, increased insensible water loss, and their limited ability to communicate thirst. Hence, hyponatremia is not uncommon in hospitalized children and pediatric patients presenting at the Emergency Department. Hyponatremia in children is most often caused by gastroenteritis and water intoxication, the former leading to hypovolemic volume state and requiring fluid administration. Other underlying diseases that can be accompanied by either euvolemic or hypervolemic hyponatremia are CHF, liver diseases, adrenal insufficiency, and renal disorders. The syndrome of inappropriate secretion of antidiuretic hormone (SIADH) is often associated with central nervous system or pulmonary conditions and also malignancies. An excess of arginine vasopressin (AVP) excretion with impaired free water excretion can lead to hyponatremia in febrile children and approximately 30% of these hospitalized children have SIADH. In addition, several drugs such as thiazide diuretics, antidepressants, anticonvulsants, and chemotherapeutics have been associated with SIADH.

The United States (US) Food and Drug Administration (FDA) has required pediatric trials be conducted for tolvaptan for the indication of hyponatremia. This trial will assess the short-term safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) of tolvaptan in children and adolescent subjects with euvolemic or hypervolemic hyponatremia.

#### 1.1 Nonclinical Data

Tolvaptan is a vasopressin antagonist that blocks the binding of AVP at the  $V_2$  receptors of the distal portions of the nephron, thereby inducing water diuresis (aquaresis) without depletion of electrolytes. In vitro binding studies demonstrated that tolvaptan has affinity

for the human vasopressin  $V_2$  and  $V_{1a}$  receptors but not  $V_{1b}$  receptors. The receptor selectivity potential of tolvaptan for human  $V_2$  receptors (inhibition constant  $[K_i] = 0.43 \text{ nmol/L}$ ) is approximately 30 times that for human  $V_{1a}$  receptors  $(K_i = 12.3 \text{ nmol/L})$  and at concentrations not achieved clinically. Several tolvaptan metabolites (DM-4110, DM-4111, and MOP-21826) have affinity for the human  $V_2$  or  $V_{1a}$  receptors but to a lesser degree than tolvaptan. None of the metabolites appear to have affinity for  $V_{1b}$  receptors. Tolvaptan is 1.8 times more potent in binding activity than native AVP.

In vivo pharmacology experiments using water loaded, alcohol-anesthetized rats indicated that tolvaptan at 3 to 30 µg/kg intravenous (IV) dose-dependently antagonized the antidiuretic action of exogenous vasopressin. In conscious mice, rats, and dogs, tolvaptan at 0.3, 1, 3, and 10 mg/kg by mouth (PO) caused dose-dependent water diuresis (aquaresis), ie, an increase in urine volume and a decrease in urine osmolality. The dose required to triple the urine output (ED<sub>3</sub>) within 2 hours post dosing in rats was estimated to be 0.54 mg/kg and the ED<sub>3</sub> after 6 hours in dogs was estimated to be 1.1 mg/kg PO. In the rat model of acute progressive hyponatremia, tolvaptan (0, 1, 3, and 10 mg/kg PO) produced a clear dose-dependent aquaresis over the dosing duration, which resulted in a gradual increase in plasma sodium concentration and a decrease in the mortality rate. In severe hyponatremia, mortality rate decreased from 47% in 1-deamino-8-D-arginine vasopressin (DDAVP) and water loaded rats to 38% in the 1 mg/kg dose group, and no deaths were seen in the 3 and 10 mg/kg dose groups of tolvaptan-treated rats. In the rat model of chronic hyponatremia induced by DDAVP infusion (1 ng/h subcutaneous) and liquid diet, plasma sodium concentration was reduced to about 110 mEq/L and maintained at that level without any deaths. Oral dose titration of tolvaptan from 0.25 to 8 mg/kg gradually increased plasma sodium concentration to the normal levels, and improved the wet weight of kidney and water content in the brain and heart, which were increased by sustained hyponatremia. 13,14

In a dog model of pacing-induced congestive heart failure (CHF), tolvaptan alone exerted aquaretic effects without activation of sympathetic and renin-angiotensin-aldosterone systems and produced a significant decrease in cardiac preload without affecting cardiac afterload or renal functions. Tolvaptan did not affect the human ether-a-go-go-related gene channel current at the tested concentration up to  $2 \times 10^{-6}$  mol/L, which was the solubility limit for the external solution. In conscious dogs, tolvaptan at doses of up to 1,000 mg/kg PO showed no significant changes in the ST segment, QRS width, QT interval, and QTc interval when compared to the control group. In an action potential

duration study in the guinea pig ventricular papillary muscle, tolvaptan did not affect any of the parameters studied (resting membrane potential, action potential amplitude, maximum aortic velocity, action potential duration at 30%, 60%, and 90% repolarization) at tested concentrations of up to  $3 \times 10^{-5}$  mol/L, which was about 30-fold higher than the maximum serum concentrations in humans at an oral clinical dose of 60 mg of the spray-dried formulation.

Based on results from single-dose toxicity studies, the approximate lethal dose of tolvaptan is higher than 2,000 mg/kg in rats and dogs. The nontoxic dose of the compound is estimated to be 1,000 mg/kg/day in the males, and 100 mg/kg/day in the females in a 26-week repeated oral dose study in rats and 100 mg/kg/day in both males and females in a 52-week repeated oral dose study in dogs. The exposures in animals at these nontoxic dose levels are 4.0 to 13.1 times higher than that in humans following administration of the compound at a dose of 60 mg/day.

No deleterious changes in copulation or fertility were seen in the fertility studies in rats. No male-factor effects were exhibited in offspring of treated male rats. No increases in fetal mortality or malformation were seen in embryo-fetal development studies in pregnant female rats at up to 1,000 mg/kg and in pregnant female rabbits at up to 100 mg/kg. However, an additional embryo-fetal development study in pregnant female rabbits showed high fetal mortality and a marginal increase in malformations at 1,000 mg/kg/day. A prenatal and postnatal development study in rats showed increased perinatal death and body weight suppression during the lactation period and after weaning in the offspring at 1,000 mg/kg/day. Drug exposure in the rabbits based on area under the concentration-time curve (AUC) values of 3.882 and 16.924 µg·h/mL at doses of 100 and 1,000 mg/kg/day, respectively, was approximately 1.2- and 5.2-fold higher than the AUC value of 3.2376 µg·h/mL seen in man receiving a 60-mg/day dose. No genotoxicity of the compound was observed and no antigenicity was evident in guinea pigs. No increases in mortality and tumor incidence were seen in the 2-year carcinogenicity study in male mice at doses up to 60 mg/kg/day, in female mice at doses up to 100 mg/kg/day, and in rats at doses up to 1,000 mg/kg/day.

Exposure to metabolites present in humans (including DM-4103, which, while inactive at the AVP receptors, has the highest human exposure) was adequate in animal models for estimation of effects on toxicity, reproduction, and carcinogenicity. No evidence of long-term pharmacologic or toxicologic effects was seen.

Toxicology data suggested that tolvaptan may be safe in humans. No male-factor effects were seen; however, appropriate precautions should be implemented for the inclusion of women of childbearing potential in clinical trials. Additional information relating to

nonclinical studies conducted with tolvaptan can be found in the current version of the Investigator's Brochure (IB). 14

#### 1.1.1 Juvenile Animal Toxicity Data

Six-week repeated oral dose toxicity study of tolvaptan was conducted in juvenile Sprague-Dawley rats (Crl:CD[SD], 25 days of age at the start of administration, 10 animals of each sex for 30 and 100 mg/kg groups, and 15 animals of each sex for the control and 1,000 mg/kg groups) at daily dose levels of 0 (1% [w/v] hypromellose solution), 30, 100, or 1,000 mg/kg. The reversibility of any effects was also assessed following a 4-week untreated recovery period using 5 animals of each sex in the control and 1,000 mg/kg groups. In addition, serum concentrations of tolvaptan and its 2 metabolites (DM-4103 and DM-4107) were determined after dosing on the first day (Day 1) and last day (Day 42) of administration. No deaths occurred during the administration or recovery period. No test article-related effects were noted in clinical observation, detailed clinical observation, sensory functional examination, or necropsy. Based on the above results, the no observed adverse effect level was judged to be 100 mg/kg/day for both males and females. <sup>14</sup>

A 1-week dose range-finding study was conducted in rat pups at 4 or 7 days of age and results showed tolvaptan to be lethal at 1000 mg/kg/day and tolerable at 100 mg/kg/day and lower.

In another study, male and female rat pups at 4 days of age were orally administered tolvaptan for 9 weeks at doses of 10, 30, and 100 mg/kg/day. Similar to the above study, pharmacologically mediated changes were noted in urine volume, water consumption, and urine electrolytes at all doses. Dilated renal pelvis considered to be attributable to increased urine volume during very early infancy was noted in males at 30 mg/kg/day and higher and females at 100 mg/kg/day. Toxicities were noted at 100 mg/kg/day, including death in one male, suppressed body weight gain and food consumption in males and females, and delayed balanopreputial separation and prolonged prothrombin time in males. Except for prolonged prothrombin time, all changes noted during the administration period showed reversibility after a 4-week recovery period. The no observed adverse effect level in both males and females was judged to be 30 mg/kg/day.<sup>14</sup>

#### 1.2 Clinical Data

Tolvaptan was approved by the United States (US) Food and Drug Administration (FDA) on 19 May 2009, by the European Medicines Agency (EMA) on 03 Aug 2009, and

subsequently in 10 other countries for the treatment of specific forms of hyponatremia. Tolvaptan was approved by the Japanese Ministry of Health, Labour, and Welfare on 27 Oct 2010 for the adjunct treatment of volume overload in HF when adequate response is not obtained with other diuretics; in September 2013 for body fluid retention in hepatic cirrhosis when adequate response is not obtained with other diuretics; and in March 2014 for suppression of progression of autosomal dominant polycystic kidney disease (ADPKD) with increased kidney volume and a rapid rate of increase. Phase 3 development for hepatic edema has been completed in China. Tolvaptan is also being developed for the treatment of ADPKD in the US and multinationally; for the adjunct treatment of chronic renal failure treated with peritoneal dialysis and hematodialysis or hemodiafiltration, for carcinomatous edema in Japan, and for cardiac edema in China and Taiwan. Tolvaptan, under the brand name Jinarc®, is approved to treat ADPKD in Canada and the European Union. As of 31 Mar 2015, the tolvaptan clinical development program consists of 105 trials; 97 trials had been completed worldwide, 4 trials were terminated because of slow enrollment, and 8 trials were ongoing. More information is available in the IB. 14

#### 1.2.1 Pharmacokinetics

Since inception of the program, a total of 53 clinical pharmacology trials have been completed with tolvaptan (as of 31 Mar 2015) in healthy subjects or special populations in Japan, the United Kingdom, China, Korea, Argentina, and the US.

In healthy subjects, following IV dosing, the terminal-phase elimination half-life  $(t_{1/2,z})$  of tolvaptan is about 3 hours. Following single oral tablet doses, the  $t_{1/2,z}$  of tolvaptan increases with increasing dose with mean values around 3 hours for a 15-mg dose and 12 hours for 120- to 480-mg doses. Tolvaptan is very insoluble, with solubility being 0.00005 w/v% at 25°C and is pH independent. At lower doses, tolvaptan is mostly absorbed from the upper GI tract so the decline of the terminal portion of the concentration curve reflects elimination process only. With increasing dose, there is continued absorption of tolvaptan from the GI tract such that the rate of decline of the terminal portion of the concentration curve is reflective of both absorption and elimination processes. <sup>14</sup>

The limited early absorption of tolvaptan is exemplified by the fact that the maximum (peak) plasma concentration ( $C_{max}$ ) values show less than dose proportional increases from 30 to 240 mg and then a plateau at doses from 240 to 480 mg. Despite the changes in tolvaptan absorption, tolvaptan AUC values increase proportionally with increasing

dose and apparent clearance of drug from plasma after extravascular administration (CL/F) values are unchanged for single doses of 30 to 480 mg. <sup>14</sup>

Tolvaptan concentrations do not accumulate following once daily dosing. Following 300-mg doses,  $C_{max}$  and AUC during the dosing interval at steady state (AUC<sub> $\tau$ </sub>) were only 4.2- and 6.4-fold higher, respectively, when compared with the 30-mg dose. This indicates bioavailability decreases with increasing dose. Mean (range) absolute bioavailability of tolvaptan when administered as a 30-mg tablet was 56% (42% to 80%).

In healthy subjects, tolvaptan pharmacokinetics following a 15 mg dose as a 1 mg/mL suspension shows a more rapid absorption (the median  $t_{max}$  is shorter, 1.00 versus 2.00 hours respectively), when compared to a 15 mg tablet. The geometric mean ratio (90% CI), for suspension over the tablet, for  $C_{max}$  is 1.614 (1.484 to 1.754) but AUC is unchanged.<sup>14</sup>

Trials in subjects with hyponatremia secondary to liver disease showed that following a single oral dose, tolvaptan concentrations increase dose proportionally from 5 to 60 mg. The clearance following single oral doses of tolvaptan was independent of the dose and similar to clearance in healthy subjects. Following multiple oral doses, tolvaptan concentrations accumulated 2-fold and clearance was decreased about 50%. <sup>14</sup>

Once a day dosage regimen trials in CHF subjects with extracellular volume expansion showed that tolvaptan concentrations increased less than proportionally with dose upon multiple dosing regimens (10, 15, 30, 60, 90, and 120 mg once daily for 13 days) in this subject population. The  $t_{1/2,z}$  and CL/F were unchanged across dose groups. Compared to healthy subjects, the disposition of tolvaptan is slower with longer  $t_{1/2,z}$  (7.8 to 11.1 hours) and smaller CL/F (0.9 to 3.3 mL/min/kg). The  $C_{max}$  was 2- to 2.5-fold greater than that of healthy subjects (at 60- and 90-mg doses). The median volume of distribution following extravascular administration of tolvaptan ranged from 1 to 2.5 L/kg and was not different from healthy subjects.

Tolvaptan is a sensitive substrate for cytochrome P450 (CYP) 3A4 and has no inhibitory activity at CYP3A4. Tolvaptan administration does not produce clinically significant changes in amiodarone, warfarin (or its 7-hydroxy and 10-hydroxy metabolites), lovastatin, furosemide, or hydrochlorothiazide plasma concentrations. Steady state digoxin concentrations were increased approximately 20% (as determined by  $AUC_{\tau}$ ).

When administered with the potent CYP3A4 inhibitor ketoconazole, the ketoconazole + tolvaptan/tolvaptan alone ratio for tolvaptan mean  $C_{max}$  and AUC from

time zero to infinity values were 3.48 and 5.40, respectively. Therefore, a 4-fold reduction in tolvaptan dose is recommended when initiating tolvaptan therapy in subjects using potent CYP3A4 inhibitors and a 2-fold reduction in tolvaptan dose is recommended for subjects using moderate CYP3A4 inhibitors. Lovastatin increases tolvaptan  $C_{max}$  by approximately 20% but CL/F is unchanged. Tolvaptan  $C_{max}$  and AUC calculated to the last observable concentration at time t (AUC<sub>t</sub>) are increased 1.9- and 1.6-fold, respectively, when tolvaptan is coadministered with grapefruit juice. Following coadministration with 600 mg once daily rifampin at steady state, tolvaptan  $C_{max}$  and AUC<sub>t</sub> are decreased 83% and 87%, respectively.

When 30- or 60-mg tablet doses were given following a standard high-fat, high-calorie meal, no clinically significant differences in urine output were observed. <sup>15</sup>

Following multiple oral doses, the tolvaptan metabolite DM-4103 was found to accumulate. This metabolite has no pharmacological activity and has shown an acceptable toxicity profile. The metabolite has not been shown to accumulate in nonclinical toxicokinetic studies; however, in a 26-week study in rats, DM-4103 plasma concentrations greater than those expected at the dose used in this trial revealed no evidence of time-dependent toxicological effects. <sup>14</sup>

## 1.2.2 Pharmacodynamics

Tolvaptan increases urine excretion rate at concentrations around 20 ng/mL and maximal urine excretion rates are reached between 100 and 150 ng/mL. A single oral dose trial in healthy subjects using doses from 60 to 240 mg showed that there were 1) no further increases in urine excretion rate with doses beyond 180 mg; 2) no further increases in zero to 24 hour urine excretion with doses beyond 180 mg; and 3) as dose was increased, increases in urine excretion were sustained over time. Tolvaptan elevated electrolyte-free water clearance to a positive value, increased serum sodium and serum osmolality, and increased plasma AVP concentrations and renin activity, but no dose-related increases were observed for any other parameter.

When compared to a 15-mg spray-dried tablet, the pharmacodynamic profiles of urine excretion rate, cumulative urine volume, free water clearance, urine osmolality, and serum sodium were not different for 15-mg of the suspension.<sup>14</sup>

Details of the currently available PK/PD data for the compound are available in the IB. 14

## 1.2.3 Clinical Efficacy

Thirteen trials involving either exclusive evaluation of adult subjects with hyponatremia (10 trials in which all subjects have hyponatremia and a long-term extension trial) or substantial subpopulations of subjects with hyponatremia (3 CHF trials - not all subjects in these trials had hyponatremia) have been conducted.

Briefly, in clinical trials, tolvaptan has consistently been shown to improve or normalize serum sodium concentrations in hyponatremic subjects, regardless of etiology. In clinical trials in subjects with volume overload and hyponatremia, the effect of tolvaptan on serum sodium is combined with a reduction in fluid overload, as shown by greater decreases in body weight compared to placebo. Additionally, subjects with liver disease responded to higher doses of tolvaptan with reductions in body weight.<sup>14</sup>

Data from two phase 3, multicenter, randomized, double-blind, placebo-controlled trials evaluating tolvaptan in euvolemic and hypervolemic hyponatremia subjects (Study of Ascending Levels of Tolvaptan in Hyponatremia [SALT] 1 and 2 trials) served as the basis for approval in the US and Europe. A total of 448 subjects were randomized in these trials (oral placebo n = 223 and tolvaptan n = 225) for a 30-day treatment period. The first single daily dose (15 mg) was monitored in-hospital with optional fluid restriction. Subjects were discharged and fluid intake and tolvaptan (30 or 60 mg) were titrated as clinically indicated.

The primary efficacy endpoints for the SALT 1 and 2 trials were the average daily AUC of change from baseline in serum sodium concentration up to Day 4 and up to Day 30. For both primary endpoints, the difference between the treatment groups were highly statistically significant (p < 0.0001), and demonstrated that serum sodium concentrations increased more with tolvaptan than placebo over the first 4 days and the entire 30 days. Significance was seen in both mild and severe hyponatremia subgroups (p < 0.001). When tolvaptan therapy was stopped, serum sodium concentrations fell to the level of placebo concentrations (Figure 1.2.3-1), but recovered upon resumption of tolvaptan therapy (Figure 1.2.3-2).



Figure 1.2.3-1 Mean (Standard Error) Changes From Baseline in Serum Sodium Concentration Following Tolvaptan or Placebo Treatment for 30 Days and at 7 Days Following Withdrawal of Therapy (Trials 156-02-235 and 156-03-238 [SALT 1 and 2] Combined)

7DFU = 7-day follow-up.



BSL = Baseline, 7FU = 7-day follow-up, FU = follow-up; SALTWATER = Safety and sodium Assessment of Long-term Tolvaptan With hyponatremia: A year-long, open-label Trial to gain Experience under Real-world conditions.

Figure 1.2.3-2 Mean (Standard Error) Serum Sodium Concentration Over Time From the Parent Trials (156-02-235 and 156-03-238 [SALT 1 and 2]) to the Open-label Extension Trial (156-03-244 [SALTWATER]); All Subjects (Observed Case)

Details of the currently available efficacy data for tolvaptan are available in the IB. 14

#### 1.3 Known and Potential Risks and Benefits

As of 31 Mar 2015, pooled exposure data are available from 93 trials, including 7373 subjects worldwide who were exposed to oral doses of tolvaptan. The extent of exposure to oral tolvaptan by dose in the pooled database (N = 7373) comprises 3115 subjects in trials for heart failure (HF), 511 subjects in trials for hyponatremia, 961 subjects in the pivotal long-term ADPKD trial, 270 subjects in short-term trials for ADPKD or renal impairment, 437 subjects in trials for cardiac edema, 855 subjects in trials for hepatic edema 43 subjects in trials for chronic renal failure, 43 subjects in a trial for carcinomatous edema, 37 subjects with renal impairment in a phase 1 trial, and 1101 healthy subjects in clinical pharmacology trials. As of 31 Mar 2014, additionally, 14 healthy adult subjects were also exposed to the tolvaptan suspension formulation. 14

The most commonly reported treatment-emergent adverse events (TEAEs; by > 10% incidence and greater than placebo) in healthy subjects treated with tolvaptan were thirst, pollakiuria, and headache. Headache was the most commonly reported TEAE in the placebo subjects.

The hyponatremia program comprised 835 subjects from 12 short-term trials involving either exclusive evaluation of subjects with hyponatremia (9 trials) or substantial subpopulations of subjects with hyponatremia (3 CHF trials). The 511 subjects in the hyponatremia trials were exposed to oral tolvaptan doses ranging from 5 to 60 mg, for a total of 8339 days of exposure. In the 9 hyponatremia trials, the most commonly reported TEAEs (> 5% incidence) in the tolvaptan subjects were thirst, dry mouth, peripheral oedema, nausea, dizziness, fatigue, constipation, headache, ascites, diarrhoea, pollakiuria, asthenia, hypotension, pyrexia, and hypokalaemia. The most commonly reported TEAE (> 5% incidence) in the placebo subjects were peripheral oedema, diarrhoea, headache, ascites, vomiting, dyspnoea, nausea, and hypotension. The IB provides a review of the adverse events (AEs) experienced with the spray-dried tablet and suspension formulation of tolvaptan during clinical trials. <sup>14</sup>

There is the potential for osmotic diarrhea due to the sorbitol content in the suspension. D-Sorbitol is a hexahydric sugar alcohol that naturally occurs in fruits and animal tissue. The daily per capita consumption of sorbitol as a food ingredient is approximately 200 mg. The compound is about 35-60% as sweet as sugar, and has been the impetus as a substitute for sugar to reduce caloric intake and prophylactic measures against the formation of dental caries. Absorption of sorbitol by humans is limited by its rate of diffusion from the GI tract and by laxation that may occur after ingestion of high doses. Typically, 25-50 g in adults may cause osmotic diarrhea. The corresponding dose in children is thought to be 10 g and higher, but is dependent on body weight and types of foods ingested. Similar findings are also observed with other sugar alcohols, eg, xylitol. <sup>16</sup>

Following a single 15 mg tolvaptan dose of the suspension, containing 8 g of sorbitol, in healthy adults, no diarrhea was reported. 14

Therefore, in this trial, suspension dosing is limited to subjects who weigh  $\leq$  30 kg; the maximum dose of sorbitol is expected to be approximately 9.6 grams in a 0.6 mg/kg dose for a subject who weighs 30 kg. Subjects will be started on the lowest dose for their weight and titrated to higher doses as appropriate for their clinical condition. Subjects will be in a hospital setting during titration and will be closely monitored for rate of sodium correction and signs of dehydration including diarrhea.

Analyses of the completed 3-year pivotal Trial 156-04-251 (double-blind, placebo-controlled trial to determine long-term safety and efficacy of oral tolvaptan in adult subjects with ADPKD) have revealed new and important safety information. In this trial, a new signal for imbalanced elevations of liver transaminases in ADPKD subjects

receiving tolvaptan compared with placebo was detected and formally adjudicated by an expert panel blinded to treatment.

Based on the analyses of combined central and local laboratory data, a total of 3 tolvaptan subjects in the ADPKD program (2 in Trial 156-04-251 and one in the ongoing extension Trial 156-08-271) were identified as meeting Hy's Law laboratory criteria (ie, alanine transaminase [ALT] or aspartate transaminase [AST] > 3 times the upper limit of normal [ULN] accompanied by total bilirubin >  $2 \times ULN$  with the elevated total bilirubin occurring within 30 days after the transaminase elevation). Based on review of the data from the adjudicated subjects, the transaminase elevations associated with tolvaptan treatment were reversible (ie, returned to  $\le 3 \times ULN$  typically within 1 to 4 months), and were not associated with fulminant liver failure, or permanent liver injury or dysfunction.

No association with tolvaptan dose or exposure was found. The results do not appear to suggest an association between tolvaptan and age or gender with respect to an increased risk of potential liver injury.

Retrospective evaluation of data from the hyponatremia and HF clinical development programs did not reveal an imbalance of subjects with elevated ALT between tolvaptan and placebo groups. In addition, no signal of tolvaptan-induced hepatotoxicity has been detected in the review of the postmarketing experience to date for any non-ADPKD indication. However, these data are not adequate to exclude the possibility that subjects treated with tolvaptan are at a potential increased risk for liver injury. Further details regarding this issue can be found in the IB. <sup>14</sup>

In clinical trials, tolvaptan consistently has shown a beneficial effect in hyponatremic subjects by improving serum sodium concentrations, in many cases to normalization. In subjects with HF, tolvaptan has consistently shown a beneficial effect by improving fluid balance through the induction of increased urine volume. In subjects with volume overload and hyponatremia receiving optimal standard HF therapy, the effect of tolvaptan on serum sodium is combined with a reduction in fluid overload, as shown by greater decreases in body weight as compared with placebo. In subjects hospitalized with worsening HF and symptoms of fluid overload, tolvaptan treatment, in addition to continued conventional therapy including diuretics, increased weight reduction, improved subject-assessed dyspnea and pedal edema, normalized serum sodium concentrations in subjects with hyponatremia, and maintained renal function in comparison to placebo.

Additional safety information can be found in the IB. <sup>14</sup> To date, no clinical trials in children have been completed with tolvaptan.

# 2 Trial Rationale and Objectives

#### 2.1 Trial Rationale

The purpose of this trial is to establish the effects of tolvaptan on serum sodium concentration as well as the safety of use of tolvaptan in children and adolescents with euvolemic or hypervolemic hyponatremia secondary to

In addition, blood samples will be taken to determine tolvaptan PK specific to a pediatric population, as the absorption, distribution, metabolism, and elimination of drugs in children and adolescents can vary from that of adults. These differences can be due to differences in physiology based on maturity status (eg, GI transit times are faster, the ratio of total body water to body fat is shifting, and the expression of drug metabolizing enzymes change) or based on underlying disease state. Hyponatremia alone does not appear to affect tolvaptan PK; however, tolvaptan exposure is 2-fold greater in adult subjects with CHF compared to healthy adult subjects and clearance appears to decrease about 50% in subjects with moderate to severe hepatic failure (Child-Pugh score > 6). As the primary pharmacodynamic effect of tolvaptan is to produce an increase in urine output (aquaresis), urine output and fluid intake will be determined as PD endpoints.

The proposed population size of 100 subjects is expected to yield 70 subjects who respond to tolvaptan (henceforth termed "responders"), which has adequate power (> 90%) to test for statistical significance in the primary endpoint. Enrollment is expected to take approximately 3 years using approximately 60 sites globally. Additional blood sampling will be included across populations to provide PK information.

Even with a limited size, recruitment for such a trial is expected to be challenging due to the low frequency of AVP-mediated hyponatremia in children. Therefore, the trial will be organized at major pediatric referral centers to access the largest patient population.

It is recognized that the pediatric population is a vulnerable subgroup and there are risks in conducting a clinical trial in the pediatric population. However, given the possible serious and life-threatening consequences of untreated hyponatremia, it is necessary to study hyponatremia treatment in children. Children have different physiology and metabolisms from adults and, therefore, it is not sufficient to study hyponatremia treatment in the adult population to determine the proper course of treatment for hyponatremia in the pediatric population. A clear understanding of exposure-response in adults that can be applied to pediatrics (or from one pediatric group to another) has not yet been established, furthering the need for this trial. <sup>18</sup>

Every effort will be made to anticipate and reduce known risks. This trial was designed to minimize the number of participants and the number of procedures, consistent with good study design. <sup>19</sup> Children will be continuously monitored for signs of distress during this trial. The risk threshold for subjects will be constantly monitored by the investigator. A detailed list and description of the safety monitoring to be conducted during this trial can be found in Section 3.7.4.

#### 2.1.1 Dosing Rationale

Enrolled subjects will be dosed based on formulation type, age, weight, and the use of CYP3A4 inhibitors.

In the pivotal hyponatremia trials <sup>14,20,21</sup> the starting 15-mg dose was administered to adult subjects weighing 34.0 to 164.7 kg; in terms of mg/kg, the starting dose of tolvaptan ranged from 0.09 to 0.44 mg/kg. The weight cutoffs for use of tolvaptan tablets in this trial were selected to produce mg/kg doses of tolvaptan within the range observed for the adult trials. Table 2.1.1-1 outlines the mg/kg dose ranges for tolvaptan tablet doses and body weights of 10, 20, 50, 70 (standard adult man), and 100 kg.

| <b>Table 2.1.1-1</b> | Starting Tolvaptan Tablet Doses as mg/kg of Body Weight | | | | |
|---|---|---|---|---|---|
| Tolvaptan | Tolvaptan Doses as mg/kg | | | | |
| Tablets | BW of 10 kg | BW of 20 kg | BW of 50 kg | BW of 70 kg | BW of 100 kg |
| 3.75 mg | 0.375 | 0.19 | - | - | - |
| 7.5 mg | - | 0.375 | 0.15 | - | - |
| 15 mg | = | = | 0.30 | 0.21 | 0.15 |

BW = body weight.

Tolvaptan is metabolized by the CYP3A isozyme. At birth, the amount of CYP3A per gram of liver is less than in an adult, but adult levels of CYP3A are reached by 2 years of age. A physiologically-based pharmacokinetic model of adult tolvaptan concentrations was modified to estimate tolvaptan concentrations in subjects from  $\geq 4$  weeks (or  $\geq 44$  weeks of adjusted gestational age) to < 2 years of age and in subjects  $\geq 2$  to < 4 years of age. It was estimated that doses of 0.1 mg/kg and 0.15 mg/kg, respectively, of the suspension would produce peak tolvaptan concentrations similar to those produced by a 15 mg tablet in an adult subject. However, overall exposure for the suspension as determined by AUC would be 33% and 13% lower, respectively, for subjects < 2 years of age and subjects  $\geq 2$  to < 4 years of age when compared to a 15 mg tablet in an adult. It is expected that a 0.15 mg/kg starting dose of tolvaptan suspension would also be suitable for children > 4 years of age, as CYP3A expression would be the same as for children  $\geq 2$  to 4 years of age. Suspension will only be administered to

children who weigh 30 kg or less to limit the amount of sorbitol administered; a 30 kg child titrated to a 0.6 mg/kg dose of tolvaptan suspension would receive 18 mL of tolvaptan suspension, containing approximately 9.6 g of sorbitol.

Tolvaptan is a sensitive CYP3A4 substrate; plasma concentrations increased approximately 4-fold when tolvaptan was administered with the potent CYP3A4 inhibitor ketoconazole. Where appropriate dose reductions are possible, tolvaptan doses may be coadministered with potent or moderate CYP3A4 inhibitors. Table 3.2.3-1 outlines starting dose adjustments when tolvaptan is administered concurrently with potent or moderate CYP3A inhibitors.

#### 2.2 Trial Objectives

## 2.2.1 Primary Objective

The primary objective is to demonstrate that tolvaptan effectively and safely increases and maintains serum sodium concentrations in children and adolescent subjects with euvolemic or hypervolemic hyponatremia.

### 2.2.2 Secondary Objectives

The key secondary objective is to assess the PK of tolvaptan and the effect on fluid balance in children and adolescent subjects with euvolemic or hypervolemic hyponatremia.

# 3 Trial Design

## 3.1 Type/Design of Trial

This is an open-label, multicenter, multiple-dose, randomized withdrawal, parallel-group trial of tolvaptan in children and adolescents hospitalized with chronic euvolemic or hypervolemic hyponatremia (serum sodium < 130 mEq/L [mmol/L]) persisting despite initial standard therapy. A schematic of the trial design is provided in Figure 3.1-1.


**PI = Principal investigator.** 

Figure 3.1-1 Trial Design Schematic

#### 3.1.1 Trial Phases

Screening should be performed on Days -2 to -1 to confirm eligibility, followed by the 3 trial phases described in Section 3.7.1.

#### 3.1.1.1 Treatment Phase A

All subjects will initially receive tolvaptan once daily on Days 1 and 2. If a subject's serum sodium level has not increased by at least 4 mEq/L (mmol/L) by Day 2, an additional day of treatment is required and is referred to as Day 2a. If subjects do not achieve an increase in serum sodium concentration of  $\geq$  4 mEq/L (mmol/L) on Day 2a, they will be defined as nonresponders. If subjects achieve an increase in serum sodium concentration of  $\geq$  4 mEq/L (mmol/L) on Day 2 (or 2a) they will be defined as responders.

#### 3.1.1.2 Treatment Phase B

On Day 3 responders will be randomized (Section 3.1.1.2.1) to either the Early Withdrawal group or the Late Withdrawal group. Nonresponders will not be randomized.

For nonresponders from Treatment Phase A, the investigator will determine if the subject is to either:

- Continue treatment with study drug or
- Prescribe treatment per local standard of care for Days 3 and 4.

#### 3.1.1.2.1 Randomization

Responders will be randomized to either:

- Late Withdrawal group subjects continue tolvaptan treatment on Days 3 and 4
- Early Withdrawal group subjects do not receive additional tolvaptan treatment on Days 3 and 4.



Subjects randomized to the Early Withdrawal group will be observed to determine whether additional intervention is required to maintain appropriate serum sodium levels. Subjects whose serum sodium declines by  $\geq 4$  mEq/L (mmol/L) or whose overall clinical condition requires further treatment to raise serum sodium levels should be treated per local standard of care. Any intervention intended to raise serum sodium concentration during the first 48 hours of the Early Withdrawal phase (including fluid restriction) will be defined as rescue therapy. Subjects receiving rescue therapy will be considered to

Protocol 156-08-276

have reached their clinical endpoint, and their data will be censored from that time forward.

# 3.1.1.3 Follow-up Phase C

All subjects will have an additional serum sodium measurement at 72 ( $\pm$  4) hours post-last dose and 7 ( $\pm$  1) days post-last dose. A final safety follow-up telephone contact/visit will be performed 14 ( $\pm$  2) days post-last dose.

#### 3.2 Trial Treatments

### 3.2.1 Tablet Formulation

Tolvaptan tablets will be administered orally once daily, preferably in the morning hours, with a dose proportional amount of water, as follows:

- Doses of  $\geq$  15 mg tolvaptan will be given with 240 mL of water.
- Doses of 7.5 mg tolvaptan will be given with 120 mL of water.
- Doses of 3.75 mg of tolvaptan will be given with 60 mL of water.

The treatment duration will be up to 5 days. Any initiation or titration of tolvaptan must occur in a hospital setting.

The maximum starting doses, by weight, age, and CYP3A inhibitor, for subjects are shown in Table 3.2.3-1 and are within the range previously used in trials involving adult hyponatremic subjects.

The investigator has the option of performing a swallow test and providing coaching on swallowing techniques using placebo tablets if it is unknown if the subject is able to swallow tablets. Placebo tablets will be provided for use in performing this test during screening.

# 3.2.2 Suspension Formulation

Tolvaptan suspension, 1 mg/mL (0.1% w/v), will be administered orally once daily, preferably in the morning hours. The treatment duration will be up to 5 days. Any initiation or titration of tolvaptan must occur in a hospital setting.

The maximum starting doses for subjects, by weight, age, and CYP3A inhibitor are shown in Table 3.2.3-1.

# 3.2.3 Dosing Guidelines

Subjects will be administered tolvaptan on a formulation, age- and weight-based scale.

Table 3.2.3-1 outlines starting tolvaptan doses and adjustments when tolvaptan is administered concurrently with potent or moderate CYP3A inhibitors. Tolvaptan doses will be reduced 75% and 50% if a potent or moderate inhibitor, respectively, is being concurrently administered. As the smallest volume of suspension that can be administered is 0.3 mL (0.3 mg), subjects weighing < 3 kg, < 6 kg and taking a moderate or a potent CYP3A4 inhibitor, or weighing < 12 kg and taking a potent CYP3A4 inhibitor may not be enrolled. Suspension should be administered with the syringes provided.

| Table 3.2.3-1 Starting Tolvaptan Doses With or Without Potent or Moderate CYP3A Inhibitors | | | | |
|---|---|---|---|---|
| Age/Weight | Can subject swallow a tablet? | Starting Dose: No<br>CYP Inhibitor | Starting Dose:<br>Moderate CYP<br>Inhibitor | Starting Dose:<br>Potent CYP<br>Inhibitor |
| $\geq$ 4 wk (or ≥ 44 wk<br>adjusted gestational<br>age) to < 2 y AND<br>$\geq$ 3 kg to < 6 kg <sup>c</sup> | N/A | 0.1 mg/kg<br>suspension a,b | Not eligible for treatment | Not eligible for treatment |
| $\geq$ 4 wk (or $\geq$ 44 wk<br>adjusted gestational<br>age) to < 2 y AND<br>$\geq$ 6 to < 12 kg <sup>c</sup> | N/A | 0.1 mg/kg<br>a,b<br>suspension | 0.05 mg/kg<br>suspension | Not eligible for treatment |
| $\geq 2 \text{ y to } \leq 6 \text{ y AND}$<br>$\leq 30 \text{ kg}^{\text{c}}$ | N/A | 0.15 mg/kg<br>suspension | 0.08 mg/kg suspension | 0.04 mg/kg<br>suspension |
| > 6 y AND ≤ 30 kg | No | 0.15 mg/kg<br>suspension | 0.08 mg/kg<br>suspension | 0.04 mg/kg<br>suspension |
| > 6 y AND 20 to 50 kg | Yes | 7.5 mg tablet | 3.75 mg tablet | 1.90 mL suspension |
| > 6 y AND > 50 kg | Yes | 15 mg tablet | 7.5 mg tablet | 3.75 mg tablet |

<sup>&</sup>lt;sup>a</sup> The smallest volume of suspension that may be administered is 0.3 mL (0.3 mg), therefore dose reductions cannot be accommodated for children < 6 kg taking moderate inhibitors and for children < 12 kg taking potent inhibitors.

Titration of tolvaptan doses can occur once daily and will be based on serum sodium levels assessed at > 20 hours following initiation of therapy and each subsequent dose; titration may not occur within 24 ( $\pm$  4) hours of the previous dose. Up-titration is limited to no more than twice the previous dose.

- Subjects  $\geq$  4 weeks (or  $\geq$  44 weeks adjusted gestational age) to < 2 years of age and weighing  $\geq$  3 kg to < 6 kg will receive 0.1 mg/kg of the suspension on Day 1 with possible up-titration to 0.2 mg/kg and 0.4 mg/kg doses.
- Subjects ≥ 4 weeks (or ≥ 44 weeks adjusted gestational age) to < 2 years of age and weighing ≥ 6 kg to < 12 kg will receive 0.1 mg/kg of the suspension on Day 1 with possible up-titration to 0.2 mg/kg and 0.4 mg/kg doses.

b Tolvaptan suspension is provided in a concentration of 1 mg/mL.

<sup>&</sup>lt;sup>c</sup> Suspension required (pediatric subjects  $\leq$  6 years of age and  $\leq$  30 kg body weight).

- Subjects ≥ 2 to ≤ 6 years of age, weighing ≤ 30 kg will receive a 0.15 mg/kg dose of the suspension on Day 1 with possible up-titration to 0.3 mg/kg and 0.6 mg/kg doses.
- Subjects > 6 years of age, weighing ≤ 30 kg and who cannot safely swallow a tablet, will receive a 0.15 mg/kg dose of the suspension on Day 1 with possible up-titration to 0.3 mg/kg and 0.6 mg/kg doses.
- Subjects > 6 years of age and weighing 20 to 50 kg, inclusive, will receive a 7.5 mg tablet on Day 1 with possible up-titration to 15-mg and 30-mg doses.
- Subjects > 6 years of age and weighing > 50 kg, will receive a 15 mg tablet on Day 1 with possible up-titration to 30-mg and 60-mg doses.

Following their initial tolvaptan dose in the trial, subjects will continue dosing according to the titration scheme (see Section 3.2.4), targeting a final serum sodium concentration between 135 and 140 mEq/L (mmol/L). Titration guidelines are designed to achieve a change in serum sodium concentration of at least 4 to 8 mEq/L (mmol/L)/24 hours but not

# 3.2.4 Titration Guidelines and Rescue Therapy

Initiation and titration of tolvaptan must occur in a hospital setting. Up titration can only take place on Treatment Day 2 (or 2a). Titration (up or down) may not occur within 20 hours of the previous dose. Up-titration is limited to no more than twice the previous dose.

The medical monitor should be contacted at any point if questions arise regarding titration or initiation of rescue therapy. The rationale for any up- or down-titration of tolvaptan must be documented. The evaluation of serum sodium levels, management of tolvaptan titration, and rescue therapy is described in Figure 3.2.4-1.



Figure 3.2.4-1 Titration and Rescue Therapy Scheme

1 mEq/L = 1 mmol/L.

Figure 3.2.4-1 Titration and Rescue Therapy Scheme

### **3.2.4.1** Titration

Tolvaptan dose titration (after the initial dose) should be based on changes in serum sodium levels as follows:

• If the serum sodium level increases by  $\leq 4$  mEq/L (mmol/L)/24 hours and the subject is still below the therapeutic target for serum sodium level

- (135 mEq/L [mmol/L]), then the tolvaptan dose may be titrated up to the next scheduled dose appropriate for the subject's body weight.
- If the serum sodium level increases > 4 to  $\le 8$  mEq/L (mmol/L)/24 hours in response to tolvaptan treatment and the serum sodium is  $\le 140$  mEq/L (mmol/L), then the dose of tolvaptan should remain the same for the subsequent day.
- If the serum sodium level increases > 8 mEq/L (mmol/L)/24 hours or reaches a concentration of > 140 mEq/L (mmol/L), then the next dose of tolvaptan should not be given and the medical monitor should be contacted to consider options (ie, down-titration, tolvaptan interruption, concomitant medication adjustment, fluid supplementation and/or withdrawal).
- If serum sodium level increases by following dosing, or, at any time after dosing, the serum sodium level is
   145 mEq/L (mmol/L), the next dose of tolvaptan should not be given and the medical monitor should be contacted immediately to consider options.

# 3.2.4.2 Rescue Therapy

Rescue therapy is defined as any treatment, eg, hypertonic saline, isotonic saline (with or without diuretic for purpose of increasing the serum sodium level), plasmapheresis/dialysis, demeclocycline, urea, lithium, or commercially available vaptans intended to raise the level of serum sodium during the trial. Subjects who develop worsening hyponatremia symptoms may receive rescue therapy at any time during the trial.

If at any point during the trial serum sodium levels or hyponatremia symptoms worsen or fail to improve adequately and definitive therapy (eg, isotonic or hypertonic saline) is required, the subject will be withdrawn from trial treatment to receive rescue therapy Please see Section 4.2 for further details. These subjects will continue to Follow-up Phase C for collection of safety information.

Additional guidelines for rescue therapy concerning hyponatremia symptoms and decreasing serum sodium level:

- If a subject has worsening symptoms and/or has a serum sodium level at or below the baseline value, repeat serum sodium [STAT] to confirm level, and begin rescue therapy.
- If a subject is asymptomatic and serum sodium has decreased by ≥ 4 mEq/L (mmol/L), but is still above the baseline value, consider need for rescue therapy according to local standard of care.
- If a subject is asymptomatic and serum sodium has decreased by ≤ 3 mEq/L (mmol/L), but is still above the baseline value, no action is required.

Subjects who are randomized to the Early Withdrawal group will initially be observed to determine whether additional intervention is required to maintain appropriate serum sodium levels. For those subjects whose serum sodium declines by  $\geq 4$  mEq/L (mmol/L) or whose overall clinical condition requires further treatment to increase serum sodium, the investigator may consider rescue therapy per local standard of care. Any intervention intended to raise serum sodium level during the first 48 hours in the responder Early Withdrawal group (including fluid restriction) will be defined as rescue therapy. These subjects will be considered to have reached their clinical endpoint, and their data will be censored from that time forward.

Subjects randomized to the Late Withdrawal group who receive rescue therapy will be considered treatment failures. A subject requiring rescue therapy at any time after starting tolvaptan will be discontinued from trial treatment and will proceed to Follow-up Phase C.

### 3.2.4.3 Fluid Restriction Considerations

In subjects with chronic hyponatremia, fluid restriction coadministered with initiation of treatment with a vaptan has the potential to accentuate the rate of sodium correction and to cause overly rapid correction or over correction of hyponatremia. Therefore, during treatment, subjects must have access to water and maintain fluid intake levels per institutional guidelines. Fluid restriction at any time during the trial including during the first 48 hours after discontinuation of tolyaptan will be considered rescue therapy.

## 3.3 Trial Population

This trial will include approximately 100 male and female subjects aged  $\geq 4$  weeks (or  $\geq 44$  weeks adjusted gestational age) to < 18 years who have been diagnosed with euvolemic or hypervolemic hyponatremia (< 130 mEq/L [mmol/L]) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). Age groups will be enrolled such that at least 50% of these subjects will be < 10 years old and at least 25% of subjects < 6 years old. Subjects who are defined as responders will be further stratified by the magnitude of serum sodium response to tolvaptan ( $\leq 7$  and  $\geq 7$  mEq/L [mmol/L]), age, and underlying etiology of hyponatremia.

## Hyponatremia Etiology in Children and Adolescents

Children with Factor V Leiden or Factor VII abnormalities may be eligible for treatment only if the benefit is judged to outweigh any risk. Tolvaptan may be administered to children with hepatocellular disease (including cirrhosis) who have platelet counts

Protocol 156-08-276

between 50,000 and  $100,000/\mu L$  if the need to treat is felt to outweigh the increased risk of GI bleeding.

Children can develop symptomatic hyponatremia more frequently than adults and at less severe levels of hyponatremia because of the large brain volumes in relatively small skulls. The most serious consequence of hyponatremia is hyponatremic encephalopathy, which occurs in over 50% of children with serum sodium < 125 mmol/L.<sup>24</sup>

Hyponatremic encephalopathy is seen in hospitalized children and adolescents in association with SIADH or in the postoperative period. Hyponatremic encephalopathy is a medical emergency that requires immediate intervention; <sup>25,26,27</sup> thus, subjects with known risk factors for developing hyponatremic encephalopathy may be ineligible for tolvaptan treatment (eg, hypoxia, infection, brain injury, neurosurgery, uncontrolled seizure disorders, cerebritis, encephalopathy, central nervous system disorders such as cytotoxic and vasogenic cerebral edema, unstable space-occupying brain lesion, or elevated AVP levels).

Symptoms include headache, nausea and vomiting, weakness, confusion, altered consciousness, and lethargy and may progress to more advanced symptoms, including seizures, coma, and death, if untreated. Subjects with overt symptoms of hyponatremia that require immediate intervention to raise serum sodium acutely will be ineligible for tolvaptan treatment; this syndrome is rapidly reversible with hypertonic saline administration.

Additionally, those subjects who are at risk of developing cerebral demyelination will be ineligible for tolvaptan treatment, including subjects who have severe hyponatremia ≤ 120 mEq/L (mmol/L), hypernatremia, hypoxemia, severe liver disease, alcoholism, severe burns, severe malnutrition, hypokalemia, diabetes, or renal failure. <sup>24,25</sup>

Subjects eligible for treatment with tolvaptan will be identified based on serum sodium concentrations that persist at levels < 130 mEq/L (mmol/L). Upon determination of eligibility, each subject's serum sodium will be reassessed just before tolvaptan administration to confirm it remains below this threshold prior to intended treatment initiation.

If any serum sodium value obtained during the pretreatment baseline period for tolvaptan treatment is  $\geq 130$  mEq/L (mmol/L), the subject will be ineligible for tolvaptan administration at that time.

Sorbitol is metabolized to fructose.<sup>28</sup> Subjects who have hereditary fructose intolerance (HFI) who continue to ingest fructose containing products can develop hepatic and renal

dysfunction.<sup>29</sup> The tolvaptan suspension formulation contains sorbitol. Therefore, children who have HFI should not take the tolvaptan suspension formulation.

Hereditary fructose intolerance is typically diagnosed in young children upon the introduction of solid foods containing fructose, sucrose and/or sorbitol (eg, fruits and vegetables). It is not commonly diagnosed in children who are fed exclusively on breast milk. Clinical symptoms can include vomiting, nausea, restlessness, pallor, sweating, lethargy, coagulation disturbances and in some cases, apathy, coma, and convulsions. Laboratory abnormalities may include signs of acute liver failure (eg, elevated serum transaminases, hyperbilirubinemia, abnormal blood clotting factors) or renal failure (eg, proteinuria, generalized hyperaminoaciduria, metabolic acidosis). Continued exposure to fructose can result in hypoglycemia, hepatomegaly, jaundice, steatosis, coagulation disturbances, edema, ascites and signs of proximal renal tubular dysfunction. If HFI is suspected, a thorough history that emphasizes nutritional complaints including the timing of the introduction of fruits and vegetables to the diet should be obtained as well as the appropriate laboratory assessment for confirmation of diagnosis.

For children aged > 2 years, a detailed history with regard to HFI symptoms has to be taken prior to trial entry.

# 3.3.1 Subject Eligibility by Hyponatremia Etiology

#### 3.3.1.1 General Guidelines

Investigators should assess subjects' appropriateness to receive tolvaptan. Investigators should ultimately use their medical judgment to make the final determination. It remains the responsibility of the investigator to determine the etiology of hyponatremia and to assess the volume status for each subject using diagnostic tests (eg, fractional excretion of sodium [FENa], fractional excretion of urea [FE urea], urine osmolality, serum osmolality) employed in the usual clinical course of care.

# 3.3.1.2 Specific Guidelines by Etiology

- Subjects diagnosed with hyponatremia secondary to SIADH will be evaluated specifically to ensure appropriate volume status. Hypovolemic states are not compatible with tolvaptan administration. Plasma and urine sodium, potassium, creatinine, and urea should be assessed in order to calculate and evaluate FENa and FE urea prior to dosing to ensure safety of tolvaptan administration.
- For hyponatremia due to hepatocellular disease (including cirrhosis), in addition to the above guidelines, the underlying etiology of hepatocellular disease must be documented.
- For hyponatremia due to HF:
  - 1) A definitive diagnosis of HF by a cardiologist must be documented.

2) Loop diuretic use should be assessed and minimized where possible. Steady doses of diuretics are acceptable. Thiazide diuretics must be stopped before tolvaptan administration; the time that these medications must be stopped prior to the first tolvaptan dose depends on the half-life of the diuretic. At least 1 day or a minimum of 3 half-lives are required for washout.

The medical monitor should be contacted if there are questions. The guidelines listed in Table 3.3.1.2-1 are to help guide the medical judgment of the investigator.

| Table 3.3.1.2-1 | Screening Algorithms by Hyponatremia Etiology |
|---|---|
| Etiology | Instruction |
| All etiologies | Two documented serum sodium assessments of < 130 mEq/L (mmol/L) at least 12 hours apart |
| | One serum sodium assessment of < 130 mEq/L (mmol/L) within 2-4 hours prior to tolvaptan administration |
| | Screen subjects for AKI criteria per exclusion criteria |
| | Collect labs <sup>a</sup> |
| | Calculate serum osmolality, FENa, and FE urea at pretreatment baseline only |
| HF | Cardiologist documented diagnosis of HF |
| | Discontinue or stabilize diuretic use prior to tolvaptan administration |
| Hepatocellular disease (including cirrhosis) | The underlying etiology of hepatocellular disease must be documented |

AKI = acute kidney injury.

#### 3.4 Eligibility Criteria

#### 3.4.1 Informed Consent/Assent

Written informed consent and assent, as appropriate, will be freely obtained from the subject's parent/legal guardian or legally acceptable representative, as applicable for local laws, in accordance with requirements of the trial center's institutional review board/independent ethics committee (IRB/IEC). The subject, as required by the trial center's IRB/IEC, must provide informed assent at screening and as such must be able to understand that he or she can withdraw from the trial at any time.

Age-appropriate assent documents will be created and subjects who are able will be required to reconsent or assent as appropriate if they matriculate from one age group to another. Subjects who became legal adults during the trial will be required to provide written informed consent as soon as they reach legal age.

Consent and assent will be documented on a written informed consent form (ICF). The ICF will be approved by the same IRB/IEC that approves this protocol. Each ICF will comply with the International Conference on Harmonisation (ICH) Good Clinical

<sup>&</sup>lt;sup>a</sup>Refer to Table 3.7.4.2.3-1 for complete lists of laboratory assessments.

Protocol 156-08-276

Practice (GCP) Guideline<sup>30</sup> and local regulatory requirements. The investigator will review any written ICF/assent used in the trial, prior to submission to the IRB/IEC.

Investigators may discuss trial availability and the possibility for entry with a potential subject and his/her family without first obtaining consent and assent, as applicable. However, informed consent/assent (as applicable) must be obtained and documented prior to initiation of any procedures that are performed solely for the purpose of determining eligibility for this trial, including withdrawal from current medication(s).

Once appropriate essential information has been provided and fully explained in layman's language to the subject and his/her parent/legal guardian or legally acceptable representative by the investigator (or a qualified designee), the IRB/IEC-approved written ICF will be signed and dated by both the subject's parent/legal guardian or legally acceptable representative and the person obtaining consent (investigator or designee), as well as by any other parties required by the IRB/IEC. In addition, the subject, as required by the trial center's IRB/IEC, must provide informed assent by signing the appropriate form for their age group. The subject's parent/legal guardian or legally acceptable representative will receive a copy of the signed ICF and assent form (as applicable); the originals shall be kept on file by the investigator.

Subjects' parents/legal guardian(s) or legally acceptable representative(s) may be asked to sign additional ICFs if the protocol is amended to significantly add or change procedures. Subjects who are able may be asked to re-assent as appropriate if the protocol is amended to significantly add or change procedures.

## 3.4.2 Inclusion Criteria

Subjects are required to meet the inclusion criteria presented in Table 3.4.2-1.

| Tab | le 3.4.2-1 Inclusion Criteria |
|---|---|
| 1. | Male and female subjects $\geq$ 4 weeks (or $\geq$ 44 weeks adjusted gestational age) to $<$ 18 years old |
| 2. | Subjects hospitalized with euvolemic or hypervolemic hyponatremia resistant to initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist) and who are |
| | deemed by the investigator as likely to benefit from a therapy that raises serum sodium levels |
| 3. | Persistent euvolemic or hypervolemic hyponatremia defined as being documented as present for at least 48 hours, evidenced by at least 2 serum sodium assessments < 130 mEq/L (mmol/L) drawn at least 12 hours apart (these values can be documented using historical values previously obtained per standard of care); a third (STAT) serum sodium assessment < 130 mEq/L (mmol/L), which will |
| | serve as the baseline value for final trial qualification and clinical management strategy, is to be obtained within 2-4 hours prior to the first dose of tolvaptan |
| 4. | Ability to take oral medication |
| 5. | Ability to maintain adequate fluid intake whether orally or via IV support with adequate monitoring |
| 6. | Ability to comply with all requirements of the trial |
| 7. | Trial-specific written informed consent/assent obtained from a parent/legal guardian or legally acceptable representative, as applicable per age of subject or local laws, prior to the initiation of any protocol-required procedures. In addition, the subject as required by local laws must provide informed assent at Screening and must be able to understand that he or she can withdraw from the trial at any time. All informed consent/assent procedures must be in accordance with the trial center's IRB/IEC and local regulatory requirements |
| 8. | Ability to commit to remain fully abstinent (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] or withdrawal are not acceptable methods of contraception) or practice double-barrier birth control during the trial and for 30 days following the last dose of IMP for sexually active females of childbearing potential |

IMP = investigational medicinal product.

## 3.4.3 Exclusion Criteria

Subjects will be excluded if they meet any of the exclusion criteria in Table 3.4.3-1.

| Tab | ole 3.4.3-1 Exclusion Criteria |
|---|---|
| 1. | Has evidence of hypovolemia or intravascular volume depletion (eg, hypotension, clinical evidence of volume depletion, response to saline challenge); if the subject has systolic blood pressure or heart rate outside of the normal range for that age volume status should be specifically clinically assessed to rule out volume depletion. |
| 2. | Has serum sodium < 120 mEq/L (mmol/L), with or without associated neurologic impairment (ie, symptoms such as apathy, confusion, or seizures) |
| 3. | Current use or expected use during the trial of a potent CYP3A4 inhibitor in subjects weighing < 12 kg or a moderate CYP3A4 inhibitor in subjects weighing < 6 kg |
| 4. | Lacks free access to water (inability to respond to thirst) or without ICU-level fluid monitoring and management |
| 5. | Has a history or current diagnosis of nephrotic syndrome |
| 6. | Has transient hyponatremia likely to resolve (eg, head trauma or post-operative state) |
| 7. | Has hyperkalemia defined as serum potassium above the ULN for the appropriate pediatric age range |

| Tab | le 3.4.3-1 Exclusion Criteria |
|---|---|
| 8. | Has eGFR < 30 mL/min/1.73 m <sup>2</sup> calculated by the following equation: |
| ٥. | |
| | eGFR (mL/min/1.73 m <sup>2</sup> ) = $0.413 \times \text{height (cm)/serum creatinine (mg/dL)}$ |
| 9. | Has AKI defined as: |
| | • Increase in serum creatinine by $\ge 0.3 \text{ mg/dL}$ ( $\ge 26.5 \mu\text{mol/L}$ ) within 48 hours; or |
| | • Increase in serum creatinine to ≥ 1.5 times baseline, which is known or presumed to have occurred within the prior 7 days; or |
| | • Urine volume < 0.5 mL/kg/h for 6 hours |
| 10. | Has severe or acute neurological symptoms requiring other intervention (eg, hyperemesis, obtundation, seizures) |
| 11. | Has had treatment for hyponatremia with: |
| | <ul> <li>Hypertonic saline (including normal saline challenge) within 8 hours of qualifying serum<br/>sodium assessments;</li> </ul> |
| | • Urea, lithium, demeclocycline, conivaptan, or tolvaptan within 4 days of qualifying serum sodium assessments; |
| | <ul> <li>Other treatment for the purpose of increasing serum sodium concurrent with dosing of trial<br/>medication</li> </ul> |
| 12. | Has anuria or urinary outflow obstruction, unless the subject is, or can be, catheterized during the trial |
| 13. | Has a history of drug or medication abuse within 3 months prior to Screening or current alcohol abuse |
| 14. | Has a history of hypersensitivity and/or idiosyncratic reaction to benzazepine or benzazepine derivatives (such as benzazepil) |
| 15. | Has psychogenic polydipsia (subjects with other psychiatric illness may be included per medical monitor approval) |
| 16. | Has uncontrolled diabetes mellitus, defined as fasting glucose > 300 mg/dL (16.7 mEq/L [mmol/L]) |
| 17. | Has screening liver function values $> 3 \times ULN$ |
| 18. | Subjects who have cirrhosis and meet any of the following conditions: a major GI bleed within the past 6 months, evidence of active bleeding (eg, epistaxis, petechiae/purpura, hematuria, or hematochezia), platelet count $< 50,000/\mu L$ , or use of concomitant medications known to increase |
| | bleeding risk |
| 19. | Has hyponatremia due to the result of any medication that can safely be withdrawn (eg, thiazide diuretics) |
| 20. | Has hyponatremia (eg, hyponatremia in the setting of adrenal insufficiency, untreated hypothyroidism, or hypotonic fluid administration) that is most appropriately corrected by alternative therapies |
| 21. | Is currently pregnant or breastfeeding |
| 22. | Has any medical condition that, in the opinion of the investigator, could interfere with evaluation of the trial objectives or safety of the subjects. |
| 23. | Is deemed unsuitable for trial participation in the opinion of the investigator |
| 24. | Participation in another investigational drug trial within the past 30 days, without prior approval from the sponsor medical monitor |
| 25. | Subjects who weigh < 3 kg |
| 26. | Unable to swallow tablets if the suspension formulation is unavailable |
| 27. | Subjects who require the suspension formulation and have Hereditary Fructose Intolerance |

eGFR = estimated glomerular filtration rate; ICU = intensive care unit.

Use of the suspension formulation is at the discretion of the local regulatory authorities and IRB/IECs.

#### 3.5 Outcome Variables

# 3.5.1 Primary Efficacy Outcome Variable

For subjects with serum sodium level increases of  $\geq 4$  mEq/L (mmol/L) (ie, responders), change in serum sodium concentration from Day 2 (or 2a) at the end of Treatment Phase A to the end of Treatment Phase B for Early compared to Late Withdrawal groups.

## 3.5.2 Key Secondary Efficacy Outcome Variable

For all subjects, the key secondary endpoint is the change in serum sodium concentration at the end of Day 2 (or 2a) in Treatment Phase A from baseline.

## 3.5.3 Other Secondary Outcome Variables

## 3.5.3.1 Safety Variables

The safety endpoints for all subjects include:

- Percentage of subjects with overly rapid increase in serum sodium level
- Change in serum sodium level from 24 hours post-last dose to 7 days post-last dose
- Percentage of subjects requiring rescue therapy (other than fluid restriction) during Treatment Phase A and Treatment Phase B
- Percentage of subjects requiring fluid restriction during Treatment Phase A and Treatment Phase B
- Vital signs, blood pressure, clinical laboratory tests, body weight, and neurological examinations

#### 3.5.3.2 Pharmacokinetic Variables

Pharmacokinetic endpoints are tolvaptan  $C_{max}$ , time to maximum (peak) plasma concentration ( $t_{max}$ ), and AUC from time zero to 24 hours (AUC<sub>0-24h</sub>) on Day 1.

## 3.5.3.3 Pharmacodynamic Variables

Pharmacodynamic endpoints are fluid intake, urine output, and fluid balance (intake minus output) every 6 hours on Days 1 and 2 in Treatment Phase A.

### 3.5.4 Exploratory Variables

• Efficacy will be assessed in nonresponders continuing on tolvaptan therapy by change from baseline in serum sodium concentration at the end of Treatment Phase B compared to the end of Treatment Phase A

- In all subjects, 24-hour excretion of sodium, creatinine, and urine osmolality on Days 1 and 2
- 24-hour sodium clearance on Day 1
- Quality of life (QoL) assessments

## 3.6 Measures to Minimize/Avoid Bias

This is an open-label trial. Subjects defined as responders from Treatment Phase A will be randomized to either the Early Withdrawal group or the Late Withdrawal group in Treatment Phase B. Treatment assignments for Treatment Phase B will be based on a computer-generated randomization code provided by Otsuka Pharmaceutical Development & Commercialization, Inc. (OPDC) Biometrics Department.

#### 3.7 Trial Procedures

Treatment in this trial will last up to 5 days. Any initiation or titration of tolvaptan must occur in a hospital setting. Parent(s)/legal guardian(s) or legally acceptable representative(s) must provide informed consent and subjects must provide informed assent (as appropriate) and be screened 1 or 2 days prior to dosing.

In Treatment Phase A, subjects who meet the inclusion and exclusion criteria will be enrolled and will be administered tolvaptan doses based on age, weight, ability to swallow a tablet, and the use of CYP3A4 inhibitors. At the end of Day 2 (or 2a) in Treatment Phase A, subjects who are responders will be randomized to either continue treatment with tolvaptan for 2 additional days (Late Withdrawal) or to discontinue tolvaptan treatment (Early Withdrawal).

In Treatment Phase B, subjects who are nonresponders may continue on tolvaptan therapy for 2 additional days or may be withdrawn from tolvaptan to be treated per the investigator's preferred standard of care. During Treatment Phase B, subjects in the Late Withdrawal group and nonresponders continuing treatment will continue to receive tolvaptan for 2 additional days and all subjects will have serum sodium levels measured at  $12 \pm 4$  hours postdose and at trough  $(24 \pm 4)$  hours post-previous dose) each day. Subjects in the Early Withdrawal group should be monitored for the first 48 hours postlast dose

In Follow-up Phase C, all subjects will be monitored and will have an additional serum sodium measurement at 72 ( $\pm$  4) hours post-last dose as well as at 7 ( $\pm$  1) days post-last dose. A final safety follow-up telephone contact/visit will be performed 14 ( $\pm$  2) days post-last dose.

#### Protocol 156-08-276

Trial assessment time points are summarized in Table 3.7-1. Section 3.7.1 provides a flow overview that describes the sequence of assessments during a visit. Section 3.7.2 provides details around efficacy assessments, Section 3.7.3 provides details around pharmacokinetic/pharmacodynamic assessments and Section 3.7.4 provides details around safety assessments.

Pharmacokinetic samples will be obtained for all subjects on Day 1 at 2 and 8 hours post-first dose and at trough (24  $[\pm 4]$  hours post-previous dose) on Days 1, 2, 3, and 4 for all subjects dosed with tolvaptan on Days 1, 2, 3, and 4, respectively, regardless of responder status. Once adequate PK data are obtained, PK sampling will be discontinued for all subjects.

Subjects will be required to be in a hospital setting during initiation or titration of tolvaptan. A subject is allowed to be discharged, if they:

- 1) Continue to come to the clinic for daily study assessments and
- 2) Are either:
  - a) A nonresponder on standard of care or
  - b) On a stable dose of study drug, or
  - c) In the early withdrawal group without study treatment.

Follow-up for all subjects may occur in the hospital if the subject has not been discharged or the subject may return for outpatient visits if the subject has been discharged from the hospital.

| Table 3.7-1 Schedule of Assessments | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening Treatment Phase A | | | Phase A | Treatment Phase B | | | Follow-up Phase C | | | |
| | Day -2 to -1 | Day 1 | Day 2 | Day 2a<br>(optional) | Day 3 | Day 4 | Day 5 <sup>a</sup> | 72 (±4) h<br>post last<br>dose | 7 (+1)<br>days post-<br>last dose | 14 (+2)<br>days post-<br>last dose | Early<br>Termin-<br>ation (ET) |
| Informed Consent/Assent | X | | | | | | | | | | |
| Inclusion/exclusion criteria | X | X | | | | | | | | | |
| Demographic information | X | | | | | | | | | | |
| Medical and hyponatremia history | X | | | | | | | | | | |
| Vital signs <sup>c</sup> | X | X | X | X | X | X | X | X | X | | X |
| 12-lead ECG | X | | | | | | | | | | |
| Height | X | | | | | | | | | | |
| Body weight <sup>d,e</sup> | X | X | X | X | X | X | X | X | X | | X |
| Physical examination f | X | X | X | X | X | X | | X | X | | X |
| Tanner staging | X | | | | | | | | | | |
| Neurological examination | X | X <sup>g</sup> | X | | X | X | | X | X | | X |
| Clinical status h assessment | X | X | X | X | X | X | | X | X | | X |
| Quality of life assessment | X | | | | | X | | | X | | |
| Alcohol/drug screen | X | | | | | | | | | | |
| Pregnancy test (if | X | | | | | | | | X | | |
| applicable) <sup>J</sup> | | | | | | | | | | | |
| Fluid intake <sup>k</sup> | | X | X | | | | | | | | |
| Urine volume | | X | X | | | | | | | | |
| Urinalysis | X | | | | | | | X | | | X |
| Urine chemistry k,l | X | X | X | | | | | | | | |
| Serum sodium <sup>m</sup> | X | X | X | X | X | X | <u></u> | X | X | | X |

| Table 3.7-1 Schedule of Assessments | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening | Treatment Phase A | | Treatment Phase B | | | Follow-up Phase C | | | | |
| | Day -2 to -1 | Day 1 | Day 2 | Day 2a<br>(optional) | Day 3 | Day 4 | Day 5 <sup>a</sup> | 72 (±4) h<br>post last<br>dose | 7 (+1)<br>days post-<br>last dose | 14 (+2)<br>days post-<br>last dose | Early<br>Termin-<br>ation (ET) |
| Hematology, coagulation, | X | | | | | | | X | | | X |
| and serum chemistry <sup>n</sup> | | | | | | | | | | | |
| Serum osmolality, FENa, and FE urea | X | | | | | | | | | | |
| TSH and cortisol <sup>o</sup> | X | | | | | | | | | | |
| PK plasma samples <sup>p</sup> | | X | X | | X | X | | | | | X |
| Tolvaptan dosing q | | X | X | X | X | X | | | | | |
| Swallow test | x <sup>r</sup> | | | | | | | | | | |
| Assessment for response to tolvaptan | | | X | X | | | | | | | |
| Palatability and acceptability assessment | | | X | | | | | | | | |
| Randomization | | | | | X | | | | | | |
| Follow-up phone call or visit | | | | | | | | | | X | |
| Vital status <sup>s</sup> | | | | | | | | | | | X |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X |

ECG = electrocardiogram; eCRF = electronic case report form; TSH = thyroid-stimulating hormone.

<sup>&</sup>lt;sup>a</sup>The Day 5 visit is only for Late Withdrawal subjects and nonresponders continuing on tolvaptan treatment.

<sup>&</sup>lt;sup>b</sup>Inclusion/exclusion criteria will be checked at screening and predose on Day 1.

<sup>&</sup>lt;sup>c</sup>Vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be assessed after the subject has been supine for ≥ 3 minutes and prior to any blood draws. Vital signs are to be assessed at 4 hours and 8 hours postdose on Day 1 and, on Days 2 through 4, at trough (24 [± 4] hours post-previous dose, but prior to the next dose).

d Record growth percentiles at screening only.

<sup>&</sup>lt;sup>e</sup>Weight will be taken predose.

- Screening: 2 assessments should be taken, at least 12 hours apart (may be part of medical history). One assessment can be combined with the serum chemistry panel.
- Treatment Phase A: Baseline (STAT) assessment will be within 2-4 hours prior to first dose. Post-first dose assessments: 8 (-1 to + 0.25) hours and trough (24 [± 4] hours postdose [STAT assessment]). Then every 12 (± 4) hours thereafter (alternating 12 hours postdose and at trough [24 (± 4) hours postdose; STAT assessment])
- Treatment Phase B: Assessments to be taken every 12 (± 4) hours (alternating 12 hours postdose and at trough [24 (± 4) hours postdose; STAT assessment])
- Treatment Phase C: Assessments to be taken at 72 (± 4) hours post-last dose (can be combined with the serum chemistry panel) and at the 7 (+1) days post-last dose visit.

In addition to serum sodium samples obtained for trial qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, on Day 1 at 4 to 6 hours postdose and at 18 ( $\pm$  1) hours postdose, and on Day 2 (and Day 2a, if applicable) at 6 (-1 to + 0.25) hours postdose as well as at 18 ( $\pm$  1) hours postdose. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if they can be combined with standard of care labs).

The initial physical examination should be a full physical. Subsequent physical examinations can be directed physical examinations that are focused on hyponatremia-related signs and symptoms as well as any major changes from baseline. A physical examination should include a fontanelle assessment as age appropriate.

<sup>&</sup>lt;sup>g</sup>A neurological examination will be performed predose and at 8 hours post-first dose.

<sup>&</sup>lt;sup>h</sup>Clinical status assessment must be performed predose on Day 1. It is preferred that clinical status assessments be performed predose during subsequent visits. Clinical status assessments will be performed per inpatient standard of care, ie, review subject chart entries (including hyponatremia assessment notes and laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate overall subject eligibility in terms of hyponatremia state. Volume status will be assessed every 6 hours prior to trial entry and every 6 hours during Treatment Phase A.

<sup>&</sup>lt;sup>1</sup>Alcohol/drug screen is performed per clinical judgment and institutional guidelines.

<sup>&</sup>lt;sup>J</sup>A serum or urine pregnancy test will be performed on female subjects ≥ 12 years of age and all female subjects < 12 years of age if menstruation has started. In the case of a positive urine pregnancy test result, a serum pregnancy test will be performed as confirmatory.

k. Intervals starting immediately after dosing at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours).

Samples within a collection interval are to be refrigerated and pooled. An aliquot for urine chemistry tests will be taken for each collection interval. Urine urea is to be measured at screening only.

<sup>&</sup>lt;sup>m</sup>Serum sodium assessments are closely tied to dosing time points and PK blood draws.

<sup>&</sup>lt;sup>n</sup>Serum chemistry panel includes serum sodium and assessments can be combined for visits where both assessments are indicated.

OResults of these tests will further characterize hyponatremia etiology for the Hyponatremia History eCRF and are not required to determine eligibility. Subjects who have clinically relevant TSH or cortisol levels may not respond properly to tolvaptan and will be withdrawn from the trial.

<sup>p</sup>PK samples are closely tied to dosing time points and serum sodium assessments. An early termination (ET) sample will be taken for any subject who is receiving tolvaptan.

- In Treatment Phase A, PK samples should be collected on Day 1 at 2 hours (± 5 minutes) and 8 hours post-first dose and assessed at trough (24 [± 4] hours post-first dose). A PK sample should be assessed on Day 2 at trough (24 [± 4] hours post-previous dose, but prior to the next dose). On Day 2a no PK samples are taken.
- In Treatment Phase B, PK will be assessed in subjects continuing treatment with tolvaptan (Late Withdrawal group and nonresponders continuing on tolvaptan) at trough (24 [± 4] hours post-previous dose, but prior to the next dose) on Days 3 and 4.

If there are restrictions in the allowable total daily blood volumes per local guidelines and subject age, the PK assessment schedule should be the following:

- Day 1at 2 hours postdose (± 5 minutes)
- Day 2 at 8 (± 2) hours postdose (may be concurrent with serum sodium or other blood sampling)
- Days 3 and 4 at trough (24 [± 4] hours post-previous dose, but prior to the next dose and concurrent with serum sodium sample)

<sup>&</sup>lt;sup>q</sup>The tolvaptan dose will be titrated based on serum sodium levels as described in Section 3.2.4.

Optional swallow test for subjects for whom it is unknown if they are able to swallow tablets, at the investigator's discretion.

<sup>&</sup>lt;sup>S</sup>Vital status will be collected at 14 days post-last dose only for subjects who discontinued early and did not withdraw consent.

#### 3.7.1 Schedule of Assessments

# 3.7.1.1 Screening

The procedures listed below will be performed during the Screening Visit (Days -2 to -1) to ensure that the subject qualifies for the trial.

- Trial procedures and information regarding the nature of the trial will be reviewed and written informed consent/assent will be obtained prior to any trial-related procedures.
  - a) Informed consent will be obtained from each subject's parent/legal guardian or legally acceptable representative prior to any trial procedures being conducted.
  - b) Each subject who is able will indicate willingness to participate in the trial by signing or marking an assent form (as applicable) supplied for this purpose.
- 2) Inclusion and exclusion criteria will be reviewed.
- 3) Demographic information will be collected.
- 4) Medical and hyponatremia history will be recorded.
  - a) Medical history should include the subject's current list of medical problems that impacts the subject's current hospital stay.
  - b) The hyponatremia medical history should include the etiology of subject's hyponatremia (see Section 3.3.1) and what treatment was administered prior to trial enrollment. A detailed history specific to etiology of hyponatremia will also be recorded.
  - c) Any observable symptoms of hyponatremia will be assessed and recorded.
- 5) Vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be assessed prior to blood draws.
- 6) A resting 12-lead electrocardiogram (ECG) will be performed after the subject has been supine and at rest  $\geq$  10 minutes.
- 7) Body height and weight will be measured. Growth percentiles will be recorded.
- 8) The initial physical examination should be a full physical. Subsequent physical examinations can be directed physical examinations that are focused on hyponatremia-related signs and symptoms as well as any major changes from baseline.
- 9) Tanner staging will be performed.
- 10) A neurological examination will be performed.
- 11) Quality-of-life (QoL) assessment will be performed, as appropriate by age and where available.
- 12) Clinical status assessments will be performed per inpatient standard of care, eg, subject chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings,

- medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state.
- 13) Alcohol/drug screen is performed per clinical judgment and institutional guidelines.
- 14) A serum or urine pregnancy test will be performed on all female subjects ≥ 12 years of age and all female subjects < 12 years of age if menstruation has started. In the case of a positive urine pregnancy test result, a serum pregnancy test will be performed as confirmatory.
- 15) Urinalysis and urine chemistry laboratory samples will be collected for analysis.
- 16) Two blood samples for serum sodium testing will be collected at least 12 hours apart and can be part of the recent medical history to document chronic hyponatremia. (One of these blood draws can be combined with the serum chemistry panel as appropriate to minimize blood draws.)
- 17) Hematology, coagulation, and serum chemistry laboratory samples will be collected for analysis.
- 18) Serum osmolality, FENa, and FE urea will be calculated.
- 19) Thyroid-stimulating hormone (TSH) and cortisol blood samples will be collected to determine possible need for alternate mode of therapy.
- 20) Concomitant medications will be recorded.
- 21) Adverse events will be recorded.
- 22) Optional swallow test for subjects for whom it is unknown if they are able to swallow tablets, at the investigator's discretion. Placebo tablets will be provided for use in performing this test at screening.

#### 3.7.1.2 Treatment Phase A

During Treatment Phase A every effort should be made to have accurate dosing time points and follow the sequence of assessments specified below as PK/PD assessments and serum sodium blood draws are closely tied to dosing time points.

# 3.7.1.2.1 Day 1

The procedures listed below will be performed on Day 1 for all subjects.

#### **Predose**

1) Any observable symptoms of hyponatremia will be assessed within 2 hours prior to first dose to confirm eligibility as part of a clinical status assessment. Clinical status assessments will be performed per inpatient standard of care, eg, subject chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state.

#### Protocol 156-08-276

- 2) Vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be assessed prior to blood draws.
- 3) A blood sample for STAT serum sodium testing will be collected within 2 to 4 hours prior to dosing.
- 4) Body weight will be measured.
- 5) A directed physical examination will be performed.
- 6) A neurological examination will be performed.
- 7) Inclusion and exclusion criteria will be reviewed and confirmed.

# **Dosing**

8) Tolvaptan will be administered.

## <u>Postdose</u>

- 9) A blood sample will be collected at 2 hours (± 5 minutes) post-first dose for PK analysis of tolvaptan (central laboratory).
- 10) Vital signs will be assessed at 4 and 8 hours post-first dose. Blood pressure, heart rate, respiratory rate, and temperature will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be assessed prior to blood draws at 8 hours.
- 11) Fluid intake will be recorded at 6-hour intervals starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours).
- 12) Urine will be collected at 6-hour intervals starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours). Subjects should be asked to void just prior to the end time of each collection interval, as possible.
  - a) Urine volume will be determined from urine voids made during the 6-hour collection intervals which will be pooled prior to determination of final volume.
  - b) A urine chemistry sample will be collected and assessed from each 6-hour volume interval starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours).
- 13) Blood samples will be collected concurrently at 8 hours (-1 to + 0.25) post-first dose for:
  - a) Serum sodium testing
  - b) PK analysis
- 14) A neurological examination will be performed at 8 hours post-first dose.
- 15) In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, on Day 1 at 4 to 6 hours postdose and at  $18 (\pm 1)$  hours postdose. This sodium safety assessment will be repeated at 6 (-1 to + 0.25) and  $18 (\pm 1)$  hours postdose each day for the remainder of titration. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if they can be combined with standard of care labs).

- 16) Blood samples will be collected concurrently at trough (24 [ $\pm$  4] hours post-first dose) for:
  - a) A blood sample for STAT serum sodium testing should be taken and the results known prior to subsequent tolvaptan dosing.
  - b) A blood sample for PK analysis.

## Throughout the visit

- 17) Concomitant medications will be recorded.
- 18) Adverse events will be assessed.

# 3.7.1.2.2 Day 2

The following procedures will be performed on Day 2 for all subjects.

# Trough (24 [ $\pm$ 4] hours post-first dose)

- 1) Vital signs will be assessed. Blood pressure, heart rate, respiratory rate, and temperature will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be performed predose and prior to blood draws.
- 2) Clinical status assessments will be performed per inpatient standard of care, eg, subject chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state.
- 3) Complete fluid intake and urine volume collection for specified intervals prior to next dosing with tolvaptan.
- 4) A directed physical examination will be performed.
- 5) Body weight will be measured.
- 6) A neurological examination will be performed.

## **Dosing**

7) Tolvaptan will be administered. If the subject's serum sodium concentration is < 135 mEq/L (mmol/L) and a ≤ 4 mEq/L (mmol/L) increase, tolvaptan dose should be adjusted per the titration guidelines (Section 3.2.4) for the assigned weight group.

#### Postdose

- 7) Assess palatability and acceptability of the tolvaptan dose for subjects immediately after dosing and again between 15 to 20 minutes after dosing.
- 8) Fluid intake will be recorded at 6-hour intervals starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours).
- 9) Urine will be collected at 6-hour intervals starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours). Subjects should be asked to void just prior to the end time of each collection interval, as possible.

- a) Urine volume will be determined from urine voids made during the 6-hour collection intervals which will be pooled prior to determination of final volume
- b) A urine chemistry sample will be collected and assessed from each 6-hour volume interval starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours).
- 10) A blood sample will be collected for serum sodium testing at 12 ( $\pm$  4) hours postdose.
- 12) In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, at 6 and 18 hours postdose. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if they can be combined with standard of care labs).
- 13) At the end of the Day 2 visit subjects will be assessed for response to tolvaptan treatment. Subjects who are:
  - a) Responders (serum sodium level increase of  $\geq 4$  mEq/L [mmol/L]) will proceed to Treatment Phase B (see Section 3.7.1.3) for randomization.
  - b) Not responding to tolvaptan treatment (serum sodium level increase of < 4 mEq/L [mmol/L]) will proceed to Day 2a (see Section 3.7.1.2.3).
- 14) Blood samples will be collected concurrently at trough (24 [ $\pm$  4] hours post-previous dose) for:
  - a) STAT serum sodium testing and the results known prior to subsequent tolvaptan dosing.
  - b) PK analysis of tolvaptan.

## Throughout the visit

- 15) Concomitant medications will be recorded.
- 16) Adverse events will be assessed.

# 3.7.1.2.3 Day 2a (optional)

The following procedures will be performed on Day 2a for all subjects who are not responsive to tolvaptan treatment at the end of Day 2.

#### Trough (24 [ $\pm$ 4] hours post-previous dose)

- 1) Vital signs will be assessed at 24 hours post-previous dose. Blood pressure, heart rate, respiratory rate, and temperature will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be performed predose and prior to blood draws
- 2) Clinical status assessments will be performed per inpatient standard of care, eg, subject chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings,

#### Protocol 156-08-276

medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state.

#### Predose

- 3) A directed physical examination will be performed.
- 4) Body weight will be measured.

# **Dosing**

5) Tolvaptan will be administered.

If the subject's serum sodium concentration is < 135 mEq/L (mmol/L) and a
≤ 4 mEq/L (mmol/L) increase, tolvaptan dose should be adjusted per the titration guidelines (Section 3.2.4) for the assigned weight group.

#### Postdose

- 6) A blood sample will be collected for serum sodium testing at 12 ( $\pm$  4) hours postdose.
- 7) In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, at 6 and 18 hours postdose. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if they can be combined with standard of care labs).
- 8) At the end of the Day 2a visit subjects will be assessed for response to tolvaptan treatment. Subjects who are:
  - a) Responders (serum sodium level increase of  $\geq 4$  mEq/L [mmol/L]) will proceed to Treatment Phase B (see Section 3.7.1.3) for randomization.
  - b) Nonresponders (serum sodium level increase of < 4 mEq/L [mmol/L]) will continue to Treatment Phase B where they either continue on tolvaptan therapy for 2 additional days or are withdrawn from tolvaptan to be treated per the investigator's preferred standard of care.
- 9) A blood sample will be collected for serum sodium testing at trough (24 [ $\pm$  4] hours postdose).

## Throughout the visit

- 10) Concomitant medications will be recorded.
- 11) Adverse events will be assessed.

#### 3.7.1.3 Treatment Phase B

# 3.7.1.3.1 Day 3

The following procedures will be performed on Day 3. Some assessments are required for all subjects while other assessments only apply to certain subsets of subjects as indicated

#### For all subjects

At trough (24 [ $\pm$  4] hours post-previous dose) the following assessments will be performed:

- 1) Vital signs will be assessed. Blood pressure, heart rate, respiratory rate, and temperature will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be performed predose and prior to blood draws.
- 2) Clinical status assessments will be performed per inpatient standard of care, eg, subject chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state.

#### For all subjects classified as Responders at the end of Treatment Phase A

1) Randomize the subject to the Early or Late Withdrawal group using the trial's interactive web response system (IWRS).

# For subjects receiving tolvaptan (Late Withdrawal group and nonresponders with continuing treatment)

- 1) Body weight will be measured predose.
- 2) A directed physical examination will be performed predose.
- 3) A neurological examination will be performed.
- 4) Tolvaptan will be administered.
- 5) A blood sample will be collected for serum sodium testing at 12 ( $\pm$  4) hours postdose.
- 6) Blood samples will be collected concurrently at trough (24 [ $\pm$  4] hours post-previous dose) for:
  - a) STAT serum sodium testing and the results known prior to subsequent tolvaptan dosing.
  - b) PK analysis of tolvaptan.
- 8) Concomitant medications will be recorded.
- 9) Adverse events will be assessed.

# For subjects not receiving tolvaptan treatment (Early Withdrawal group and nonresponders treated with standard of care)

- 1) Early Withdrawal subjects will be observed to determine whether additional intervention is required to maintain appropriate serum sodium levels.
- 2) Nonresponders discontinuing tolvaptan will be treated per the investigator's preferred standard of care.
- 3) A directed physical examination will be performed.
- 4) A neurological examination will be performed.
- 5) A blood sample will be collected for serum sodium testing at 12 ( $\pm$  4) hours post the nominal dosing time.
- 6) A blood sample will be collected for serum sodium testing at 24 ( $\pm$  4) hours post the nominal dosing time.
- 7) Concomitant medications will be recorded.
- 8) Adverse events will be assessed.

## 3.7.1.3.2 Day 4

The following procedures will be performed on Day 4. Some assessments are required for all subjects while other assessments only apply to certain subsets of subjects as indicated.

# For all subjects

At trough (24 [ $\pm$  4] hours post-previous dose) the following assessments will be performed:

- 1) Vital signs will be assessed. Blood pressure, heart rate, respiratory rate, and temperature will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be performed predose and prior to blood draws.
- 2) Clinical status assessments will be performed per inpatient standard of care, eg, subject chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state.

# For subjects receiving tolvaptan (Late Withdrawal group and nonresponders with continuing treatment)

- 1) Body weight will be measured predose.
- 2) A directed physical examination will be performed predose.
- 3) A neurological examination will be performed.
- 4) Tolvaptan will be administered.

- 5) A blood sample will be collected for serum sodium testing at 12 ( $\pm$  4) hours postdose.
- 6) A QoL assessment will be conducted.
- 7) Blood samples will be collected concurrently at trough (24 [ $\pm$  4] hours post-previous dose) for:
  - a) STAT serum sodium testing and the results known prior to subsequent tolvaptan dosing.
  - b) PK analysis of tolvaptan.
- 8) Concomitant medications will be recorded.
- 9) Adverse events will be assessed.

# For subjects not receiving tolvaptan treatment (Early Withdrawal group and nonresponders treated with standard of care)

- 1) Early Withdrawal subjects will be observed to determine whether additional intervention is required to maintain appropriate serum sodium levels.
- 2) Nonresponders discontinuing tolvaptan will continue to be treated per the investigator's preferred standard of care.
- 3) A directed physical examination will be performed.
- 4) A neurological examination will be performed.
- 5) A blood sample will be collected for serum sodium testing at 12 ( $\pm$  4) hours post the nominal dosing time.
- 6) A QoL assessment will be conducted.
- 7) Concomitant medications will be recorded.
- 8) Adverse events will be assessed.

## 3.7.1.3.3 Day 5

The following procedures will be performed on Day 5.

# For subjects receiving tolvaptan (Late Withdrawal group and nonresponders with continuing tolvaptan treatment)

# At trough (24 [± 4] hours post-previous dose)

- 1) Vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be performed prior to blood draws.
- 2) Body weight will be measured.

## Throughout the visit

3) Concomitant medications will be recorded.

4) Adverse events will be assessed.

# For subjects not receiving tolvaptan treatment (Early Withdrawal group and nonresponders treated with standard of care)

1) Proceed to Follow-up Phase C, as for these subjects the 72-hour post-last dose time point (Section 3.7.1.4.1) falls on the morning of Day 5.

## 3.7.1.4 Follow-up Phase C

### 3.7.1.4.1 72 Hours Post-last Dose or ET

The following procedures will be performed for all subjects at 72 ( $\pm$  4) hours post-last dose or at early termination (ET).

- 1) Vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be assessed after the subject has been supine for  $\geq 3$  minutes. Vital signs should be performed prior to blood draws.
- 2) Hematology, coagulation, and serum chemistry laboratory samples will be collected.
- 3) For Early Termination only:
  Blood sample for PK analysis of tolvaptan will be collected for all subjects on tolvaptan. The sample is to be taken concurrently with the serum sodium sample (part of the serum chemistry panel).
- 4) A directed physical examination will be performed.
- 5) A neurological examination will be performed.
- 6) Body weight will be measured.
- 7) A urinalysis laboratory sample will be collected.
- 8) Clinical status assessments will be performed per inpatient standard of care, eg, subject chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state.
- 9) For Early Termination:
  Subjects will be monitored and treated as clinically warranted per the investigator's preferred standard of care for up to 3 additional days after the last dose of tolvaptan.
- 10) Concomitant medications will be recorded.
- 11) Adverse events will be assessed.
- 12) If a subject terminates early from the trial and agrees to continued telephone contact, the subject or parent/legal guardian or legally acceptable representative will be contacted by telephone at 14 days post-last dose for vital status.

# 3.7.1.4.2 7 Days Post-last Dose

Subjects will be assessed for maintenance of normal or target serum sodium concentration at 7 (+ 1) days post-last dose. All clinical labs will be performed locally. If the subject was discharged, he/she should return to the clinic for this visit.

- 1) Vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be assessed after the subject has been supine for  $\geq 3$  minutes. Vital signs should be performed prior to blood draws.
- 2) A blood sample for serum sodium testing will be collected.
- 3) A serum or urine pregnancy test will be performed on all female subjects ≥ 12 years of age and all female subjects < 12 years of age if menstruation has started. In the case of a positive urine pregnancy test result, a serum pregnancy test will be performed as confirmatory.
- 4) A OoL assessment will be conducted.
- 5) A directed physical examination will be performed.
- 6) A neurological examination will be performed.
- 7) Clinical status assessments will be performed per inpatient standard of care, eg, subject chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state.
- 8) Body weight will be measured.
- 9) Concomitant medications will be recorded.
- 10) Adverse events will be assessed.

### **3.7.1.4.3 14 Days Post-last Dose**

Subjects or their parent(s)/legal guardian(s) or legally acceptable representative(s) will be contacted via telephone or will be asked to come back to the clinic for a visit at 14 (+2) days post-last dose to assess any new or ongoing AEs and to collect information on any medications administered since the last visit. Ongoing follow-up may be required after a subject's trial completion for health status before the analysis of all trial results is completed.

# 3.7.2 Efficacy Assessments

Efficacy will be assessed through determination of overall serum sodium concentrations and clinical status assessments.

#### 3.7.2.1 Serum Sodium Concentrations

Monitoring frequency of serum sodium is at the discretion of the clinical investigator; however, the minimum sample collection required for all subjects is described in Section 3.7.1 and Section 3.7.4.2.1.

In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, on Day 1 at 4 to 6 hours postdose and at 18 hours postdose. This sodium safety assessment will be repeated at 6 and 18 hours postdose each day for the remainder of titration. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if they can be combined with standard of care labs).

In order to qualify for this trial, subjects must have documentation of chronic dilutional hyponatremia (serum sodium < 130 mEq/L [mmol/L]) that is present for  $\geq$  48 hours. Specifically, each subject must have 2 blood samples collected at least 12 hours apart over a minimum of 48 hours for assessment of baseline serum sodium level to determine subject eligibility. These can be either part of the recent medical history concerning the current hospital stay or prospectively collected as part of this trial.

On Day 1, a third (STAT) serum sodium sample should be drawn within 2-4 hours prior to dosing; the results must be verified to be < 130 mmol/L prior to the first dose. Serum sodium assessments should be performed at 8 hours post-first dose and at trough (24 [±4] hours post-first dose; this assessment will fall on Day 2 predose).

On Day 2 (or 2a), Day 3, and Day 4 (through the following morning on Day 5):

- For all subjects receiving tolvaptan (Late Withdrawal and nonresponders continuing on tolvaptan) serum sodium assessments will be performed at trough (24 [±4] hours post-previous dose) and 12 (± 4) hours postdose each day during Treatment Phase A and Treatment Phase B.
- For all subjects not receiving tolvaptan (Early Withdrawal and nonresponders treated with standard of care) serum sodium assessments will be performed every 12 (± 4) hours throughout Treatment Phase A and Treatment Phase B.

For all subjects final serum sodium assessments will be taken at 72 ( $\pm$  4) hours post-last dose and 7 days post-last dose.

The serum sodium assessments schedule is presented in Table 3.7.2.1-1.

| Table 3.7.2.1-1 Serum Sodium Assessments | | | | |
|---|---|---|---|---|
| | | | Blood Draws for So | erum Sodium |
| Phase | Visit | Day | Efficacy | Supplemental Safety |
| Treatment<br>Phase A | Screening | −2 to −1 | 2 blood samples, at least<br>12 hours apart | - |
| | Titration | 1 | Within 2 to 4 hours prior to dosing (STAT) | - |
| | | | 8 (-1 to + 0.25) hours<br>post-first dose | 4 to 6 hours postdose |
| | | | 24 (± 4) hours post-first dose (STAT) | 18 (± 1) hours<br>postdose |
| | | 2 | 12 (± 4) hours postdose | 6 (-1 to + 0.25) and<br>18 (± 1) hours<br>postdose |
| | | | 24 (± 4) hours post-previous<br>dose (trough) (STAT) | - |
| | | 2a<br>(Optional) | 12 (± 4) hours postdose | 6 (-1 to + 0.25) and<br>18 (± 1) hours |
| | | | 24 (± 4) hours post-previous<br>dose (trough) (STAT) | postdose<br>- |
| Treatment | Late Withdrawal | 3 | 12 (± 4) hours postdose | - |
| Phase B | group and nonresponders with | | 24 (± 4) hours post-previous<br>dose (trough) (STAT) | - |
| | continuing treatment | 4 | 12 (± 4) hours postdose | - |
| | | | 24 (± 4) hours post-previous dose (trough) | - |
| | Early Withdrawal group and | 3 | 12 (± 4) hours post nominal dosing | - |
| | nonresponders treated with standard of care | | 24 (± 4) hours post nominal dosing | - |
| | | 4 | 12 (± 4) hours post nominal dosing | - |
| Follow-up | Follow-up | - | 72 ( $\pm$ 4) hours post-last dose | - |
| Phase C | | - | 7 (+ 1) days post-last dose | - |

## 3.7.2.2 Clinical Assessments

Clinical status assessment must be performed predose on Day 1. It is preferred that clinical status assessments be performed predose during subsequent visits. Clinical assessments will be performed per inpatient standard of care and should include review of subject chart entries, including hyponatremia assessment notes, trial- and nontrial-specific laboratory results, any examination findings, medical problem list changes, and fluid intake and output to evaluate overall subject eligibility in terms of hyponatremia state. The clinical assessment will focus on symptoms and signs which will inform treatment decisions (eg, the need to switch to rescue therapy, or the ability to safely discharge a subject from the hospital). The clinical assessment should be

performed by a trial investigator who will be aware of laboratory and other clinical response data.

## 3.7.2.3 Quality of Life Assessments

Two patient-reported outcomes instruments (acute versions with 7 day recall period) will be used to assess subject quality of life: PedsQL Generic Core Scale and PedsQL Multidimensional Fatigue Scale. Both instruments are appropriate for ≥ 2 years of age, however availability may be limited for certain ages and languages. The age groups covered by these assessments are Toddler (2–4 years), Young child (5–7 years), Child (8–12 years), and Adolescent (13–18 years). Depending on the subject's age, the questionnaire may be completed by either the subject, subject and parent/caregiver, or the parent/caregiver, as appropriate.

The PedsQL Generic Core Scale consists of 23 items encompassing physical, emotional, social, and school domains.

The PedsQL Multidimentional Fatigue Scale consists of 18 items in 3 subscales: general fatigue, sleep/rest fatigue, and cognitive fatigue. The instrument focuses on the domains of processing speed, attention/vigilance, visual and working memory.

The assessment time points are at screening, Day 4 and 7 days post-last dose.

## 3.7.3 Pharmacokinetic/Pharmacodynamic Assessments

#### 3.7.3.1 Pharmacokinetic Assessments

#### 3.7.3.1.1 Blood Collection Times

Blood samples will be taken so that tolvaptan and metabolite concentrations can be determined. Samples will be taken at the following times:

- On Day 1 at 2 hours (± 5 minutes) and 8 hours (concurrent with 8 h serum sodium sample) post-first dose.
- On Days 1, 2, 3, and 4 samples will be taken at trough (24 [± 4] hours post-previous dose) (prior to the subsequent dose), concurrent with serum sodium samples, for subjects dosed with tolvaptan on Days 1, 2, 3, and 4, respectively, regardless of status as responder/nonresponder.
- An early termination (ET) sample will be taken for any subject who is receiving tolvaptan.

On Day 2a no PK samples are taken.

For each PK blood sample collected volumes are not expected to exceed 1.2 mL. Total volume per sample may be lower depending on finalization of blood collection supplies.

Serum sodium assessments and other clinically necessary blood samples take priority; therefore, due to restrictions in allowable total daily blood volumes based on local guidelines and subject age, it may not be possible to take more than one PK sample per day. If so, the PK sampling should be changed to:

- Day 1: 2 hours postdose (± 5 minutes)
- Day 2: 8 (± 2) hours postdose (may be concurrent with serum sodium or other blood sampling)
- Day 3 at trough, ie, predose/24 hours post prior dose (concurrent with serum sodium sample)
- Day 4 at trough, ie, predose/24 hours post prior dose (concurrent with serum sodium sample)

The PK profiles will be evaluated on an ongoing basis to determine the variability between subjects. Based on the findings, PK sampling will continue for as long as necessary to establish suitable estimates of clearance with a 90% CI similar to that observed in the adult populations. Once these estimates are achieved, sampling will be discontinued in subsequent subjects.

For each subject all samples will be collected according to local guidelines and best practices for pediatric care. If a sample is missing due to limitations in allowable blood volumes based on local regulations or local practice this will not count as a protocol deviation.

## 3.7.3.1.2 Sample Handling and Processing

All blood samples will be shipped to the testing facility for analysis. Detailed handling and shipping instructions are provided in Appendix 3.

### 3.7.3.2 Pharmacodynamic Assessments

#### 3.7.3.2.1 Fluid Intake

Fluid intake (both oral and IV) will be measured at the times presented in the schedule of assessments (Section 3.7.1). The fluid content of foods with significant water content (eg, soup) should be added to the total fluid intake. Fluid intake will be monitored per institutional guidelines.

#### 3.7.3.2.2 Urine Volume

Urine volume will be determined in urine samples that will be collected at the intervals presented in the schedule of assessments, Section 3.7.1. All urine voids within a collection interval should be kept refrigerated and pooled according to the size of
available collection containers. At the end of the collection interval all samples should be pooled and the urine volume determined.

# 3.7.3.2.3 Urine Chemistry

Urine chemistry will be determined from pooled urine samples collected for the intervals presented in the schedule of assessments, Section 3.7.1. An aliquot will be taken for each collection interval according to the procedures of the local clinical chemistry laboratory. The list of urine chemistry tests to be conducted is presented in Table 3.7.4.2.3-1.

## 3.7.3.2.4 Palatability and Acceptability Assessment

A questionnaire will be administered immediately after dosing to assess palatability to rate flavor/taste, smell, sweetness, and overall liking of the study medication. Subjects will also be asked about the ease of swallowing the study medication. Between 15 to 20 minutes after dosing, a questionnaire will be administered to subjects again to assess overall liking of the study medication. This assessment will only be done in subjects aged 3 years to 18 years.

# 3.7.4 Safety Assessments

Safety will be assessed through the monitoring of AEs, clinical laboratory tests, vital signs, body weight, directed physical examinations, neurological examinations, rescue therapy, and fluid restriction.

The monitoring frequency of safety assessments is at the discretion of the clinical investigator; however, the trial requires the minimum sample collection for all subjects noted in Section 3.7.1 and Section 3.7.4.2.1.

#### 3.7.4.1 Adverse Events

Refer to Section 5, Reporting of Adverse Events.

In addition, active monitoring is required for:

- Absolute serum sodium level ≥ 145 mEq/L (mmol/L) or an overly rapid rise in serum sodium level (an increase in serum sodium of > 8 mEq/L [mmol/L] over a 10-hour period, ≥ 12 mEq/L [mmol/L] over a 24-hour period, or a rate of increase in serum sodium concentration that the investigator deems too rapid), neurological symptoms, or other signs or symptoms suggestive of osmotic demyelination (see Section 0 for more details).
- Elevations in AST or ALT that are  $\geq 2 \times \text{ULN}$  or levels that increase  $\geq 2$  times their previously observed level. If this occurs, a total bilirubin level should also be evaluated. See Section 3.7.4 for more information and Section 5.4.1 for detailed instructions on how this type of event should be captured.
- Worsening symptoms of hyponatremia
- Hypovolemia or hypotension requiring intervention

## 3.7.4.2 Clinical Laboratory Assessments

#### 3.7.4.2.1 Serum Sodium

In addition to serum sodium samples obtained for trial qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, on Day 1 at 4 to 6 (-1 to + 0.25) hours postdose and at 18 ( $\pm$  1) hours postdose. This sodium safety assessment will be repeated at 6 (-1 to + 0.25) and 18 ( $\pm$  1) hours postdose each day for the remainder of Treatment Phase A. A point of care assessment unit is preferred since it is expected to reduce overall daily blood volume needed for assessments (expected 0.5 mL for regular blood draws versus up to several drops for a point of care assessment, depending on the device used); however, regular blood draws may be used (especially if they can be combined with standard of care labs).

Additional unscheduled serum sodium assessments may be performed at the discretion of the clinical investigator and other physicians of record, depending on the local standards and subject's clinical condition. All unscheduled serum sodium concentrations collected as part of standard of care will be reported as unscheduled sodium assessments in the electronic case report form (eCRF) through the follow-up sodium assessments.

# 3.7.4.2.2 Serum Osmolality

Serum osmolality will be calculated to help guide dosing. Local site personnel will determine serum osmolality using one of the following equations:

a) Where Na, glucose, and blood urea nitrogen (BUN) are measured in mg/dL:

Serum Osmolality (mOsm/kg) = 2 Na + BUN / 2.8 + (glucose / 18)

b) Where Na, glucose, and urea are measured in mmol/L:

Serum Osmolality (mOsm/kg) = 2 Na + glucose + urea

## 3.7.4.2.3 Clinical Lab Tests

Table 3.7.4.2.3-1 presents required clinical laboratory assessments (serum chemistry, hematology, coagulation, urinalysis, and urine chemistry). All clinical laboratory tests will be performed by local laboratories. Serum cortisol and TSH will be measured during screening using the remaining blood sample obtained for serum chemistry. If these results are obtained as part of the standard of care for the subject, a trial-specific sample should be obtained and sent to the local laboratory for analysis per the schedule of assessments (Section 3.7.1). Urine urea will be measured during screening for calculation of FE urea.

It is recognized that there may be limitations based on age and weight of children for the amount of blood that can be drawn at a single time point, per day, and the overall conduct of the trial. Wherever possible, it is encouraged to combine standard of care samples that would be taken regardless of trial participation with those samples required for the trial.

In case of limited blood or urine volume availability, the bolded assessments in Table 3.7.4.2.3-1 take priority. Serum sodium and liver function tests are essential to the conduct of the trial.

| T 11 2 7 4 2 2 1 CP 1 1 1 1 1 T 1 1 1 D C 1 1 H | |
|---|---|
| Table 3.7.4.2.3-1 Clinical Laboratory Tests to be Performed Locally | |
| Hematology: | Serum Chemistry: |
| WBC count with differential | ALT |
| RBC count | Alkaline phosphatase |
| Hematocrit | AST |
| Hemoglobin | Bicarbonate (or carbon dioxide) |
| Mean corpuscular volume | Bilirubin, total |
| Mean corpuscular hemoglobin concentration | Urea or Blood urea nitrogen (BUN) |
| Platelet count | Calcium |
| RBC volume distribution width | Chloride |
| Additional Tests: | Cholesterol, total |
| TSH | Creatinine |
| Serum cortisol | Gamma glutamyl transferase |
| Sei uni coi tisoi | Glucose |
| Coagulation: | Lactic dehydrogenase |
| International normalized ratio | Potassium |
| Platelets | Protein, total |
| Prothrombin time | Triglycerides |
| Activated partial thromboplastin time | Uric acid |
| | Efficacy: |
| | Serum sodium |
| Urinalysis: | Drug Screen (all items in urine): |
| Color | Alcohol |
| Appearance | Amphetamines |
| Bilirubin | Barbiturates |
| Glucose | Benzodiazepines |
| Ketones | Cannabinoids |
| Leukocytes | Cocaine |
| Nitrites | Methadone |
| Occult blood | Opiates |
| Protein | Phencyclidine |
| Urobilinogen | |
| Microscopic analysis of RBC/WBC (per high | Additional Drug Screen Test: |
| powered field) | Alcohol (breath) |
| Urine Chemistry: | |
| Osmolality | |
| Sodium | |
| Potassium | |
| Creatinine | |
| Urea | |
| Orca | |
| Additional Test: | |
| Serum or urine pregnancy test (if applicable) | |
| became of arme pregnancy test (if applicable) | |

WBC = white blood cell; RBC = red blood cell.

In case of limited blood or urine volume availability the **bolded** assessments take priority. Serum Sodium and liver function tests are essential to the conduct of the trial.

# 3.7.4.2.4 Monitoring of Liver Transaminases

Long-term use of tolvaptan has demonstrated the potential to cause a clinically significant elevation in laboratory tests of liver function. Based on previous research in the adult

polycystic kidney disease population, the expected onset of the elevation, if it occurs, is between 3 and 14 months of chronic treatment with tolvaptan.

For a subject who experiences an elevation in AST or ALT that is  $\geq 2 \times ULN$  or whose levels increase  $\geq 2$  times their previous observed value, a total bilirubin level should also be evaluated. These elevated values should be confirmed by retesting. If total bilirubin is  $\geq 2 \times ULN$  or  $\geq 2$  times their previous observed value, an immediately reportable event (IRE) form with all values listed should be completed and also reported as an AE on the eCRFs. See Section 5.4.1 for detailed instructions on how this type of event should be captured.

## 3.7.4.3 Physical Examination

Full and directed physical examinations will be performed and documented according to the schedule of assessments (Section 3.7.1). The initial physical examination should be a full physical. Subsequent physical examinations can be directed physical examinations that are focused on hyponatremia-related signs and symptoms as well as any major changes from baseline.

The principal investigator or his/her appointed designee is primarily responsible to perform the physical examination. If the appointed designee is to perform the physical examination, he/she must be permitted by local regulations. Whenever possible, the same individual should perform all physical examinations for a given subject. Any condition present at the post-treatment directed physical examination that was not present at Screening should be documented as an AE and followed to a satisfactory conclusion.

Full physical examination assessments should include assessments of all major body systems, including but not limited to, ears, nose, and throat, the thorax area, abdomen, urogenital, extremities, and skin and mucosae. Directed physical examinations should be focused on hyponatremia-related signs and symptoms as well as any major changes from baseline. Physical examination will include a fontanelle assessment as age appropriate. Neurological examinations will be performed in an age-appropriate manner per Section 3.7.4.3.1.

Body weight will be measured predose each day throughout Treatment Phase A, Treatment Phase B and at each clinic visit in Follow-up Phase C, as possible. Every effort should be made to ensure that body weight measurements are performed in a reproducible and consistent manner. Body weight measurements should be performed at the clinical site always using the same scale. Subjects should wear the same type of clothes at each measurement, preferably a gown and no shoes. All body weight measurements should be taken post void.

# 3.7.4.3.1 Neurological Examination

A neurological examination will be performed as part of the directed physical exam per the schedule of assessments (Section 3.7.1). It will include an evaluation of mental status, cranial nerves, muscle tone, muscle strength/symmetry, reflexes, neonatal primitive reflexes, sensory system, gait, and finger to nose, as age appropriate.

## 3.7.4.4 Tanner Staging

Tanner Staging must be completed together with the physical examination by the same trial-affiliated clinician in the most inconspicuous manner for the subject as possible. Tanner Staging could be completed by the trial affiliated pediatrician or family practitioner (additionally physician's assistant or nurse practitioner where licensing permits). Sites should make attempts to have examiners of both sexes. Attempts should be made to have the examination performed by the same sex personnel as the subject. Otherwise, trial-affiliated personnel of the same sex as the subject (ie, nurse) should be in the same examination room as the subject.

Tanner Staging assessment consists of 2 domains (pubic hair and breast development) for girls and 3 domains (pubic hair, penis development, and testes development) for boys. The Tanner Staging assessment as a reference for the completing clinician is included in Appendix 4. The investigator will arrive at a single score summarizing the domains (not individual domain scores) when evaluating the subject.

# 3.7.4.5 Vital Sign Assessments

Vital signs (including supine blood pressure, heart rate, respiratory rate, and temperature) will be assessed at time points according to Section 3.7.1 of this protocol. Supine vital signs will be taken when the subject has been lying down (bed positioned < 45 degree angle) for  $\ge$  3 minutes. All assessments for vital signs should be performed around the time of the formal hyponatremia assessment (sodium blood draw) during Screening, Treatment Phase A and Treatment Phase B and anytime during the Follow-up Period consistent with the timing of other trial assessments. All vital sign assessments should be performed predose and prior to the blood draw at the nominal time point.

## 3.7.4.6 Electrocardiogram Assessments

One ECG will be recorded at screening, prior to any blood draws. Twelve-lead ECGs will be recorded with the subject supine and at rest (for at least 10 minutes). Heart rate, PR interval, QRS duration, and QT interval will be recorded. The principal investigator or designee will review, sign, and date each ECG reading. Any abnormalities should be reported as part of the medical history. Whenever possible, the same reviewer should

evaluate, sign, and date the ECGs. A paper copy of the ECG will be sent for storage to a central ECG storage facility.

# 3.7.4.7 Hyponatremia History

Each subject's hyponatremia medical history will be recorded at screening. The hyponatremia history should include the etiology of subject's hyponatremia (including assessments per Section 3.2.4.2) and what treatment was administered prior to trial enrollment. Symptoms potentially attributable to hyponatremia should be specifically assessed for prior history. The hyponatremia assessment at Screening will consist of documentation of hyponatremia etiology (eg, HF, hepatocellular disease [including cirrhosis], SIADH/other), prior fluid intake and output, and prior hyponatremia treatment, ie, fluid restriction, if applicable. A detailed history specific to etiology of hyponatremia will also be recorded.

#### 3.7.4.8 Volume Status Assessment

Volume status will be assessed every 6 hours prior to trial entry and every 6 hours during Treatment Phase A.

## 3.7.4.9 Vital Status

An assessment of vital status will be conducted on subjects who terminate prior to the last study visit, and do not withdraw consent for continued telephone contact. The telephone contact will be made 14 days post-last dose, and will be conducted with a reliable informant; either the subject and/or the parent/guardian, per investigator discretion. Vital status collected and recorded will be:

- Subject alive
- Subject deceased (date of death, cause of death)

## 3.7.5 End of Trial

The End of Trial Date is defined as the last Date of Contact or the Date of Final Contact Attempt from the Post-treatment Follow-up eCRF page for the last subject completing or withdrawing from the trial.

## 3.7.6 Independent Data Monitoring Committee

An independent data monitoring committee (IDMC) will be established for this trial. This committee will meet on a regular basis to ensure the safe and ethical treatment of trial subjects, ensure the scientific integrity of the trial, and to ensure the trial is conducted within the bounds of ethical medical practice. It may make recommendations

to the sponsor and trial steering committee to amend or terminate the trial based on grounds of safety, futility, or greater than expected efficacy as defined by the accepted statistical practices and procedures to be detailed in their charter. The specific duties of the IDMC will be detailed in a separate IDMC charter document.

## 3.8 Stopping Rules, Withdrawal Criteria and Procedures

# 3.8.1 Entire Trial or Treatment Arm(s)

If the sponsor terminates or suspends the trial for safety or unanticipated other reasons, prompt notification will be given to investigators, IRBs/IECs, and regulatory authorities in accordance with regulatory requirements.

#### 3.8.2 Individual Site

The investigator will notify the sponsor promptly if the trial is terminated by the investigator or the IRB/IEC at the site.

# 3.8.3 Individual Subject Discontinuation

If a subject discontinues from the trial prematurely, the reason must be fully evaluated and recorded appropriately in source documents and the eCRF. If the subject is being withdrawn because of an AE, that AE should be indicated as the reason for withdrawal.

All subjects have the right to withdraw at any point during treatment without prejudice. The investigator can discontinue a subject's participation in the trial at any time if medically necessary. In addition, subjects meeting the following criteria following the first dose of tolvaptan must be withdrawn from the trial:

- a) Occurrence of any AE, intercurrent illness, or abnormality in a laboratory assessment which, in the opinion of the investigator, warrants the subject's permanent withdrawal from the trial;
- Treatment with a prohibited concomitant medication other than the use of appropriate medications for the treatment of AEs under direction of the investigator;
- c) Subject noncompliance, defined as refusal or inability to adhere to the trial schedule or procedures (eg, blood draw requirements); see Section 3.12, Subject Compliance);
- d) At the request of the subject, investigator, OPDC or designee, or regulatory authority;
- e) Subject becomes pregnant; or
- f) Subject is lost to follow-up.

#### Protocol 156-08-276

Subjects who have clinically relevant TSH or cortisol levels may not respond properly to tolvaptan and will be withdrawn from the trial.

In addition, subjects meeting the following criteria should have results confirmed with a repeat test (if the result is confirmed, the medical monitor should be contacted to consider options of down-titration, dose interruption, concomitant medication adjustment, fluid supplementation, and/or withdrawal):

- Subject's serum sodium level increases by > 8 mEq/L [mmol/L] in any 10-hour period following dosing on Day 1
- Subject's serum sodium level increases by ≥ 12 mEq/L [mmol/L] in the 24-hour period following dosing
- At any time after dosing, the subject's serum sodium is  $\geq 145 \text{ mEq/L} \text{ [mmol/L]}$

Subjects who require IV infusion of isotonic or hypertonic saline for hyponatremia or who receive another approved/off-label therapy (rescue therapy) for hyponatremia before completion of the trial will be withdrawn from trial treatment; these subjects should continue to Phase C to be followed. Subjects, who are randomized to the Early Withdrawal group, whose serum sodium level declines by  $\geq 4$  mEq/L (mmol/L), or whose overall clinical condition requires further treatment to increase serum sodium level will be treated per the investigator's preferred standard of care. Any intervention intended to raise serum sodium during the first 48 hours of the Early Withdrawal phase (including fluid restriction) will be defined as rescue therapy. The subject will be considered to have reached their clinical endpoint, and their data will be censored from that time forward.

The sponsor and the medical monitor should be notified promptly when a subject requires treatment other than trial treatment for the purpose of raising serum sodium. Subjects receiving rescue therapy are to continue to be monitored per protocol (to discharge or death). Subjects terminated prior to completion will not be re-enrolled.

The investigator will notify the sponsor promptly when a subject is withdrawn.

When a subject or parent/legal guardian or legally responsible representative decides to withdraw from the trial they will be asked to indicate whether they wish to discontinue from the trial as a whole, or still allow telephone contact. If they agree to continued telephone contact, they will be contacted 14 days after the last study visit for vital status (Section 3.7.4.9).

#### 3.9 Screen Failures

A screen failure subject is one from whom informed consent/assent (if applicable) has been obtained and is documented in writing (ie, the subject's parent/legal guardian or legally acceptable representative signs an ICF), but who is not enrolled into the trial. If a subject's serum sodium level during the Screening period is  $\geq 130$  mEq/L [mmol/L], that subject will be determined a screen failure. Subjects who are deemed screen failures may be rescreened for possible participation if they have not taken a dose of IMP.

# 3.10 Definition of Completed Subjects

The treatment period is defined as the time period during which subjects are evaluated for primary and/or secondary objectives of the trial irrespective of whether or not the subject actually consumed all doses of the tolvaptan.

For purposes of this trial, subjects who are randomized responders and who complete required trial assessments (including their assigned trial treatment) through the end of the trial will be defined as responder trial completers.

For purposes of this trial, subjects who are nonresponders (not randomized) but who complete required trial assessments through the end of the trial will be defined as nonresponder trial completers.

Subjects who discontinue tolvaptan prior to the end of Treatment Phase B, but who continue in the trial and complete some or all of their required assessments to the end of the trial, will be considered "early" end of treatment (EEOT) completers.

# 3.11 Definition of Lost to Follow-up

Subjects or subjects' parent(s)/legal guardian(s) or legally acceptable representative(s) who cannot be contacted on or before the final Follow-up Contact at 14 days post-last dose prior to the trial termination date, who do not have a known reason for discontinuation (eg, withdrew consent or AE) and for whom a current health status at the end of the trial cannot be determined will be classified as "lost to follow-up" as the reason for discontinuation. Current health status can be determined from a variety of sources, either by obtaining acceptable documentation for death (ie, death certificate, medical records, public records, or statement by a family member or primary care physician) or acceptable documentation for life (ie, direct contact with the subject, medical records, successful telephone contact with the subject, statement by a family member or primary care physician, or public records).

The site will make 3 documented attempts to contact the subject by telephone and in the event the site is unable to reach the subject by telephone, the site will attempt to contact

Protocol 156-08-276

the subject via certified mail or an alternative similar method, where appropriate, before assigning a "lost to follow-up" status.

# 3.12 Subject Compliance

All subjects in this trial who deviate from assigned treatment will be considered noncompliant.

Compliance will be ensured by watching the subject take his/her tolvaptan while the subject is hospitalized or during clinical trial site visits. For nonclinical trial site days, compliance will be assessed by the number of tablets remaining when the subject returns the blister cards at the next visit. This information will be recorded on the appropriate eCRF and on the Drug Accountability Forms.

#### 3.13 Protocol Deviations

In the event of a significant deviation from the protocol due to an emergency, accident, or mistake (eg, violation of informed consent/assent process, IMP dispensing or subject dosing error, subject enrolled in violation of eligibility criteria or concomitant medication criteria), the investigator or designee will contact INC Research at the earliest possible time by telephone. The investigator and INC Research will come as quickly as possible to a joint decision regarding the subject's continuation in the trial. This decision will be documented by the investigator and INC Research, and reviewed by the site monitor.

## 4 Restrictions

#### 4.1 Prohibited Medications

Continuous or short term use of other medications, while not prohibited, may be restricted by the investigator because of their potential for interference with tolvaptan metabolism. Tolvaptan is a sensitive CYP3A4 substrate; plasma concentrations increased approximately 4-fold when tolvaptan was administered with the potent CYP3A4 inhibitor ketoconazole. Where appropriate dose reductions are possible, tolvaptan doses may be coadministered with potent or moderate CYP3A4 inhibitors (see Section 2.1.1 and Table 3.2.3-1).

A partial list of CYP3A4 inhibitors is provided in Table 4.1-1.

| <b>Table 4.1-1</b> | List of Cytochrome P450 3A4 Inhibitors (Partial List) |
|---|---|
| boceprevir | nefazodone |
| clarithromycin | nelfinavir |
| clotrimazole (oral) | posaconazole |
| conivaptan | ritonavir |
| indinavir | saquinavir |
| itraconazole | telaprevir |
| ketoconazole | telithromycin |
| lopinavir | voriconazole |
| mibefradil | |

## 4.2 Other Restrictions

The ingestion of pomelo, grapefruit, grapefruit juice, products containing Seville oranges, and St. John's Wort is prohibited from 72 hours prior to dosing until 24 hours post-last dose of IMP. In addition, the use of alcohol within 72 hours prior to dosing and during the trial is prohibited.

Other treatment for the purpose of increasing serum sodium, eg with urea, lithium, demeclocycline, conivaptan or tolvaptan, concurrent with dosing of trial medication or within 4 days of qualifying serum sodium assessments at screening is prohibited.

The use of saline in this population should be closely monitored. The use of hypertonic saline (3% or greater), including normal saline challenge within 8 hours of the qualifying screening serum sodium laboratory assessment is prohibited. The use of hypertonic saline (3% or greater) is prohibited during tolvaptan treatment. Routine use of hypertonic saline, while prohibited, may be considered only if used emergently (ie, with a severe symptomatic episode) and with the understanding that free water clearance may be stimulated if tolvaptan had been administered in the prior 24 hours, based on the medical judgment of the investigator.

The use of normal saline (0.9%) is allowed during screening until the beginning of Treatment Phase A; normal saline use can resume in Phase C. Subjects should no longer be on maintenance fluids containing normal saline during treatment with tolvaptan. Subjects may be administered IV solutions containing hypotonic saline (eg, half-normal [0.45%] saline), if necessary, for fluid management. The medical monitor should be contacted at any point if questions arise regarding the use of saline during the trial.

# 5 Reporting of Adverse Events

## 5.1 Definitions

An AE is defined as any untoward medical occurrence in a patient or clinical trial subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. AEs would not include information recorded as medical history at screening for pre planned procedures for which the underlying condition was known and no worsening occurred. An adverse reaction is any untoward and unintended response to an IMP related to any dose administered.

A suspected adverse reaction is any AE for which there is a reasonable possibility that the IMP caused the AE. For the purpose of Investigational New Drug (IND) safety reporting, "reasonable possibility" means there is evidence to suggest a causal relationship between the IMP and the AE. Suspected adverse reaction implies a lesser degree of certainty about causality.

An SAE includes any event that results in any of the following outcomes:

- Death
- Life-threatening; ie, the subject was, in the opinion of the investigator, at immediate risk of death from the event as it occurred. It does not include an event that, had it occurred in a more severe form, might have caused death.
- Persistent or significant incapacity/disability or substantial disruption of the ability to conduct normal life functions.
- Requires in-patient hospitalization or prolongs hospitalization.
  - Hospitalization itself should not be reported as an SAE; whenever possible the reason for the hospitalization should be reported.
  - Hospitalizations or prolonged hospitalizations for social admissions (ie, those required for reasons of convenience or other non-medical need) are not considered SAEs.
- Congenital anomaly/birth defect.
- Other medically significant events that, based upon appropriate medical
  judgment, may jeopardize the subject and may require medical or surgical
  intervention to prevent one of the outcomes listed above; eg, allergic
  bronchospasm requiring intensive treatment in an emergency room or home,
  blood dyscrasias or convulsions that do not result in hospitalization, or the
  development of drug dependency or drug abuse.

Nonserious adverse events are all AEs that do not meet the criteria for a "serious" AE. Immediately Reportable Event (IRE):

- Any SAE.
- Any AE related to occupational exposure.
- Potential Drug Induced Liver Injury (DILI) case (see Section 5.4).
- Pregnancies are also defined as IREs. Although normal pregnancy is not an AE, it will mandate IMP discontinuation and must be reported on an IRE form to the sponsor. Pregnancy will only be documented on the AE eCRF if there is an abnormality or complication.

Clinical Laboratory Test Value Changes: It is the investigator's responsibility to review the results of all laboratory tests as they become available. This review will be documented by the investigator's dated signature on the laboratory report. For each abnormal laboratory test result, the investigator needs to ascertain if this is an abnormal (ie, clinically significant) change from baseline for that individual subject. This determination, however, does not necessarily need to be made the first time an abnormal value is observed. The investigator may repeat the laboratory test or request additional tests to verify the results of the original laboratory tests. If this laboratory value is considered medically relevant by the investigator (subject is symptomatic, requiring corrective treatment or further evaluation), or if the laboratory value leads to discontinuation, and/or fulfills a seriousness criterion, this is considered an AE.

<u>Severity:</u> Adverse events will be graded on a 3-point scale and reported as indicated on the eCRF. The intensity of an adverse experience is defined as follows:

**1 = Mild:** Discomfort noticed, but no disruption to daily activity.

**2 = Moderate:** Discomfort sufficient to reduce or affect normal daily activity.

**3 = Severe:** Inability to work or perform normal daily activity.

<u>IMP Causality:</u> Assessment of causal relationship of an AE to the use of the IMP is defined as follows:

**Related**: There is a reasonable possibility of a temporal and causal

relationship between the IMP and the AE.

**Not Related**: There is no temporal or causal relationship between the IMP and

the AE

# 5.2 Eliciting and Reporting Adverse Events

The investigator will periodically assess subjects for the occurrence of AEs. To avoid bias in eliciting AEs, subjects should be asked the non-leading question: "How have you

felt since yesterday/last time we spoke?" <u>All AEs</u> (serious and nonserious) reported by the subject must be recorded on the source documents and eCRFs provided by the sponsor. Serious AE collection is to begin after a subject has signed the ICF.

Use medical terminology in AE reporting. Adverse events should be reported as a single unifying diagnosis whenever possible or, in the absence of a unifying diagnosis, as individual signs or symptoms. Exacerbation or disease progression should be reported as an AE only if there are unusual or severe clinical features that were not present, or experienced earlier, or not expected based on the course of the condition.

In addition, the sponsor must be notified immediately by telephone, fax, or e-mail of any IREs according to the procedure outlined below, in Section 5.3. Special attention should be paid to recording hospitalization and concomitant medications.

## 5.3 Immediately Reportable Events

The investigator must immediately report after either the investigator or site personnel become aware of any <u>SAE</u>, <u>DILI</u>, <u>or confirmed pregnancy</u>, by telephone, fax, or e-mail to INC Research as outlined in <u>Appendix 1</u>. An IRE form must be completed and sent by e-mail, fax, or overnight courier to INC Research. (Please note that the IRE form is NOT the AE eCRF.)

Subjects experiencing SAEs should be followed clinically until their health has returned to baseline status, or until all parameters have returned to normal or have otherwise been explained. It is expected that the investigator will provide or arrange appropriate supportive care for the subject and will provide prompt updates on the subject's status to INC Research.

# 5.3.1 Hyponatremia-related Adverse Events

## 5.3.1.1 Rapid Correction of Serum Sodium

When tolvaptan is not administered with adequate fluid intake, overly rapid correction of serum sodium may occur. Rapid correction of serum sodium level may lead to osmotic demyelination syndrome, a condition that can lead to severe brain damage and even death. Age-appropriate neurological examinations will be performed during administration of tolvaptan to monitor changes in health status in addition to serum sodium. This protocol is designed to provide adequate vigilance during the administration of tolvaptan to ensure that over rapid correction does not occur in this pediatric population.

Rapid correction of hyponatremia is defined as any increase in serum sodium.

If this change is observed during the trial, it should be reported as an IRE following the instructions detailed in Section 5.3 of the protocol.

# 5.3.1.2 Other Hyponatremia-related Adverse Events

Other events related to hyponatremia should be monitored closely and reported as appropriate depending on their severity:

- Absolute serum sodium level ≥145 mEq/L
- Any increase in serum sodium > 8 mEq/L [mmol/L] over a 10-hour period
- Neurological symptoms or other signs or symptoms suggestive of osmotic demyelination
- Worsening symptoms of hyponatremia
- Hypovolemia or hypotension requiring intervention
- Signs and symptoms of dehydration

All AEs must be monitored until symptom resolution or until the condition stabilizes.

# 5.4 Potential Drug-induced Liver Injury

For a subject who experiences an elevation in AST or ALT that is  $\geq 2 \times ULN$  or whose levels increase  $\geq 2$  times their initial baseline value, a total bilirubin level should also be evaluated. Elevated values should be confirmed via retest. If the total bilirubin is  $\geq 2 \times ULN$  or  $\geq 2$  times their baseline value, an IRE form should be completed with all values listed and also should be reported as an AE on the eCRFs.

If hepatic injury is suspected, tolvaptan should be promptly discontinued, appropriate treatment should be instituted, and investigations should be performed to determine probable cause. Such an event should be reported and followed until resolution.

#### 5.4.1 Liver Transaminase Elevations

Management of abnormal liver function test results should be based on the investigator's clinical judgment. A liver function test result that is  $2 \times ULN$  is generally accepted as a medically significant occurrence across various medical disciplines.

For a subject that experiences an elevation in AST or ALT that is  $\geq 2 \times ULN$  or whose levels increase  $\geq 2$  times their initial baseline value in subjects with an elevated baseline value, a total bilirubin level should also be evaluated. If the total bilirubin is  $\geq 2 \times ULN$  or  $\geq 2$  times their baseline value in subjects with an elevated baseline value, an IRE form with all values listed should be completed and also reported as an AE on the eCRFs.

#### Protocol 156-08-276

The following guideline for repeat testing may be used by investigators as a reference for any subject with an ALT or AST  $\geq 2 \times ULN$ :

- 1) ALT, AST, alkaline phosphatase, and total bilirubin should be repeated within 48 to 72 hours (needed to confirm abnormalities and determine if they are increasing or decreasing).
- 2) Inquiries should be made about symptoms (fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, and/or rash) and signs like jaundice, yellowish discoloration of sclera, etc.
- 3) If discharged or transferred, the subjects should be retested locally and results given to the investigator immediately, along with that laboratory's normal ranges.
- 4) Close observation is required if symptoms persist or repeat testing shows ALT or AST ≥ 3 × ULN for subjects with normal baseline measures OR 2-fold increases above baseline values for subjects with elevated values before drug exposure. If close monitoring is not possible, the drug should be interrupted until such monitoring is possible or the drug should be permanently discontinued.
- 5) All trial subjects with evidence of possible drug-induced liver injury should be followed until all abnormalities return to normal or to the baseline state.

## Close observation may involve:

- 1) Repeating liver enzymes and serum bilirubin tests 2 or 3 times weekly.
- 2) Frequency of retesting can decrease to once a week or less if abnormalities stabilize or if the trial drug has been interrupted/discontinued and the subject is asymptomatic.
- 3) Obtaining a more detailed history of symptoms and prior or concurrent diseases.
- 4) Obtaining a history of concomitant drug use (including non-prescription medications and herbal and dietary supplement preparations), alcohol use, recreational drug use, special diets, and change in diet.
- 5) Ruling out acute viral hepatitis types A, B, C, D, and E; autoimmune or alcoholic hepatitis, nonalcoholic steatohepatitis; hypoxic/ischemic hepatopathy; and biliary tract disease.
- 6) Obtaining a history of exposure to environmental chemical agents.
- 7) Obtaining additional tests to evaluate liver function, as appropriate (eg, international normalized ratio [INR], direct bilirubin).
- 8) Considering gastroenterology or hepatology consultations.

# 5.4.1.1 Criteria for Discontinuation Due to Liver Transaminase Elevations

A subject must be discontinued from the trial on confirmation of any of the following criteria:

- 1) ALT or AST  $\geq 8 \times ULN$
- 2) ALT or AST  $\geq$  5 × ULN for more than 2 weeks
- 3) ALT or AST  $\geq 3 \times$  ULN AND (total bilirubin  $\geq 2 \times$  ULN or INR > 1.5)
- 4) ALT or AST  $\geq$  3 × ULN with appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and/or eosinophilia (> 5%) and signs of jaundice

If there is any question about how to proceed with a particular subject's case, do not hesitate to contact your regional medical monitor to discuss. The FDA has issued a guidance for industry regarding this topic. This guidance is not specific to hyponatremia. Otsuka is integrating many of the recommendations in this guidance into all of its clinical research programs. Links to this guidance and information from the FDA regarding drug-induced liver injury are provided in the references. 31,32

# 5.5 Pregnancy

Women of childbearing potential (WOCBP) are defined as female subjects for whom menstruation has started and who are not documented as sterile (ie, have had a bilateral oopherectomy and/or hysterectomy or who have been postmenopausal for at least 12 months).

For WOCBP and for males who are sexually active, there must be a documented agreement that the subject and/or their partner will take effective measures (ie, double-barrier method) to prevent pregnancy during the course of the trial and for 30 days after the last dose of IMP. Unless the subject is sterile (ie, women who have had a bilateral oophorectomy and/or hysterectomy or who have been postmenopausal for at least 12 consecutive months) or remains fully abstinent (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] or withdrawal are not acceptable methods of contraception), 2 of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, condom with spermicide, or sponge with spermicide. The following 3 contraceptive methods are not allowed in this trial: birth control pills, birth control depot injection, and birth control implant. Any single method of birth control, including vasectomy and tubal ligation, may

Protocol 156-08-276

fail, leading to pregnancy. The contraceptive method will be documented at each trial visit.

Before enrolling WOCBP in this clinical trial, investigators must review the below guidelines about trial participation with all WOCBP. The topics should generally include:

- General information
- ICF/assent form, as applicable
- Pregnancy prevention information
- Drug interactions with hormonal contraceptives
- Contraceptives in current use
- Guidelines for the follow-up of a reported pregnancy

Before trial enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. The subject or the subject's parent/legal /guardian or legally acceptable representative must sign an ICF stating that the above-mentioned risk factors and the consequences were discussed with the subject and/or the parent/legal guardian or legally acceptable representative.

A urine and/or serum pregnancy test for human chorionic gonadotropin (hCG) will be performed at screening on all WOCBP and female subjects  $\geq$  12 years of age and all female subjects  $\leq$  12 years of age, if menstruation has started. If a urine test is performed and is positive, the investigator will follow up with a confirmatory serum test.

During the trial, all WOCBP should be instructed to contact the investigator immediately if they suspect they might be pregnant (eg, missed or late menstrual cycle).

If a subject is suspected to be pregnant before she receives IMP, the IMP administration must be withheld until the results of serum pregnancy tests are available. If the pregnancy is confirmed, the subject must not receive the IMP and must not be enrolled in the trial. If pregnancy is suspected while the subject is taking IMP, the IMP must be withheld immediately (if reasonable, taking into consideration any potential withdrawal risks) until the result of the pregnancy is known. If pregnancy is confirmed, the IMP will be permanently discontinued in an appropriate manner (eg, dose tapering if necessary for subject safety) and the subject will be withdrawn from the trial. (Exceptions to trial discontinuation may be considered for life-threatening conditions only after consultations with INC Research [see Appendix 1 for contact information].)

The investigator must immediately notify INC Research of any pregnancy associated with IMP exposure during the trial and for 30 days after the last dose of IMP, and record the event on the IRE form and forward it to INC Research. INC Research will forward Pregnancy Surveillance Form(s) for monitoring the outcome of the pregnancy.

Protocol-required procedures for trial discontinuation and follow-up must be performed on the subject unless contraindicated by pregnancy (eg, x-ray trials). Other appropriate pregnancy follow-up procedures should be considered, if indicated. In addition, the investigator must report to INC Research on appropriate Pregnancy Surveillance form(s), follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome. Infants will be followed for a minimum of 6 months from the date of birth.

## 5.6 Procedure for Breaking the Blind

Not applicable as this is an open-label trial.

## 5.7 Follow-up of Adverse Events

For this trial, information on AEs will be followed for up to 14 days post-last dose for all subjects or until resolution, whichever is longer.

# 5.7.1 Follow-up of Nonserious Adverse Events

Nonserious AEs that are identified at any time during the trial must be recorded on the AE eCRF with the current status noted. If a subject has an AE or has not recovered from an AE at the last scheduled contact, follow-up contacts will be scheduled at least every 4 weeks until resolution of the AE is confirmed or the condition is considered clinically stable. All nonserious events that are ongoing at the last scheduled contact will be recorded as ongoing on the eCRF. For any AE having been identified throughout the trial, during analysis, additional relevant medical history information may be requested to further ascertain causality (including, but not limited to, information such as risk-related behavior, family history and occupation).

# 5.7.2 Follow-up of Serious Adverse Events

This trial requires that subjects be actively monitored for SAEs up to 14 days post-last dose or until resolution of the SAE, whichever is longer.

Serious AEs that are **identified or ongoing at the last scheduled contact** must be recorded on the AE eCRF page and reported to INC Research according to the reporting procedures outlined in Section 5.3. This may include **unresolved previously reported SAEs, or new SAEs.** The investigator will follow SAEs until the events are resolved,

stabilized, or the subject is lost to follow-up. Resolution means that the subject has returned to the baseline state of health and stabilized means that the investigator does not expect any further improvement or worsening of the subject's condition. The investigator will continue to report any significant follow-up information to INC Research up to the point the event has been resolved.

# 5.7.3 Follow-up and Reporting of Serious Adverse Events Occurring After Last Scheduled Contact

Any new SAEs reported by the subject to the investigator that occur **after the last scheduled contact**, and are determined by the investigator to be reasonably associated with the use of the IMP, should be reported to INC Research. This may include SAEs that are captured on follow-up telephone contact or at any other time point after the defined trial period (ie, up to last scheduled contact). The investigator should follow serious related AEs identified after the last scheduled contact until the events are resolved, or the subject is lost to follow-up. The investigator should continue to report any significant follow-up information to INC Research up to the point the event has been resolved

# 6 Pharmacokinetic/Pharmacodynamic Analyses

# 6.1 Pharmacokinetic Analysis

A population analysis will be performed and reported separately.

# 6.2 Pharmacodynamic Analysis

Urine volume will be summarized by 6-hour intervals using descriptive statistics. Fluid intake and the calculated value of fluid balance will be summarized for each 6-hour period and for the 24-hour daily interval on Days 1 and 2 in Treatment Phase A using descriptive statistics. A subgroup analysis by the disease etiology of hyponatremia or by

Protocol 156-08-276

fluid status (euvolemic, hypervolemic) may be conducted if there are sufficient subjects in each category.

Urine osmolality and urine creatinine, potassium, and sodium concentrations will be summarized by collection interval and for zero to 24 hours on Days 1 and 2 in Treatment Phase A using descriptive statistics.

Missing urine concentrations or volumes will not be imputed. All calculations will use nominal times.

If urine volume during a collection interval is zero, then the amount excreted for that interval will be set to missing; values for 24 hours will be determined.

Correlations between urine output or fluid balance and change in serum sodium concentration may be explored graphically.

Correlations between tolvaptan AUC values and urine output on Day 1 may be explored graphically.

# 7 Statistical Analysis

# 7.1 Sample Size

# 7.1.1 Sample Size for Efficacy

A total of 70 randomized subjects will provide 90% power to detect a treatment difference of 4 mEq/L (mmol/L) in change in serum sodium from Day 2 (or 2a) at the end of Treatment Phase A to the end of Treatment Phase B using a 2-sided alpha of 0.05. An SD of 5 in change of serum sodium was used for the sample size calculation. After the end of Treatment Phase A at Day 2 (or 2a), subjects will be randomized at a ratio of 1:1 to either continue treatment with tolvaptan for 2 additional days (Late Withdrawal) or to discontinue tolvaptan treatment (Early Withdrawal). Sample size re-estimation will be conducted when 90% of the subjects finish (complete or discontinue) the trial. The trial must include no fewer than 60 subjects on IMP for the assessment of safety based on regulatory feedback.

# 7.1.2 Sample Size for Pharmacokinetic Parameters



order to establish a 95% CI within 60% and 140% of the point estimate for the geometric mean estimate of clearance in an age group (age < 10 or  $\ge 10$  years), under the assumption that the geometric means estimates of clearance are equal between adult and pediatric subjects, CIs of the ratio of geometric means of pediatrics and adults will be constructed. Twenty pediatric subjects and 80 adult subjects are needed to have 90% power to establish a 95% CI of the ratio of geometric means within 0.71 and 1.40. In the actual analysis, all 81 adult subjects' data will be used.

## 7.2 Datasets for Analysis

The following samples are defined for this trial:

- Enrolled Sample consists of all subjects for whom an ICF/assent form was signed for the trial.
- Treatment Phase A Safety Sample consists of all subjects who receive at least one dose of IMP in Treatment Phase A of the trial.
- Treatment Phase B Safety Sample consists of all randomized late withdrawal subjects who receive at least one dose of IMP in Treatment Phase B of the trial and all randomized early withdrawal subjects.
- Treatment Phase A Efficacy Sample consists of all subjects who are in Treatment Phase A Safety Sample and have baseline and at least one post-baseline efficacy evaluation in Treatment Phase A.
- Treatment Phase B Efficacy Sample is based on the intent-to-treat (ITT) principle; the full analysis dataset will be composed of all subjects who are in the Treatment Phase B Safety Sample and have both baseline and at least one post-baseline efficacy evaluation in Treatment Phase B.

Core dataset for efficacy analyses will be based on the ITT population. In order to handle missing data and restrictions imposed by different types of analyses (eg, change from baseline analysis), datasets derived from the ITT dataset will be used for the efficacy analyses.

# 7.3 Handling of Missing Data

For the primary endpoint analysis, missing data will be handled by analysis of mixed-model repeated measures (MMRM) methodology under the assumption of missing at random. The MMRM analysis will be performed based on the observed cases (OC) data. In order to assess sensitivity of results due to missing data, last observation carried forward (LOCF) analysis will be performed as a sensitivity analysis. In contrast to the OC dataset, which will consist of the actual observations recorded at each visit, the LOCF dataset will include data recorded at a scheduled visit (ie, all OC data, or, if no observation is recorded at that visit, data carried forward from the previously scheduled

visit). Baseline data will not be carried forward to impute missing values for the LOCF dataset.

# 7.4 Primary and Secondary Outcome Analysis

# 7.4.1 Primary Outcome Analysis

The primary endpoint in this trial is the change in serum sodium level for responders from Day 2 (or 2a) at the end of Treatment Phase A (where all subjects receive tolvaptan) to the end of Treatment Phase B for the Early compared to Late Withdrawal groups. The null hypothesis of this comparison is that there is no difference between the Late and the Early Withdrawal groups in change of serum sodium level from Day 2 (or 2a) at the end of Treatment Phase A to the end of Treatment Phase B. The analysis of the primary endpoint is based on the Treatment Phase B Efficacy Sample. Once a subject is randomized to Treatment Phase B, any additional therapies for the purpose of raising serum sodium, including fluid restriction, will be considered rescue therapy. Upon receipt of rescue therapy, a subject's endpoint data will be collected and then censored thereafter. The primary analysis of this protocol is based on the data collected in this manner.

A sensitivity analysis will be provided to include serum sodium data collected while an Early Withdrawal subject is under fluid restriction for the analysis of the primary endpoint. This sensitivity analysis would become the primary analysis if at least 30% of the Early Withdrawal subjects do not have serum sodium data at 24 and 48 hours post-randomization due to application of fluid restriction in the withdrawal phase of the protocol.

| The MMRM analysis with an unstructured var | riance covariance structure based on the OC |
|---|---|
| dataset will be performed on the primary endp | point. The MMRM model will include |
| fixed effect of treatment, age subgroup | , serum |
| sodium response subgroup ( | ), underlying etiology ( |
| | , visit, treatment visit |
| interaction, and covariate of baseline and baseline visit interaction. Statistical test of the | |
| least squares (LS) mean differences between treatment groups at the end of Treatment | |
| Phase B of the MMRM analysis will serve as the primary analysis. | |

As a sensitivity analysis, analysis of covariance with baseline value as covariate and treatment, age subgroup, serum sodium response subgroup, and underlying etiology of hyponatremia as factors will be applied to the LOCF dataset. Treatment comparison between the Late and Early Withdrawal groups will be conducted by comparing LS means.

For the primary endpoint analysis, baseline is the last evaluation of serum sodium level in Treatment Phase A prior to randomization.

# 7.4.2 Secondary Outcome Analyses

# 7.4.2.1 Secondary Efficacy Outcome Analyses

For all subjects, the key secondary endpoint is the change in serum sodium concentration at the end of Day 2 (or 2a) at the end of Treatment Phase A. The analysis of the key secondary endpoint will be based on the Treatment Phase A Efficacy Sample.

A paired Student's t-test will be used to analyze the key secondary endpoint.

For the key secondary efficacy analysis, a hierarchical testing procedure will be used to maintain the overall experiment-wise type I error rate at 0.05. Thus, if the primary efficacy analysis yields a statistically significant result at alpha level of 0.05 (2-sided), then the paired t-test will be performed at an alpha level of 0.05 for the key secondary endpoint.

Baseline for the key secondary analysis is the last evaluation prior to first dose of IMP in Treatment Phase A.

# 7.4.2.2 Secondary Safety Outcome Analyses

Other secondary endpoints include:

- Percentage of subjects with overly rapid increase in serum sodium level
- Change in serum sodium level from 24 hours post-last dose to 7 days post-last dose.
- Percentage of subjects requiring rescue therapy (other than fluid restriction) during Treatment Phase A and Treatment Phase B.
- Percentage of subjects requiring fluid restriction during Treatment Phase A and Treatment Phase B.
- Other secondary safety outcomes to be assessed are presented in Section 3.5.3.1 (Vital signs, blood pressure, clinical laboratory tests, body weight, and neurological examinations)

Descriptive statistics along with 2-sided 95% CIs will be applied for percentage of subjects with overly rapid increase in serum sodium and percentage of subjects requiring rescue therapy or fluid restriction.

The change in serum sodium level from 24 hours post-last dose to 7 days post-last dose will be summarized using a paired Student's t-test.

#### 7.4.2.3 Pharmacokinetic Parameters

Previously obtained PK data from 81 adult subjects who received a 30-mg dose of tolvaptan will be included in the analysis to show the similarity for PK parameter estimates between adult and pediatric subjects. An analysis of variance model will be performed on the natural-log transformed PK parameters using the MIXED procedure in SAS, in which only one fixed effect of subject group (pediatric and adult groups) is included in the model. The anti-logs of the difference of LS means and the confidence limits will provide the estimate and 90% CI for the ratio of the geometric means of pediatric group and adult group. Similarity of a PK parameter between pediatrics and adults will be indicated if the 90% CI for the ratio of the population geometric means is contained within the equivalence limits of 0.6 to 1.4.

## 7.4.3 Exploratory Outcome Analyses

Details will be provided in the statistical analysis plan.

The change in serum sodium concentration in nonresponders continuing on tolvaptan therapy by change from baseline at the end of Treatment Phase B compared to the end of Treatment Phase A will be analyzed using a paired Student's t-test.

The procedure for the analysis of data for the QoL assessments will be provided in the statistical analysis plan (SAP).

The analysis for the following exploratory PD endpoints is described in Section 6.2:

- In all subjects, 24-hour excretion of sodium, creatinine, and osmolality on Days 1 and 2
- 24-hour sodium clearance on Day 1

## 7.4.4 Interim Analysis

It was recommended by the FDA that the sample size should be re-estimated when approximately 90% of the subjects had finished the trial. The sample size re-estimation will assess the variability of change from Day 2 (or 2a) at the end Treatment Phase A to the end of Treatment Phase B in serum sodium level by using the pooled variance of the 2 treatment groups. At the trial planning stage, an SD of 5 was used to detect a treatment difference of 4, resulting in a sample size of 70 with a 2-sided alpha of 0.05 and 90% power. In case the variance ratio (equal to the observed pooled variance divided by 25, the square of 5 as an SD used in the sample size calculation) is  $\leq$  1, no sample size increase will be made, and the trial will proceed to finish enrollment of 70 randomized subjects. In case the variance ratio is  $\geq$  1, the sample size re-estimation will be equal to

70 multiplied by the variance ratio, then rounded up to the nearest even number. Table 7.4.4-1 provides an example of the sample size re-estimation under different variance ratios.

| <b>Table 7.4.4-1</b> | Sample Size Re-estimation |
|----------------------|---------------------------|
| Variance Ratio | Sample Size |
| 1.1 | 78 |
| 1.2 | 84 |
| 1.3 | 92 |
| 1.4 | 78 |
| 1.5 | 106 |

# 7.5 Analysis of Demographic and Baseline Characteristics

Demographic characteristics and medical history at Screening will be summarized by descriptive statistics, eg, proportion, mean, median, SD, minimum, and maximum values. These summary statistics will be reviewed to identify any potential lack of balance between the groups.

## 7.6 Safety Analysis

Safety analysis will be conducted based on the Safety Samples, which are defined in Section 7.2. Safety variables (in addition to those listed in Section 7.4.2.2) to be analyzed include AEs, clinical laboratory data, and vital signs. In general, summary statistics will be provided for safety variables based on all available data.

Safety analyses will be performed for Treatment Phase A and Treatment Phase B separately.

#### 7.6.1 Adverse Events

All AEs will be coded by system organ class and Medical Dictionary for Regulatory Activities (MedDRA) preferred term. The incidence of the following events will be summarized by treatment group:

- Treatment-emergent AEs (TEAEs)
- TEAEs by severity
- TEAEs potentially causally related to the IMP
- TEAEs with an outcome of death
- Serious TEAEs
- TEAEs leading to discontinuation of the IMP

The above summaries will also be prepared for TEAEs potentially causally related to the IMP.

# 7.6.2 Clinical Laboratory Assessment Data

Summary statistics for changes from baseline in the clinical laboratory measurements will be provided. Potentially clinically significant results in laboratory tests will also be summarized. Shift tables will be produced for assessing changes from baseline in clinical laboratory measurements in low-normal-high scale.

# 7.6.3 Physical Examination and Vital Signs Data

In general, summary statistics for changes from baseline in vital signs will be provided. Potentially clinically significant results in vital signs will also be summarized. No analysis will be performed on physical examination data. Physical examination data will be listed.

# 8 Management of Investigational Medicinal Product

# 8.1 Packaging and Labeling

The IMP will be provided to the investigator(s) by the sponsor (or designated agent). The IMP will be supplied as 3.75-, 7.5-, 15-, and 30-mg spray-dried tablets in blister packs or as 60 mL bottles containing 1 mg/mL (0.1% w/v) tolvaptan suspension. Each blister pack and suspension bottle used in the dosing period will be labeled to clearly disclose the compound ID, trial number, the sponsor's name and address, instructions for use, route of administration, appropriate precautionary statements, and other information required by local regulatory authorities. Each site will be supplied with bottle(s) containing placebo tablets to use for subject screening purposes. Each placebo bottle will be labeled to clearly disclose the compound ID, trial number, instruction for use, route of administration, appropriate precautionary statement, and other information required by the local regulatory authorities. For dosing suspension, syringes and bottle adaptors will be made available to the sites.

## 8.2 Storage

The IMP will be stored in a securely locked cabinet or enclosure. Access will be limited to the investigators and their designees. Neither investigators nor any designees may provide trial drugs to any subject not participating in this protocol.

The IMP blister packs will be stored at 25°C (77°F) or below, with excursions allowed from 15 to 30°C (59 to 86°F). The IMP suspension bottles will be stored at 2 to 8°C (35.6 to 46.4°F) and protected from light. The clinical site staff or designated personnel will maintain a temperature log in the IMP storage area recording the temperature at least once each working day.

# 8.3 Accountability

The investigator, or designee, must maintain an inventory record of IMP received, dispensed, administered, and returned.

#### 8.4 Returns and Destruction

Upon completion or termination of the trial, all unused and/or partially used IMP must be returned to OPDC (or a designated contractor).

All IMP returned to OPDC must be accompanied by the appropriate documentation and be clearly identified by protocol number and trial site number on the outermost shipping container. Returned supplies should be in the original containers. The assigned trial monitor should facilitate the return of unused and/or partially used IMP.

# 8.5 Reporting of Product Quality Complaints

A product quality complaint (PQC) is any written, electronic, or verbal communication by a healthcare professional, consumer, subject, medical representative, Competent Authority, regulatory agency, partner, affiliate, or other third party that alleges deficiencies or dissatisfaction related to identity, quality, labeling, packaging, reliability, safety, durability, tampering, counterfeiting, theft, effectiveness, or performance of a drug product or medical device after it is released for distribution. Examples include, but are not limited to, communications involving:

- Failure/malfunction of a product to meet any of its specifications
- Incorrect or missing labeling
- Packaging issues (eg, damaged, dirty, crushed, missing product)
- Blister defects (eg, missing, empty blisters)
- Bottle defects (eg, under/over-fill, no safety seal)
- Vial defects
- Product defect (eg., odor, chipped, broken, embossing illegible)
- Loss or theft of product

# 8.5.1 Eliciting and Reporting Product Quality Complaints

The investigator or designee must record all PQCs identified through any means from the receipt of the IMP from the sponsor through and including reconciliation and up to destruction, including subject dosing. The investigator or designee must notify the sponsor (or sponsor's designee) within 24 hours of becoming aware of the PQC by e-mail or telephone and according to the procedure outlined below.

- Online Send information required for reporting purposes (listed below) to OAPI-EQCProductComplaints@Otsuka-us.com
- Phone Rocky Mountain Call Center at +1-800-438-6055

Identification of a PQC by the subject should be reported to the site investigator, who should then follow one of the reporting mechanisms above.

# 8.5.2 Information Required for Reporting Purposes

Information required for reporting purposes include:

- Description of complaint
- Reporter identification (eg, subject, investigator, site)
- Reporter contact information (eg, address, phone number, e-mail address)
- ID of material (product/compound name, coding)
- Clinical protocol reference (number and/or trial name)
- Dosage form/strength (if known)
- Pictures (if available)
- Availability for return

#### 8.5.3 Return Process

During the report of the PQC, it should be indicated whether the complaint sample is available for return. If the complaint sample is available for return, the sample should be returned in the product retrieval package, which will be provided by Otsuka America Pharmaceutical, Inc.-Ethics, Quality and Compliance (OAPI-EQC).

It should be documented in the site accountability record that a complaint sample for a dispensed kit has been forwarded to OAPI-EQC for complaint investigation.

#### 8.5.4 Assessment/Evaluation

Assessment and evaluation of PQCs will be handled by OAPI EQC-QM group.

# 9 Records Management

#### 9.1 Source Documents

Source documents are defined as the results of original observations and activities of a clinical investigation. Source documents will include but are not limited to progress notes, electronic data, screening logs, and recorded data from automated instruments. All source documents pertaining to this trial will be maintained by the investigators and made available for direct inspection by authorized persons.

Investigator(s)/institution(s) will permit trial-related monitoring, audits, IRB/IEC review, and regulatory inspection(s) by providing direct access to source data/documents by authorized persons as defined in the ICF. In all cases, subject confidentiality must be maintained in accordance with local regulatory requirements.

#### 9.2 Data Collection

During each subject's visit to the clinic, a clinician participating in the trial will record progress notes to document all significant observations. At a minimum, these notes will contain:

- Documentation of the informed consent process, including any revised consents;
- Documentation of the investigator's decision to enroll the subject into the trial, the review of all inclusion/exclusion criteria prior to IMP administration, and confirmation of the subject's actual participation in the trial;
- The date of the visit and the corresponding Visit or Day in the trial schedule;
- General subject status remarks, including any *significant* medical findings. The severity, frequency, duration, action taken, and outcome of any AEs and the investigator's assessment of relationship to IMP must also be recorded;
- Any changes in concomitant medications or dosages;
- A general reference to the procedures completed:
- The signature (or initials) and date of each clinician (or designee) who made an entry in the progress notes.

In addition, any contact with the subject via telephone or other means that provides significant clinical information will also be documented in the progress notes as described above. Any changes to information in the trial progress notes and other source documents will be <u>initialed and dated on the day the change is made</u> by a site trial staff member authorized to make the change. Changes will be made by striking a single line through erroneous data (so as not to obliterate the original data), and clearly entering the

correct data (eg, wrong data right data). If the reason for the change is not apparent, a brief explanation for the change will be written in the source documentation by the clinician. If electronic data systems are being utilized, a full audit trail of changes must be maintained.

Information from the trial progress notes and other source documents will be promptly and LEGIBLY transcribed to eCRFs for transmission to the sponsor. Changes will be entered by investigative site personnel directly onto electronic CRFs in the sponsor's electronic data capture (EDC) system. Changes to the data will be captured by an automatic audit trail.

# 9.3 File Management at the Trial Site

The investigator will ensure that the trial site file is maintained in accordance with Section 8 of the ICH GCP Guideline E6<sup>30</sup> and as required by applicable local regulations. The investigator/institution will take measures to prevent accidental or premature destruction of these documents.

#### 9.4 Records Retention at the Trial Site

Regulatory requirements for the archival of records for this trial necessitate that participating investigators maintain detailed clinical data for the longest of the following 3 periods:

- A period of at least 2 years following the date on which approval to market the drug is obtained (or if IMP development is discontinued, the date regulatory authorities were notified of discontinuation); OR
- A period of at least 3 years after the sponsor notifies the investigator that the final report has been filed with regulatory authorities; OR
- Longer, region-specific storage requirements, if applicable.

The investigator must not dispose of any records relevant to this trial without either (1) written permission from the sponsor or (2) provision of an opportunity for sponsor to collect such records. The investigator will be responsible to maintain adequate and accurate electronic or hard copy source documents of all observations and data generated during this trial including any data clarification forms received from the sponsor. Such documentation is subject to inspection by the sponsor and relevant regulatory authorities. If the investigator withdraws from the trial (eg, due to relocation or retirement), all trial-related records should be transferred to a mutually agreed upon designee within a sponsor-specified timeframe. Notice of such transfer will be given to the sponsor in writing.

# 10 Quality Control and Quality Assurance

## 10.1 Monitoring

The sponsor has ethical, legal, and scientific obligations to follow this trial in accordance with established research principles, the ICH E6 GCP: Consolidated Guidance, and applicable regulatory requirements and local laws. As part of a concerted effort to fulfill these obligations (maintain current personal knowledge of the progress of the trial), the sponsor's monitors will visit the site during the trial, as well as communicate frequently via telephone, e-mail, and written communications. In addition, all investigators and clinical site personnel will undergo initial and ongoing training for this particular trial, and this training will be clearly documented.

## 10.2 Auditing

The sponsor's Quality Assurance Unit (or representative) may conduct trial site audits. Audits will include, but are not be limited to, IMP supply, presence of required documents, the informed consent process, and comparison of eCRFs with source documents. The investigator agrees to participate with audits.

Regulatory authorities may inspect the investigator during or after the trial. The investigator will cooperate with such inspections and will contact the sponsor immediately if such an inspection occurs.

# 11 Ethics and Responsibility

This trial must be conducted in compliance with the protocol, ICH GCP Guideline (E6), international ethical principles derived from the Declaration of Helsinki and Council for International Organizations of Medical Science guidelines, and applicable local laws and regulations. Each trial site will seek approval/favorable opinion by an IRB or IEC according to regional requirements, and the investigator will provide that documentation to the sponsor. The IRB/IEC will evaluate the ethical, scientific, and medical appropriateness of the trial. Further, in preparing and handling eCRFs, the investigator, subinvestigator, and their staff will take measures to ensure adequate care in protecting subject privacy. To this end, a subject number and subject identification code will be used to identify each subject.

Financial aspects, subject insurance, and the publication policy for the trial will be documented in the agreement between the sponsor and the investigator.

# 12 Confidentiality

All information generated in this trial will be considered confidential and will not be disclosed to anyone not directly concerned with the trial without the sponsor's prior written permission. Subject confidentiality requirements of the region(s) where the trial is conducted will be met. However, authorized regulatory officials and sponsor personnel (or their representatives) may be allowed full access to inspect and copy the records, consistent with local requirements. All IMPs, subject bodily fluids, and/or other materials collected shall be used solely in accordance with this protocol, unless otherwise agreed to in writing by the sponsor.

Subjects will be identified only by unique subject numbers in eCRFs. If further subject identification is required, subjects' full names may be made known to a regulatory agency or other authorized officials if necessary, subject to local regulations.

# 13 Amendment Policy

The investigator will not make any changes to this protocol without the sponsor's prior written consent and subsequent approval/favorable opinion by the IRB/IEC. Any permanent change to the protocol, whether an overall change or a change for specific trial site(s), must be handled as a protocol amendment. Any amendment will be written by the sponsor. Each amendment will be submitted to the IRB/IEC, as required by local regulations. Except for "administrative" or "non-substantial" amendments, investigators will wait for IRB/IEC approval/favorable opinion of the amended protocol before implementing the change(s). Administrative amendments are defined as having no effect on the safety of subjects, conduct or management of the trial, trial design, or the quality or safety of IMP(s) used in the trial. A protocol change intended to eliminate an apparent immediate hazard to subjects should be implemented immediately after agreement by the sponsor and investigator, followed by IRB/IEC notification within local applicable timelines. The sponsor will submit protocol amendments to the applicable regulatory agencies within local applicable timelines.

When the IRB/IEC, investigators, and/or the sponsor conclude that the protocol amendment substantially alters the trial design and/or increases the potential risk to the subject, the currently approved written ICF will require similar modification. In such cases, after approval/favorable opinion of the new ICF by the IRB/IEC, repeat written informed consent will be obtained from subjects enrolled in the trial before expecting

continued participation and before the amendment-specified changes in the trial are implemented.

# 14 Publication Authorship Requirements

Authorship for any Otsuka-sponsored publications resulting from the conduct of this trial will be based on International Committee of Medical Journal Editors (ICMJE) authorship criteria (http://www.icmje.org/recommendations). According to ICMJE guidelines, one may be considered an author only if the following criteria are met:

- 1. Substantial contributions to the conception or design of the work; or the acquisition, analysis, or interpretation of data for the work; AND
- 2. Drafting the work or revising it critically for important intellectual content; AND
- 3. Final approval of the version to be published; AND
- 4. Agreement to be accountable for all aspects of the work in ensuring that questions related to the accuracy or integrity of any part of the work are appropriately investigated and resolved.

All authors must meet the above criteria, and all who qualify for authorship based on the above criteria should be listed as authors.

Investigators or other trial participants who do not qualify for authorship may be acknowledged in publications resulting from the trial. By agreeing to participate in the trial, investigators or other trial participants consent to such acknowledgement in any publications resulting from its conduct.

# 15 References

- Totapally BR, Raszynski A. Hyponatremia in pediatric practice. Int Pediatrics. 2006;21(1):37-50.
- Eulmesekian PG, Perez A, Minces, PG, Bohn D. Hospital-acquired hyponatremia in postoperative pediatric patients: Prospective observational study. Pediatr Crit Care Med. 2010;11(4):479-83.
- Hanna M, Saberi MS. Incidence of hyponatremia in children with gastroenteritis treated with hypotonic intravenous fluids. Pediatr Nephrol. 2010;25:1471-5.
- Moritz ML, Ayus JC. New aspects in the pathogenesis, prevention, and treatment of hyponatremic encephalopathy in children [Review]. Pediatr Nephrol. 2010;25:1225-38.
- Adrogue HJ. Consequences of inadequate management of hyponatremia. Am J Nephrol. 2005;25:240-9.

- Miller M, Morley JE, Rubenstein LZ. Hyponatremia in a nursing home population. J Am Geriatr Soc. 1995;43(12):1410-3.
- Schrier RW. Pathogenesis of sodium and water retention in high-output and low-output cardiac failure, nephrotic syndrome, cirrhosis, and pregnancy. (Second of two parts). N Engl J Med. 1988;319(17):1127-34.
- <sup>8</sup> Chen L-K, Lin M-H, Hwang S-J, Chen T-W. Hyponatremia among the institutionalized elderly in two long-term care facilities in Taipei. J Chin Med Assoc. 2006;69(3):115-9.
- Huda MSB, Boyd A, Skagen K, Wile D, Van Heyningen C, Watson I, et al. Investigation and management of severe hyponatraemia in a hospital setting. Postgrad Med J. 2006;82:216-9.
- Wald R, Jaber BL, Price LL, Updahyay A, Madias N. Impact of hospital-associated hyponatremia on selected outcomes. Arch Int Med. 2010;170(3):294-302.
- Adrogue HJ, Madias NE. Hyponatremia. N Engl J Med. 2000;342:1581-9.
- Hasegawa H, Okubo S, Ikezumi Y, Uchiyama K, Hirokawa T, Hirano H, et al. Hyponatremia due to an excess of arginine vasopressin is common in children with febrile disease. Pediatr Nephrol. 2009;24(3):507-11.
- 13 experimental SIADH model. Otsuka Study No. 019174, Otsuka Report No. 015404, 2003.
- Otsuka Pharmaceutical Development & Commercialization, Inc. OPC-41061 Investigator's Brochure, edition 21. Otsuka Report, issued 25 Aug 2015.
- An open-label, randomized, three-period crossover study of the pharmacokinetics and pharmacodynamics of oral tolvaptan tablets under fasting and non-fasting conditions in subjects of Caucasian and Japanese descent. Otsuka Clinical Study Report for Protocol 156-03-242, issued 08 Oct 2004.
- Makinen K. 1984. Effect of long-term, peroral administration of sugar alcohol on man. Swed. Dent. J. 8:113-124.
- National Center for Health Statistics, National Center for Chronic Disease Prevention and Health Promotion. Clinical Growth Charts [available on the Internet]. Last updated Nov 2000.
- U.S. Food and Drug Administration. Guidance for Industry. Pediatric Study Plans: Content of and Process for Submitting Initial Pediatric Study Plans and Amended Pediatric Study Plans [report on the internet]. 2013 Jul [cited 05 Jul 2013].
- US Department of Health and Human Services: Guidance for Industry: E11 Clinical Investigation of Medicinal Products in the Pediatric Population. ICH December 2000.
- Multicenter, randomized, double-blind, placebo-controlled, efficacy and safety study of the effects of titrated oral tolvaptan tablets in patients with hyponatremia. Otsuka Clinical Study Report for Protocol 156-02-235, issued 07 Aug 2006.
- International, multicenter, randomized, double-blind, placebo-controlled, efficacy and safety study of the effects of titrated oral tolvaptan tablets in patients with hyponatremia. Otsuka Clinical Study Report for Protocol 156-03-238, issued 25 Jul 2006.
- 22 Physiologically-based pharmacokinetic modeling of tolvaptan for the prediction of syrup suspension doses in pediatric subjects from 4 Weeks to 4 years of age. Otsuka Clinical Study Report for Protocol 156-13-214, issued 27 Feb 2014, amended 13 Mar 2014.
- A Randomized Double-Blind Study to Assess the Safety and Pharmacokinetics of Concomitant Administration of Orally Administered OPC 41061 Tablets and Ketoconazole in Healthy Adult Male and Female Volunteers. Otsuka Clinical Study Report for Protocol 156-98-201, issued 07 Dec 2000, amended 15 Feb 2001, 28 May 2003, and 03 Mar 2004.
- Moritz ML, Ayus JC. Preventing neurological complications from dysnatremias in children. Pediatr Nephrol. 2005;20:1687-700.
- Moritz ML, Ayus JC. New aspects in the pathogenesis, prevention, and treatment of hyponatremic encephalopathy in children [Review]. Pediatr Nephrol. 2010;25(7):1225-38.
- Verbalis JG, Goldsmith SR, Greenberg A, Schrier RW, Sterns RH. Hyponatremia treatment guidelines 2007: expert panel recommendations. Am J Med. 2007;120(11 Suppl 1):S1-S21.
- Karp BI, Laureno R. Pontine and extrapontine myelinolysis; a neurologic disorder following rapid correction of hyponatremia. Medicine. 1993;72:359-73.
- El-Kabbani O, Darmanin C, Chung RP. Sorbitol dehydrogenase: structure, function and ligand design. Curr Med Chem. 2004 Feb;11(4):465-76.
- Mayatepek E, Hoffmann B, Meissner T. Inborn errors of carbohydrate metabolism. Best Practice & Research Clinical Gastroenterology. 2010;24:607-618.
- International Conference on Harmonisation (ICH) [homepage on the Internet]. E6: Good Clinical Practice: Consolidated Guideline [finalized 1996 May, corrected 1996 Jun 1996; cited 2005 Dec 6].
- U.S. Food and Drug Administration. Guidance for Industry. Drug-induced liver injury: premarketing clinical evaluation [report on the Internet]. 2009 Jul [cited 15 Feb 2014].
- U.S. Food and Drug Administration. [homepage on the Internet]. Silver Spring: [updated 05 Aug 2015; cited 12 Nov 2015].

## **Appendix 1** Names of Sponsor Personnel

Report Immediately Reportable Events (serious adverse events, potential drug-induced liver injuries, and pregnancies) as follows:

| Country | INC Research Safety Fax | INC Research Safety Fax Numbers |
|---|---|---|
| Belgium | | |
| Canada | (primary) or | (alternative) |
| Czech Republic | - | |
| Germany | | |
| Italy | | |
| Poland | | |
| Romania | | |
| Spain | | |
| Turkey | No toll free number available; please dial | (primary) or |
| | (alterna | ative) |
| United Kingdom | | |
| United States | (primary) or | (alternative) |



#### **Institutions Concerned With the Trial** Appendix 2

Institutions concerned with this trial are: Sponsor **Medical Monitoring** Otsuka Pharmaceutical Development & **INC** Research Commercialization, Inc. 3201 Beechleaf Court, Suite 600 2440 Research Boulevard Raleigh, North Carolina 27604-1547, USA Rockville, Maryland 20850, USA Phone: Fax: Phone: **Medical Monitor:** Phone ; Mobile Fax: E-Mail: **Electronic Data Capture Trial Management & Clinical** Monitoring MediData Solutions **INC** Research 79 Fifth Avenue, 8th Floor 3201 Beechleaf Court, Suite 600 New York, New York 10003, USA Raleigh, North Carolina 27604-1547, USA Phone: Fax: Phone: **Investigational Materials Study Communications & Patient/Site** Fisher Clinical Services **Support** Matthews Media Group 7554 Schantz Road Allentown, Pennsylvania 18106, USA 700 King Farm Boulevard, Suite 500 Phone: Rockville, MD 20850, USA Fax: Phone: Central ECG Storage **IRT Systems (treatment randomization)** S-CLINICA eResearch Technology, Inc. 1500 Market Street 1818 Market Street Philadelphia, Pennsylvania 19103, USA 12th Floor East Tower Philadelphia, Pennsylvania 19102, USA Phone: Phone: Clinical Laboratory Supplies **Central Laboratory (PK)** Covance Central Laboratory Services ICON Development Solutions, Inc. 8211 SciCor Drive 8282 Halsey Road Indianapolis, Indiana 46214, USA Whitesboro, New York 13492, USA

Phone:

Phone:

# IDMC Support

Chiltern (formerly Theorem Clinical Research)
1016 West Ninth Avenue
King of Prussia, PA 19406, USA
Phone:

Fax:

#### **Appendix 3** Handling and Shipment of Bioanalytical Samples

All tubes must be labeled such that the protocol number, subject number, date of collection, and time can be verified. The OPDC Bioanalytical Scientist must approve the labels, prior to use. It is important to note the exact time of the blood collection on the eCRF, not the scheduled time for the drawing. The exact time of dosing should also be noted.

#### Plasma Samples for Tolvaptan

Blood will be collected into tubes containing lithium heparin anticoagulant. The tubes should be gently inverted 3 to 4 times and then centrifuged at 2,000 to 3,000 rpm for at least 10 to 15 minutes at 4°C. The rpm should be kept at a constant setting throughout the trial. Plasma should be stored in a freezer at -20°C or colder or on dry ice. Samples should be shipped after a subject has completed treatment and the final PK sample has been drawn and processed so as to include the entire set of samples for each subject within one shipment.

#### **Shipment of Plasma**

The label on each tube must correspond to the requisition sheet and must be firmly attached with transparent tape and should include the protocol number, subject number, date of collection, and sample protocol time elapsed postdose. Samples must be neatly packed and retained in an insulated container (place container supplied within a cardboard box) with enough dry ice to last 72 hours (ie, at least 15 to 20 pounds). Boxes should be completely filled with dry ice to avoid air spaces that will allow evaporation of the dry ice. The container should be sealed with tape and placed in a cardboard box. The recipient must be alerted of shipments. Packages will not be shipped on Thursdays, Fridays, Saturdays, or any day prior to a holiday. Shipments will be via an overnight carrier.

# Appendix 4 Tanner Staging

# **Classification of Sex Maturity Stages in Girls**

| Stage | Pubic Hair | Breasts |
|---|---|---|
| 1 | Preadolescent | Preadolescent |
| 2 | Sparse, lightly pigmented, straight, medial | Breast and papilla elevated as small mound; |
| | border of labia | areolar diameter increased |
| 3 | Darker, beginning to curl, increased amount | Breast and areola enlarged, no contour |
| | | separation |
| 4 | Coarse, curly, abundant but amount less than | Areola and papilla form secondary mound |
| | adult | |
| 5 | Adult feminine triangle, spread to medial | Mature; nipple projects, areola part of the |
| | surface of thighs | general breast contour |

# **Classification of Sex Maturity Stages in Boys**

| Stage | Pubic Hair | Penis | Testes |
|---|---|---|---|
| 1 | Preadolescent | Preadolescent | Preadolescent |
| 2 | Scanty, long, slightly pigmented | Slight enlargement | Enlarged scrotum, pink texture altered |
| 3 | Darker, starts to curl, small amount | Longer | Larger |
| 4 | Resembles adult type but less in quantity; coarse, curly | Larger; glans and breadth increase in size | Larger, scrotum dark |
| 5 | Adult distribution, spread to medial surface of thighs | Adult size | Adult size |

#### **Appendix 5 Protocol Amendments**

Amendment Number: 1

**Issue Date:** 04 Nov 2013

#### **PURPOSE:**

- To update the clinical management representative for this trial
- To remove the serum chemistry assessment at 7 ( $\pm$  1) days post-randomization
- To change the sample size from 80 to 70 responders
- To clarify that subjects who cannot safely swallow the tablet are excluded until a liquid formulation is available
- To add neurological exam as an exploratory variable
- To update the dosing rationale based on starting doses (mg/kg) used for hyponatremia trials of tolvaptan in adults
- To change early termination from the 7-day Follow-up Visit to Day 5/6
- To clarify that Phase B (Randomization Phase) applies to all subjects
- To correct the definition of a rapid correction of serum sodium
- To update the interim analysis
- To update the contact list for reporting an IRE

**BACKGROUND:** This protocol is being amended to provide a more developed argument for the dosing rationale. The statistical section has also been updated.

#### MODIFICATIONS TO PROTOCOL:

- **Bold and underlined text:** Changed Text
- Bold and strike through text: Deleted Text
- **Bold and italicized text:** Added Text

#### **COVER PAGE**

#### **Added and Changed Text:**

#### **REVISED** CLINICAL PROTOCOL

Clinical Management t
Phone ; Fax



Date of Amendment 1: 04 Nov 2013

FOOTER

**Changed Text:** 

Final 03 Jul 2013 Amendment 1: 04 Nov 2013

SYNOPSIS TRIAL DESIGN

#### **Deleted Text:**

Phase C (Follow-up Phase): All subjects will be monitored and treated as clinically warranted per the investigator's preferred standard of care for up to 3 additional days after the last dose of tolvaptan (note: the Early Withdrawal group should be monitored for the first 48 hours post-last dose). All subjects will have an additional serum sodium measurement at 72 ( $\pm$  4) hours post randomization and 7 ( $\pm$  1) days post-randomization. An additional chemistry panel will also be collected 7 ( $\pm$  1) days post-randomization. A final safety follow-up telephone contact/visit will be performed 14 ( $\pm$  2) days post-last dose.

#### SYNOPSIS SUBJECT POPULATION

#### **Changed Text:**

This trial will include up to 100 male and female subjects aged  $\geq 4$  weeks (or  $\geq 44$  weeks adjusted gestational age for premature births) to < 18 years who have been diagnosed with euvolemic or hypervolemic hyponatremia (< 130 mmol/L) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). It is expected that **80 70** subjects will have a serum sodium increase of  $\geq 4$  mmol/L (ie, responders).

Eighty Seventy randomized subjects will provide 90% power to detect a treatment difference of 4 mmol/L in change in serum sodium from randomization (at the end of Day 2/3 [Phase A]) to the end of Day 4/5 (2 days after randomization [Phase B]). Age groups will be stratified such that half (40 35) of these subjects will be < 10 years old with at least 25% (20 17) of subjects < 6 years old. Subjects who are

defined as responders will be further stratified by the magnitude of serum sodium response to tolvaptan ( $\leq 7$  and > 7 mmol/L) and underlying etiology of hyponatremia.

# SYNOPSIS INVESTIGATIONAL MEDICINAL PRODUCT, DOSE, FORMULATION, MODE OF ADMINISTRATION

#### **Changed Text:**

• Subjects < 2 years of age, or weighing < 10 kg, or who cannot safely swallow the tablet will be excluded until the availability of a liquid formulation. Dosing information will be available at that time.

#### SYNOPSIS CRITERIA FOR EVALUATION

#### **Added Text:**

#### **Exploratory Endpoints:**

#### Efficacy:

• In nonresponders continuing on tolvaptan therapy, change in trough serum sodium concentration on Day 6 compared to Day 4

#### Safety:

• Neurological examinations

#### Pharmacodynamic:

- In all subjects, 24-hour excretion of sodium, creatinine, and osmoles on Days 1 and 2
- 24-hour sodium clearance

#### LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

#### **Added Text:**

BW Body weight

#### Section 2.1 TRIAL RATIONALE

#### **Changed Text:**

The proposed population size of 100 subjects should provide **80** <u>70</u> responders, which has adequate power (> 90%) to test for statistical significance in the primary endpoint. Enrollment is expected to take 3 years using up to 50 sites globally. Additional blood sampling will be included across populations to provide PK information.

#### Section 2.1.1 DOSING RATIONALE

#### **Added and Changed Text:**

Enrolled subjects will be dosed based on age, weight, and the use of CYP3A4 inhibitors. Subjects < 2 years of age or < 10 kg will be excluded until the availability of a liquid formulation. Subjects  $\ge 2$  years of age and weighing  $\ge 10$  to < 20 kg will receive an oral once daily dose of tolvaptan starting as a 3.75-mg spray-dried tablet. Subjects weighing 20 to 50 kg, inclusive, will receive an oral once daily dose of tolvaptan starting as a 7.5 mg spray-dried tablet. Subjects weighing > 50 kg will receive an oral once daily dose of tolvaptan starting as a 15-mg spray-dried tablet. For subjects weighing  $\ge 20$  kg and taking moderate inhibitors of CYP3A4, a half dose will be used (3.75 or 7.5 mg, by weight). For subjects weighing > 50 kg and taking potent inhibitors of CYP3A4, a one quarter dose will be used (3.75 mg). Subjects weighing < 20 kg and who are taking any CYP3A4 inhibitors will be excluded from the trial until such time that an alternate dosing formulation is available.

It is estimated that subjects 6 years of age weigh approximately 25 kg. <sup>17</sup> A 7.5-mg dose in a subject weighing 25 kg would be 0.3 mg/kg. For a subject weighing 50 kg, a 7.5-mg dose would be a 0.15-mg/kg dose. For a 15-mg dose, the corresponding body weights for 0.3- and 0.15-mg/kg doses would be 50 to 100 kg.

In the pivotal hyponatremia trials, <sup>13,18,19</sup> the starting 15-mg dose was administered to adult subjects weighing 34.0 to 164.7 kg; in terms of mg/kg, the starting dose of tolvaptan ranged from 0.09 to 0.44 mg/kg. The weight cutoffs for this trial were selected to produce mg/kg doses of tolvaptan within the range observed for the adult trials. Table 2.1.1-1 outlines the mg/kg dose ranges for tolvaptan tablet doses and body weights of 10, 20, 50, 70 (standard adult man), and 100 kg.

| <b>Table 2.1.1-1</b> | Table 2.1.1-1 Proposed Tolvaptan Doses as mg/kg of Body Weight | | | | |
|---|---|---|---|---|---|
| <b>Tolvaptan</b> | Tolvaptan Doses as mg/kg | | | | |
| <b>Tablets</b> | BW of 10 kg | BW of 20 kg | BW of 50 kg | BW of 70 kg | BW of 100 kg |
| <u>15 mg</u> | _ | = | 0.30 | 0.21 | 0.15 |
| 7.5 mg | _ | 0.375 | 0.15 | = | = |
| 3.75 mg | 0.375 | 0.19 | = | = | Ξ |

**BW** = body weight.

Tolvaptan is a sensitive CYP3A4 substrate; plasma concentrations increased approximately 4-fold when tolvaptan was administered with the potent CYP3A4 inhibitor ketoconazole. Where appropriate dose reductions are possible, tolvaptan doses may be coadministered with potent or moderate CYP3A4 inhibitors.

#### Section 3.1 TYPE/DESIGN OF TRIAL

#### **Deleted Text:**

Phase C (Follow-up Phase): All subjects will be monitored and treated as clinically warranted per the investigator's preferred standard of care for up to 3 additional days after the last dose of tolvaptan (note: the Early Withdrawal group should be monitored for the first 48 hours post-last dose). All subjects will have an additional serum sodium measurement at 72 ( $\pm$  4) hours post randomization and 7 ( $\pm$  1) days post randomization. An additional chemistry panel will also be collected 7 ( $\pm$  1) days post-randomization. A final safety follow-up telephone contact/visit will be performed 14 ( $\pm$  2) days post-last dose.

Figure 3.1-1 TRIAL DESIGN SCHEMATIC

#### Added Text:

<sup>a</sup>Subjects must be  $\geq 2$  years of age *and weigh*  $\geq 10$  kg until development of a liquid formulation is complete.

#### Section 3.2 TREATMENTS

#### Added Text:

Subjects who cannot take an oral tablet are currently excluded due to their inability to safely swallow the spray-dried tablet. Subjects weighing < 10 kg are also excluded as that weight has not been studied in previous PK trials and, therefore, the dose of tolvaptan being delivered is not confirmed. To support the enrollment of these subjects, an age and weight appropriate suspension formulation is being developed. Once available, the protocol will be amended to include the formulation.

Consequently, the maximum starting dose for subjects weighing > 50 kg is slightly less than 0.30 mg/kg; starting doses for subjects weighing 20 to 50 kg, inclusive, range from 0.38 to 0.15 mg/kg; starting doses for subjects weighing  $\geq 10$  to < 20 kg range from 0.375 mg/kg to slightly greater than 0.19 mg/kg. Therefore, the maximum starting doses planned for this pediatric trial are in the range previously used in adult hyponatremic subjects.

#### **Deleted Text:**

Some very young subjects will not be able to safely swallow the spray-dried tablet. To support the enrollment of these subjects, an age appropriate suspension formulation is being developed. Once available, the protocol will be amended to include the formulation.

#### Section 3.3 TRIAL POPULATION

#### **Changed Text:**

This trial will include up to 100 male and female subjects aged  $\geq$  4 weeks (or  $\geq$  44 weeks adjusted gestational age for premature births) to < 18 years, who have been diagnosed with euvolemic or hypervolemic hyponatremia (< 130 mmol/L) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). It is expected that **80** <u>70</u> subjects will have a serum sodium increase of  $\geq$  4 mmol/L (ie, responders).

Age groups will be stratified such that half (40 <u>35</u>) of these subjects will be age < 10 years with at least 25% (<u>20 17</u>) of subjects < 6 years old. Subjects who are defined as responders will be further stratified by the magnitude of serum sodium response to tolvaptan ( $\leq 7$  and  $\geq 7$  mmol/L) and underlying etiology of hyponatremia.

Section 3.5.3.2 SAFETY VARIABLE

**Added Text:** 

3.5.3.2 Safety Variable

The other safety variable is neurological examinations.

Section 3.7 TRIAL PROCEDURES

#### **Deleted Text:**

Treatment in this trial will be up to 5 days. Any initiation or titration of tolyaptan must occur in a hospital setting. Parents or legal guardians will consent and subjects will assent (as appropriate) and be screened up to 24 hours prior to dosing. Subjects who meet the inclusion and exclusion criteria will be enrolled and will be administered a 3.75-, 7.5-, or 15-mg dose based on age, weight, and the use of CYP3A4 inhibitors. At the end of Treatment Day 2 (optionally Day 3 [Phase A]), subjects who are responders will be randomized to either continue treatment with tolvaptan for 2 additional days (Late Withdrawal) or to discontinue tolvaptan treatment (Early Withdrawal). Subjects who are nonresponders may continue on tolvaptan therapy for 2 additional days at their highest dose or may be withdrawn from tolvaptan to be treated per the investigator's preferred standard of care. During Phase B, subjects in the Late Withdrawal group and nonresponders continuing treatment will continue treatment with tolvaptan for 2 additional days and all subjects will have serum sodium measured every 12 ( $\pm$  4) hours post-randomization. In Phase C, or Follow-up Phase, subjects will be monitored and treated as clinically warranted per the investigator's preferred standard of care for up to 3 additional days after the last dose of tolvaptan (note: the Early Withdrawal group should be monitored for the first 48 hours post-last dose) and will have an additional serum

sodium concentration measurement at 72 ( $\pm$  4) hours post randomization and 7 ( $\pm$  1) days post-randomization. **An additional chemistry panel will also be collected at 7 (\pm 1) days post-randomization.** A final safety follow-up telephone contact/visit will be performed 14 ( $\pm$  2) days post-last dose.

Table 3.7-1 SCHEDULE OF ASSESSMENTS

# **Changed Text:**

| Procedures | | Phase A | Phase B | | Phase C | |
|---|---|---|---|---|---|---|
| | Screening/<br>Baseline Visit<br>Days -2 to -1 | Initial Treatment Phase<br>Days 1 and 2/3 | Randomization<br>Phase<br>Days 3/4 and 4/5 | Follow-up<br>Phase<br>Day 5/6 <u>or ET</u> | Follow-up<br>(7 [± 1] days<br>post-random.)<br>or ET | Follow-up<br>Phone Call/Visit<br>(14 [+ 2] days<br>post-random.) |
| Informed consent and assent | X | | | | | |
| Review inclusion/exclusion criteria | X | Day 1: predose | | | | |
| Demographic information | X<br>X | | | | | |
| Medical and hyponatremia history | X | | | | | |
| Alcohol and drug screen | X | | | | | |
| Pregnancy test (if applicable) <sup>a</sup> | X | | | | | |
| Serum chemistry | X | | | X | X | |
| Serum osmolality, FeNa, and Fe urate | X | | | | | |
| TSH and cortisol <sup>b</sup> | X | | | | | |
| Hematology and coagulation | X | | | X | | |
| Urinalysis | X | | | X | | |
| Urine chemistry | X | Days 1 and 2 only: 6-hour intervals starting at Hour 0 | | | | |
| Serum sodium <sup>c</sup> | 2 assessments at<br>least 12 hours<br>apart | Baseline (Hour 0; within 3 ±1 hours of dosing), 12 hours post-first dose, and 24 (± 4) hours post-previous dose | 12, 24, 36, and<br>48 (± 4) hours<br>post-random. | 72 (± 4) hours post-random. | X | |

| Procedures | | Phase A | Phase B | | Phase C | |
|---|---|---|---|---|---|---|
| | Screening/<br>Baseline Visit<br>Days -2 to -1 | Initial Treatment Phase<br>Days 1 and 2/3 | Randomization<br>Phase<br>Days 3/4 and 4/5 | Follow-up<br>Phase<br>Day 5/6 <u>or ET</u> | Follow-up (7 [± 1] days post-random.) or ET | Follow-up<br>Phone Call/Visit<br>(14 [+ 2] days<br>post-random.) |
| Vital signs d | X | 2, 4, 8, and 24 hours post-first dose and on Day 3, if applicable | X | X | X | |
| Fluid intake and urine volume | | Days 1 and 2 only: 6-hour intervals starting at Hour 0 | | | | |
| PK plasma samples e | | 1, 2, 4, 12, and 24 hours post-first dose | 24 and 48 hours post-random. | ET only | ET only | |
| 12-lead ECG | X | | | | | |
| Directed physical examination | X | Baseline (Hour 0), 8 hours post-first dose, and Day 2/3 | Daily | X | X | |
| Neurological examination | X | Baseline (Hour 0), 8 hours post-first dose, and Day 2/3 | Daily | X | X | |
| Body height and weight f | X | Daily (predose): weight only | Daily (predose):<br>weight only | Weight only | Weight only | |
| Clinical assessment <sup>g</sup> | X | End of Day 2/3 | Day 4/5 | X | X | |
| Randomization | | Responders: End of Day 2 (optionally Day 3) | | | | |
| Tolvaptan dosing h | | Once daily | Once daily | | | |
| Follow-up phone call | | | | | | X |
| Concomitant medications | < | | | | | > |
| Adverse events | < | | | | | > |

#### Section 3.7.1.1 PHASE B: RANDOMIZATION PHASE

#### **Added Text:**

The following procedures will be performed on Days 3/4 and 4/5 *for all subjects*:

#### Section 3.7.1.3.1 FOLLOW-UP (DAY 5/6)/EARLY TERMINATION

#### Added Text:

#### 3.7.1.3.1 Follow-up (Day 5/6)/Early Termination

The following procedures will be performed on Day 5/6 *or at early termination (ET)* for all subjects:

4) A blood sample for PK analysis of tolvaptan will be collected at ET only if ET occurs before the last scheduled PK assessment (ie, 48 hours post-randomization for subjects continuing on tolvaptan).

#### Section 3.7.1.3.2 FOLLOW-UP

#### **Deleted Text:**

#### 3.7.1.3.2 Follow-up/Early Termination

Subjects will be assessed for maintenance of normal or target serum sodium concentration at  $7 (\pm 1)$  days post-randomization. If the subject was discharged, he/she should return to the clinic for the serum sodium collection. In addition, the following procedures will be performed for any subjects terminating early:

- 1) A serum chemistry laboratory sample will be collected.
- 2) A blood sample for serum sodium testing will be collected. (This blood draw can be combined with the chemistry panel as appropriate to minimize blood draws.)
- 3) A blood sample for PK analysis of tolvaptan will be collected at early termination (ET) only if ET occurs before the last scheduled PK assessment (ie, 48 hours post-randomization for subjects continuing on tolvaptan).

#### Section 3.7.4.1 ADVERSE EVENTS

#### **Changed Text:**

In particular, the following AEs must be actively monitored: absolute serum sodium level  $\geq 145$  mmol/L, overly rapid rise in serum sodium defined as an increase in serum sodium of > 8 mmol/L over a 10-hour period,  $> \geq 12$  mmol/L over a 24-hour period, or a rate of increase in serum sodium that the investigator deems too rapid,

neurological symptoms, or other signs or symptoms suggestive of osmotic demyelination (see Section 5.3.1 for more detail).

#### Section 3.8.3 INDIVIDUAL SUBJECT

#### **Changed Text:**

• The subject's serum sodium increases by > ≥ 12 mmol/L in the 24-hour period following dosing

#### Section 5.3.1.1 RAPID CORRECTION OF SERUM SODIUM

#### **Changed Text:**

Rapid correction of hyponatremia is defined as any increase in serum sodium  $\geq \geq 12 \text{ mmol/L/24}$  hours. If this change is observed during the trial, it should be reported as an IRE following the instructions detailed in Section 5.3 of the protocol.

#### Section 7.1.1 SAMPLE SIZE FOR EFFICACY

#### **Changed Text:**

A total of **80** <u>70</u> randomized subjects will provide 90% power to detect a treatment difference of 4 mmol/L in change in serum sodium from randomization (at the end of Day 2/3 [Phase A]) to the end of Day 4/5 (2 days after randomization [Phase B]) using a 2-sided alpha of 0.05. An SD of 5 in change of serum sodium was used for the sample size calculation. After the end of treatment at Day 2/3, subjects will be randomized at a ratio of 1:1 to either continue treatment with tolvaptan for 2 additional days (Late Withdrawal) or to discontinue tolvaptan treatment (Early Withdrawal). Sample size re estimation will be conducted when 90% of the subjects finish (complete or discontinue) the trial.

#### Section 7.4.2.3 PHARMACOKINETIC PARAMETERS

#### **Deleted Text:**

The PK data of 81 adult subjects with a 30-mg **tolvaptan**-dose will be included in the analysis to show the similarity for PK parameter estimates between adults and pediatrics.

#### Section 7.4.3 EXPLORATORY OUTCOME ANALYSIS

#### **Added Text:**

#### 7.4.3 Exploratory Outcome Analysis

Details will be provided in the statistical analysis plan.

Section 7.4.3.1 EFFICACY

**Added Text:** 

7.4.3.1 *Efficacy* 

The change in serum sodium concentration on Day 6 compared to Day 4 in nonresponders continuing on tolvaptan therapy will be analyzed using a paired Student's t-test.

Section 7.4.3.2 SAFETY

**Added Text:** 

7.4.3.2 Safety

Neurological examination data will be presented in the data listings.

Section 7.4.3.3 PHARMACODYNAMIC

**Added Text:** 

7.4.3.3 Pharmacodynamic

The exploratory PD endpoints include:

- In all subjects, 24-hour excretion of sodium, creatinine, and osmoles on Days 1 and 2
- 24-hour sodium clearance

These endpoints will be analyzed as described in Section 6.2.

Section 7.4.4 INTERIM ANALYSIS

**Changed Text:** 

**7.4.3 7.4.4** Interim Analysis

It was recommended that an interim analysis should be conducted by the FDA to re-estimate the sample size when about 90% of the subjects had finished the trial, in order to re-evaluate the power of this protocol and provide sample size re-estimation if needed. In this case, this protocol would be a protocol of 2-stage adaptive design, in which the first stage would provide data for sample size re evaluation and the second stage would include all data collected after the first stage. The final statistical test would combine data collected in both stages to

conclude the trial. It was further recommended that the weighted Z statistic approach outlined in Cui et al 1999 should be used as the final statistical test, due to its flexibility and being able to maintain the type I error in any cases once the weights are prespecified.<sup>23</sup>

To identify the need of sample size increase, the conditional power (CP) would be examined under the current trend in the interim analysis. Conditional power under the current trend is defined as the power of the trial of its planned sample size of 80 and the prespecified alpha of 0.05, under the assumption that the current trend observed at the interim analysis will continue to the end of the trial. Under this assumption, there is no need to increase the sample size when the CP is high or low enough, since it is expected the trial would succeed if the CP is high enough and fail if the CP is low enough. For this trial, the window for sample size increase is 50% ≤ CP < 80%. Furthermore, this window is divided into 3 intervals [50%, 60%), [60%, 70%), and [70%, and 80), and the sample size increase (or sample size needed in the Stage 2) in these 3 intervals will be determined by the sample size increase when the CP is equal to 50%, 60%, and 70%, respectively. With a designed sample size of 80, an interim analysis at 70, and the use of the weighted Z statistics proposed in Cui et al 1999, 23 in which nature weights of  $(70/80)^{1/2}$  and  $(10/80)^{1/2}$  are assigned to the Z statistics obtained in Stages 1 and 2, respectively, the estimated sample sizes based on these 3 intervals of CP are shown in Table 7.4.3 1.

| Table 7.4.3-1 Condition Power | |
|-------------------------------|-------------------------|
| Condition Power | Sample Size for Stage 2 |
| 50% ≤ CP < 60% | <del>168</del> |
| <del>60% ≤ CP &lt; 70%</del> | 130 |
| <del>70% ≤ CP &lt; 80%</del> | <del>96</del> |

Since the sample sizes needed for Stage 2 when CP falls in this window for sample size increase are very big and even bigger than the sample size planned for this trial (80), this adaptive design is very inefficient. It would be much more efficient to allow this trial to run through its planned sample size (10 additional subjects) and, if necessary, to use the information collected to design a new trial. Thus, no adaptive sample size re-estimation will be designed in this trial, and no interim analysis in this trial will be conducted for the adaptive design.

The sample size re-estimation will assess the variability of change from randomization (end of Phase A) to end of Day 4/5 (Phase B) in serum sodium by using the pooled variance of the 2 treatment groups. At the trial planning stage, an SD of 5 was used to detect a treatment difference of 4, resulting in a sample size of 70 with a 2-sided alpha of 0.05 and 90% power. In case the variance ratio (equal to the observed pooled variance divided by 25, the square of 5 as an SD used in the sample size calculation) is  $\leq 1$ , no sample size increase will be made, and the trial will proceed to finish enrollment of 70 randomized subjects. In case the variance ratio is  $\geq 1$ , the sample size re-estimation will be equal to 70

# multiplied by the variance ratio, then rounded up to the nearest even number. Table 7.4.3-1 provides an example of the sample size re-estimation under different variance ratios.

| Table 7.4.3-1 Sample Size Re-estimation | |
|-----------------------------------------|-------------|
| Variance Ratio | Sample Size |
| <u>1.1</u> | <u>78</u> |
| 1.2 | 84 |
| 1.3 | 92 |
| 1.4 | 78 |
| 1.5 | 106 |

#### Section 7.6.4 NEUROLOGICAL EXAMINATION

#### **Deleted Text:**

Neurological examination data will be presented in the listings.

#### Section 8.1 PACKAGING AND LABELING

#### **Added Text:**

The current tolvaptan tablet formulation intended for use in this trial is limited to administration to those who can easily swallow a 3.75-mg tablet (6 mm) *and weigh*  $\geq 10 \text{ kg}$ . A suspension formulation is in development that will be suitable for children who cannot swallow tablets (eg, < 4 years) and will also allow dosage adjustment for children with body weight < 20 or  $\leq$  50 kg who are taking moderate or potent inhibitors of CYP3A4, respectively. Once available, the protocol will be amended to include the details of this formulation.

#### **Section 14 REFERENCES**

#### **Added Text:**



### **Deleted Text:**

<sup>23</sup>—Cui L, Hung HMJ, Wang SJ. Modification of sample size in group sequential clinical trials. Biometrics. 1999;55:1551-62.

Appendix 1 NAMES OF SPONSOR PERSONNEL

# Replaced table:

| Country | Safety Fax Numbers |
|-------------------|--------------------|
| Taiwan | |
| Philippines | |
| Malaysia | |
| Singapore | |
| <b>Thailand</b> | |
| Hong Kong | |
| Australia | |
| Czech Republic | |
| Netherlands | |
| Belgium | |
| <del>Italy</del> | |
| Romania | |
| Spain | |
| Poland | |
| Russia | |
| Ukraine | |
| Israel | |
| South Africa | |
| Germany | |
| France | |
| <del>Serbia</del> | |
| United Kingdom | |
| Finland | |
| <del>Peru</del> | _ |
| Columbia | |
| Argentina | |
| Mexico | |
| US | (primary) or |
| | (alternative) |
| Canada | (primary) or |
| | (alternative) |

| Country | Safety Fax Numbers | |
|------------------|--------------------|---------------|
| United States | (primary) or | (alternative) |
| Argentina | | |
| <u>Australia</u> | _ | |
| <u>Belgium</u> | | |
| <u>Canada</u> | (primary) or | (alternative) |
| <u>Colombia</u> | | |
| Czech Republic | | |
| Finland | | |

| France | |
|--------------------|------------------------------------------------------|
| Georgia | No toll free number available; please dial (primary) |
| | or (alternative) |
| Germany | |
| Hong Kong | |
| Israel | |
| <u>Italy</u> | |
| <b>Korea</b> | |
| <u>Latvia</u> | |
| <u>Malaysia</u> | |
| Mexico | |
| <b>Netherlands</b> | |
| <b>Philippines</b> | |
| <u>Peru</u> | |
| <b>Poland</b> | |
| Romania | |
| Russia | |
| <u>Serbia</u> | |
| <b>Singapore</b> | |
| South Africa | |
| <u>Spain</u> | |
| <u>Taiwan</u> | |
| <u>Thailand</u> | |
| <u>Turkey</u> | No toll free number available; please dial (primary) |
| | or (alternative) |
| <u>Ukraine</u> | |
| United Kingdom | |

## **Changed Text:**



**ADDITIONAL RISK TO THE SUBJECT:** There is no additional risk to the subjects.

**Amendment Number: 2** 

**Issue Date:** 19 May 2014

#### **PURPOSE:**

• To increase the consistency of this protocol with other tolvaptan pediatric hyponatremia protocols

- To add neurocognitive and quality-of-life assessments as exploratory endpoints
- To clarify study design, procedures, and assessments
- To better define study phases and associated visits
- To provide greater detail about clinical laboratory tests
- To add Tanner staging to the assessments performed during the physical examination
- To better define completers and stopping rules
- To incorporate newly revised definitions of IMP causality

**BACKGROUND:** As several protocols in the tolvaptan hyponatremia pediatric development program were being conceived through negotiations with both US and European regulatory agencies, it became apparent that they needed to be aligned more closely in order to achieve as much consistency in data collection and to allow for data to be generated that could be synthesized and analyzed across studies.

#### **SECTIONAL REVISIONS:**

| Location: | Old Text: | New Text: |
|---|---|---|
| Title Page: | Medical Director: | |
| | | Date of Amendment 2: 19 May 2014 |
| Protocol | To assess the pharmacokinetics (PK) of | To assess tolvaptan's pharmacokinetics |
| Synopsis/ | tolvaptan and the effect on fluid balance in | (PK) and its effect on fluid balance in |
| Secondary | children and adolescent subjects with | children and adolescent subjects with |
| Objective: | euvolemic or hypervolemic hyponatremia. | euvolemic or hypervolemic hyponatremia. |
| Trial Design: | Subjects will undergo a treatment phase (2 to 5 days of tolvaptan) and a follow-up phase post-randomization of 14 days. <b>Phase A</b> (Treatment Phase): All subjects will initially receive tolvaptan once daily for the first 2 days. If a subject has not reached the desired sodium target improvement per the investigator's judgment (ie, the subject is a nonresponder) after Day 2 of tolvaptan | The trial will be conducted in two stages. The first stage will be conducted using the available tablet formulation of tolvaptan whereas the second stage will expand to the use of a suspension once that formulation becomes available Subjects will be required to be in a hospital setting during initiation and titration of |

#### Location: Old Text: New Text: administration (post 2 doses), a third day of tolvaptan. treatment is permitted. Overall, in this trial, subjects will undergo At the end of Day 2 (optionally Day 3), treatment (2 to 5 days of tolvaptan among 2 subjects who are responders will be treatment phases) and a post-last dose randomized to either the Early or Late follow-up phase of 14 days. Withdrawal group. Responders will be defined as those subjects who achieve an Treatment Phase A After screening, all subjects will initially increase in serum sodium by $\geq 4$ mmol/L. receive tolvaptan once daily for 2 days. If Early or Late Withdrawal assignment will the desired serum sodium level target be stratified by age improvement is not reached after Day 2 of ), serum sodium response tolvaptan administration (post 2 doses), a , and underlying etiology third day (Day 2a) of treatment is required. of hyponatremia. If the subject remains a At the end of Day 2 (or 2a), subjects will be nonresponder to tolvaptan at the end of Day assessed for a serum sodium level change of 3, the investigator is permitted to continue $\geq$ 4 mEg/L (mmol/L). At that time, subjects tolvaptan for 2 additional days at the highes who are responders will be randomized to dose or to discontinue tolvaptan and treat either the Early Withdrawal group or Late the subject per the investigator's preferred Withdrawal group. Responders are defined standard of care. as those subjects who achieve an increase in serum sodium concentration of Phase B (Randomization Phase): Subjects who are randomized to the Late Withdrawal $\geq$ 4 mEq/L (mmol/L); nonresponders are defined as subjects who do not achieve an group and nonresponders continuing treatment after Day 3 will continue increase in serum sodium concentration of treatment with tolvaptan for 2 additional $\geq$ 4 mEq/L (mmol/L). days. Subjects who are randomized to the Early Withdrawal group and nonresponders Treatment Phase B discontinuing treatment after Day 3 will Responders discontinue tolvaptan treatment Responders from Treatment Phase A will be immediately after randomization. randomized to either the: Late Withdrawal group - subjects Nonresponders will be treated per the continue tolyaptan treatment on Days 3 investigator's preferred standard of care during Days 3/4 and 4/5 (treatment day is Early Withdrawal group - subjects do dependent upon the number of doses that a not receive additional tolvaptan subject receives during Phase A). treatment on Days 3 and 4. Randomization will include stratification by Those subjects whose serum sodium age declines by $\geq 4 \text{ mmol/L}$ or whose overall serum sodium response clinical condition requires further treatment , and underlying etiology of to increase serum sodium will be treated per hyponatremia. the investigator's preferred standard of care. Any intervention intended to raise serum Those subjects whose serum sodium level sodium during the first 48 hours of the declines by $\geq 4$ mEq/L (mmol/L), or whose Early Withdrawal phase (including fluid overall clinical condition requires further restriction) will be defined as rescue treatment to increase serum sodium level, therapy; the subject will be considered to will be treated per the investigator's have reached their clinical endpoint, and

forward

their data will be censored from that time

measured at 12, 24, 36, and 48 ( $\pm$  4) hours

All subjects will have serum sodium

preferred standard of care. Any

intervention intended to raise serum sodium

level during the first 48 hours of the Early Withdrawal phase (including fluid

restriction) will be defined as rescue

therapy. Subjects who receive rescue

#### Location: Old Text: New Text: post-randomization. Serum sodium therapy will be considered to have reached their clinical endpoint, and their data will be assessment time points for nonresponders censored from that time forward. will follow the same schedule, but the values will be reported separately from the primary efficacy analysis. For analysis Nonresponders purposes, these assessments for If the subject remains a nonresponder at the nonresponders will be referred to as end of Day 2 (or 2a), the investigator decides to either (a) continue tolvaptan for 2 "post-randomization." additional days, or (b) discontinue tolvaptan Phase C (Follow-up Phase): All subjects and treat the subject per the investigator's will be monitored and treated as clinically preferred standard of care during Days 3 and warranted per the investigator's preferred 4. Subjects will continue to follow standard of care for up to 3 additional days scheduled assessments regardless of after the last dose of tolvaptan (note: the treatment. Early Withdrawal group should be monitored for the first 48 hours post-last All Subjects dose). All subjects will have an additional All subjects will have serum sodium levels measured at 8, 12, and 24 hours post-first serum sodium measurement at dose and thereafter every 12 hours through 72 ( $\pm$ 4) hours post-randomization and $7 (\pm 1)$ days post-randomization. A final completion of Treatment Phase B. safety follow-up telephone contact/visit will Follow-up Phase C be performed 14 (+ 2) days All subjects will have an additional serum post-randomization. sodium assessment at 72 ( $\pm$ 4) hours post-Pharmacokinetic samples will be obtained last dose and 7 ( $\pm$ 1) days post-last dose. A on Day 1 (Phase A) and, for tolvaptanfinal safety follow-up telephone treated subjects, at 24 and 48 hours contact/visit will be performed 14 (+ 2) post-randomization in Phase B. The PK days post-last dose. profiles will be evaluated on an ongoing basis to determine the variability between Pharmacokinetic Sampling subjects. Based on the findings, PK Blood samples for pharmacokinetic (PK) sampling will continue for as long as analysis will be obtained at 2 and 8 hours necessary to establish suitable estimates of post-first dose, and at trough on Days 2, 3, 4 clearance with a 90% confidence interval and 5 for all subjects when dosed with (CI) similar to that observed in the adult tolvaptan on Days 1, 2, 3, and 4, respectively, regardless of responder status. populations. Once these estimates are achieved, sampling will be discontinued in PK profiles will be evaluated on an ongoing subsequent subjects in order to minimize basis to determine variability among blood draws in this population. subjects. Based on the findings, PK sampling will continue for as long as Subjects will be required to be in the necessary to establish suitable estimates of hospital during initiation or up-titration of clearance with a 90% confidence interval administration of tolvaptan. If a subject is (CI), similar to that observed in adult in the withdrawal phase or is not expected subject populations. Once these estimates to receive a higher dose of tolvaptan, are achieved, sampling will be discontinued continued administration can be done in subsequent subjects in order to minimize outside of the hospital setting. Follow-up blood draws in this pediatric population. for all subjects may occur in the hospital if the subject has not been discharged or the subject may return for outpatient visits if the subject has been discharged from the hospital. This trial will include up to 100 male and This trial will include up to 100 male and Subject Population: female subjects aged $\geq 4$ weeks (or $\geq 44$ female subjects aged $\geq 4$ weeks (or $\geq 44$

| Location: | Old Text: | New Text: |
|---|---|---|
| | weeks adjusted gestational age for | weeks adjusted gestational age) to < 18 |
| | premature births) to < 18 years who have | years who have been diagnosed with |
| | been diagnosed with euvolemic or | euvolemic or hypervolemic hyponatremia |
| | hypervolemic hyponatremia | (< 130 mEq/L [mmol/L]) that persists |
| | (< 130 mmol/L) that persists despite initial | despite initial standard background therapy |
| | standard background therapy (including | (including fluid restriction and excluding a |
| | fluid restriction and excluding a vasopressin | vasopressin antagonist). Age groups will be |
| | antagonist). It is expected that 70 subjects | enrolled such that 50% of these subjects |
| | will have a serum sodium increase of $\geq 4$ | will be < 10 years old and at least 25% of |
| | mmol/L (ie, responders). | subjects < 6 years old. |
| | Subjects with euvolemic or hypervolemic | Subjects with acute hyponatremia or |
| | hyponatremia eligible to be screened for | hyponatremia expected to resolve |
| | participation in this trial include, but are not | spontaneously will be excluded from the |
| | limited to, those diagnosed and admitted to | trial |
| | a hospital for treatment of heart failure, | |
| | hepatocellular disease (including cirrhosis), | |
| | or syndrome of inappropriate secretion of | |
| | antidiuretic hormone (SIADH). Subjects | |
| | with acute hyponatremia or hyponatremia | |
| | expected to resolve spontaneously will be | |
| | excluded from the trial | |
| | Seventy randomized subjects will provide | |
| | 90% power to detect a treatment difference | |
| | of 4 mmol/L in change in serum sodium | |
| | from randomization (at the end of Day 2/3 | |
| | [Phase A]) to the end of Day 4/5 (2 days | |
| | after randomization [Phase B]). | |
| | Subjects who are defined as responders will | |
| | be further stratified by the magnitude of | |
| | serum sodium response to tolvaptan | |
| | and underlying etiology of | |
| | hyponatremia. | |
| | All subjects will be initially identified based | |
| | on serum sodium concentrations that persist | |
| | at levels < 130 mmol/L despite initial | |
| | standard background therapy (including | |
| | fluid restriction and excluding a vasopressin | |
| | antagonist). Upon determination of | |
| | eligibility, each subject's serum sodium will | |
| | be reassessed just before tolvaptan | |
| | administration to confirm that it remains | |
| | persistent below this threshold prior to | |
| | intended treatment initiation. | |
| Inclusion/ | Key inclusion criteria: | Key inclusion criteria: |
| Exclusion | • Male and female subjects $\geq 4$ weeks (or | • Male and female subjects ≥ 4 weeks (or |
| Criteria: | ≥ 44 weeks adjusted gestational age for | ≥ 44 weeks adjusted gestational age) to |
| | premature births) to < 18 years old | < 18 years old |
| | Persistent euvolemic or hypervolemic | Persistent euvolemic or hypervolemic |

| Location: | Old | l Text: | Ne | ew Text: |
|---|---|---|---|---|
| | | hyponatremia defined as being | | hyponatremia defined as being |
| | | documented as present for at least 48 | | documented as present for at least 48 |
| | | hours, evidenced by at least 2 serum | | hours, evidenced by at least 2 serum |
| | | sodium assessments < 130 mmol/L | | sodium assessments < 130 mEq/L |
| | | drawn at least 12 hours apart (these | | (mmol/L) drawn at least 12 hours apart |
| | | values can be documented using | | (these values can be documented using |
| | | historical values previously obtained | | historical values previously obtained |
| | | per standard of care); a third (STAT) | | per standard of care); a third (STAT) |
| | | serum sodium assessment < 130 | | serum sodium assessment < 130 mEq/L |
| | | mmol/L, which will serve as the | | (mmol/L), which will serve as the |
| | | baseline value for efficacy endpoints, is | | baseline value for efficacy endpoints, is |
| | | to be obtained within 3 ( $\pm$ 1) hours of | | to be obtained 2-4 hours prior to the |
| | | the first dose of trial medication | 17 | first dose of tolvaptan |
| | Key | y exclusion criteria: | Ke | ey exclusion criteria: |
| | • | Has evidence of hypovolemia or | • | Has evidence of hypovolemia or |
| | | intravascular volume depletion (eg, | | intravascular volume depletion (eg, |
| | | hypotension, clinical evidence of | | hypotension, clinical evidence of |
| | | volume depletion, response to saline | | volume depletion, response to saline |
| | | challenge); if the subject has systolic | | challenge); if the subject has systolic |
| | | blood pressure < 90 mmHg or pulse > | | blood pressure or heart rate outside of<br>the normal range for that age, then |
| | | 120 bpm, then volume status should be | | volume status should be specifically |
| | | specifically clinically assessed to rule | | clinically assessed to rule out volume |
| | | out volume depletion | | depletion |
| | • | Has serum sodium < 120 mmol/L, with or without associated neurologic | | Has serum sodium level < 120 mEq/L |
| | | impairment (ie, symptoms such as | | (mmol/L), with or without associated |
| | | apathy, confusion, or seizures) | | neurologic impairment (ie, symptoms |
| | • | Has a history or current diagnosis of | | such as apathy, confusion, or seizures) |
| | | nephrotic syndrome | • | Has estimated glomerular filtration rate |
| | • | Has transient hyponatremia likely to | _ | $(eGFR) < 30 \text{ mL/min/1.73 m}^2$ |
| | | resolve (eg, head trauma or post- | • | Has had treatment for hyponatremia |
| | | operative state) | | with: |
| | • | Has hyperkalemia defined as serum | • | Uncontrolled diabetes mellitus defined |
| | | potassium above the upper limit of | | as fasting glucose > 300 mg/dL (16.7 |
| | | normal (ULN) for the appropriate | | mEq/L [mmol/L]) |
| | | pediatric age range | • | Screening liver function values |
| | • | Has estimated glomerular filtration rate | | >3×ULN |
| | | $(eGFR) < 30 \text{ mL/min/1.73 m}^2$ | • | Deficient coagulation (eg, cirrhotic at |
| | | calculated by the following equation: | | risk of gastrointestinal [GI] bleed), |
| | | eGFR (mL/min/1.73 m <sup>2</sup> ) = $0.413 \times$ | | including subjects who meet any of the |
| | | height (cm)/serum creatinine (mg/dL) | | following criteria: a major GI bleed |
| | • | Has severe or acute neurological | | within the past 6 months, evidence of |
| | | symptoms requiring other intervention | | active bleeding (eg, epistaxis, |
| | | (eg, hyperemesis, obtundation, seizures) | | petechiae/purpura, hematuria, or |
| | • | Has had treatment for hyponatremia | | hematochezia), platelet count |
| | | with: | | $< 50,000/\mu L$ , or use of medications |
| | • | Has psychogenic polydipsia (subjects | | known to increase bleeding risk |
| | | with other psychiatric illness may be | | |
| | | included per medical monitor approval) | | |
| | • | Has uncontrolled diabetes mellitus | | |
| | | defined as fasting glucose > 300 mg/dL | | |
| | | (16.7 mmol/L) | | |
| | • | Has Screening liver function values > 3 | | |
| | | × ULN | | |

| Location: | Old Text: | New Text: |
|---|---|---|
| | Has deficient coagulation (eg, cirrhotic | |
| | at risk of gastrointestinal [GI] bleed), including subjects who meet any of the | |
| | following criteria: a major GI bleed | |
| | within the past 6 months, evidence of | |
| | active bleeding (eg, epistaxis, | |
| | petechiae/purpura, hematuria, or | |
| | hematochezia), platelet count < | |
| | 50,000/μL, or use of concomitant | |
| | medications known to increase bleeding | |
| | risk | |
| | Has hyponatremia due to the result of | |
| | any medication that can safely be | |
| | withdrawn (eg, thiazide diuretics) | |
| | Has hyponatremia (eg, hyponatremia in the | |
| | setting of adrenal insufficiency, untreated | |
| | hypothyroidism, or hypotonic fluid | |
| | administration) that is most appropriately corrected by alternative therapies | |
| Investigational | Upon the availability of a liquid | Upon the availability of an oral |
| Medicinal | formulation, the protocol will be amended | suspension formulation, the protocol will be |
| Product, Dose, | to reflect additional dosing options. | amended to reflect additional dosing |
| Formulation, | are seemed and are seemed at the seemed at t | options. |
| Mode of | Up-titration of tolvaptan doses will be | 1 |
| Administration | based on serum sodium levels at > 20 hours | Up-titration of tolvaptan doses will be |
| | following initiation of therapy; a change in | based on serum sodium levels at > 20 hours |
| | serum sodium ≤ 4 mmol/L from baseline | following initiation of therapy and at >20 |
| | should warrant up-titration, which is limited | hours following each additional dose; a |
| | to no more than twice the previous dose. | change in serum sodium ≤ 4 mEq/L |
| | | (mmol/L) from baseline should warrant |
| | • Subjects < 2 years of age, weighing < 10 | up-titration, which is limited to no more than twice the previous dose. |
| | kg, or who cannot safely swallow the tablet will be excluded until the | than twice the previous dose. |
| | availability of a liquid formulation. | • Subjects < 2 years of age, weighing < 10 |
| | Dosing information will be available at | kg, or who cannot safely swallow the |
| | that time. | tablet will be excluded until the |
| | | availability of a suspension formulation. |
| | The subjects will continue dosing according | |
| | to a titration scheme targeting a final | The subjects will continue dosing according |
| | sodium concentration between 135 and 140 | to a titration scheme targeting a final serum |
| | mmol/L. Titration will ideally achieve a | sodium concentration between 135 and 140 |
| | change in serum sodium concentration of at least 4 to 8 mmol/L/24 hours but not | mEq/L (mmol/L). Titration will ideally |
| | exceeding 12mmol/L/24 hours. | achieve a change in serum sodium concentration of at least 4 to 8 mEq/L |
| | CACCOMING 12 IIIIIIO II LI 27 IIOUIS. | (mmol/L)/24 hours but not exceeding |
| | At the end of Day 2 (optionally Day 3 | |
| | [Phase A]), subjects with a serum sodium | |
| | increase of $\geq$ 4 mmol/L will be randomized | |
| | to either continue treatment with tolvaptan | |
| | for 2 additional days (Late Withdrawal) or | |
| | to discontinue tolvaptan treatment (Early | |
| | Withdrawal). Early or Late Withdrawal | |
| | assignment will be stratified by age | |
| | , serum | |

| Location: | Old Text: | New Text: |
|---|---|---|
| | sodium response , and | |
| | underlying etiology of hyponatremia. | |
| | Nonresponders will be allowed to be treated | |
| | with tolvaptan for 2 additional days at the | |
| | highest dose or to discontinue tolvaptan and | |
| | be treated per the investigator's preferred | |
| 7D • 1 | standard of care. | DI 1: .: / 1 1 : |
| Trial | Pharmacokinetic/pharmacodynamic: | Pharmacokinetic/pharmacodynamic: |
| Assessments: | Blood sampling for tolvaptan plasma<br>concentrations | Blood sampling for tolvaptan and match clita plasma concentrations |
| | | metabolite plasma concentrations |
| | • Fluid balance | • Fluid intake |
| | Urine output and urine chemistry | • Urine output |
| | Safety: | Urine chemistry Safety: |
| | <ul> <li>Physical examinations, including body</li> </ul> | <ul> <li>Physical examinations, including body</li> </ul> |
| | weight | weight and neurological examinations |
| | <ul> <li>Neurological examinations</li> </ul> | weight and neurological examinations |
| | 1 (Curological examinations | |
| | Screening/Baseline: | |
| | <ul> <li>Clinical laboratory tests (hematology,</li> </ul> | |
| | coagulation, chemistry, urinalysis) | |
| | • Electrocardiogram | |
| | Medical and hyponatremia history | |
| | Thyroid-stimulating hormone and | |
| | cortisol tests | |
| | <ul> <li>Plasma osmolality, fractional excretion</li> </ul> | |
| | of sodium, and fractional excretion of | |
| | urate | |
| | <ul> <li>Alcohol and drug screen</li> </ul> | |
| | <ul> <li>Pregnancy test</li> </ul> | |
| Criteria for | Primary Endpoints: | Primary Efficacy Endpoint |
| <b>Evaluation:</b> | Efficacy: | <ul> <li>For subjects with serum sodium level</li> </ul> |
| | <ul> <li>For subjects with serum sodium</li> </ul> | increases of $\geq$ 4 mEq/L (mmol/L) (ie, |
| | increases of $\geq 4 \text{ mmol/L}$ (ie, | responders), change in serum sodium |
| | responders), change in serum sodium | concentration from Day 2 (or 2a) at the |
| | concentration from randomization (at | end of Treatment Phase A to the end of |
| | the end of Day 2/3 [end of Phase A]) to | Treatment Phase B for Early compared |
| | the end of Day 4/5 (Phase B) for Early | to Late Withdrawal groups. |
| | compared to Late Withdrawal groups | |
| | | Key Secondary Efficacy Endpoint |
| | Secondary Endpoints: | • For all subjects, the key secondary |
| | <ul><li>Efficacy:</li><li>For all subjects, change in serum</li></ul> | endpoint is the change in serum sodium concentration at the end of Day 2 (or |
| | sodium concentration at the end of | 2a) in Treatment Phase A from |
| | Day 2/3 from baseline in Phase A | baseline. |
| | Safety: | bascinic. |
| | <ul> <li>Percentage of subjects with overly rapid</li> </ul> | |
| | increase in serum sodium | Other Secondary Endpoints Safety: |
| | <ul> <li>Percentage of subjects requiring rescue</li> </ul> | <ul> <li>Percentage of subjects with overly rapid</li> </ul> |
| | medication during Phase A and Phase B | increase in serum sodium level |
| | of the trial | moreuse in serum souldin level |
| | • Change in serum sodium from 24 hours | ) |

| Location: | Old Text: | New Text: |
|---|---|---|
| | post-last dose to 14 days post- | • Change in serum sodium level from 24 |
| | randomization | hours post-last dose to 7 days post-last |
| | • Vital signs, blood pressure, clinical | dose |
| | laboratory tests, and body weight | <ul> <li>Percentage of subjects requiring rescue</li> </ul> |
| | Pharmacokinetic: | therapy (other than fluid restriction) |
| | • On Day 1, tolvaptan maximum (peak) | during Treatment Phase A and |
| | plasma concentration ( $C_{max}$ ), time to | Treatment Phase B |
| | maximum (peak) plasma concentration | Percentage of subjects requiring fluid |
| | (t <sub>max</sub> ), and area under the concentration-time curve from time | restriction during Treatment Phase A and Treatment Phase B |
| | zero to 24 hours (AUC <sub>0-24h</sub> ) | Vital signs, blood pressure, clinical |
| | Pharmacodynamic: | laboratory tests, body weight, and |
| | • Fluid intake, urine output, and fluid | neurological examinations |
| | balance (intake – output) every 6 hours | Pharmacokinetic: |
| | on Days 1 and 2 (Phase A) | • On Day 1 in Treatment Phase A, |
| | | tolvaptan maximum (peak) plasma |
| | Exploratory Endpoints: | concentration ( $C_{max}$ ), time to maximum |
| | Efficacy: | (peak) plasma concentration $(t_{max})$ , and |
| | <ul> <li>In nonresponders continuing on</li> </ul> | area under the concentration-time curve |
| | tolvaptan therapy, change in trough | from time zero to 24 hours (AUC <sub>0-24h</sub> ) |
| | serum sodium concentration on Day 6 | Pharmacodynamic: |
| | compared to Day 4 | • Fluid intake, urine output, and fluid |
| | Safety: | balance (intake minus output) every 6 |
| | Neurological examinations Phograph and depositions | hours on Days 1 and 2 in Treatment |
| | Pharmacodynamic: In all subjects 24-hour excretion of | Phase A |
| | • In all subjects, 24-hour excretion of sodium, creatinine, and osmoles on | <ul><li>Exploratory Endpoints</li><li>Efficacy will be assessed in</li></ul> |
| | Days 1 and 2 | nonresponders continuing on tolvaptan |
| | • 24-hour sodium clearance | therapy by change from baseline in |
| | 21 Hour sourchin electronice | serum sodium concentration at the end |
| | | of Treatment Phase B compared to the |
| | | end of Treatment Phase A. |
| | | • In all subjects, 24-hour excretion of |
| | | sodium, creatinine, and osmolality on |
| | | Days 1 and 2 |
| | | • 24-hour sodium clearance on Day 1 |
| | | <ul> <li>Neurocognition test battery</li> </ul> |
| | | Quality of life (QoL) assessments |
| List of | | Abbreviation Definition |
| Abbreviations | | BUN Blood urea nitrogen |
| and Definitions of Terms | | FENa Fractional excretion of sodium |
| or rerins | | FE urate Fractional excretion of |
| | | urate |
| | | HF Heart failure |
| | | SAP Statistical analysis plan |
| 1.2 Clinical | Tolvaptan was approved in adults by the US | Tolvaptan is approved for (a) the treatment |
| Data | FDA, in the European Union, and 9 other | of specific forms of hyponatremia in adults |
| | countries for the treatment of specific forms | by the European Medicines Agency (EMA), |
| | of hyponatremia, and by the Japanese | United States (US) Food and Drug |
| | Ministry of Health, Labour, and Welfare for | |
| | volume overload in heart failure. Tolvaptan | |
| | is currently being developed for the | volume overload in heart failure (HF) by the |
| | treatment of autosomal dominant polycystic | papanese Ministry of Health, Labour, and |

| Location: | Old Text: | New Text: |
|---|---|---|
| | kidney disease (ADPKD), and for the | Welfare. Tolvaptan is currently being |
| | treatment of hepatic edema and | investigated for the treatment of autosomal |
| | carcinomatous edema. As of 31 Mar 2013, | dominant polycystic kidney disease |
| | 83 trials have been completed, 2 trials were | (ADPKD) and the treatment of hepatic |
| | terminated due to slow enrollment, and 12 | edema and carcinomatous edema. As of 31 |
| | trials are ongoing. | Mar 2013, 83 trials have been completed, 2 |
| | | trials were terminated due to slow |
| | | enrollment, and 12 trials were ongoing. |
| | | More information is available in the IB.1 |
| 2.1 Trial | The purpose of this trial various | The purpose of this trial HF, |
| Rationale | etiologies As the primary physiological | hepatocellular disease (including cirrhosis), |
| | effect of tolvaptan | and SIADH/other As the primary |
| | The proposed population size of 100 | pharmacodynamic effect of tolvaptan |
| | subjects should provide 70 responders, | The proposed population size of 100 |
| | | subjects is expected to yield 70 subjects |
| | | who respond to tolvaptan (henceforth |
| | | termed "responders"), |
| 2.2.2 Secondary | The secondary objective is to assess the PK | The key secondary objective is to assess the |
| Objective | of tolvaptan and the effect on fluid balance | PK of tolvaptan and the effect on fluid |
| | in children and adolescent subjects with | balance in children and adolescent subjects |
| | euvolemic or hypervolemic hyponatremia. | with euvolemic or hypervolemic |
| | | hyponatremia. |
| 3 Trial Design | 3.1 Type/Design of Trial | 3.1 Type of Trial |
| | See Figure 3.1-1 for a schematic of the trial | This is an open-label, multicenter, multiple- |
| | design. | dose, randomized withdrawal, |
| | | parallel-group trial of tolvaptan in children |
| | This will be an open-label, multicenter, | and adolescents hospitalized with chronic |
| | multiple-dose, randomized withdrawal, | euvolemic or hypervolemic hyponatremia |
| | parallel-group trial of tolvaptan in children | (serum sodium < 130 mEq/L [mmol/L]) |
| | and adolescent subjects hospitalized with | persisting despite initial standard therapy. |
| | euvolemic or hypervolemic hyponatremia. | A schematic of the trial design is provided |
| | Pediatric and adolescent subjects who are | in Figure 3.1-1. |
| | diagnosed with euvolemic or hypervolemic | |
| | hyponatremia (serum sodium < 130 | This is the first clinical trial of tolvaptan in |
| | mmol/L) that persists despite initial | a pediatric population, and the majority of |
| | standard background therapy (eg, including | subjects may require only short-term |
| | fluid restriction) are eligible to be screened | treatment of hyponatremia, however some |
| | for participation in this trial. Subjects who | subjects may require prolonged treatment |
| | demonstrate prior resistance to vasopressin | and additional follow-up information on |
| | antagonist therapy will be excluded. All | their response to tolvaptan may be desired |
| | potential subjects must also be deemed by | to better understand its long-term safety |
| | the investigator as likely to benefit from a | profile in this pediatric population. Hence, |
| | therapy that raises serum sodium levels. | all subjects (responders and nonresponders) |
| | Since hyponatremia in this patient | who complete this trial will be eligible for |
| | population can often be transient and/or | enrollment into an extension trial |
| | may be secondary to hypovolemic states, | (156-11-294) to continue receiving |
| | potential subjects will be screened for | tolvaptan, as clinically appropriate, until it |
| | hyponatremic histories as well as clinically | is approved and available locally. If |
| | evaluated to rule out such cases. For the | eligible, subjects could continue therapy |
| | purpose of this protocol, persistent | with tolvaptan in that trial after completing |
| | hyponatremia will be defined as serum | the 14 (+2) day Follow-up Visit and |
| | sodium assessments < 130 mmol/L | completion of this trial. (The extension |
| | documented as present for at least 48 hours. | study will also provide long-term post- |
| | | treatment safety follow-up information for a |

| Location: | Old Text: | New Text: |
|---|---|---|
| | Specifically, subjects must have at least | minimum of 6 months.) |
| | 2 serum sodium assessments < 130 mmol/L | |
| | drawn at least 12 hours apart. These values | The trial will be conducted in two stages. |
| | can be documented using historical values | The first stage will be conducted using the |
| | previously obtained as per standard of care. | available tablet formulation of tolvaptan |
| | | whereas the second stage will expand to the |
| | A third (immediate [STAT]) serum sodium | use of a suspension once that formulation |
| | assessment < 130 mmol/L, which will serve | becomes available. |
| | as the baseline value for efficacy endpoints, | |
| | is to be obtained within 3 ( $\pm$ 1) hours of the | |
| | first dose of trial medication. | |
| | As stated above, all subjects will be | |
| | evaluated to determine a minimal 48-hour | |
| | history of hyponatremia to establish | |
| | chronicity. However, it remains the | |
| | responsibility of the investigator to | |
| | determine the etiology of the hyponatremia | |
| | and to assess the volume status for each | |
| | subject using diagnostic tests (eg, fractional | |
| | excretion of sodium [FeNa], fractional | |
| | excretion of urate [Fe urate], urine | |
| | osmolality, plasma osmolality) employed in | |
| | the usual clinical course of care. | |
| | Additionally, the following considerations | |
| | should be noted per underlying etiology: | |
| | <ul> <li>Subjects diagnosed with hyponatremia</li> </ul> | |
| | secondary to SIADH will be evaluated | |
| | specifically to ensure appropriate | |
| | volume status. Hypovolemic states are | |
| | not compatible with tolvaptan | |
| | administration. Plasma and urine | |
| | sodium, potassium, creatinine, and uric | |
| | acid will be assessed in order to | |
| | calculate and evaluate the FeNa and the | |
| | Fe urate prior to dosing to ensure safety | |
| | of tolvaptan administration. | |
| | Subjects diagnosed with hyponatremia CHE are required to have | |
| | secondary to CHF are required to have a definitive diagnosis of CHF by a | |
| | cardiologist and must have any diuretic | |
| | regimen evaluated to ensure it is not | |
| | contraindicated with tolvaptan | |
| | administration. | |
| | <ul> <li>Subjects diagnosed with hyponatremia</li> </ul> | |
| | due to hepatocellular disease must have | |
| | stable disease. | |
| | <ul> <li>All subjects must meet appropriate</li> </ul> | |
| | acute kidney injury (AKI) criteria per | |
| | the exclusion criteria. | |
| | The first dose of trial medication will be | |
| | administered upon successful completion of | |

| Location: | Old Text: | New Text: |
|---|---|---|
| | all screening procedures. | |
| | Subjects will undergo a treatment phase (2 | |
| | to 5 days of tolvaptan) and a follow-up | |
| | phase post-randomization of 14 days. | |
| | Phase A (Treatment Phase): All subjects | |
| | will initially receive tolvaptan once daily for | |
| | the first 2 days. If a subject has not reached the desired sodium target improvement per | |
| | the investigator's judgment (ie, the subject | |
| | is a nonresponder) after Day 2 of tolvaptan | |
| | administration (post 2 doses), a third day of | |
| | treatment is permitted. | |
| | At the end of Day 2 (optionally Day 3), | |
| | subjects who are responders will be | |
| | randomized to either the Early or Late | |
| | Withdrawal group. Responders will be | |
| | defined as those subjects who achieve an | |
| | increase in serum sodium by $\geq 4$ mmol/L. | |
| | Randomized withdrawal assignment will be | |
| | stratified by age | |
| | , by serum sodium response | |
| | , and by underlying | |
| | etiology of hyponatremia. If the subject | |
| | remains a nonresponder to tolvaptan at the | |
| | end of Day 3, the investigator is permitted | |
| | to continue tolvaptan for 2 additional days | |
| | at the highest dose or to discontinue | |
| | tolvaptan and treat the subject per the investigator's preferred standard of care. | |
| | Phase B (Randomization Phase): Subjects | |
| | who are randomized to the Late Withdrawal | |
| | group and nonresponders continuing | |
| | treatment after Day 3 will continue | |
| | treatment with tolvaptan for 2 additional | |
| | days. Subjects who are randomized to the | |
| | Early Withdrawal group and nonresponders | |
| | discontinuing treatment after Day 3 will | |
| | discontinue tolvaptan treatment | |
| | immediately after randomization. | |
| | Nonresponders will be treated per the | |
| | investigator's preferred standard of | |
| | care during Days 3/4 and 4/5 | |
| | (treatment day is dependent upon the | |
| | number of doses that a subject | |
| | receives during Phase A). | |
| | Subjects who are randomized to the Early | |
| | Withdrawal group will initially be observed | |
| | to determine whether additional intervention | |
| | is required to maintain appropriate serum | |
| | sodium levels. Those subjects whose serum | |
| | sodium declines by $\geq 4 \text{ mmol/L}$ or whose | |

| Location: | Old Text: | New Text: |
|-----------|-----------------------------------------------|-----------|
| | overall clinical condition requires further | |
| | treatment to increase serum sodium will be | |
| | treated per the investigator's preferred | |
| | standard of care. Any intervention intended | |
| | to raise serum sodium during the first 48 | |
| | hours of the Early Withdrawal phase | |
| | (including fluid restriction) will be defined | |
| | as rescue therapy; the subject will be | |
| | considered to have reached their clinical | |
| | endpoint, and their data will be censored | |
| | from that time forward. | |
| | All subjects will have sorum sodium | |
| | All subjects will have serum sodium | |
| | measured at 12, 24, 36, and 48 (± 4) hours | |
| | post-randomization. Serum sodium | |
| | assessment time points for nonresponders | |
| | will follow the same schedule, but the | |
| | values will be reported separately from the | |
| | primary efficacy analysis. For analysis | |
| | purposes, these assessments for | |
| | nonresponders will be referred to as "post- | |
| | randomization." | |
| | Phase C (Follow-up Phase): All subjects | |
| | will be monitored and treated as clinically | |
| | warranted per the investigator's preferred | |
| | standard of care for up to 3 additional days | |
| | after the last dose of tolvaptan (note: the | |
| | Early Withdrawal group should be | |
| | monitored for the first 48 hours post-last | |
| | dose). All subjects will have an additional | |
| | serum sodium measurement at | |
| | 72 ( $\pm$ 4) hours post-randomization and | |
| | $7 (\pm 1)$ days post-randomization. A final | |
| | safety follow-up telephone contact/visit will | |
| | be performed 14 (+ 2) days | |
| | post-randomization. | |
| | Pharmacokinetic samples will be obtained | |
| | on Day 1 (Phase A) and, for tolvaptan- | |
| | treated subjects, at 24 and 48 hours post- | |
| | randomization in Phase B. The PK profiles | |
| | will be evaluated on an ongoing basis to | |
| | determine the variability between subjects. | |
| | Based on the findings, PK sampling will | |
| | continue for as long as necessary to | |
| | establish suitable estimates of clearance | |
| | with a 90% confidence interval (CI) similar | |
| | to that observed in the adult populations. | |
| | Once these estimates are achieved, sampling | |
| | will be discontinued in subsequent subjects | |
| | in order to minimize blood draws in this | |
| | population. | |

| Location: | Old Text: | New Text: |
|-----------|-------------------------------------------------|-----------|
| | Subjects will be required to be in the | |
| | hospital during initiation or up-titration of | |
| | the administration of tolvaptan. If a subject | |
| | is in the withdrawal phase or is not expected | |
| | to receive a higher dose of tolvaptan, | |
| | continued administration can be done | |
| | outside of the hospital setting. Follow-up | |
| | for all subjects may occur in the hospital if | |
| | the subject has not been discharged or the | |
| | subject may return for outpatient visits if the | |
| | subject has been discharged from the | |
| | hospital. | |
| | Subjects who do not improve on tolvaptan | |
| | may receive rescue therapy per the | |
| | investigator's judgment (see Section 3.2.2). | |
| | These subjects will be withdrawn from trial | |
| | treatment and will continue to Phase C to be | |
| | followed as per protocol. | |
| | While understanding that the majority of | |
| | hyponatremia in this patient population may | |
| | only require short-term treatment, it is | |
| | recognized that some subjects may require | |
| | prolonged treatment. Hence, all subjects | |
| | (responders and nonresponders) who | |
| | complete this trial may be eligible to be | |
| | enrolled for an additional (planned) open- | |
| | label use trial (156-11-294) to enable | |
| | continued use of tolvaptan or to be | |
| | clinically followed. If deemed eligible, | |
| | these subjects could continue therapy with | |
| | tolvaptan after the 14-day Follow-up Visit | |
| | and completing this trial. | |

#### **Old Text:**

#### 3.1: Type of Trial



**Figure 3.1-1 Trial Design Schematic**
# **New Text:**

Figure 3.1: Type of Trial



**Figure 3.1-1 Trial Design Schematic** 

#### Location: Old Text: New Text: 3.1.1 Trial Phases Subjects must be $\geq 2$ years of age and Screening should be performed on Days -2 weigh $\geq 10$ kg until development of a liquid formulation is complete. and -1 to confirm eligibility, followed by the 3 trial phases described in Section 3.7.1. 3.2 Treatments 3.1.1.1 Treatment Phase A Tolvaptan will be administered once daily All subjects will initially receive tolvaptan orally, preferably in the morning hours, once daily on Days 1 and 2. If a subject's with a dose proportional amount of water. serum sodium level has not increased by at The acceptability and palatability of least 4 mEg/L (mmol/L) by Day 2, an tolvaptan tablets will be recorded on the additional day of treatment is required and case report form (CRF). Doses of $\geq 15$ mg is referred to as Day 2a. If subjects achieve tolvaptan will be given with 240 mL of an increase in serum sodium concentration water... of $\geq 4$ mEq/L (mmol/L) on Day 2 (or 2a) ...Up-titration of tolvaptan doses can occur they will be defined as responders. If once daily and will be based on serum subjects do not achieve an increase in sodium levels at > 20 hours following serum sodium concentration of $\geq 4 \text{ mEq/L}$ initiation of therapy and each subsequent (mmol/L) on Day 2 (or 2a) they will be dose; up-titration may not occur within 20 defined as nonresponders. hours of the previous dose. A change in serum sodium ≤ 4 mmol/L from baseline 3.1.1.2 Treatment Phase B should warrant up-titration, which is On Day 3 responders will be randomized limited to no more than twice the previous (Section 3.1.1.2.1) to either the Early dose. Withdrawal group or the Late Withdrawal Subjects < 2 years of age or weighing < group. Nonresponders will not be 10 kg are excluded until a liquid randomized. formulation is available. Tolvaptan For nonresponders from Treatment Phase metabolism is primarily mediated by A, the investigator will determine if the CYP3A4 and intestinal and hepatic subject is to either: concentrations of this enzyme increase Continue treatment with study drug or following birth. Developmental information from PK models of Prescribe treatment per local standard of care for Days 3 and 4. midazolam and cisapride, other CYP3A4 substrates, in neonates and 3.1.1.2.1 Randomization infants will be used to provide dosing Responders will be randomized to either: recommendations for the liquid formulation when available. Late Withdrawal group - subjects continue tolyaptan treatment on Days 3 Subjects $\geq 2$ years of age and weighing $\geq$ 10 to $\leq$ 20 kg will be given a 3.75 -mg tablet on Day 1 with possible • Early Withdrawal group - subjects do up-titration to 7.5- and 15 -mg tablet not receive additional tolvaptan treatment on Days 3 and 4. doses. Randomization will be stratified by age (< Subjects weighing 20 to 50 kg. inclusive, will be given a 7.5 -mg tablet ), serum on Day 1 with possible up-titration to sodium response , and underlying hyponatremia 15- and 30 -mg tablet doses. etiology Subjects weighing > 50 kg will be given a 15 -mg tablet on Day 1 with possible up-titration to 30- and 60 -mg tablet doses. Subjects randomized to the Early Withdrawal group will be observed to determine whether additional intervention Subjects who cannot take an oral tablet are is required to maintain appropriate serum currently excluded due to their inability to safely swallow the spray-dried tablet. sodium levels. Subjects whose serum

Subjects weighing < 10 kg are also

sodium declines by  $\geq 4$  mEq/L (mmol/L) or

# Location: O

### Old Text:

excluded as that weight has not been studied in previous PK trials and, therefore, the dose of tolvaptan being delivered is not confirmed. To support the enrollment of these subjects, an age and weight appropriate suspension formulation is being developed. Once available, the protocol will be amended to include the formulation. Table 3.2-1 presents starting doses of tolvaptan (15, 7.5, or 3.75 mg) when adjusted for body weight.

Consequently, the maximal starting dose for subjects weighing > 50 kg is slightly less than 0.30 mg/kg; starting doses for subjects weighing 20 to 50 kg, inclusive, range from 0.38 to 0.15 mg/kg; starting doses for subjects weighing  $\geq 10 \text{ to} < 20 \text{ kg}$  range from 0.375 mg/kg to slightly greater than 0.19 mg/kg. Therefore, the maximal starting doses planned for this pediatric trial are in the range previously used in adult hyponatremic subjects.

For subjects weighing  $\geq 20$  kg and taking moderate inhibitors of CYP3A4, a half dose will be used (3.75 or 7.5 mg, by weight).... The subjects will continue dosing according to a titration scheme (Section 3.2.1) targeting a final sodium concentration between 135 and 140 mmol/L. Titration guidelines are designed to ideally achieve a change in serum sodium concentration of at least 4 to 8 mmol/L/24 hours but not exceeding 12 mmol/L/24 hours.

At the end of Day 2 (optionally Day 3 [Phase A]), subjects with a serum sodium increase of  $\geq 4$  mmol/L will be randomized to either continue treatment with tolvaptan for 2 additional days (Late Withdrawal) or to discontinue tolvaptan treatment (Early Withdrawal). Early or Late Withdrawal assignment will be stratified by the ages of

, serum

sodium response

underlying etiology of hyponatremia. Subjects with serum sodium response of < 4 mmol/L may continue on tolvaptan therapy for 2 additional days at their highest dose or may be withdrawn from tolvaptan to be treated per the investigator's preferred standard of care.

### New Text:

whose overall clinical condition requires further treatment to raise serum sodium levels should be treated per local standard of care. Any intervention intended to raise serum sodium concentration during the first 48 hours of the Early Withdrawal phase (including fluid restriction) will be defined as rescue therapy. Subjects receiving rescue therapy will be considered to have reached their clinical endpoint, and their data will be censored from that time forward.

### 3.1.1.3 Follow-up Phase C

All subjects will have an additional serum sodium measurement at 72 ( $\pm$  4) hours post-last dose and 7 ( $\pm$  1) days post-last dose. A final safety follow-up telephone contact/visit will be performed 14 ( $\pm$  2) days post-last dose.

### 3.2.1 Tablet Formulation

Tolvaptan tablets will be administered orally once daily, preferably in the morning hours, with a dose proportional amount of water. Doses of ≥ 15 mg tolvaptan will be given with 240 mL of water...

The maximum starting doses, by weight, for subjects are shown in Table 2.1.1-1 and are within the range previously used in trials involving adult hyponatremic subjects.

The palatability of tolvaptan tablets will be assessed.

### 3.2.2 Suspension Formulation

Additional information on the proposed suspension formulation of tolvaptan (currently in development) will be added to the protocol in an amendment when available. Until that time, subjects < 2 years of age or weighing < 10 kg and those unable to swallow tablets, are excluded from the trial.

### **3.2.3 Dosing Guidelines**

...Titration of tolvaptan doses can occur once daily and will be based on serum sodium levels assessed at > 20 hours following initiation of therapy and each subsequent dose; titration may not occur within 20 hours of the previous dose. Up-titration is limited to no more than twice the previous dose.

#### New Text: Location: Old Text: 3.2.1 Titration Guidelines Subjects < 2 years of age or weighing < The titration scheme is presented in Figure 10 kg are excluded until an oral suspension formulation is available. Subjects $\geq 2$ years of age and weighing If serum sodium increases > 4 to < 8 $\geq$ 10 to $\leq$ 20 kg will receive a 3.75 mg mmol/L/24 hours, then the dose of tablet on Day 1 with possible tolvaptan should remain the same. If up-titration to 7.5 mg and 15 mg tablet serum sodium increases ≥ 8 mmol/L/24 doses. hours or reaches a concentration $\geq 140$ Subjects weighing 20 to 50 kg, mmol/L, then the dose of tolvaptan inclusive, will receive a 7.5 mg tablet should be held and the medical monitor on Day 1 with possible up-titration to should be called. If serum sodium 15 mg and 30 mg tablet doses. changes by $\leq 4 \text{mmol/L/24}$ hours and the Subjects weighing > 50 kg will receive subject is still below the therapeutic a 15 mg tablet on Day 1 with possible target for serum sodium (135mmol/L), up-titration to 30 mg and 60 mg tablet then the tolvaptan dose may be titrated up to the next scheduled dose For subjects weighing $\geq 20 \text{ kg}$ and taking appropriate to the subject's body weight. moderate inhibitors of CYP3A4, one half of If at any point serum sodium or the standard dose will be used (3.75 or 7.5 symptoms worsen or fail to improve and mg, by weight).... definitive therapy (eg, isotonic or Following their initial tolvaptan dose in the hypertonic saline) is required, the trial subjects will continue dosing subject will be withdrawn from the trial according to the titration scheme (see to receive "rescue therapy." These Section 3.2.4), targeting a final serum subjects will be withdrawn from trial sodium concentration between 135 and 140 treatment and will continue to Phase C mEg/L (mmol/L). Titration guidelines are to be followed as per protocol. The designed to achieve a change in serum medical monitor should be contacted at sodium concentration of at least 4 to any point if questions arise regarding 8 mEq/L (mmol/L)/24 hours but not titration. The rationale for any up-or exceeding down-titration of tolvaptan must be documented. Any initiation or titration 3.2.4 Titration Guidelines and Rescue of tolvaptan must occur in a hospital Therapy setting. Initiation and titration of tolvaptan must occur in a hospital setting. Up titration can 3.2.1.1 Rescue Therapy only take place on Treatment Day 2 (or 2a). Subjects with worsening hyponatremia Down titration can occur at any point in the symptoms during the trial may receive trial but should be discussed with the rescue therapy. ....commercial vaptans, or medical monitor. Titration (up or down) any treatment intended to raise the level of may not occur within 20 hours of the serum sodium. previous dose. Up-titration is limited to no Subjects who are randomized to the Early more than twice the previous dose. Withdrawal group will initially be observed The medical monitor should be contacted at to determine whether additional any point if questions arise regarding intervention is required to maintain titration or initiation of rescue therapy. The appropriate serum sodium levels. Those rationale for any up- or down-titration of subjects whose serum sodium declines by ≥ tolvaptan must be documented. The 4 mmol/L or whose overall clinical evaluation of serum sodium levels. condition requires further treatment to management of tolvaptan titration and increase serum sodium will be treated per rescue therapy is described in Figure 3.2.4the investigator's preferred standard of care. Any intervention intended to raise

the Early Withdrawal phase (including fluid | Tolvaptan dose titration (after the initial

3.2.4.1 Titration

serum sodium during the first 48 hours of

| Location: | Old Text: | New Text: |
|---|---|---|
| | restriction) will be defined as rescue | dose) should be based on changes in serum |
| | therapy. The subject will be considered to | sodium levels as follows: |
| | have reached their clinical endpoint, and<br>their data will be censored from that time<br>forward. | • If the serum sodium level increases by ≤ 4 mEq/L (mmol/L)/24 hours and the subject is still below the therapeutic |
| | Subjects receiving rescue therapy will be considered treatment failures. A subject | target for serum sodium level (135 mEq/L [mmol/L]), then the tolvaptan dose may be titrated up to the |
| | requiring rescue therapy at any time after enrollment will be discontinued from the trial treatment and will continue to Phase C | next scheduled dose appropriate for the subject's body weight. • If the serum sodium level increases > 4 |
| | to be followed as per protocol. | to ≤ 8 mEq/L (mmol/L)/24 hours in response to tolvaptan treatment and the serum sodium is ≤ 140 mEq/L (mmol/L), then the dose of tolvaptan should remain the same for the subsequent day. |
| | | If the serum sodium level increases > 8 mEq/L (mmol/L)/24 hours or reaches a concentration of > 140 mEq/L (mmol/L), then the next dose of tolvaptan should not be given and the medical monitor should be contacted to |
| | | consider options (ie, down-titration, tolvaptan interruption, concomitant medication adjustment, fluid supplementation and/or withdrawal). |
| | | If serum sodium level increases by period following dosing, or, at any time after dosing, the serum sodium level is 145 mEq/L (mmol/L), the next dose of tolvaptan should not be given and the medical monitor should be contacted immediately to consider options. |
| | | 3.2.4.2 Rescue Therapy Subjects with worsening hyponatremia symptoms or whose serum sodium level declines may receive rescue therapycommercially available vaptans, or any treatment intended to raise the level of serum sodium at any time during the trial. If at any point during the trial serum sodium levels or hyponatremia symptoms worsen or fail to improve adequately and definitive therapy (eg, isotonic or |
| | | hypertonic saline) is required, the subject will be withdrawn from trial treatment to receive rescue therapy. These subjects will continue to Follow-up Phase C for collection of safety information. Additional guidelines for rescue therapy concerning hyponatremia symptoms and |

| Location: | Old Text: | New Text: |
|---|---|---|
| | | decreasing serum sodium level: |
| | | <ul> <li>If a subject has worsening symptoms and/or has a serum sodium level at or below the baseline value, repeat serum sodium [STAT] to confirm level, and begin rescue therapy.</li> <li>If a subject is asymptomatic and serum sodium has decreased by ≥ 4 mEq/L (mmol/L), but is still above the baseline value, consider need for rescue therapy.</li> <li>If a subject is asymptomatic and serum sodium has decreased by ≤ 3 mEq/L (mmol/L), but is still above the baseline value, no action is required.</li> </ul> |
| | | Subjects who are randomized to the Early Withdrawal group will initially be observed to determine whether additional intervention is required to maintain appropriate serum sodium levels. Those subjects whose serum sodium declines by ≥ 4 mEq/L (mmol/L) or whose overall clinical condition requires further treatment to increase serum sodium will be treated per standard of care. Any intervention intended to raise serum sodium level during the first 48 hours in the responder Early Withdrawal group (including fluid restriction) will be defined as rescue therapy. These subjects will be considered to have reached their clinical endpoint, and their data will be censored from that time forward. |
| | | Subjects randomized to the Late Withdrawal group who receive rescue therapy will be considered treatment failures. A subject requiring rescue therapy at any time after starting tolvaptan will be discontinued from trial treatment and will proceed to Follow-up Phase C. |
| | | 3.2.4.3 Fluid Restriction Considerations In subjects with chronic hyponatremia, fluid restriction coadministered with initiation of treatment with a vaptan has the potential to accentuate the rate of sodium correction and to cause overly rapid correction or over correction of hyponatremia. Therefore, during treatment, subjects must have access to water and maintain fluid intake levels per institutional guidelines. Fluid restriction at any time |

| <b>Location:</b> | Old Text: | New Text: |
|---|---|---|
| | | during the trial including during the first 48 |
| | | hours after discontinuation of tolvaptan will |
| | | be considered rescue therapy. |

# **Old Text: 3.7 Trial Procedures**



**Figure 3.2.1-1 Titration Scheme** 



### **New Text: 3.7 Trial Procedures**

Figure 3.2.4-1 Titration and Rescue Therapy Scheme

| Locatio | Old Text: | New Text: |
|---|---|---|
| n: | | |
| 3.3 | This trial will include up to | This trial will include up to 100 male and female subjects aged |
| Trial | 100 male and female | $\geq$ 4 weeks (or $\geq$ 44 weeks adjusted gestational age) to $<$ 18 years |
| Populati | subjects aged ≥ 4 weeks (or | who have been diagnosed with euvolemic or hypervolemic |
| on | ≥ 44 weeks adjusted gestational age for premature births) to < 18 years, who have been diagnosed with euvolemic or hypervolemic hyponatremia (< 130 mmol/L) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin | hyponatremia (< 130 mEq/L [mmol/L]) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). Age groups will be enrolled such that 50% of these subjects will be < 10 years old and at least 25% of subjects < 6 years old. Subjects who are defined as responders will be further stratified by the magnitude of serum sodium response to tolvaptan (≤ 7 and > 7 mEq/L [mmol/L]), and underlying etiology of hyponatremia. Subjects with euvolemic or hypervolemic hyponatremia eligible to be screened for participation in this trial include, but are not |
| | antagonist). It is expected | limited to, those diagnosed and admitted to a hospital for |
| | that 70 subjects will have a | treatment of HF, hepatocellular disease (including cirrhosis), or |
| | serum sodium increase of ≥ | SIADH/other |
| | 4 mmol/L (ie, responders). | |

| Locatio<br>n: | Old Text: | New Text: |
|---|---|---|
| 11. | The trial will be conducted | All potential subjects must have chronic (≥ 48 hours) dilutional |
| | at up to 50 centers globally. | hyponatremia (euvolemic or hypervolemic) associated with HF, |
| | Subjects with euvolemic or hypervolemic hyponatremia | hepatocellular disease (including cirrhosis), or SIADH/other and |
| | eligible to be screened for | be deemed by the investigator as likely to benefit from a therapy |
| | participation in this trial | that raises serum sodium levels. The etiology of hyponatremia (presumed cause) must be documented and evaluated per |
| | include, but are not limited | Section 3.3.1. Those subjects who have acute or transient |
| | to, those diagnosed and | hyponatremia, have overt symptoms of hyponatremia requiring |
| | admitted to a hospital for | immediate intervention, or who are at increased risk for |
| | treatment of heart failure, | developing hyponatremic encephalopathy or osmotic |
| | hepatocellular disease | demyelination are excluded from this trial. |
| | (including cirrhosis), or | |
| | SIADH | Since hyponatremia in this patient population can often be |
| | Hospitalized hyponatremic | transient and/or may be secondary to hypovolemic states, |
| | encephalopathy is seen in | potential subjects will be screened for hyponatremic histories as |
| | association with SIADH or | well as clinically evaluated to rule out such cases. For the |
| | in the post-operative period. | purpose of this protocol, persistent hyponatremia will be defined |
| | Hyponatremic | as serum sodium level < 130 mEq/L (mmol/L) documented as |
| | encephalopathy is a medical | present for at least 48 hours. Specifically, subjects must have at |
| | emergency that requires | least 2 serum sodium assessments < 130 mEq/L (mmol/L) drawn |
| | immediate intervention;<br>thus, subjects with known | at least 12 hours apart. These values can be documented using |
| | risk factors for developing | historical values previously obtained as per standard of care. A third (STAT) serum sodium assessment < 130 mEq/L (mmol/L), |
| | hyponatremic | which will serve as the baseline value for efficacy endpoints, is to |
| | encephalopathy will be | be obtained within 2-4 hours prior to the first dose of trial |
| | excluded from this trial (ie, | medication. |
| | hypoxia, infection, brain | |
| | injury, neurosurgery, seizure | If a subject's serum sodium level during the screening period is ≥ |
| | disorders, cerebritis, | 130 mEq/L (mmol/L), the subject will be determined to be a |
| | encephalopathy, central | screen failure. Subjects deemed screen failures may be |
| | nervous system disorders | rescreened, as appropriate. Subjects who receive a randomization |
| | such as cytotoxic and | number may not be rescreened regardless of whether they receive |
| | vasogenic cerebral edema, | trial medication |
| | space-occupying brain | |
| | lesion, or elevated AVP levels). <sup>22</sup> | Hospitalized hyponatremic encephalopathy is seen in association |
| | levels). | with SIADH or in the immediate post-operative period. |
| | Age groups will be stratified | Hyponatremic encephalopathy is a medical emergency that requires immediate intervention; thus, subjects with known risk |
| | such that half (35) of these | factors for developing hyponatremic encephalopathy will be |
| | subjects will be age < | excluded from this trial (ie, hypoxia, infection, brain injury, |
| | 10 years with at least 25% | neurosurgery, active seizure disorders, cerebritis, encephalopathy, |
| | (17) of subjects < 6 years | central nervous system disorders such as cytotoxic and vasogenic |
| | old. Subjects who are | cerebral edema, space-occupying brain lesion, or elevated AVP |
| | defined as responders will be | levels). <sup>22</sup> |
| | further stratified by the | |
| | magnitude of serum sodium | 3.3.1.1 General Guidelines |
| | response to tolvaptan | Investigators should assess subjects' appropriateness to receive |
| | $(\le 7 \text{ and} > 7 \text{ mmol/L})$ and | tolvaptan. Investigators should ultimately use their medical |
| | underlying etiology of | judgment to make the final determination. It remains the |
| | hyponatremia. | responsibility of the investigator to determine the etiology of |
| | All subjects will be initially identified based on serum | hyponatremia and to assess the volume status for each subject |
| | sodium concentrations that | using diagnostic tests (eg, fractional excretion of sodium [FENa], fractional excretion of urate [FE urate], urine osmolality, serum |
| | persist at levels | osmolality) employed in the usual clinical course of care. |

| Locatio<br>n: | Old Text: | | New Text: | |
|---|---|---|---|---|
| | < 130 mmol/L despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). Upon determination of eligibility, each subject's serum sodium will be reassessed just before tolvaptan administration to confirm it remains persistent below this threshold prior to intended treatment initiation. If any result, during the Screening period is ≥ 130 mmol/L, the subject will be determined a screen failure. Subjects deemed screen failures may be rescreened, as appropriate. Subjects who receive a randomization number may not be rescreened regardless of whether they receive trial medication or complete the trial. | | Subjects will be a status. I administ creatining calculate ensures a seriology For hype cirrhosise etiology For hype doc 7) Control of the stop half | sific Guidelines by Etiology so diagnosed with hyponatremia secondary to SIADH evaluated specifically to ensure appropriate volume Hypovolemic states are not compatible with tolvaptan tration. Plasma and urine sodium, potassium, ne, and uric acid should be assessed in order to e and evaluate FENa and FE urate prior to dosing to eafety of tolvaptan administration. conatremia due to hepatocellular disease (including s), in addition to the above guidelines, the underlying of hepatocellular disease must be documented. conatremia due to HF: definitive diagnosis of HF by a cardiologist must be enumented. Op diuretic use should be assessed and minimized ere possible. Steady doses of diuretics are acceptable. azide diuretics must be stopped before tolvaptan ministration; the time that these medications must be oped prior to the first tolvaptan dose depends on the f-life of the diuretic. monitor should be contacted if there are questions. less listed in Table 3.3.1-1 are to help guide the genent of the investigator. |
| | 3.3.1 Tolvaptan | | | -1 Screening Algorithms by |
| | Administration<br>Hyponatremia I | | | mia Etiology |
| | Investigators sho<br>subjects' appropring receive tolyaptan<br>investigator shou<br>ultimately use the<br>judgment to mak<br>determination. T | uld assess<br>riateness to<br>. Each<br>ld<br>eir medical<br>e the final<br>'he | All etiologies | Instruction Two documented serum sodium assessments of < 130 mEq/L (mmol/L) at least 12 hours apart One serum sodium assessment of < 130 mEq/L (mmol/L) within 2-4 hours prior to |
| | guidelines listed 3.3.1-1 are to hel medical judgmen investigator. Table 3.3.1-1 So | p guide the<br>it of each | | tolvaptan administration Screen subjects for AKI criteria per exclusion criteria Collect labs <sup>a</sup> Calculate serum osmolality, |
| | Algorithms by<br>Hyponatremia I<br>SIADH/ CHF | Hepatoc | HF | FENa, and FE urate at pretreatment baseline only Cardiologist documented |
| | Two Two<br>serum serum<br>sodium sodium | ellular Disease Two serum sodium | ITIF | diagnosis of HF Discontinue or stabilize diuretic use prior to tolvaptan administration |

| Locatio<br>n: | Old Text: | | | New Text: |
|---|---|---|---|---|
| | 12 hours | | at least<br>12 hours | <sup>a</sup> Refer to Table 3.7.4.2-1 for complete lists of laboratory assessments. |
| | apart | hours<br>apart | apart | |
| | One | One | One | |
| | serum | serum | serum | |
| | 11 | sodium | sodium | |
| | assessm | | assessme | |
| | ent 3 (± | | nt 3 (± 1) | |
| | 1) hours | | hours | |
| | before | before | before | |
| | _ | _ | tolvaptan | |
| | n | n | administ | |
| | administ | | ration of | |
| | ration of | | < 130 | |
| | < 130 | of < 130 | mmol/L | |
| | mmol/L | | | |
| | Screen | Screen | Screen | |
| | subjects | | subjects | |
| | per AKI | | per AKI | |
| | criteria | criteria | criteria | |
| | per | per | per | |
| | exclusio | | exclusio | |
| | n | n | n criteria | |
| | | criteria | C-114 | |
| | Collect | Collect | Collect | |
| | | labs <sup>a</sup> | labs <sup>a</sup> | |
| | Calculat | | Calculat | |
| | e plasma | | e plasma | |
| | osmolali | osmolal | osmolalit | |
| | ty,<br>FENa, | ity, | y, FENa,<br>and FE | |
| | | FENa, | urate at | |
| | 1 1 | and FE | pretreat | |
| | pretreat | urate at | ment | |
| | ment | pretreat | baseline | |
| | baseline | | only | |
| | only | baseline | ) | |
| | | only | | |
| | | Cardiol | | |
| | | ogist | | |
| | | docume | | |
| | | nted | | |
| | | diagnosi | | |
| | | s of | | |
| | | Disconti | | |
| | | nue or | | |
| | | stabilize | | |
| | | diuretic | | |
| | | use | | |
| | | prior to | | |
| | | tolvapta | | |

| Locatio n: | Old Text: | New Text: |
|------------|-----------------------------------------------------|-----------|
| 11. | n | |
| | adminis | |
| | tration | |
| | <sup>a</sup> Refer to Table 3.7-1 and | |
| | Table 3.7.4.2-1 for a | |
| | complete list of | |
| | laboratory | |
| | assessments. | |
| | 3.3.1.1 Hyponatremia due | |
| | to Syndrome of | |
| | Inappropriate Secretion of | |
| | Antidiuretic Hormone | |
| | Evidence of low serum | |
| | sodium should be | |
| | demonstrated for at least 48 | |
| | hours prior to scheduled | |
| | tolvaptan administration. | |
| | Two serum sodium | |
| | assessments of < 130 | |
| | mmol/L should be collected | |
| | at least 12 hours apart. One | |
| | serum sodium assessment of | |
| | < 130 mmol/L should be | |
| | collected 3 ( $\pm$ 1) hours | |
| | before the initial tolvaptan | |
| | administration. If any result, | |
| | during the Screening period | |
| | is $\geq 130 \text{ mmol/L}$ , the subject | |
| | will be determined a screen | |
| | failure. Subjects determined | |
| | screen failures may be | |
| | rescreened, as appropriate. | |
| | Subjects who receive a | |
| | randomization number may | |
| | not be rescreened regardless | |
| | of whether they receive trial | |
| | medication or complete the | |
| | trial. At Screening/Baseline, | |
| | urine chemistry should be | |
| | assessed and the plasma | |
| | osmolality, FENa, and FE urate should be calculated | |
| | for all subjects prior to the | |
| | first dose of tolvaptan. | |
| | Please see Table 3.7-1 for a | |
| | full schedule of assessments | |
| | and timing. | |
| | Subjects must be screened | |
| | per the AKI criteria detailed | |
| | in the exclusion criteria | |
| | (Section 3.4.3). | |

| Locatio<br>n: | Old Text: | New Text: |
|---|---|---|
| | Hyponatremia due to | |
| | Congestive Heart | |
| | Failure | |
| | Evidence of low serum | |
| | sodium should be | |
| | demonstrated for at least 48 | |
| | hours prior to scheduled | |
| | tolvaptan administration. | |
| | Two serum sodium | |
| | assessments of < 130 | |
| | mmol/L should be collected | |
| | at least 12 hours apart. One | |
| | serum sodium assessment of | |
| | < 130 mmol/L should be | |
| | collected 3 (± 1) hours | |
| | before the initial tolvaptan | |
| | administration. If any result, | |
| | during the Screening period | |
| | is $\geq 130 \text{ mmol/L}$ , the subject | |
| | will be determined a screen | |
| | failure. Subjects determined screen failures may be | |
| | rescreened, as appropriate. | |
| | Subjects who receive a | |
| | randomization number may | |
| | not be rescreened regardless | |
| | of whether they receive trial | |
| | medication or complete the | |
| | trial. At Screening/Baseline, | |
| | urine chemistry should be | |
| | assessed and the plasma | |
| | osmolality, FENa, and FE | |
| | urate should be calculated | |
| | for all subjects prior to the | |
| | first dose of tolvaptan. | |
| | Please see Table 3.7-1 for a | |
| | full schedule of assessments | |
| | and timing. | |
| | 5) Loop diuretic use should | |
| | be assessed and | |
| | minimized where | |
| | possible. Steady doses of diuretics are | |
| | acceptable. Thiazide | |
| | diuretics must be | |
| | stopped before tolvaptan | |
| | administration; the time | |
| | that these medications | |
| | must be stopped prior to | |
| | the first tolvaptan dose | |
| | depends on the half-life | |
| | of the diuretic. The | |
| | medical monitor should | |

| Locatio<br>n: | Old Text: | New Text: |
|---|---|---|
| - | be contacted if there are | |
| | questions. | |
| | A definitive diagnosis of | |
| | CHF by a cardiologist must | |
| | be documented. | |
| | Subjects must be screened | |
| | per the AKI criteria detailed | |
| | in the exclusion criteria (Section 3.4.3). | |
| | 3.3.1.2 Hyponatremia due | |
| | to Hepatocellular Disease | |
| | Evidence of low serum | |
| | sodium should be | |
| | demonstrated for at least 48 | |
| | hours prior to scheduled | |
| | tolvaptan administration. | |
| | Two serum sodium | |
| | assessments of < 130 | |
| | mmol/L should be collected | |
| | at least 12 hours apart. One | |
| | serum sodium assessment of < 130 mmol/L should be | |
| | collected 3 (± 1) hours | |
| | before the initial tolvaptan | |
| | administration. If any result, | |
| | during the Screening period | |
| | is $\geq 130 \text{ mmol/L}$ , the subject | |
| | will be determined a screen | |
| | failure. Subjects determined | |
| | screen failures may be | |
| | rescreened, as appropriate. | |
| | Subjects who receive a | |
| | randomization number may | |
| | not be rescreened regardless | |
| | of whether they receive trial medication or complete the | |
| | trial. At Screening/Baseline, | |
| | urine chemistry should be | |
| | assessed and the plasma | |
| | osmolality, FENa, and FE | |
| | urate should be calculated | |
| | for all subjects prior to the | |
| | first dose of tolvaptan. | |
| | Please see Table 3.7-1 for a | |
| | full schedule of assessments | |
| | and timing. | |
| | Subjects must be screened | |
| | per the AKI criteria detailed | |
| | in the exclusion criteria | |
| | (Section 3.4.3). | |
| | The underlying etiology of | |
| | hepatocellular disease must | |

| Locatio | Old Text: | New Text: |
|---|---|---|
| n: | be documented. | |
| 3.4 | be documented. | Eligible subjects must satisfy all informed consent requirements, |
| Eligibili | | as well as meet all inclusion and exclusion criteria. Subjects who |
| ty | | do not meet all of these requirements are to be defined as screen |
| Criteria | | failures and may rescreen, if eligible, at a later date. |
| 3.4.2 | Eligible subjects must satisfy all informed consent | |
| Inclusio<br>n | requirements, as well as | |
| Criteria | meet all inclusion criteria | |
| Crittia | and none of the exclusion | |
| | criteria. It is required to | |
| | have documentation of | |
| | chronic hyponatremia, | |
| | defined by serum sodium < | |
| | 130 mmol/L persisting for | |
| | ≥ 48 hours duration and | |
| | assessed at least 12 hours | |
| | apart. Finally, there must be a final serum sodium | |
| | assessed STAT prior to the | |
| | initial dose of tolvaptan. | |
| | This final serum sodium | |
| | screening assessment must | |
| | be verified to be < 130 | |
| | mmol/L prior to the initial | |
| | dose. Subjects who do not | |
| | meet all of these | |
| | requirements are to be defined as screen failures | |
| | and may rescreen if eligible | |
| | at a later date | |
| 3.5 | 3.5.1 Primary Outcome | 3.5.1 Primary Efficacy Outcome Variable |
| Outcom | Variables | For subjects with serum sodium level increases of ≥ 4 mEq/L |
| e | 3.5.2 Efficacy Variables | (mmol/L) (ie, responders), change in serum sodium concentration |
| Variabl | For subjects with serum | from Day 2 (or 2a) at the end of Treatment Phase A to the end of |
| es | sodium increases of | Treatment Phase B for Early compared to Late Withdrawal |
| | ≥ 4mmol/L (ie, responders), | groups. |
| | the primary endpoint is the change in serum sodium | 3.5.2 Key Secondary Efficacy Outcome Variable |
| | concentration from | For all subjects, the key secondary endpoint is the change in |
| | randomization (at the end of | serum sodium concentration at the end of Day 2 (or 2a) in |
| | Day 2/3 [end of Phase A]) to | Treatment Phase A from baseline. |
| | the end of Day 4/5 (Phase B) | |
| | for Early compared to Late | 3.5.3.1 Safety Variables |
| | Withdrawal groups. | Percentage of subjects with overly rapid increase in serum |
| | 3.5.3 Secondary Outcome | sodium level ( |
| | Variables | • Change in serum sodium level from 24 hours post-last dose to |
| | 3.5.4 Efficacy Variables | 7 days post-last dose |
| | For all subjects, the key | Percentage of subjects requiring rescue therapy (other than |
| | secondary endpoint is the | fluid restriction) during Treatment Phase A and Treatment |
| | change in serum sodium | Phase B |
| | concentration at the end of | Percentage of subjects requiring fluid restriction during |

| Locatio | Old Text: | New Text: |
|---|---|---|
| Location: | Day 2/3 from baseline in Phase A. 3.5.4.1 Safety Variables • Percentage of subjects with overly rapid increase in serum sodium (≥ 12mmol/L in 24 hours after first dose). • Percentage of subjects requiring rescue medication during Phase A and Phase B of the trial. • Change in serum sodium from 24 hours post-last dose to 14 days post-randomization. • Vital signs, blood pressure, clinical laboratory tests, and body weight. 3.5.4.3 Pharmacodynamic Variables Pharmacodynamic endpoints are fluid intake, urine output, and fluid balance (intake − output) every 6 hours on Days 1 and 2 (Phase A). 3.5.5 Exploratory Variables • The other efficacy endpoint in nonresponders continuing on tolvaptan therapy is the change in trough serum sodium concentration on Day 6 compared to Day 4. 3.5.5.2 Safety Variable The other safety variables is neurological examinations. 3.5.5.3 Pharmacodynamic Variables | Treatment Phase A and Treatment Phase B Vital signs, blood pressure, clinical laboratory tests, body weight, and neurological examinations 3.5.3.3 Pharmacodynamic Variables Pharmacodynamic endpoints are fluid intake, urine output, and fluid balance (intake minus output) every 6 hours on Days 1 and 2 in Treatment Phase A. 3.5.4 Exploratory Variables Efficacy will be assessed in nonresponders continuing on tolvaptan therapy by change from baseline in serum sodium concentration at the end of Treatment Phase B compared to the end of Treatment Phase A In all subjects, 24-hour excretion of sodium, creatinine, and urine osmolality on Days 1 and 2 24-hour sodium clearance on Day 1 Neurocognition test battery QoL assessments |
| | The other PD endpoints include: | |

| Locatio | Old Text: | New Text: |
|---|---|---|
| n: | • In all subjects, 24-hour | |
| | excretion of sodium, creatinine, and osmoles | |
| | on Days 1 and 2. | |
| | • | |
| 3.6<br>Measur | This is an open-label trial. Subjects defined as | This is an open-label trial. Subjects defined as responders from |
| es to | responders (serum sodium | Treatment Phase A will be randomized to either the Early Withdrawal group or the Late Withdrawal group in Treatment |
| Minimiz | increase of $\geq 4 \text{ mmol/L}$ ) will | Phase B. Treatment assignments for Treatment Phase B will be |
| e/void | be randomized to either the | based on a computer-generated randomization code provided by |
| Bias | Early Withdrawal group or the Late Withdrawal group. | OPDC Biometrics Department. |
| | The assignments will be | |
| | stratified by age (< 10 and ≥ | |
| | 10 to < 18 years), magnitude | |
| | of serum sodium response (≤ 7 and > 7 mmol/L), and | |
| | underlying etiology of | |
| | hyponatremia. The dose of | |
| | the investigational medicinal | |
| | product (IMP) assigned to a subject is determined by the | |
| | subject's age, weight, and | |
| | the use of CYP3A4 | |
| 2.5 | inhibitors. | |
| 3.7<br>Trial | Treatment in this trial will be up to 5 days. Any initiation | Treatment in this trial will last up to 5 days. Any initiation or titration of tolvaptan must occur in a hospital setting. Parents or |
| Procedu | or titration of tolvaptan must | legal guardians must provide informed consent and subjects must |
| res | occur in a hospital setting. | provide informed assent (as appropriate) and be screened up to |
| | Parents or legal guardians | 24 hours prior to dosing. |
| | will consent and subjects will assent (as appropriate) | In Treatment Phase A, subjects who meet the inclusion and |
| | and be screened up to | exclusion criteria will be enrolled and will be administered a |
| | 24 hours prior to dosing. | 3.75-, 7.5-, or 15-mg dose tablet based on age, weight, and the use |
| | Subjects who meet the inclusion and exclusion | of CYP3A4 inhibitors. At the end of Day 2 (or 2a) in Treatment Phase A, subjects who are responders will be randomized to either |
| | criteria will be enrolled and | continue treatment with tolvaptan for 2 additional days (Late |
| | will be administered a 3.75-, | Withdrawal) or to discontinue tolvaptan treatment (Early |
| | 7.5-, or 15-mg dose based on | Withdrawal). |
| | age, weight, and the use of CYP3A4 inhibitors. | In Treatment Phase B, subjects who are nonresponders may |
| | C 11 5A4 minotors. | continue on tolvaptan therapy for 2 additional days or may be |
| | At the end of Treatment Day | withdrawn from tolvaptan to be treated per the investigator's |
| | 2 (optionally Day 3 [Phase | preferred standard of care. During Treatment Phase B, subjects in |
| | A]), subjects who are responders will be | the Late Withdrawal group and nonresponders continuing treatment will continue to receive tolvaptan for 2 additional days |
| | randomized to either | and all subjects will have serum sodium levels measured at 12 (± |
| | continue treatment with | 4) hours post-dose and at trough each day. Subjects in the Early |
| | tolvaptan for 2 additional | Withdrawal group should be monitored for the first 48 hours post- |
| | days (Late Withdrawal) or to discontinue tolvaptan | last dose. |
| | treatment (Early | In Follow-up Phase C, all subjects will be monitored and will |
| | Withdrawal). Subjects who | have an additional serum sodium measurement at 72 (± 4) hours |

| Locatio<br>n: | Old Text: | New Text: |
|---|---|---|
| | are nonresponders may continue on tolvaptan therapy for 2 additional days at their highest dose or may be withdrawn from tolvaptan to be treated per the investigator's preferred standard of care. During Phase B, subjects in the Late Withdrawal group and nonresponders continuing treatment will continue treatment with tolvaptan for 2 additional days and all subjects will have serum sodium measured every 12 (± 4) hours post-randomization. In Phase C, or Follow-up Phase, subjects will be monitored and treated as clinically warranted per the investigator's preferred standard of care for up to 3 additional days after the last dose of tolvaptan (note: the Early Withdrawal group should be monitored for the first 48 hours post-last dose) and will have an additional serum sodium concentration measurement at 72 (± 4) hours post-randomization. A final safety follow-up telephone contact/visit will be performed 14 (+ 2) days post-randomization. Trial assessment time points are summarized in Table 3.7-1. Pharmacokinetic samples will be obtained on Day 1 (Phase A) for all subjects and at 24 and 48 hours post-randomization for tolvaptantreated subjects in Phase B, including subjects who are | post-last dose as well as at 7 (± 1) days post-last dose. A final safety follow-up telephone contact/visit will be performed 14 (+ 2) days post-last dose. Trial assessment ime points are summarized in Table 3.7-1. Section 3.7.1 provides a flow overview that describes the sequence of assessments during a visit. Section 3.7.2 provides details around efficacy assessments, Section 3.7.3 provides details around pharmacokinetic/pharmacodynamic assessments and Section 3.7.4 provides details around safety assessments. Pharmacokinetic samples will be obtained for all subjects on Day 1 at 2 and 8 hours post-first dose and at trough on Days 2, 3, 4 and 5 for all subjects when dosed with tolvatpan on Days 1, 2, 3, and 4, respectively, regardless of responder status. Once adequate PK data are obtained, PK sampling will be discontinued for all subjects. Subjects will be required to be in a hospital setting during initiation or titration of tolvaptan. A subject is allowed to be discharged, if they: 1) Continue to come to the clinic for daily study assessments and 2) Are either: a) A nonresponder on standard of care or b) On a stable dose of study drug, or c) In the early withdrawal group without study treatment. Follow-up for all subjects may occur in the hospital if the subject has not been discharged or the subject may return for outpatient visits if the subject has been discharged from the hospital. |

# Protocol 156-08-276

| Locatio | Old Text: | New Text: |
|---|---|---|
| n: | | |
| | deemed nonresponders and continue on tolvaptan. Once adequate PK data are obtained, PK sampling will be discontinued for all subjects. | |

# Old Text:

# **3.7 Trial Procedures**

| Table 3.7-1 Schedule of Assess | ments | | | | | |
|---|---|---|---|---|---|---|
| Procedures | | Phase A | Phase B | Phase C | | |
| | Screening/<br>Baseline Visit<br>Days -2 to -1 | Initial Treatment Phase<br>Days 1 and 2/3 | Randomization<br>Phase<br>Days 3/4 and 4/5 | Follow-up<br>Phase<br>Day 5/6 or ET | Follow-up<br>(7 [± 1] days<br>post-random.) | Follow-up<br>Phone Call/Visit<br>(14 [+ 2] days<br>post-random.) |
| Informed consent and assent | X | | | | | |
| Review inclusion/exclusion criteria | X | Day 1: predose | | | | |
| Demographic information | X | | | | | |
| Medical and hyponatremia history | X | | | | | |
| Alcohol and drug screen | X | | | | | |
| Pregnancy test (if applicable) <sup>a</sup> | X | | | | | |
| Serum chemistry | X | | | X | | |
| Plasma osmolality, FeNa, and Fe urate | X | | | | | |
| TSH and cortisol <sup>b</sup> | X | | | | | |
| Hematology and coagulation | X | | | X | | |
| Urinalysis | X | | | X | | |
| Urine chemistry | X | Days 1 and 2 only: 6-hour intervals starting at Hour 0 | | | | |
| Serum sodium <sup>c</sup> | 2 assessments at<br>least 12 hours<br>apart | Baseline (Hour 0; within 3 ±1 hours of dosing), 12 hours post-first dose, and 24 (± 4) hours post-previous dose | 12, 24, 36, and<br>48 (± 4) hours<br>post-random. | 72 (± 4) hours post-random. | X | |
| Vital signs d | X | 2, 4, 8, and 24 hours post-first dose and on Day 3, if applicable | X | X | X | |
| Fluid intake and urine volume | | Days 1 and 2 only: 6-hour | | | | |

| Table 3.7-1 Schedule of Assess | ments | | | | | |
|---|---|---|---|---|---|---|
| Procedures | | Phase A | Phase B | Phase C | | |
| | Screening/<br>Baseline Visit<br>Days -2 to -1 | Initial Treatment Phase<br>Days 1 and 2/3 | Randomization<br>Phase<br>Days 3/4 and 4/5 | Follow-up<br>Phase<br>Day 5/6 or ET | Follow-up<br>(7 [± 1] days<br>post-random.) | Follow-up<br>Phone Call/Visit<br>(14 [+ 2] days<br>post-random.) |
| | | intervals starting at Hour 0 | | | | |
| PK plasma samples e | | 1, 2, 4, 12, and 24 hours post-first dose | 24 and 48 hours post-random. | ET only | | |
| 12-lead ECG | X | | | | | |
| Directed physical examination | X | Baseline (Hour 0), 8 hours post-first dose, and Day 2/3 | Daily | X | X | |
| Neurological examination | X | Baseline (Hour 0), 8 hours post-first dose, and Day 2/3 | Daily | X | X | |
| Body height and weight f | X | Daily (predose): weight only | Daily (predose):<br>weight only | Weight only | Weight only | |
| Clinical assessment <sup>g</sup> | X | End of Day 2/3 | Day 4/5 | X | X | |
| Randomization | | Responders: End of Day 2 (optionally Day 3) | | | | |
| Tolvaptan dosing h | | Once daily | Once daily | | | |
| Follow-up phone call | | | | | | X |
| Concomitant medications | < | | | | | > |
| Adverse events | < | | | | | > |

ECG = electrocardiogram; ET = early termination; post-random. = post-randomization; TSH = thyroid-stimulating hormone.

Note: See Table 3.7.4.2-1 for further details regarding laboratory tests.

<sup>&</sup>lt;sup>a</sup>Pregnancy tests will be performed on female subjects  $\geq$  12 years of age and all female subjects  $\leq$  12 years of age if menstruation has started.

<sup>&</sup>lt;sup>b</sup>Results of these tests will further characterize hyponatremia etiology for the Hyponatremia History CRF and are not required to determine eligibility.

<sup>&</sup>lt;sup>c</sup>Results of the serum sodium from the chemistry panel are sufficient for the protocol. It is not necessary to collect a separate serum sodium concentration.

<sup>&</sup>lt;sup>d</sup>Vital signs to be assessed include supine blood pressure, heart rate, respiratory rate, and temperature. Vital signs should be assessed prior to any blood draws per protocol.

<sup>&</sup>lt;sup>e</sup>An ET sample will be collected only if ET is before the last scheduled PK assessment. The PK samples in Phase B will be collected for all subjects who are on tolvaptan, including subjects who are deemed nonresponders and continue on tolvaptan. Pharmacokinetic blood samples should be taken within ± 5 minutes for each draw up to 2 hours postdose and ± 30 minutes for later time points.

Weight will be taken predose as possible during administration of tolvaptan.

<sup>&</sup>lt;sup>g</sup>Subject clinical status assessments will be performed per inpatient standard of care, ie, review patient chart entries (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate overall subject eligibility in terms of hyponatremia state.

h The dose will be titrated at a minimum of 24 (± 4)-hour intervals from 3.75 to 7.5 to 15 mg for subjects ≥ 2 years of age and weighing ≥ 10 to < 20 kg, from 7.5 to 15 to 30 mg for subjects weighing 20 to 50 kg, inclusive, or from 15 to 30 to 60 mg for subjects weighing > 50 kg. Subjects starting at lower doses may be sequentially titrated to the maximal dose allowed for their weight group. Each upward titration may not exceed twice the previous dose.

<sup>•</sup> In Phase B, tolvaptan will only be administered to subjects randomized to the Late Withdrawal group and to nonresponders who are continuing on tolvaptan. Subjects randomized to the Late Withdrawal group will receive the same dose that they received on Day 2/3; nonresponders may continue on tolvaptan therapy for 2 additional days at their highest dose at the discretion of the investigator.

# **New Text:**

# **3.7 Trial Procedures**

| Table 3.7-1 Schedule of As | ssessments | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening Treatment Phase A | | Trea | tment Phas | se B | Follow-up Phase C | | | | | |
| | Day -2<br>and -1 | Day 1 | Day 2 | Day 2a<br>(optional) | Day 3 | Day 4 | Day 5 | 72 (±4) h<br>post last<br>dose | 7 (±1)<br>days post-<br>last dose | 14 (+2)<br>days post-<br>last dose | Early<br>Termin-<br>ation (ET) |
| Informed Consent/Assent | X | | | | | | | | | | |
| Inclusion/exclusion criteria <sup>a</sup> | X | X | | | | | | | | | |
| Demographic information | X | | | | | | | | | | |
| Medical and hyponatremia history | X | | | | | | | | | | |
| Vital signs <sup>b</sup> | X | X | X | X | X | X | X | X | X | | X |
| 12-lead ECG | X | | | | | | | | | | |
| Height | X | | | | | | | | | | |
| Body weight <sup>c</sup> | X | X | X | X | X | X | X | X | X | | X |
| Directed physical examination | X | X | X | X | X | X | | X | X | | X |
| Tanner staging | X | | | | | | | | | | |
| Neurological examination | X | X | X | | X | X | | X | X | | X |
| Neurocognitive assessment <sup>d</sup> | X | X | X | X | X | X | X | X | X | | X |
| Quality of life assessment | X | | | | | X | | | X | | |
| Clinical status assessment <sup>e</sup> | X | X | X | X | X | X | | X | X | | X |
| Alcohol/drug screen | X | | | | | | | | | | |
| Pregnancy test (if applicable) <sup>f</sup> | X | | | | | | | | | | |
| Fluid intake <sup>g</sup> | | X | X | | | | | | | | |
| Urine volume <sup>g</sup> | | X | X | | | | | | | | |
| Urinalysis | X | | | | | | | X | | | X |
| Urine chemistry <sup>g,h</sup> | X | X | X | | | | | | | | |
| Serum sodium <sup>1</sup> | X | X | X | X | X | X | X | X | X | | X |

| Table 3.7-1 Schedule of As | ssessments | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening | Treatment Phase A | | Treatment Phase B | | Follow-up Phase C | | | | | |
| | Day -2<br>and -1 | Day 1 | Day 2 | Day 2a<br>(optional) | Day 3 | Day 4 | Day 5 | 72 (±4) h<br>post last<br>dose | 7 (±1)<br>days post-<br>last dose | 14 (+2)<br>days post-<br>last dose | Early<br>Termin-<br>ation (ET) |
| Hematology, coagulation, and serum chemistry <sup>j</sup> | X | | | | | | | X | | | X |
| Serum osmolality, FENa, and FE urate | X | | | | | | | | | | |
| TSH and cortisol <sup>k</sup> | X | | | | | | | | | | |
| PK plasma samples | | X | X | | X | X | X | | | | X |
| Tolvaptan dosing <sup>m</sup> | | X | X | X | X | X | | | | | |
| Assessment for response to tolvaptan | | | X | X | | | | | | | |
| Palatability assessment | | | X | | | | | | | | |
| Randomization | | | | | X | | | | | | |
| Follow-up phone call or visit | | | | | | | | | | X | |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X |

ECG = electrocardiogram; TSH = thyroid-stimulating hormone.

<sup>i</sup>Serum sodium assessments are closely tied to neurocognitive assessments, dosing time points and PK blood draws.

• Screening: 2 assessments should be taken, at least 12 hours apart (may be part of medical history). 1 assessment can be combined with the serum chemistry panel.

<sup>&</sup>lt;sup>a</sup>Inclusion/exclusion criteria will be checked at screening and predose on Day 1.

<sup>&</sup>lt;sup>b</sup>Vital signs to be assessed include supine blood pressure, heart rate, respiratory rate, and temperature. Vital signs should be assessed prior to any blood draws.

<sup>&</sup>lt;sup>c</sup>Weight will be taken predose as possible.

<sup>&</sup>lt;sup>d</sup>Neurocognitive assessments are closely tied to serum sodium assessments and should be done within 1 hour of sodium blood draws.

<sup>&</sup>lt;sup>e</sup>Clinical status assessments will be performed per inpatient standard of care, ie, review patient chart entries (including hyponatremia assessment notes and laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate overall subject eligibility in terms of hyponatremia state.

 $<sup>^{\</sup>mathrm{f}}$ Urine pregnancy tests will be performed on female subjects  $\geq$  12 years of age and all female subjects  $\leq$  12 years of age if menstruation has started.

<sup>&</sup>lt;sup>g</sup>Intervals starting immediately after dosing at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours).

<sup>&</sup>lt;sup>h</sup>Samples within a collection interval are to be refrigerated and pooled. An aliquot for urine chemistry tests will be taken for each collection interval. Uric acid is to be measured at screening only.

- Treatment Phase A: Baseline [STAT] assessment will be at 2-4 hours prior to first dose. Post-first dose assessments: 8 and 24 (trough) hours. Then every 12 hours thereafter (alternating 12 hours post-dose and at trough)
- Treatment Phase B: Assessments to be taken every 12 hours (alternating 12 hours post-dose and at trough)
- Treatment Phase C: Assessments to be taken at 72 (± 4) hours post-last dose (can be combined with the serum chemistry panel) and at the 7 day post-last dose visit.

<sup>J</sup>Serum chemisty panel includes serum sodium and assessments can be combined for visits where both assessments are indicated.

<sup>1</sup>PK samples are closely tied to dosing time points and serum sodium assessments. An ET sample will be collected only if ET is before the last scheduled PK assessment.

- In Treatment Phase A PK samples should be collected at 2 and 8 hours and at trough post-first dose.
- In Treatment Phase B PK will be assessed in subjects continuing treatment with tolvaptan (Late Withdrawal group and nonresponders continuing on tolvaptan) at trough on Days 3, 4 and 5.

<sup>m</sup>The tolvaptan dose will be titrated based on serum sodium levels as described in Section 3.2.4.

<sup>&</sup>lt;sup>k</sup>Results of these tests will further characterize hyponatremia etiology for the Hyponatremia History CRF and are not required to determine eligibility. Subjects who have clinically relevant TSH or cortisol levels may not respond properly to tolvaptan and will be withdrawn from the trial.

| Location: | Old Tex | · · · | New To | ovt. |
|---|---|---|---|---|
| 3.7.1 Schedule | | Phase A: Treatment Phase | | 3.7.1.1 Screening |
| of Assessments | | Screening/Baseline | | ocedures listed below will be |
| of Assessments | | owing procedures will be | | ned during the Screening Visit |
| | | ed during the Screening/Baseline | | -2 to -1) to ensure that the subject |
| | | ays -2 to -1 prior to dosing) to | ` - | es for the trial. |
| | | | 1) | |
| | | he subject qualifies for the trial: | , | Trial procedures and information |
| | | Trial procedures and information | | regarding the nature of the trial will be reviewed and written |
| | | regarding the nature of the trial will be reviewed and written | | informed consent/assent will be |
| | | informed consent/assent will be | | |
| | | | | obtained prior to any trial-related |
| | | obtained prior to any trial-related | | procedures. |
| | | procedures. | | a) Informed consent will be |
| | | a) Informed consent will be | | obtained from each subject's |
| | | obtained from each subject's | | parent or legal guardian prior |
| | | parent or legal guardian prio | | to any trial procedures being |
| | | to any trial procedures being conducted. | | conducted. |
| | | | | b) Each subject who is able will indicate willingness to |
| | | b) Each subject who is able wil | | <u> </u> |
| | | indicate willingness to | | participate in the trial by |
| | | participate in the trial by | | signing or marking an assent |
| | | signing or marking an assent | | form (as applicable) supplied |
| | | form (as applicable) supplied | II. | for this purpose. |
| | 2) | for this purpose. | 2) | Inclusion and exclusion criteria will be reviewed. |
| | 2) | Inclusion and exclusion criteria | 2) | |
| | 2) | will be reviewed. | 3) | Demographic information will be collected. |
| | 3) | Demographic information will be collected. | | |
| | | | 4) | Medical and hyponatremia history will be recorded. |
| | | a) Medical and hyponatremia history will be recorded | | a) Medical history should |
| | | separately. Medical history | | include the subject's current |
| | | should include the subject's | | list of medical problems that |
| | | current list of medical | | impacts the subject's current |
| | | problems that impacts the | | hospital stay. |
| | | subject's current hospital sta | 17 | b) The hyponatremia medical |
| | | b) The hyponatremia medical | у. | history should include the |
| | | history should include the | | etiology of subject's |
| | | etiology of subject's | | hyponatremia (see |
| | | hyponatremia (including test | 8 | Section 3.2.1) and what |
| | | per protocol) and what | 3 | treatment was administered |
| | | treatment was administered | | prior to trial enrollment. A |
| | | before trial enrollment. A | | detailed history specific to |
| | | detailed history specific to | | etiology of hyponatremia will |
| | | etiology of hyponatremia wi | 1 | also be recorded. |
| | | also be recorded. | | c) Any observable symptoms of |
| | | c) Any observable symptoms o | f | hyponatremia will be assessed |
| | | hyponatremia will be assessed | | and recorded. |
| | | and recorded separately. | 5) | Vital signs (blood pressure, heart |
| | 4) | Alcohol and drug screens will be | | rate, respiratory rate, and |
| | '' | performed. | 1 | temperature) will be assessed after |
| | 5) | A urine or serum pregnancy test | | the subject has been supine for $\geq 3$ |
| | | will be performed on all female | | minutes. Vital signs should be |
| | | subjects $\geq 12$ years of age and all | | assessed prior to blood draws. |
| | | female subjects < 12 years of age | | A resting 12-lead |
| | | if menstruation has started. | | electrocardiogram (ECG) will be |
| | 6) | Two samples for serum sodium | 1 | performed after the subject has |
| | L 0) | 1 wo samples for serum soutuin | | performed after the subject has |

| Location: | Old Text: | New Text: |
|---|---|---|
| | testing will be collected at least 12 | |
| | hours apart. (These blood draws | minutes. |
| | can be combined with the serum | 7) Body height and weight will be |
| | chemistry panel as appropriate to | measured. |
| | minimize blood draws.) | 8) A directed physical examination |
| | 7) Urinalysis and urine chemistry | will be performed. |
| | laboratory samples will be | 9) Tanner staging will be performed. |
| | collected. | 10) A neurological examination will |
| | 8) Plasma osmolality, FENa, and FE | be performed. |
| | urate will be calculated. | 11) A neurocognitive assessment will |
| | 9) Thyroid-stimulating hormone | be performed, as appropriate by |
| | (TSH) and cortisol blood samples | age and where available. |
| | will be collected to determine need | |
| | for alternate mode of therapy. | will be performed, as appropriate |
| | 10) Vital signs (blood pressure, heart | by age and where available. |
| | rate, respiratory rate, and | 13) Clinical status assessments will be |
| | temperature) will be assessed after | 1 1 |
| | the subject has been supine for ≥ 3 | of care. |
| | minutes. Vital signs should be | 14) Alcohol and drug screens will be performed, as age appropriate. |
| | performed prior to the blood draws. | 15) A urine pregnancy test will be |
| | 11) A resting 12-lead | performed on all female subjects |
| | electrocardiogram (ECG) will be | ≥ 12 years of age and all female |
| | performed after the subject has | subjects < 12 years of age if |
| | been supine and at rest $\geq 10$ | menstruation has started. |
| | minutes. | 16) Urinalysis and urine chemistry |
| | 12) A directed physical examination | laboratory samples will be |
| | will be performed. | collected for analysis. |
| | 13) A neurological examination will | 17) Two blood samples for serum |
| | be performed. | sodium testing will be collected at |
| | 14) Body height and weight will be | least 12 hours apart and can be |
| | measured and body mass index | part of the recent medical history |
| | will be calculated. | to document chronic |
| | 15) Clinical status assessments will be | hyponatremia. (One of these |
| | performed per inpatient standard | blood draws can be combined |
| | of care, ie, patient chart entries | with the serum chemistry panel as |
| | will be reviewed (including | appropriate to minimize blood |
| | hyponatremia assessment notes, | draws.) |
| | including laboratory results [trial and nontrial specific], any | 18) Hematology, coagulation, and serum chemistry laboratory |
| | examination findings, medical | samples will be collected for |
| | problem list changes, and fluid | analysis. |
| | intake and output) to evaluate | 19) Serum osmolality, FENa, and FE |
| | overall subject eligibility in terms | urate will be determined. |
| | of hyponatremia state. | 20) Thyroid-stimulating hormone |
| | 16) Concomitant medications will be | (TSH) and cortisol blood samples |
| | recorded. | will be collected to determine |
| | 17) Adverse events will be assessed. | possible need for alternate mode |
| | | of therapy. |
| | 3.7.1.2.1 Day 1 | 21) Concomitant medications will be |
| | The following procedures will be | recorded. |
| | performed on Day 1 for all subjects: | 22) Adverse events will be recorded. |
| | Inclusion and exclusion criteria | l |
| | will be reviewed prior to dosing to | |
| | confirm eligibility. | During Treatment Phase A every effort |

| Location: | Old Tex | at: | New Te | xt: |
|---|---|---|---|---|
| | 2) | Blood samples for STAT serum | should b | be made to have accurate dosing |
| | | sodium testing will be collected at | time poi | ints and follow the sequence of |
| | | baseline (Hour 0; within 3 [± | assessm | ents specified below as PK/PD |
| | | 1] hours prior to dosing) and 12 | assessm | ents, serum sodium blood draws |
| | | hours post-first dose per protocol, | and neu | rocognitive assessments are closely |
| | | but can be assessed as often as | tied to d | osing time points. |
| | | desired per clinician preference. | | |
| | 3) | | 3.7.1.2.1 | |
| | | and 8 hours post-first dose. Blood | The pro- | cedures listed below will be |
| | | pressure, heart rate, respiratory | perform | ed on Day 1 for all subjects. |
| | | rate, and temperature will be | <u>Predose</u> | |
| | | assessed after the subject has been | 1) | Any observable symptoms of |
| | | supine for $\geq 3$ minutes. Vital signs | | hyponatremia will be assessed |
| | | should be performed prior to the | | within 2 hours prior to first dose |
| | | blood draws at each nominal time | | to confirm eligibility as part of a |
| | | point. | | clinical status assessment. |
| | 4) | Fluid intake and urine volume will | 2) | Vital signs (blood pressure, heart |
| | | be recorded at 6-hour intervals | | rate, respiratory rate, and |
| | | starting at Hour 0. | | temperature) will be assessed after |
| | 5) | Urine chemistry will be assessed | | the subject has been supine for $\geq 3$ |
| | | using 6-hour collection intervals | | minutes. Vital signs should be |
| | | starting at Hour 0. | | assessed prior to blood draws. |
| | 6) | Any observable symptoms of | 3) | A blood sample for STAT serum |
| | | hyponatremia will be assessed at | | sodium testing will be collected |
| | | baseline (prior to dosing) to | | within 2 to 4 hours prior to dosing. |
| | | confirm eligibility. | 4) | A neurocognitive assessment will |
| | 7) | A directed physical examination | | be performed, as appropriate by |
| | | will be performed at baseline | _, | age and where available. |
| | | (prior to dosing) and 8 hours post- | 5) | Body weight will be measured. |
| | 0) | first dose. | 6) | A directed physical examination |
| | 8) | A neurological examination will | 7) | will be performed. |
| | | be performed at baseline (prior to | 7) | A neurological examination will |
| | 0) | dosing) and 8 hours post-first dose. | 9) | be performed. Inclusion and exclusion criteria |
| | 9) | Body weight will be measured | 8) | will be reviewed and confirmed |
| | 10) | predose as possible. | Dogina | will be reviewed and commined |
| | 10) | Blood samples for PK analysis of | Dosing 9) | Tolvaptan will be administered. |
| | | tolvaptan will be collected at 1, 2, 4, and 12 hours post-first dose. | Postdos | _ |
| | 11) | Tolvaptan will be administered as | | A blood sample will be collected |
| | 11) | a 3.75-, 7.5-, or 15-mg dose based | 10) | at 2 hours post-first dose for PK |
| | | on weight and the use of CYP3A4 | | analysis |
| | | inhibitors. | 11) | Vital signs will be assessed at 4 |
| | 12) | Concomitant medications will be | | and 8 hours post-first dose. Blood |
| | 12) | recorded. | | pressure, heart rate, respiratory |
| | 13) | Adverse events will be assessed. | | rate, and temperature will be |
| | | | | assessed after the subject has been |
| | 3.7.1.2.2 | 2 Day 2 (Including Day 3, if | | supine for $\geq 3$ minutes. Vital |
| | Approp | • • | | signs should be assessed prior to |
| | | owing procedures will be | | blood draws at 8 hours. |
| | | ed on Day 2/3 for all subjects: | 12) | Fluid intake will be recorded at 6- |
| | 1) | A blood sample for STAT serum | | hour intervals starting at Hour 0 |
| | | sodium testing should be taken at | | (0-6, 6-12, 12-18, and 18-24 |
| | | 24 (± 4) hours post-previous dose | | hours). |
| | | and the results known prior to | 13) | Urine will be collected at 6-hour |
| | | | | intervals starting at Hour 0 (0-6, |

| Location: | Old Tex | xt: | New Te | xt: |
|---|---|---|---|---|
| | | subsequent tolvaptan dosing. | | 6-12, 12-18, and 18-24 hours). |
| | 2) | Vital signs will be assessed at 24 | | Subjects should be asked to void |
| | | hours post-first dose and on Day 3, | | just prior to the end time of each |
| | | if applicable. Blood pressure, | | collection interval, as possible. |
| | | heart rate, respiratory rate, and | | a) Urine volume will be |
| | | temperature will be assessed after | | determined from urine voids |
| | | the subject has been supine for $\geq 3$ | | made during the 6-hour |
| | | minutes. Vital signs should be | | collection intervals which will |
| | | performed prior to the blood | | be pooled prior to |
| | | draws. | | determination of final |
| | 3) | Fluid intake and urine volume will | | volume. |
| | | be recorded at 6-hour intervals on | | b) A urine chemistry sample will |
| | | Day 2. | | be collected and assessed |
| | 4) | Urine chemistry will be assessed | | from each 6-hour volume |
| | | using 6-hour collection intervals | | interval starting at Hour 0 (0- |
| | | on Day 2. | | 6, 6-12, 12-18, and 18-24 |
| | 5) | A directed physical examination | | hours). |
| | | will be performed. | 14) | Blood samples will be collected |
| | 6) | A neurological examination will | | concurrently at 8 hours post-first |
| | | be performed. | | dose for: |
| | | c) Body weight will be measured | | a) Serum sodium testing |
| | | predose daily during | | b) PK analysis |
| | | administration of tolvaptan as | 15) | A neurocognitive assessment will |
| | | possible. | | be performed within 1 hour of the |
| | | d) A blood sample for PK | | serum sodium sample. |
| | | analysis of tolvaptan will be | 16) | A neurological examination will |
| | | collected at 24 hours post-first | | be performed at 8 hours post-first |
| | | dose. | | dose. |
| | 7) | If the subject's serum sodium | | nout the visit |
| | | concentration is < 135 mmol/L and | 17) | Concomitant medications will be |
| | | $a \le 4$ -mmol/L increase, tolvaptan | | recorded. |
| | | should be titrated per the titration | 18) | Adverse events will be assessed. |
| | | guidelines (Section 3.2.1) for the | | |
| | | assigned weight group. | 3.7.1.2.2 | |
| | 8) | Clinical status assessments will be | | owing procedures will be |
| | | performed at the end of Day 2/3 | | ed on Day 2 for all subjects. |
| | | per inpatient standard of care, ie, | | (24 hours post-first dose) |
| | | patient chart entries will be | | th the following assessments will be |
| | | 8 71 | perform | |
| | | assessment notes, including | 1) | Vital signs will be assessed. |
| | | laboratory results [trial and | | Blood pressure, heart rate, respiratory rate, and temperature |
| | | nontrial specific], any examination | | |
| | | findings, medical problem list | | will be assessed after the subject |
| | | changes, and fluid intake and | | has been supine for ≥ 3 minutes. |
| | | output) to evaluate overall subject | | Vital signs should be performed prior to blood draws. |
| | | eligibility in terms of hyponatremia state. | 2) | Blood samples will be collected |
| | 2) | Concomitant medications will be | 2) | concurrently at 24 ( $\pm$ 4) hours for: |
| | 2) | recorded. | | a) A blood sample for STAT |
| | 3) | Adverse events will be assessed. | | serum sodium testing should |
| | | a) At the end of Day 2 | | be taken and the results |
| | | (optionally Day 3), subjects | | known prior to subsequent |
| | | who are responders (serum | | tolvaptan dosing. |
| | | sodium increase of $\geq 4$ | | b) A blood sample for PK |
| | | Socium mercase of 2 4 | | analysis of tolvaptan (at a |
| [ | 1 | | ı | anaryono or torraptain (at a |

| Location: | Old Tex | | New Te | |
|---|---|---|---|---|
| | | mmol/L) will be randomized | | central lab) will be collected |
| | | to the Early or Late | | at 24 hours post-first dose. |
| | | Withdrawal group. | 3) | A neurocognitive assessment will |
| | 11) | Subjects who are nonresponders at | | be performed within 1 hour of the |
| | | the end of Day 3 may continue on | | serum sodium sample. |
| | | tolvaptan therapy for 2 additional | <b>Predose</b> | |
| | | days at their highest dose or may | 4) | Complete fluid intake and urine |
| | | be withdrawn from tolvaptan to be | | volume collection for specified |
| | | treated per the investigator's | | intervals prior to next dosing with |
| | | preferred standard of care. | | tolvaptan. |
| | | 1 | 5) | Fluid intake will be recorded at 6- |
| | 3.7.1.3 1 | Phase B: Randomization Phase | - / | hour intervals starting at Hour 0 |
| | | owing procedures will be | | (0-6, 6-12, 12-18, and 18-24 |
| | | ed on Days 3/4 and 4/5 for all | | hours). |
| | subjects | | 6) | Urine will be collected at 6-hour |
| | 1) | A blood sample for STAT serum | 0) | intervals starting at Hour 0 (0-6, |
| | 1) | | | |
| | | sodium testing should be taken 12, | | 6-12, 12-18, and 18-24 hours). Subjects should be asked to void |
| | | 24, 36, and 48 ( $\pm$ 4) hours post- | | 2 |
| | | randomization and the results | | just prior to the end time of each |
| | | known prior to subsequent | | collection interval, as possible. |
| | - | treatment. | | a) Urine volume will be |
| | 2) | Vital signs (blood pressure, heart | | determined from urine voids |
| | | rate, respiratory rate, and | | made during the 6-hour |
| | | temperature) will be assessed daily | | collection intervals which will |
| | | after the subject has been supine | | be pooled prior to |
| | | for $\geq 3$ minutes. Vital signs should | | determination of final |
| | | be performed prior to the blood | | volume. |
| | | draws. | | b) A urine chemistry sample will |
| | 3) | A directed physical examination | | be collected and assessed |
| | ĺ | will be performed daily. | | from each 6-hour volume |
| | 4) | A neurological examination will | | interval starting at Hour 0 (0- |
| | , | be performed daily. | | 6, 6-12, 12-18, and 18-24 |
| | 5) | Body weight will be measured | | hours). |
| | | predose daily during | 7) | A directed physical examination |
| | | administration of tolvaptan as | ., | will be performed. |
| | | possible. | 8) | Body weight will be measured. |
| | 6) | Blood samples for PK analysis of | 9) | A neurological examination will |
| | 0) | tolvaptan will be collected at 24 | | be performed. |
| | | and 48 hours post-randomization | Dosing | - F |
| | | | | Tolvaptan will be administered. |
| | | for all subjects on tolvaptan, | | If the subject's serum sodium |
| | | including subjects who are deemed | | concentration is < 135 mEq/L |
| | | nonresponders and continue on | | - |
| | 7 | tolvaptan. | | (mmol/L) and $a \le 4 \text{ mEq/L}$ |
| | 7) | Tolvaptan will be administered | | (mmol/L) increase, tolvaptan dose |
| | | once daily to subjects randomized | | should be adjusted per the titration |
| | | to the Late Withdrawal group and | | guidelines (Section 3.2.4) for the |
| | | nonresponders continuing on | <b>.</b> | assigned weight group. |
| | | tolvaptan. | Postdose | |
| | 8) | Subjects randomized to the Early | 2) | Assess palatability of tolvaptan |
| | | Withdrawal group will be initially | | tablets for subjects. |
| | | observed to determine whether | 3) | Fluid intake will be recorded at 6- |
| | | additional intervention is required | | hour intervals starting at Hour 0 |
| | | to maintain appropriate serum | | (0-6, 6-12, 12-18, and 18-24 |
| | | sodium levels. Nonresponders | | hours). |
| | | discontinuing tolvaptan will be | 4) | Urine will be collected at 6-hour |

| Location: | Old Te | xt: | New Te | ext: |
|---|---|---|---|---|
| Locusion | 014 10 | treated per the investigator's | 11011110 | intervals starting at Hour 0 (0-6, |
| | | preferred standard of care for | | 6-12, 12-18, and 18-24 hours). |
| | | 3 additional days after the last dose | | Subjects should be asked to void |
| | | of tolvaptan. | | just prior to the end time of each |
| | 9) | Clinical status assessments will be | | collection interval, as possible. |
| | | performed on Day 4/5 per | | a) Urine volume will be |
| | | inpatient standard of care, ie, | | determined from urine voids |
| | | patient chart entries will be | | made during the 6-hour |
| | | reviewed (including hyponatremia | | collection intervals which will |
| | | assessment notes, including | | be pooled prior to |
| | | laboratory results [trial and | | determination of final |
| | | nontrial specific], any examination | | volume. |
| | | findings, medical problem list | | b) A urine chemistry sample will |
| | | changes, and fluid intake and | | be collected and assessed |
| | | | | from each 6-hour volume |
| | | output) to evaluate overall subject | | |
| | | eligibility in terms of | | interval starting at Hour 0 (0- |
| | 10) | hyponatremia state. | | 6, 6-12, 12-18, and 18-24 |
| | 10) | Concomitant medications will be | <i>E</i> ) | hours). |
| | 11) | recorded. Adverse events will be assessed. | 5) | Clinical status assessments will be |
| | 11) | Auverse events will be assessed. | | performed per inpatient standard |
| | 2714 | Dhasa Ca Fallana an Dhasa | | of care, ie, patient chart entries |
| | | Phase C: Follow-up Phase | | will be reviewed (including |
| | | 1 Follow-up (Day 5/6)/Early | | hyponatremia assessment notes, |
| | Termin | | | including laboratory results [trial |
| | | owing procedures will be | | and nontrial specific], any |
| | | ed on Day 5/6 or at early | | examination findings, medical |
| | | tion (ET) for all subjects: | | problem list changes, and fluid |
| | 1) | Hematology, coagulation, and | | intake and output) to evaluate the |
| | | serum chemistry laboratory | | subject's hyponatremia state. |
| | 2) | samples will be collected. | 6) | A blood sample will be collected |
| | 2) | A blood sample for serum sodium | | for serum sodium testing at |
| | | testing will be collected at 72 | 7) | 12 hours post-dose. |
| | | (± 4) hours post-randomization. | 7) | A neurocognitive assessment will |
| | | (This blood draw can be combined | | be performed within 1 hour of the |
| | | with the chemistry panel as | 0) | serum sodium sample. |
| | | appropriate to minimize blood | 8) | At the end of the Day 2 visit |
| | • | draws.) | | subjects will be assessed for |
| | (3) | A urinalysis laboratory sample will | | response to tolvaptan treatment. |
| | | be collected. | | Subjects who are: |
| | 4) | A blood sample for PK analysis of | | a) Responders (serum sodium |
| | | tolvaptan will be collected at ET | | level increase of ≥ 4 mEq/L |
| | | only if ET occurs before the last | | [mmol/L]) will proceed to |
| | | scheduled PK assessment (ie, <u>48</u> | | Treatment Phase B (see |
| | | hours post-randomization for | | Section 3.7.1.3) for |
| | | subjects continuing on tolvaptan). | | randomization. |
| | 5) | Vital signs (blood pressure, heart | | b) Nonresponders (serum |
| | | rate, respiratory rate, and | | sodium level increase of < 4 |
| | | temperature) will be assessed after | | mEq/L [mmol/L]) will |
| | | the subject has been supine for $\geq 3$ | | proceed to Day 2a (see |
| | | minutes. Vital signs should be | mi . | Section 3.7.1.2.3). |
| | | performed prior to the blood | | nout the visit |
| | | draws. | 9) | |
| | 6) | A directed physical examination | 10 | recorded. |
| | | will be performed. | 10) | Adverse events will be assessed. |
| | 7) | A neurological examination will | | |

| Location: | Old Text: | | New Text: | |
|---|---|---|---|---|
| | be performed. | | 3.7.1.2.3 Day 2a (optional) | |
| | 8) | Body weight will be measured as | | owing procedures will be |
| | | possible. | | ed on Day 2a for all subjects who |
| | 9) | Subjects will be monitored and | | responsive to tolvaptan treatment at |
| | | treated as clinically warranted per | | of Day 2. |
| | | the investigator's preferred | Predose | |
| | | standard of care for up to | 1) | Vital signs will be assessed at 24 |
| | | 3 additional days after the last dose | ĺ | hours post-previous dose. Blood |
| | | of tolvaptan (note: the Early | | pressure, heart rate, respiratory |
| | | Withdrawal group should be | | rate, and temperature will be |
| | | monitored for the first 48 hours | | assessed after the subject has been |
| | | post-last dose). | | supine for $\geq 3$ minutes. Vital |
| | 10) | Concomitant medications will be | | signs should be performed prior to |
| | | recorded. | | the blood draws. |
| | 11) | Adverse events will be assessed. | 2) | A blood sample for STAT serum |
| | | | ĺ | sodium testing should be taken at |
| | 3.7.1.4.2 | 2 Follow-up | | 24 ( $\pm$ 4) hours post-previous dose |
| | 1) | Subjects will be assessed for | | and the results known prior to |
| | | maintenance of normal or target | | subsequent tolvaptan dosing. |
| | | serum sodium concentration at | 3) | A neurocognitive assessment will |
| | | 7 ( $\pm$ 1) days post-randomization. | | be performed within 1 hour of the |
| | | If the subject was discharged, | | serum sodium sample. |
| | | he/she should return to the clinic | 4) | A directed physical examination |
| | | for the serum sodium collection. | ĺ | will be performed. |
| | 2) | A blood sample for serum sodium | 5) | Body weight will be measured. |
| | | testing will be collected. | Dosing | , , |
| | 3) | Vital signs (blood pressure, heart | 6) | Tolvaptan will be administered. |
| | | rate, respiratory rate, and | | If the subject's serum sodium |
| | | temperature) will be assessed after | | concentration is < 135 mEq/L |
| | | the subject has been supine for $\geq 3$ | | (mmol/L) and a $\leq$ 4 mEq/L |
| | | minutes. Vital signs should be | | (mmol/L) increase, tolvaptan dose |
| | | performed prior to the blood | | should be adjusted per the titration |
| | | draws. | | guidelines (Section 3.2.4) for the |
| | 4) | A directed physical examination | | assigned weight group. |
| | | will be performed. | Postdos | <u>e</u> |
| | 5) | A neurological examination will | 7) | Clinical status assessments will be |
| | | be performed. | | performed per inpatient standard |
| | 6) | Body weight will be measured. | | of care, ie, patient chart entries |
| | 7) | Concomitant medications will be | | will be reviewed (including |
| | | recorded. | | hyponatremia assessment notes, |
| | 8) | Adverse events will be assessed. | | including laboratory results [trial |
| | | | | and nontrial specific], any |
| | 3.7.1.4.3 | 3 Follow-up Telephone | | examination findings, medical |
| | Contact | | | problem list changes, and fluid |
| | | s (or their parents or legal | | intake and output) to evaluate the |
| | | ns) will be contacted via telephone | | subject's hyponatremia state. |
| | or via a visit 14 (+ 2) days post- | | 8) | A blood sample will be collected |
| | randomization to assess any new or | | | for serum sodium testing at |
| | ongoing AEs and to collect information on | | | 12 hours post-dose. |
| | | dications administered since the last | 9) | A neurocognitive assessment will |
| | | ngoing follow-up may be required | | be performed within 1 hour of the |
| | | al closure for health status before | | serum sodium sample. |
| | the anal | ysis of all trial results is completed. | 10) | At the end of the Day 2a visit |
| | | | | subjects will be assessed for |

| Location: | Old Text: | New Text: |
|---|---|---|
| | | response to tolvaptan treatment. |
| | | Subjects who are: |
| | | a) Responders (serum sodium |
| | | level increase of $\geq 4 \text{ mEq/L}$ |
| | | [mmol/L]) will proceed to |
| | | Treatment Phase B (see |
| | | Section 3.7.1.3) for |
| | | randomization. |
| | | b) Nonresponders (serum |
| | | sodium level increase of < 4 |
| | | mEq/L [mmol/L]) will |
| | | continue to Treatment Phase |
| | | B where they either continue |
| | | on tolvaptan therapy for |
| | | 2 additional days or are |
| | | withdrawn from tolvaptan to |
| | | be treated per the |
| | | investigator's preferred |
| | | standard of care. |
| | | Throughout the visit |
| | | 11) Concomitant medications will be |
| | | recorded. |
| | | 12) Adverse events will be assessed. |
| | | 3.7.1.3.1 Day 3 |
| | | The following procedures will be |
| | | performed on Day 3. Some assessments are |
| | | required for all subjects while other |
| | | assessments only apply to certain subsets of |
| | | subjects as indicated. |
| | | For all subjects (at trough) |
| | | 1) At trough (24 hours post-previous |
| | | dose) the following assessments |
| | | will be performed: |
| | | a) Vital signs will be assessed. |
| | | Blood pressure, heart rate, |
| | | respiratory rate, and |
| | | temperature will be assessed |
| | | after the subject has been |
| | | supine for $\geq 3$ minutes. Vital |
| | | signs should be performed |
| | | prior to blood draws. |
| | | 2) Blood samples will be collected |
| | | concurrently at 24 ( $\pm$ 4) hours for: |
| | | a) STAT serum sodium testing |
| | | and the results known prior to |
| | | subsequent tolvaptan dosing. |
| | | b) PK analysis of tolvaptan 3) A neurocognitive assessment will |
| | | 3) A neurocognitive assessment will be performed within 1 hour of the |
| | | serum sodium sample. |
| | | For all subjects classified as Desnoydors |
| | | For all subjects classified as Responders at the end of Treatment Phase A |
| | | at the chu of i reathlellt fliase A |

| Location: | Old Text: | New Text: |
|-----------|-----------|-----------------------------------------|
| | | 4) Randomize the subject to the |
| | | Early or Late Withdrawal group |
| | | using the trial's interactive |
| | | response system. |
| | | For subjects receiving tolvaptan (Late |
| | | Withdrawal group and non-responders |
| | | with continuing treatment) |
| | | 5) Body weight will be measured. |
| | | 4) Tolvaptan will be administered. |
| | | For subjects not receiving tolvaptan |
| | | treatment (Early Withdrawal group and |
| | | non-responders treated with standard of |
| | | <u>care)</u> |
| | | 6) Early Withdrawal subjects will be |
| | | observed to determine whether |
| | | additional intervention is required |
| | | to maintain appropriate serum |
| | | sodium levels. |
| | | 3) Nonresponders discontinuing |
| | | tolvaptan will be treated per the |
| | | investigator's preferred standard |
| | | of care. |
| | | For all subjects at later time points |
| | | during the visit |
| | | 4) A directed physical examination |
| | | will be performed. |
| | | 5) A neurological examination will |
| | | be performed. |
| | | 6) A blood sample will be collected |
| | | for serum sodium testing at |
| | | 12 hours post the nominal dosing |
| | | time (regardless of treatment). |
| | | 7) A neurocognitive assessment will |
| | | be performed within 1 hour of the |
| | | serum sodium sample. |
| | | 8) Clinical status assessments will be |
| | | performed per inpatient standard |
| | | of care, ie, patient chart entries |
| | | will be reviewed (including |
| | | hyponatremia assessment notes, |
| | | including laboratory results [trial |
| | | and nontrial specific], any |
| | | examination findings, medical |
| | | problem list changes, and fluid |
| | | intake and output) to evaluate the |
| | | subject's hyponatremia state. |
| | | For all subjects throughout the visit |
| | | 9) Concomitant medications will be |
| | | recorded. |
| | | 10) Adverse events will be assessed. |
| | i | <b>_</b> |

| Location: | Old Text: | New Text: |
|---|---|---|
| | | 3.7.1.3.2 Day 4 |
| | | The following procedures will be |
| | | performed on Day 4. Some assessments |
| | | are required for all subjects while other |
| | | assessments only apply to certain subsets of |
| | | subjects as indicated. |
| | | For subjects receiving tolvaptan (Late Withdrawal group and non-responders |
| | | with continuing treatment) |
| | | At trough |
| | | 1) Vital signs (blood pressure, heart |
| | | rate, respiratory rate, and |
| | | temperature) will be assessed after |
| | | the subject has been supine for $\geq 3$ |
| | | minutes. Vital signs should be |
| | | performed prior to blood draws. |
| | | 2) A blood sample for STAT serum |
| | | sodium level testing should be |
| | | taken and the results known prior |
| | | to subsequent treatment. |
| | | 3) Blood samples for PK analysis of |
| | | tolvaptan will be collected. |
| | | 4) A neurocognitive assessment will |
| | | be performed within 1 hour of the |
| | | serum sodium sample. |
| | | At later time points during the visit |
| | | 5) Body weight will be measured. 6) Tolyanton will be administered. |
| | | 6) Tolvaptan will be administered. |
| | | For subjects not receiving tolvaptan |
| | | treatment (Early Withdrawal group and |
| | | nonresponders treated with standard of |
| | | care) |
| | | For all subjects at 48 hours post last |
| | | dose 1) Vital signs (blood pressure heart |
| | | 1) Vital signs (blood pressure, heart |
| | | rate, respiratory rate, and |
| | | temperature) will be assessed after |
| | | the subject has been supine for $\geq 3$ minutes. Vital signs should be |
| | | performed prior to blood draws. |
| | | 2) A blood sample for serum sodium |
| | | level testing should be taken. |
| | | 3) A neurocognitive assessment will |
| | | be performed within 1 hour of the |
| | | serum sodium sample. |
| | | At later time points during the visit |
| | | 4) Early Withdrawal subjects will be |
| | | observed to determine whether |
| | | additional intervention is required |
| | | to maintain appropriate serum |
| | | sodium levels. |
| | | 5) Nonresponders discontinuing tolvaptan will continue to be |

| Location: | Old Text: | New Text: |
|---|---|---|
| | | treated per the investigator's |
| | | preferred standard of care. |
| | | For all subjects at later time points |
| | | during the visit |
| | | 7) A directed physical examination |
| | | will be performed. 8) A neurological examination will |
| | | be performed. |
| | | 9) A blood sample will be collected |
| | | for serum sodium testing at |
| | | 12 hours post the nominal dosing |
| | | time (regardless of treatment). |
| | | 10) A neurocognitive assessment will |
| | | be performed within 1 hour of the |
| | | serum sodium sample. |
| | | 11) A QoL assessment will be conducted. |
| | | 12) Clinical status assessments will be |
| | | performed per inpatient standard |
| | | of care, ie, patient chart entries |
| | | will be reviewed (including |
| | | hyponatremia assessment notes, |
| | | including laboratory results [trial |
| | | and nontrial specific], any |
| | | examination findings, medical |
| | | problem list changes, and fluid |
| | | intake and output) to evaluate the |
| | | subject's hyponatremia state. |
| | | For all subjects throughout the visit |
| | | 13) Concomitant medications will be |
| | | recorded. |
| | | 14) Adverse events will be assessed. |
| | | 3.7.1.3.3 Day 5 |
| | | The following procedures will be |
| | | performed on Day 5. |
| | | For subjects receiving tolyaptan (Late Withdrawal group and non-responders |
| | | with continuing tolvaptan treatment) |
| | | At trough |
| | | 1) Vital signs (blood pressure, heart |
| | | rate, respiratory rate, and |
| | | temperature) will be assessed after |
| | | the subject has been supine for $\geq 3$ |
| | | minutes. Vital signs should be |
| | | performed prior to blood draws. |
| | | 2) A blood sample for STAT serum |
| | | sodium level testing should be taken and the results known prior |
| | | to subsequent treatment. |
| | | to subsequent treatment. |
| Location: | Old Text: | New Text: |
|-----------|-----------|---------------------------------------------------|
| | | 3) A blood sample for PK analysis of |
| | | tolvaptan will be collected. |
| | | 4) A neurocognitive assessment will |
| | | be performed within 1 hour of the |
| | | serum sodium sample. |
| | | 5) Body weight will be measured. |
| | | Throughout the visit |
| | | 6) Concomitant medications will be |
| | | recorded. |
| | | 7) Adverse events will be assessed. |
| | | For subjects not receiving tolvaptan |
| | | treatment (Early Withdrawal group and |
| | | nonresponders treated with standard of |
| | | care) |
| | | 13) Proceed to Follow-up Phase C as |
| | | for these subjects the 72h post-last |
| | | dose time point (Section 3.7.1.4.1) |
| | | falls on the morning of Day 5. |
| | | 3.7.1.4 Follow-up Phase C |
| | | 3.7.1.4.1 72 Hours Post-last Dose or ET |
| | | The following procedures will be |
| | | performed for all subjects at 72 ( $\pm$ 4) hours |
| | | post-last dose or at early termination (ET). |
| | | 1) Vital signs (blood pressure, heart |
| | | rate, respiratory rate, and |
| | | temperature) will be assessed after |
| | | the subject has been supine for $\geq 3$ |
| | | minutes. Vital signs should be |
| | | performed prior to blood draws. |
| | | 2) Hematology, coagulation, and |
| | | serum chemistry laboratory |
| | | samples will be collected. |
| | | 3) For Early Termination only: |
| | | Blood sample for PK analysis of |
| | | tolvaptan will be collected at 24 |
| | | hours post-last dose for all |
| | | subjects on tolvaptan. The sample |
| | | is to be taken concurrently with |
| | | the serum sodium sample (part of |
| | | the serum chemistry panel). |
| | | 4) A neurocognitive assessment will |
| | | be performed within 1 hour of the |
| | | serum chemistry sample. |
| | | 5) A directed physical examination |
| | | will be performed. |
| | | 6) A neurological examination will |
| | | be performed. |
| | | 7) Body weight will be measured. |
| | | 8) A urinalysis laboratory sample |
| | | will be collected. |
| | | 9) For Early Termination: Subjects |
| | | will be monitored and treated as |

| Location: | Old Text: | New Text: |
|---|---|---|
| | | clinically warranted per the |
| | | investigator's preferred standard of |
| | | care for up to 3 additional days after |
| | | the last dose of tolvaptan. |
| | | 10)Concomitant medications will be |
| | | recorded. |
| | | 11) Adverse events will be assessed. |
| | | 3.7.1.4.2 7 Days Post-last Dose Subjects will be assessed for maintenance of normal or target serum sodium |
| | | concentration at 7 ( $\pm$ 1) days post-last dose. All clinical labs will be performed locally. |
| | | If the subject was discharged, he/she |
| | | should return to the clinic for this visit. |
| | | 1) Vital signs (blood pressure, heart rate, respiratory rate, and |
| | | temperature) will be assessed after |
| | | the subject has been supine for $\geq 3$ |
| | | minutes. Vital signs should be |
| | | performed prior to blood draws. |
| | | 2) A blood sample for serum sodium |
| | | testing will be collected. |
| | | 3) A neurocognitive assessment will |
| | | be performed within 1 hour of the |
| | | serum sodium sample. |
| | | 4) A QoL assessment will be |
| | | conducted. |
| | | 5) A directed physical examination will be performed. |
| | | 6) A neurological examination will be performed. |
| | | 7) Clinical status assessments will be |
| | | performed per inpatient standard |
| | | of care, ie, patient chart entries |
| | | will be reviewed (including |
| | | hyponatremia assessment notes, |
| | | including laboratory results [trial |
| | | and nontrial specific], any |
| | | examination findings, medical |
| | | problem list changes, and fluid |
| | | intake and output) to evaluate the |
| | | subject's hyponatremia state. |
| | | 8) Body weight will be measured. |
| | | 9) Concomitant medications will be |
| | | recorded. |
| | | 7) Adverse events will be assessed. |
| | | 3.7.1.4.3 14 Days Post-last Dose |
| | | Subjects (or their parents or legal |
| | | guardians) will be contacted via telephone |
| | | or will be asked to come back to the clinic |
| | | for a visit at 14 (+2) days post-last dose to |
| | | assess any new or ongoing AEs and to |
| | | collect information on any medications |

| | | administered since the last visit. Ongoing |
|---|---|---|
| | | follow-up may be required after a subject's |
| | | trial completion for health status before the |
| | | analysis of all trial results is completed. |
| 3.7.2.1 Serum N | Monitoring frequency of serum sodium is at | Monitoring frequency of serum sodium is |
| | the discretion of the clinical investigator; | at the discretion of the clinical investigator; |
| Concentration 1 | nowever, the trial requires the minimum | however, the minimum sample collection |
| | sample collection for all subjects noted in | required for all subjects is described in |
| | Section 3.7.1. | Section 3.7.1. |
| 7 | Within 48 hours of initial tolvaptan | In order to qualify for this trial, subjects |
| | administration, 2 blood samples will be | must have documentation of chronic |
| | collected at least 12 hours apart for | dilutional hyponatremia (serum sodium < |
| | assessment of baseline serum sodium to | 130 mEq/L [mmol/L]) that is present for |
| | determine subject eligibility. A third | ≥ 48 hours. Specifically, each subject must |
| | (STAT) serum sodium sample should be | have 2 blood samples collected at least |
| | drawn within 3 ( $\pm$ 1) hours prior to dosing; | 12 hours apart over a minimum of 48 hours |
| | the results must be verified to be $< 130$ | for assessment of baseline serum sodium |
| | mmol/L prior to the first dose. A STAT | level to determine subject eligibility. |
| | serum sodium sample should be drawn and | These can be either part of the recent |
| | recorded in the CRF at the time of every | medical history concerning the current |
| | hyponatremia symptoms assessment | hospital stay or prospectively collected as |
| | (Section 3.7.1). During Phase A, serum | part of this trial. |
| | sodium will be assessed at 12 hours post- | |
| | first dose and 24 ( $\pm$ 4) hours post-previous | On Day 1, a third (STAT) serum sodium |
| | dose. Serum sodium must also be assessed | sample should be drawn within 2-4 hours |
| | at 12, 24, 36, 48, and 72 (± 4) hours and | prior to dosing; the results must be verified |
| | 7 ( $\pm$ 1) days post-randomization. | to be < 130 mmol/L prior to the first dose. |
| | (± 1) days post randomization. | Serum sodium assessments should be |
| | | performed at 8 hours post-first dose and at |
| | | trough 24 hours post-first dose (this |
| | | assessment will fall on Day 2 predose). |
| | | On Day 2 (or 2a), Day 3, and Day 4 |
| | | (through the following morning on Day 5): |
| | | <ul> <li>For all subjects receiving tolvaptan</li> </ul> |
| | | (Late Withdrawal and Nonresponders |
| | | continuing on tolvaptan) serum sodium |
| | | assessments will be performed at |
| | | trough and 12 hours post-dose each day |
| | | during Treatment Phase A and |
| | | Treatment Phase B. |
| | | • For all subjects not receiving tolvaptan |
| | | (Early Withdrawal and Nonresponders |
| | | on standard of care) serum sodium |
| | | assessments will be performed every |
| | | 12 hours throughout Treatment Phase |
| | | A and Treatment Phase B. |
| | | For all subjects final serum sodium |
| | | assessments will be taken at 24 ( $\pm$ 4) and |
| | | 72 ( $\pm$ 4) hours post-last dose as well as at 7 |
| | | days post-last dose. |
| | | 3.7.2.3 Quality of Life Assessments |
| | | Two patient-reported outcomes instruments |
| | | (acute versions with 7 day recall period) |

| <b>Location:</b> | Old Text: | New Text: |
|---|---|---|
| | | will be used to assess subject quality of |
| | | life: PedsQL Generic Core Scale and |
| | | PedsQL Multidimensional Fatigue Scale. |
| | | Both instruments are appropriate for $\geq 2$ |
| | | years of age, however availability may be |
| | | limited for certain ages and languages. The |
| | | age groups covered by these assessments |
| | | are Toddler (2–4 years), Young child (5–7 |
| | | years), Child (8–12 years), and Adolescent |
| | | (13–18 years). Depending on the subject's |
| | | age, the questionnaire may be completed |
| | | by either the subject or the |
| | | parent/caregiver, as appropriate. |
| | | The PedsQL Generic Core Scale consists of |
| | | 23 items encompassing physical, |
| | | emotional, social, and school domains. The PedsQL Multidimentional Fatigue |
| | | ` |
| | | Scale consists of 18 items in 3 subscales: |
| | | general fatigue, sleep/rest fatigue, and |
| | | cognitive fatigue. The instrument focuses |
| | | on the domains of processing speed, |
| | | attention/vigilance, visual and working |
| | | memory. |
| | | The assessment time points are at |
| | | screening, Day 4 and 7 days post-last dose. |
| | | 3.7.2.4 Neurocognitive Assessments |
| | | An age-appropriate (4-18 years of age) |
| | | neurocognitive assessment will be |
| | | performed using a computerized test |
| | | battery provided by CogState Ltd. |
| | | The instruments used for this assessment |
| | | include 4 tests: the Detection Test, |
| | | Identification Test, One Card Learning |
| | | Test, One Back Test. The tests will focus |
| | | on the domains of processing speed, |
| | | attention/vigilance, visual memory and |
| | | working memory. |
| | | For subjects 6 to 18 years of age all tests |
| | | will be administered. For subjects 4 to 5 |
| | | years of age, the Detection Test and the |
| | | Identification Test will be administered. |
| | | Availability of the assessment may be |
| | | limited for certain subject ages and |
| | | languages. |
| | | The assessment time points correlate with |
| | | serum sodium assessments and should |
| | | occur within an hour of serum sodium |
| | | blood draws. |
| 3.7.3.1.1 Blood | Tolvaptan plasma concentrations will | Blood samples will be taken so that |
| Collection | | _ |
| Concenon | oc incasured. On Day 1, blood samples | porvapian and inclassific concentrations |
| Times | J / 1 | can be determined. Samples will be taken |

| Location: | Old Text: | New Text: |
|---|---|---|
| | (1 mL) for tolvaptan concentrations | on Day 1 at 2 hours (± 5 minutes) and 8 |
| | will be taken at 1, 2, 4, 12, and 24 | hours (concurrent with 8 h serum sodium |
| | hours (± 5 minutes for each draw up to | sample) post-first dose. On Days 2, 3, 4 |
| | 2 hours postdose and $\pm$ 30 minutes for | and 5 samples will be taken at trough (24 |
| | later time points) post-first dose, at | hours post previous dose but prior to the |
| | 24 and 48 hours post-randomization | subsequent dose), concurrent with serum |
| | (for subjects on tolvaptan in Phase B, | sodium samples, for subjects dosed with |
| | including subjects who are deemed | tolvaptan on Days 1, 2, 3, and/or 4, |
| | nonresponders and continue on | respectively, regardless of status as |
| | tolvaptan), or at ET, if ET is before the | responder/non-responder. An early |
| | last scheduled PK assessment. Each | termination (ET) sample will be taken if |
| | subject contributing samples to the PK | ET occurs prior to the last planned PK |
| | analysis will be required to submit a | sample. No ET sample is required if ET occurs at the same visit where a PK sample |
| | total 5 mL of blood in 24 hours and 2 | has already been obtained. |
| | additional samples after randomization. | For each PK blood sample collected |
| | All samples will be collected from each subject according to local guidelines and | volumes are not expected to exceed 1.2 |
| | best practices for pediatric care. | mL. Total volume per sample may be lower |
| | best practices for pediatric care. | depending on finalization of blood |
| | | collection supplies. |
| | | one was suppress. |
| | | Serum sodium assessments and other |
| | | clinically necessary blood samples take |
| | | priority, therefore, due to restrictions in |
| | | allowable total daily blood volumes based |
| | | on local guidelines and subject age, it may |
| | | not be possible to take more than one PK |
| | | sample per day. If so, the PK sampling |
| | | should be changed to: |
| | | • Day 1: 2 hours post dose (± 5 minutes) |
| | | • Day 2: 8 (± 2) hours post dose (may |
| | | be concurrent with serum sodium or other blood sampling) |
| | | • Day 3 at trough, ie, pre-dose/24 hours |
| | | post prior dose (concurrent with |
| | | serum sodium sample) |
| | | For each subject all samples will be |
| | | collected according to local guidelines and |
| | | best practices for pediatric care. If a |
| | | sample is missing due to limitations in |
| | | allowable blood volumes based on local regulations or local practice this will not |
| | | count as a protocol deviation. |
| 3.7.3.3 | 3.7.3.3.1 Fluid Balance (Intake/Output) | 3.7.3.2.1 Fluid Intake |
| 0.7.0.0 | Fluid intake (both oral and IV) and urine | Fluid intake (both oral and IV) will be |
| | volume will be measured at the times | measured at the times presented in the |
| | presented in the schedule of assessments | schedule of assessments (Section 3.7.1). |
| | (Section 3.7.1). The fluid content of foods | The fluid content of foods with significant |
| | with significant water content (eg, soup) | water content (eg, soup) should be added to |
| | should be added to the total fluid intake. | the total fluid intake. Fluid intake will be |
| | Fluid balance will be monitored per | monitored per institutional guidelines. |
| | institutional guidelines. | 272224 |
| | 3.7.3.3.2 Laboratory Tests | 3.7.3.2.2 Urine Volume |

| Location: | Old Text: | New Text: |
|---|---|---|
| | Urine chemistry will be determined in urine samples that will be collected at the intervals presented in the schedule of assessments, Section 3.7.1. The list of urine chemistry tests to be collected is presented in Table 3.7.4.2-1. All urine voids within a collection interval will be kept refrigerated and at the end of the collection interval, the samples pooled together, the urine volume determined, and an aliquot taken according to instructions from the clinical chemistry laboratory. | Urine volume will be determined in urine samples that will be collected at the intervals presented in the schedule of assessments, Section 3.7.1. All urine voids within a collection interval should be kept refrigerated and pooled according to the size of available collection containers. At the end of the collection interval all samples should be pooled and the urine volume determined. 3.7.3.2.3 Urine Chemistry Urine chemistry will be determined from pooled urine samples collected for the intervals presented in the schedule of assessments, Section 3.7.1. An aliquot will be taken for each collection interval according to the procedures of the local clinical chemistry laboratory. The list of urine chemistry tests to be conducted is presented in Table 3.7.4.2-1. |
| 3.7.4 Safety<br>Assessments<br>3.7.4.1 Adverse<br>Events | • In particular, the following AEs must be actively monitored: absolute serum sodium level ≥ 145 mmol/L, overly rapid rise in serum sodium defined as an increase in serum sodium of > 8mmol/L over a 10-hour period, or a rate of increase in serum sodium that the investigator deems too rapid, neurological symptoms, or other signs or symptoms suggestive of osmotic demyelination (see Section 5.3.1 for more detail). | In addition, active monitoring is required for: • Absolute serum sodium level ≥ 145 mEq/L (mmol/L) or an overly rapid rise in serum sodium level (an increase in serum sodium of |

| Location: | Old Text: | New Text: |
|---|---|---|
| | | 3.7.4.2.1 Serum Osmolality Serum osmolality will be calculated to help guide dosing. Local site personnel will determine serum osmolality using one of the following equations: a) Where Na, glucose, and BUN are measured in mg/dL: Serum Osmolality (mOsm/kg) = 2 Na + BUN / 2.8 + (glucose / 18) b) Where Na, glucose, and urea are |
| | | measured in mmol/L:<br>Serum Osmolality (mOsm/kg) = 2 Na<br>+ glucose + urea |
| 3.7.4.1.1 | Table 3.7.4.2-1 presents the protocol- | Table 3.7.4.2-1 presents required clinical |
| Clinical | required clinical laboratory results (serum | laboratory assessments (serum chemistry, |
| Laboratory<br>Tests | chemistry, hematology, coagulation, urinalysis, and urine chemistry) that will be reported as part of the trial results. Serum cortisol and TSH will be measured at the Screening/Baseline Visit using the remaining blood sample obtained for serum chemistryassessments (Table 3.7-1). | hematology, coagulation, urinalysis, and urine chemistry). All clinical laboratory tests will be performed by local laboratories. Serum cortisol and TSH will be measured during screening using the remaining blood sample obtained for serum chemistryassessments (Section 3.7.1). Uric acid will be measured during screening for calculation of FENa and FE urate. WBC = white blood cell; RBC = red blood cell. In case of limited blood or urine volume availability the bolded assessments take priority. Serum Sodium and liver function tests are essential to the conduct of the trial. Based on previous research in the adult |
| Monitoring of<br>Liver Tran-<br>saminases | polycystic kidney disease population, the expected onset of the elevation is between 3 and 14 months of chronic treatment with tolvaptan. | polycystic kidney disease population, the expected onset of the elevation, if it occurs, is between 3 and 14 months of chronic treatment with tolvaptan. |
| | For a subject that experiences an elevation in AST or ALT that is $\geq 3 \times \text{ULN}$ or whose levels increase $\geq 3$ times their previous observed value, a total bilirubin level should also be evaluated. If the total bilirubin is $\geq 2 \times \text{ULN}$ or $\geq 2$ times their previous observed value, an immediately reportable event (IRE) form with all values listed should be completed and also reported as an AE on the CRFs. See Section 5.4.1 for detailed instructions on how this type of event should be captured. | For a subject who experiences an elevation in AST or ALT that is $\geq 2 \times \text{ULN}$ or whose levels increase $\geq 2$ times their previous observed value, a total bilirubin level should also be evaluated. These elevated values should be confirmed by retesting. If total bilirubin is $\geq 2 \times \text{ULN}$ or $\geq 2$ times their previous observed value, an immediately reportable event (IRE) form with all values listed should be completed and also reported as an AE on the CRFs. See Section 5.4.1 for detailed instructions on how this type of event should be captured. |
| <b>3.7.4.3 Physical</b> | All physical examination assessments | All physical examination assessments |
| Examination | should include assessments of all major | should include assessments of all major |

| Location: | Old Text: | New Text: |
|---|---|---|
| | body systems, including but not limited to, | body systems, including but not limited to, |
| | ears, nose, and throat, the thorax area, | ears, nose, and throat, the thorax area, |
| | abdomen, urogenital, extremities, and skin | abdomen, urogenital, extremities, and skin |
| | and mucosae. Neurological examinations | and mucosae. Neurological examinations |
| | will be performed in an age-appropriate | will be performed in an age-appropriate |
| | manner per Section 3.7.4.4. | manner per Section 3.7.4.3.1 |
| | Body weight will be measured predose each | |
| | day, | Body weight will be measured predose |
| | | each day throughout Treatment Phase A, |
| | | Treatment Phase B and at each clinic visit in Follow-up Phase C |
| 3.7.4.4 Tanner | | Tanner Staging will be completed together |
| Staging | | with the physical examination by the same |
| Staging | | trial affiliated clinician in the most |
| | | inconspicuous manner for the subject as |
| | | possible. Tanner Staging assessment |
| | | consists of 2 domains (pubic hair and |
| | | breast development) for girls and 3 |
| | | domains (pubic hair, penis development, |
| | | and testes development) for boys. The |
| | | investigator will arrive at a single score |
| | | summarizing the domains (not individual |
| | | domain scores) when evaluating the |
| | | subject. |
| 3.7.4.5 Vital | Vital sign data (including supine blood | Vital signs (including supine blood |
| Sign | pressure, heart rate, respiratory rate, and | pressure, heart rate, respiratory rate, and |
| Assessments | temperature) will be performed and | temperature) will be assessed at time points |
| | documented according to Section 3.7.1 of | according to Section 3.7.1 of this protocol. |
| | this protocol. Supine vital signs will be | Supine vital signs will be taken when the |
| | taken when the subject has been lying down | subject has been lying down (bed |
| | (bed positioned < 45 degree angle) for at | positioned < 45 degree angle) for at least 3 |
| | least 3 minutes. All post-baseline | minutes. All assessments for vital signs |
| | assessments for vital signs should be | should be performed around the time of the |
| | performed around the time of the formal | formal hyponatremia assessment (sodium |
| | hyponatremia assessment during tolvaptan | blood draw) during Screening, Treatment |
| | dosing and anytime during the Follow-up | Phase A and Treatment Phase B and |
| | Visits consistent with the timing of other | anytime during the Follow-up Period |
| | trial assessments. All vital sign assessments should be performed prior to | consistent with the timing of other trial assessments. All vital sign assessments |
| | the blood draw at the nominal time point. | should be performed prior to the blood |
| | the blood draw at the nominal time point. | draw at the nominal time point. |
| 3.7.4.6 Fluid | In subjects with chronic hyponatremia, | |
| Restriction | fluid restriction coadministered with | |
| | initiation of treatment with a vaptan has the | |
| | potential to accentuate the rate of sodium | |
| | correction and to cause overly rapid | |
| | correction or over correction of | |
| | hyponatremia. Therefore, during treatment, | |
| | subjects must have access to water and | |
| | maintain fluid intake levels per institutional | |
| | guidelines. Fluid restriction during the first | |
| | 48 hours after discontinuation of tolvaptan | |
| | will be considered rescue therapy. | |
| 3.9 Screen | A screen failure subject is one from whom | A screen failure subject is one from whom |

| Location: | Old Text: | New Text: |
|---|---|---|
| Failures | informed consent/assent (if applicable) is obtained and is documented in writing (ie, the subject's parent or legal guardian signs an ICF), but who is not enrolled into the trial | informed consent/assent (if applicable) has been obtained and is documented in writing (ie, the subject's parent or legal guardian signs an ICF), but who is not enrolled into the trial. If a subject's serum sodium level during the Screening period is $\geq 130$ mEq/L [mmol/L], that subject will be determined a screen failure |
| 3.10 Definition of Completed Subjects | The treatment period is defined as the time period during which subjects are evaluated for primary and/or secondary objectives of the trial irrespective of whether or not the subject actually consumed all doses of the IMP. Subjects who are evaluated at the last scheduled visit during the treatment period will be defined as trial completers. For purposes of this trial, subjects who complete the final Follow-up Visit at 14 days post-randomization will be defined as trial completers. | The treatment period is defined as the time period during which subjects are evaluated for primary and/or secondary objectives of the trial irrespective of whether or not the subject actually consumed all doses of the tolvaptan. For purposes of this trial, subjects who are randomized responders and who complete required trial assessments (including their assigned trial treatment) through the end of the trial will be defined as responder trial completers. For purposes of this trial, subjects who are nonresponders (not randomized) but who complete required trial assessments through the end of the trial will be defined as nonresponder trial completers. Subjects who discontinue tolvaptan prior to the end of Treatment Phase B, but who continue in the trial and complete some or all of their required assessments to the end of the trial, will be considered "early" end of treatment (EEOT) completers. |
| 4.2 Other<br>Restrictions | The use of saline in this population should be closely monitored. The use of hypertonic saline (3%) within 8 hours of the initial screening laboratory collection is prohibited. Please see Section 3.4.3 for the list of prohibited medications. The use of normal saline (0.9%) is allowed during the Screening Period until the beginning of Phase A; normal saline use can resume in Phase C. Subjects should no longer be on maintenance fluids containing normal saline during treatment with tolvaptan. | Other treatment for the purpose of increasing serum sodium, eg with urea, lithium, demeclocycline, conivaptan or tolvaptan, concurrent with dosing of trial medication or within 4 days of qualifying serum sodium assessments at screening is prohibited. The use of saline in this population should be closely monitored. The use of hypertonic saline (3%), including normal saline challenge) within 8 hours of the qualifying screening serum sodium laboratory assessment is prohibited. The use of normal saline (0.9%) is allowed during screening until the beginning of Treatment Phase A; normal saline use can resume in Phase C. Subjects should no longer be on maintenance fluids containing normal saline during treatment with |

| Location: | Old Text: | New Text: |
|---|---|---|
| | | tolvaptan. |
| 5.1 Definitions | Related: There is a reasonable possibility of a causal relationship. Possibly related: There is a reasonable causal relationship between the IMP and the AE. Dechallenge is lacking or unclear. Unlikely related: There is a temporal | IMP Causality: Assessment of causal relationship of an AE to the use of the IMP: Related: There is a reasonable probability or possibility of a temporal and causal relationship between the study drug and the AE. Not Related: There is no temporal or causal relationship to the study drug administration. |
| 5.4 Potential | For a subject who experiences an elevation | The definition of Hy's Law criteria is |
| · | in AST or ALT that is $\geq 3 \times ULN$ or whose levels increase $\geq 3$ times their initial baseline value, a total bilirubin level should also be evaluated. If the total bilirubin is $\geq 2 \times ULN$ or $\geq 2$ times their baseline value, an IRE form should be completed with all values listed and also should be reported as an AE on the CRFs. | provided in Section 5.1. To err on the side of caution Otsuka decided to set a lower threshold for identification of potential Hy's Law cases. For a subject who experiences an elevation in AST or ALT that is $\geq 2 \times$ ULN or whose levels increase $\geq 2$ times their initial baseline value, a total bilirubin level should also be evaluated. Elevated values should be confirmed via retest. If the total bilirubin is $\geq 2 \times$ ULN or $\geq 2$ times their baseline value, an IRE form should be completed with all values listed and also should be reported as an AE on the CRFs. |
| 5.4.1 Liver<br>Transaminase | Management of abnormal liver function test results should be based on the investigator's | |
| Elevations | clinical judgment. A liver function test result that is 3 × ULN is generally accepted as a medically significant occurrence across various medical cultures. For a subject that experiences an elevation in AST or ALT that is ≥ 3 × ULN or whose levels increase ≥ 3 times their initial baseline value in subjects with an elevated baseline value, a total bilirubin level should also be evaluated The following guideline for repeat testing may be used by investigators as a reference for any subject with an ALT or AST ≥ 3 × ULN: 2)Inquiries should be made about symptoms (fatigue, nausea, vomiting, right upper quadrant pain or | investigator's clinical judgment. A liver function test result that is 2 × ULN is generally accepted as a medically significant occurrence across various medical disciplines. For a subject that experiences an elevation in AST or ALT that is ≥ 2 × ULN or whose levels increase ≥ 2 times their initial baseline value in subjects with an elevated baseline value, a total bilirubin level should also be evaluated The following guideline for repeat testing may be used by investigators as a reference for any subject with an ALT or AST ≥ 2 × ULN: 2) Inquiries should be made about |
| | tenderness, fever, and/or rash). | symptoms (fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, and/or rash) and signs like jaundice, |

| Location: | Old Text: | New Text: |
|---|---|---|
| | | yellowish discoloration of sclera, etc |
| <b>5.4.1.1</b> Criteria | A subject must be discontinued from the | A subject must be discontinued from the |
| for Discon- | trial on confirmation of any of the | trial on confirmation of any of the |
| tinuation Due to | following criteria: | following criteria: |
| Liver | | _ |
| Transaminase | 1) ALT or AST $\geq$ 3 × ULN with appearance | 1) ALT or AST $\geq$ 3 × ULN with |
| Elevations | of fatigue, nausea, vomiting, right upper | appearance of fatigue, nausea, vomiting, |
| | quadrant pain or tenderness, fever, rash, | right upper quadrant pain or tenderness, |
| | and/or eosinophilia (> 5%) | fever, rash, and/or eosinophilia (> 5%) and |
| | | signs of jaundice |
| | For this trial, information on AEs will be | For this trial, information on AEs will be |
| Adverse Events | followed for up to 14 days post- | followed for up to 14 days post-last dose |
| | randomization. | for all subjects or until resolution, |
| | | whichever is longer. |
| 5.7.2 Follow-up | This trial requires that subjects be actively | This trial requires that subjects be actively |
| of Post Trial | monitored for SAEs up to 14 days | monitored for SAEs up to 14 days post-last |
| Serious Adverse | post-randomization. | dose or until resolution of the SAE, |
| Events | | whichever is longer. |
| 6.1 Pharmaco- | Tolvaptan plasma concentrations will be | Tolvaptan and metabolite plasma |
| kinetic Analysis | summarized using descriptive statistics (n, | concentrations will be summarized using |
| | median, mean, standard deviation [SD], | descriptive statistics (n, median, mean, |
| | percent coefficient of variation [CV], | standard deviation [SD], percent coefficient |
| | minimum, and maximum) by dose group | of variation [CV], minimum, and |
| | and time point. | maximum) by dose group and time point. |
| 6.2 Pharmaco- | Fluid intake and the calculated value of | Fluid intake and the calculated value of |
| dynamic | fluid balance will be summarized for each | fluid balance will be summarized for each |
| Analysis | 6-hour period on Days 1 and 2 (Phase A) | 6-hour period and for the 24-hour daily |
| | using descriptive statistics | interval on Days 1 and 2 in Treatment |
| | | Phase A using descriptive statistics |
| | Urine osmolality and urine creatinine, | |
| | potassium, uric acid, and sodium | Urine osmolality and urine creatinine, |
| | concentrations will be summarized by | potassium, and sodium concentrations will |
| | collection interval and for zero to 24 hours | be summarized by collection interval and |
| | on Days 1 and 2 (Phase A) using | for zero to 24 hours on Days 1 and 2 in |
| | descriptive statistics | Treatment Phase A using descriptive |
| | | statistics |
| | | Correlations between tolvaptan AUC |
| | | values and urine output on Day 1 may be |
| <b>7116</b> | A 4-4-1 - C70 1 | explored graphically |
| 7.1.1 Sample | A total of 70 randomized subjects will | A total of 70 randomized subjects will |
| Size for Efficacy | provide 90% power to detect a treatment | provide 90% power to detect a treatment |
| | difference of 4 mmol/L in change in serum | difference of 4 mEq/L (mmol/L) in change |
| | sodium from randomization (at the end of | in serum sodium from Day 2 (or 2a) at the |
| | Day 2/3 [Phase A]) to the end of Day 4/5 (2 | end of Treatment Phase A to the end of |
| | | Treatment Phase B using a 2-sided alpha of |
| | 2-sided alpha of 0.05. An SD of 5 in change of serum sodium was used for the | 0.05. An SD of 5 in change of serum sodium was used for the sample size |
| | sample size calculation. After the end of | calculation. After the end of Treatment |
| | treatment at Day 2/3, subjects will be randomized at a ratio of 1:1 to either | Phase A at Day 2 (or 2a), subjects will be randomized at a ratio of 1:1 to either |
| | continue treatment with tolvaptan for 2 | continue treatment with tolvaptan for 2 |
| | additional days (Late Withdrawal) or to | additional days (Late Withdrawal) or to |
| | discontinue tolvaptan treatment (Early | discontinue tolvaptan treatment (Early |
| | discontinue torvapian treatment (Early | uiscommue torvapian treatment (Earry |

| Location: | Old Text: | New Text: |
|---|---|---|
| | Withdrawal). Sample size re-estimation | Withdrawal). Sample size re-estimation |
| | will be conducted when 90% of the subjects | |
| | finish (complete or discontinue) the trial. | subjects finish (complete or discontinue) |
| | | the trial. |
| 7.4.2.2 Safety | Other secondary endpoints include: | Other secondary endpoints include: |
| | <ul> <li>Percentage of subjects with overly</li> </ul> | <ul> <li>Percentage of subjects with overly</li> </ul> |
| | rapid increase in serum sodium (≥ | rapid increase in serum sodium level |
| | 12mmol/L in 24 hours after the first | |
| | dose). | ). |
| | • Percentage of subjects requiring rescue | |
| | medication during Phase A and Phase | hours post-last dose to 7 days post-last |
| | B of the trial. | dose. |
| | • Change in serum sodium from 24 hours | |
| | post-last dose to 14 days | therapy (other than fluid restriction) |
| | post-randomization. | during Treatment Phase A and |
| | Vital signs, blood pressure, clinical | Treatment Phase B. |
| | laboratory tests, and body weight. | Percentage of subjects requiring fluid |
| | | restriction during Treatment Phase A |
| | | and Treatment Phase B. |
| | | Other secondary safety outcomes to be |
| | | assessed are presented in Section |
| | | 3.5.3.1 (Vital signs, blood pressure, |
| | | clinical laboratory tests, body weight, |
| 7.4.2 | Nouvelegical agamination data will be | and neurological examinations) |
| 7.4.3 | Neurological examination data will be | The change in serum sodium concentration |
| Exploratory Outcome | presented in the data listings. | in nonresponders continuing on tolvaptan therapy by change from baseline at the end |
| Analysis | | of Treatment Phase B compared to the end |
| Allalysis | | of Treatment Phase A will be analyzed |
| | | using a paired Student's t-test. |
| | | The procedure for the analysis of data for |
| | | the neurocognitive and QoL assessments |
| | | will be provided in the SAP. |
| | | The analysis for the following exploratory |
| | | PD endpoints is described in Section 6.2: |
| | | • In all subjects, 24-hour excretion of |
| | | sodium, creatinine, and osmolality on Days |
| | | 1 and 2 |
| | | • 24-hour sodium clearance on Day 1 |
| 14 References | | 26 U.S. Food and Drug Administration. |
| | | Guidance for Industry. Drug-induced |
| | | liver injury: premarketing clinical |
| | | evaluation [report on the internet]. |
| | | 2009 Jul [cited 15 Feb 2014]; |
| | | Available from: |
| | | http://www.fda.gov/downloads/Drugs/ |
| | | GuidanceComplianceRegulatoryInfor |
| | | mation/Guidances/UCM174090.pdf. |
| | | 27 U.S. Food and Drug Administration. |
| | | [available on the internet, last updated |
| | | 22Jan2014; cited 14Feb2014]. Available from: |
| | | http://www.fda.gov/Drugs/ |
| | | ScienceResearch/ResearchAreas/ucm0 |
| | | Science Research/Research Areas/ucino |

| Location: | Old Text: | | New Text: | |
|---|---|---|---|---|
| | | | 71471.htm | |
| Appendix 1: | Country | Safety Fax Numbers | Country | Safety Fax Numbers |
| Names of | United | (primary) or | Australia | |
| Sponsor | States | (alternative) | | |
| Personnel: IRE | Argentina | | Belgium | |
| | Australia | | Canada | (primary) |
| | | <u> </u> | | or |
| | | | | (alternative) |
| | Belgium | | Czech Republic | _ |
| | Canada | (primary) or | Germany | |
| | | (alternative) | | |
| | Colombia | | Italy | _ |
| | Czech | | Netherlands | |
| | Republic | | | |
| | Finland | | Peru | |
| | France | | Poland | |
| | Georgia | No toll free number available; | Romania | |
| | | please dial | | |
| | | (primary) or | | |
| | | (alternative) | | |
| | Germany | | Spain | |
| | Hong Kong | | Turkey | No toll free number |
| | | | | available; please dial |
| | | | | (primary) |
| | | | | or |
| | | | | (alternative) |
| | Israel | | United | |
| | | | Kingdom | |
| | Italy | | United States | (primary) |
| | | | | or |
| | | | | (alternative) |
| | Korea | | | |
| | Latvia | | | |
| | Malaysia | | | |
| | Mexico | | | |
| | Netherlands | | | |
| | Philippines | | | |
| | Peru | | | |
| | Poland | | | |
| | Romania | | | |
| | Russia | | | |
| | Serbia | | | |
| | Singapore | | | |
| | South Africa | | | |
| | Spain | | | |
| | Taiwan | | | |
| | Thailand | | | |
| | Turkey | No toll free number available; | | |
| | | please dial | | |
| | | (primary) or | | |
| | | (alternative) | | |

| Location: | Old Text: | New Text: |
|---|---|---|
| | Ukraine | |
| | United | |
| | Kingdom | |
| | • | |
| Medical | | |
| Monitor: | | 2201 December Court Color (00) |
| | | 3201 Beechleaf Court, Suite 600<br>Raleigh, North Carolina 27604 USA |
| | Phone ; Mobile | Phone |
| | , week | Mobile |
| | E-Mail | E-Mail |
| | Back-up: | |
| | Phone ; Mobile | |
| | E-Mail | |
| | E /D / CW 11 | |
| | Europe/Rest of World: | |
| | Phone | |
| | E-Mail | |
| Institutions | Study Communications & Patient/Site | Study Communications & Patient/Site |
| Concerned | Support DDK Worldwide | Support Mathema Madia Cross |
| With the Trial: | BBK Worldwide<br>117 Kendrick Street, Suite 600 | Mathews Media Group<br>700 King Farm Boulevard, Suite 500 |
| | Needham, Massachusetts 02494, US | Rockville, MD 20850, USA |
| | Phone: | Phone: |
| | Central Laboratory (non-PK) | Clinical Laboratory Supplies |
| | Covance Central Laboratory Services | Covance Central Laboratory Services |
| | Covance Central Laboratory Services<br>8211 SciCor Drive | Covance Central Laboratory Services<br>8211 SciCor Drive |
| | Covance Central Laboratory Services<br>8211 SciCor Drive<br>Indianapolis, Indiana 46214, US | Covance Central Laboratory Services<br>8211 SciCor Drive<br>Indianapolis, Indiana 46214, USA |
| | Covance Central Laboratory Services<br>8211 SciCor Drive | Covance Central Laboratory Services<br>8211 SciCor Drive<br>Indianapolis, Indiana 46214, USA<br>Phone: |
| | Covance Central Laboratory Services<br>8211 SciCor Drive<br>Indianapolis, Indiana 46214, US | Covance Central Laboratory Services 8211 SciCor Drive Indianapolis, Indiana 46214, USA Phone: Neurocognitive Battery |
| | Covance Central Laboratory Services<br>8211 SciCor Drive<br>Indianapolis, Indiana 46214, US | Covance Central Laboratory Services 8211 SciCor Drive Indianapolis, Indiana 46214, USA Phone: Neurocognitive Battery Cogstate, Ltd. |
| | Covance Central Laboratory Services<br>8211 SciCor Drive<br>Indianapolis, Indiana 46214, US | Covance Central Laboratory Services 8211 SciCor Drive Indianapolis, Indiana 46214, USA Phone: Neurocognitive Battery |

Protocol 156-08-276

| Location: | Old Text: | New Text: |
|-----------|-----------|-----------|
| | | Phone: |

**ADDITIONAL RISK TO THE SUBJECT:** There is no additional risk to the subjects.

Protocol 156-08-276

**Amendment Number:** 3

**Issue Date:** 26 Feb 2015

## **PURPOSE:**

- Implementation of additional serum sodium testing during drug titration to align with the current EU label (SmPC) for the adult indication of hyponatremia. We are adding safety testing for serum sodium at interim time points during titration with the option of using a point of care device to minimize impact on total blood volume required for the trial.
- Clarification of the "baseline" assessment for trial qualification.
- Additional background data from non-clinical juvenile toxicity studies.
- Updates to clarify the titration and rescue therapy schematic.
- Clarify roll-over into extension study 156-11-294.
- Implementation of a suspension formulation for short-term use in hospitalized subjects.
- Implementation of an optional swallow test for the tablet formulation.

## **BACKGROUND:**

This protocol serves as the single trial for the Pediatric Written Request with the FDA and the Pediatric Research Equity Act (PREA) requirement for the US. The FDA has agreed to the current version of the protocol and updates have been made to address further comments from the FDA, the Medicines and Healthcare Products Regulatory (MHRA), and other regulatory agencies.

## **MODIFICATIONS TO PROTOCOL:**

**Sectional Revisions:** changes made to specific sections of the protocol are listed in the table below.

| Location | Old Text | Updated Text |
|---|---|---|
| Title Page: | Issue Date: 03 Jul 2013 Date of Amendment 1: 04 Nov 2013 Date of Amendment 2: 19 May 2014 | Issue Date: 03 Jul 2013 Date of Amendment 1: 04 Nov 201 Date of Amendment 2: 19 May 2014 Date of Amendment 3: 26 February 2015 |
| Protocol Synopsis<br>Trial Design: | This is an open-label, multicenter, multiple-dose, randomized withdrawal, parallel-group trial of tolvaptan in children and adolescent subjects hospitalized with euvolemic or hypervolemic hyponatremia. | This is an open-label, multicenter, multiple-dose, randomized withdrawal, parallel-group trial of tolvaptan in children and adolescent subjects hospitalized with euvolemic or hypervolemic hyponatremia. |
| | The trial will be conducted in two stages. The first stage will be conducted using the available tablet formulation of tolvaptan whereas the second stage will expand to include the use of a suspension once that formulation becomes available. | Since hyponatremia in this patient population can often be transient and/or may be secondary to hypovolemic states, potential subjects will be screened for hyponatremic histories as well as clinically evaluated to rule out such cases. For the purpose of this protocol, persistent hyponatremia will be defined as serum sodium assessments < 130 mEq/L (mmol/L) documented as present for at |
| | Since hyponatremia in this patient population can often be transient and/or may be secondary to hypovolemic states, potential subjects will be screened for hyponatremic histories as well as clinically evaluated to rule out such cases. For the purpose of this protocol, persistent hyponatremia will be defined as serum sodium assessments < 130 mEq/L (mmol/L) documented as present for at least 48 hours. Specifically, subjects must have at least 2 documented serum sodium assessments < 130 mEq/L (mmol/L) drawn at least 12 hours apart. These values can be documented using historical values previously obtained as per standard of care. A third | least 48 hours. Specifically, subjects must have at least 2 documented serum sodium assessments < 130 mEq/L (mmol/L) drawn at least 12 hours apart. These values can be documented using historical values previously obtained as per standard of care. A third (immediate [STAT]) serum sodium assessment < 130 mEq/L (mmol/L), which will serve as the baseline value for final trial qualification and clinical management strategy, is to be obtained within 2-4 hours prior to the first dose of tolvaptan. Additional qualification assessments will be performed as per etiology of hyponatremia. The first dose of tolvaptan will be administered upon successful completion of all screening |
| | (immediate [STAT]) serum sodium assessment < 130 mEq/L (mmol/L), which will serve as the baseline value for efficacy | procedures. |

| Location | Old Text | Updated Text |
|---|---|---|
| | endpoints, is to be obtained within 2-4 hours prior to the first dose of tolvaptan. Additional qualification assessments will be performed as per etiology of hyponatremia. The first dose of tolvaptan will be administered upon successful completion of all screening procedures. All Subjects All subjects will have serum sodium levels measured at 8, 12, and 24 hours post-first dose and thereafter every 12 hours through completion of Treatment Phase B. | All Subjects All subjects will have serum sodium levels measured at 8, 12, and 24 hours post-first dose and thereafter every 12 hours through completion of Treatment Phase B. In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment will be obtained on Day 1 at 4 to 6 hours postdose and at 18 hours postdose. This sodium safety assessment will be repeated at 6 and 18 hours postdose each day for the remainder of titration. |
| Protocol Synopsis<br>Subject Population: | This trial will include up to 100 male and female subjects aged $\geq 4$ weeks (or $\geq 44$ weeks adjusted gestational age) to < 18 years who have been diagnosed with euvolemic or hypervolemic hyponatremia (< 130 mEq/L [mmol/L]) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). Age groups will be enrolled such that 50% of these subjects will be < 10 years old and at least 25% of subjects < 6 years old. | This trial will enroll approximately 100 male and female subjects to get approximately 70 randomized subjects aged ≥ 4 weeks (or ≥ 44 weeks adjusted gestational age) to < 18 years who have been diagnosed with euvolemic or hypervolemic hyponatremia (< 130 mEq/L [mmol/L]) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). Age groups will be enrolled such that at least 50% of these subjects will be < 10 years old and at least 25% of subjects < 6 years old. |
| Protocol Synopsis<br>Inclusion/Exclusion<br>Criteria: | Key inclusion criteria: Persistent euvolemic or hypervolemic hyponatremia defined as being documented as present for at least 48 hours, | Key inclusion criteria: Persistent euvolemic or hypervolemic hyponatremia defined as being documented as present for at least 48 hours, evidenced by at |

| Location | Old Text | Updated Text |
|---|---|---|
| | evidenced by at least 2 serum sodium assessments | least 2 serum sodium assessments < 130 mEq/L (mmol/L) drawn |
| | < 130 mEq/L (mmol/L) drawn at least 12 hours apart (these | at least 12 hours apart (these values can be documented using |
| | values can be documented using historical values previously | historical values previously obtained per standard of care); a third |
| | obtained per standard of care); a third (STAT) serum sodium | (STAT) serum sodium assessment < 130 mEq/L (mmol/L), which |
| | assessment < 130 mEq/L (mmol/L), which will serve as the | will serve as the baseline value for final trial qualification and |
| | baseline value for efficacy endpoints, is to be obtained 2-4 | clinical management strategy, is to be obtained 2-4 hours prior to |
| | hours prior to the first dose of tolvaptan | the first dose of tolvaptan |
| | Key exclusion criteria: | Key exclusion criteria: |
| | Use of potent cytochrome P450 (CYP) 3A4 inhibitors in | Use of potent cytochrome P450 (CYP) 3A4 inhibitors in subjects |
| | subjects ≤ 50 kg or moderate CYP3A4 inhibitors in subjects < | < 10 kg or moderate CYP3A4 inhibitors in subjects < 6 kg |
| | 20 kg | |
| Protocol Synopsis | The trial will be conducted at up to 50 centers globally. | The trial will be conducted at approximately 60 centers globally. |
| Trial Sites: | | |
| Protocol Synopsis | Tolvaptan will initially be supplied as 3.75-, 7.5-, 15-, and | Tolvaptan will be supplied as 3.75-, 7.5-, 15-, and 30-mg |
| Investigational<br>Medicinal Product, | 30-mg spray-dried tablets. Upon the availability of an oral | spray-dried tablets and, where approved, as a 1 mg/mL (0.1% w/v) |
| Dose, Formulation, | suspension formulation, the protocol will be amended to | suspension. |
| Mode of | reflect additional dosing options. | |
| Administration: | | |
| | | Tolvaptan tablets will be administered once daily, orally with a |
| | Tolvaptan will be administered once daily orally with a dose | dose proportional amount of water. Doses of ≥ 15 mg tolvaptan |
| | proportional amount of water. Doses of $\geq 15$ mg tolvaptan | will be given with 240 mL of water, 7.5 mg tolvaptan will be |
| | will be given with 240 mL of water, 7.5 mg tolvaptan will be | given with 120 mL of water, and 3.75 mg of tolvaptan will be |
| | given with 120 mL of water, and 3.75 mg of tolvaptan will be | given with 60 mL of water. The treatment duration will be up to |
| | given with 60 mL of water. The treatment duration will be up | 5 days. Any initiation or titration of tolvaptan must occur in a |
| | to 5 days. Any initiation or titration of tolvaptan must occur | hospital setting. |
| | in a hospital setting. | |

| Location | Old Text | Updated Text |
|---|---|---|
| | | with possible up-titration to 30- and 60-mg doses. |
| Protocol Synopsis<br>Trial Duration: | Overall trial duration of enrollment is expected to be 36 months with an enrollment rate of 33 subjects per year. Nominal trial duration for each subject is up to 21 days. Treatment duration is up to 5 days with ongoing monitoring of serum sodium levels. A serum sodium assessment and AE follow-up visit will be performed 7 (± 1) days post-last dose. A final safety follow-up telephone contact or visit will be performed 14 (+ 2) days post-last dose. | Overall trial duration of enrollment is expected to be approximately 3 years with an enrollment rate of approximately 33 subjects per year. Nominal trial duration for each subject is up to 21 days. Treatment duration is up to 5 days with ongoing monitoring of serum sodium levels. A serum sodium assessment and AE follow-up visit will be performed 7 (± 1) days post-last dose. A final safety follow-up telephone contact or visit will be performed 14 (+ 2) days post-last dose. |
| List of Abbreviations and Definitions of Terms: | Added 5 terms: EMA, MHRA, PDCO, PREA, and WOCBP | EMA European Medicines Agency MHRA Medicines and Healthcare Products Regulatory PDCO Paediatric Committee PREA Pediatric Research Equity Act WOCBP Women of child-bearing potential |
| 1.1.1 Juvenile Animal | A 1-week dose range-finding study was conducted in rat pups | A 1-week dose range-finding study was conducted in rat pups at 4 |
| <b>Toxicity Data:</b> | at 4 or 7 days of age and results showed tolvaptan to be lethal | or 7 days of age and results showed tolvaptan to be lethal at 1000 |
| | at 1000 mg/kg/day and tolerable at 100 mg/kg/day and lower. | mg/kg/day and tolerable at 100 mg/kg/day and lower. |
| | | In another study, male and female rat pups at 4 days of age were orally administered tolvaptan for 9 weeks at doses of 10, 30, and 100 mg/kg/day. Similar to the above study, pharmacologically mediated changes were noted in urine volume, water consumption, and urine electrolytes at all doses. Dilated renal pelvis considered to be attributable to increased urine volume during very early infancy was noted in males at 30 mg/kg/day and higher and females at 100 mg/kg/day. Toxicities were noted at 100 mg/kg/day, including death in one male, suppressed body weight gain and food consumption in males and females, and delayed |

| Location | Old Text | Updated Text |
|---|---|---|
| | | balanopreputial separation and prolonged prothrombin time in |
| | | males. Except for prolonged prothrombin time, all changes noted |
| | | during the administration period showed reversibility after a 4- |
| | | week recovery period. The no observed adverse effect level in |
| | | both males and females was judged to be 30 mg/kg/day. 16 |
| 1.2.1 | Since inception of the program, a total of 45 phase 1 trials | Since inception of the program, a total of 53 clinical |
| Pharmacokinetics: | have been completed with tolvaptan (as of 31 Mar 2013) in | pharmacology trials have been completed with tolvaptan (as of 11 |
| | healthy subjects or special populations in Argentina, China, | Jul 2013) in healthy subjects or special populations in Argentina, |
| | Japan, Republic of Korea, the United Kingdom (UK), and the US. 16 | China, Japan, Republic of Korea, the United Kingdom (UK), and the US. 16 |
| | Following IV dosing, the terminal-phase elimination half-life | In healthy subjects, following IV dosing, the terminal-phase |
| | $(t_{1/2,z})$ of tolvaptan is about 3 hours. Following single oral | elimination half-life $(t_{1/2,z})$ of tolvaptan is about 3 hours. |
| | tablet doses, the $t_{1/2,z}$ of tolvaptan increases with increasing | Following single oral tablet doses, the $t_{1/2,z}$ of tolvaptan increases |
| | dose with mean values around 3 hours for a 15-mg dose and | with increasing dose with mean values around 3 hours for a 15-mg |
| | 12 hours for 120- to 480-mg doses. Tolvaptan is very | dose and 12 hours for 120- to 480-mg doses. Tolvaptan is very |
| | insoluble, with solubility being 0.00005 w/v% at 25°C and is | insoluble, with solubility being 0.00005 w/v% at 25°C and is pH |
| | pH independent. At lower doses, tolvaptan is mostly | independent. At lower doses, tolvaptan is mostly absorbed from |
| | absorbed from the upper GI tract so the decline of the terminal | the upper GI tract so the decline of the terminal portion of the |
| | portion of the concentration curve reflects elimination process | concentration curve reflects elimination process only. With |
| | only. With increasing dose, there is continued absorption of | increasing dose, there is continued absorption of tolvaptan from |
| | tolvaptan from the GI tract such that the rate of decline of the | the GI tract such that the rate of decline of the terminal portion of |
| | terminal portion of the concentration curve is reflective of | the concentration curve is reflective of both absorption and |
| | both absorption and elimination processes. <sup>16</sup> | elimination processes. <sup>16</sup> |
| | The limited early absorption of tolvaptan is exemplified by | The limited early absorption of tolvaptan is exemplified by the |
| | the fact that the maximum (peak) plasma concentration ( $C_{max}$ ) | fact that the maximum (peak) plasma concentration (C <sub>max</sub> ) values |
| | values show less than dose proportional increases from 30 to | show less than dose proportional increases from 30 to 240 mg and |
| | 240 mg and then a plateau at doses from 240 to 480 mg. | then a plateau at doses from 240 to 480 mg. Despite the changes |

| Location | Old Text | Updated Text |
|---|---|---|
| | Despite the changes in tolvaptan absorption, tolvaptan AUC | in tolvaptan absorption, tolvaptan AUC values increase |
| | values increase proportionally with increasing dose and | proportionally with increasing dose and apparent clearance of drug |
| | apparent clearance of drug from plasma after extravascular | from plasma after extravascular administration (CL/F) values are |
| | administration (CL/F) values are unchanged for single doses | unchanged for single doses of 30 to 480 mg. 16 |
| | of 30 to 480 mg. <sup>16</sup> | Tolvaptan concentrations do not accumulate following once daily |
| | Tolvaptan concentrations do not accumulate following once | dosing. Following 300-mg doses, C <sub>max</sub> and AUC during the |
| | daily dosing. Following 300-mg doses, C <sub>max</sub> and AUC during | dosing interval at steady state (AUC $_{\tau}$ ) were only 4.2- and 6.4-fold |
| | the dosing interval at steady state (AUC $_{\tau}$ ) were only 4.2- and | higher, respectively, when compared with the 30-mg dose. This |
| | 6.4-fold higher, respectively, when compared with the 30-mg | indicates bioavailability decreases with increasing dose. Mean |
| | dose. This indicates bioavailability decreases with increasing | (range) absolute bioavailability of tolvaptan when administered as |
| | dose. Mean (range) absolute bioavailability of tolvaptan | a 30-mg tablet was 56% (42% to 80%). |
| | when administered as a 30-mg tablet was 56% (42% to 80%). | In healthy subjects, tolvaptan pharmacokinetics following a 15 mg |
| | Trials in subjects with hyponatremia secondary to liver | dose as a 1mg/mL suspension shows a more rapid absorption (the |
| | disease showed that following a single oral dose, tolvaptan | median $t_{max}$ is shorter, 1.00 versus 2.00 hours respectively), when |
| | concentrations increase dose proportionally from 5 to 60 mg. | compared to a 15 mg tablet. The geometric mean ratio (90% CI), |
| | The clearance following single oral doses of tolvaptan was | for suspension over the tablet, for $C_{max}$ is 1.614 (1.484 to 1.754) |
| | independent of the dose and similar to clearance in healthy | but AUC is unchanged. |
| | subjects. Following multiple oral doses, tolvaptan concentrations accumulated 2-fold and clearance was decreased about 50%. <sup>16</sup> | Trials in subjects with hyponatremia secondary to liver disease showed that following a single oral dose, tolvaptan concentrations increase dose proportionally from 5 to 60 mg. The clearance |
| | Once a day dosage regimen trials in CHF subjects with extracellular volume expansion showed that tolvaptan | following single oral doses of tolvaptan was independent of the dose and similar to clearance in healthy subjects. Following |
| | concentrations increased less than proportionally with dose | multiple oral doses, tolvaptan concentrations accumulated 2-fold |
| | upon multiple dosing regimens (10, 15, 30, 60, 90, and 120 | and clearance was decreased about 50%. 16 |
| | mg once daily for 13 days) in this subject population. The $t_{1/2,z}$ and CL/F were unchanged across dose groups. Compared to healthy subjects, the disposition of tolvaptan is | Once a day dosage regimen trials in CHF subjects with extracellular volume expansion showed that tolvaptan concentrations increased less than proportionally with dose upon |

| Location | Old Text | Updated Text |
|---|---|---|
| | slower with longer $t_{1/2,z}$ (7.8 to 11.1 hours) and smaller CL/F | multiple dosing regimens (10, 15, 30, 60, 90, and 120 mg once |
| | (0.9 to 3.3 mL/min/kg). The $C_{max}$ was 2- to 2.5-fold greater | daily for 13 days) in this subject population. The $t_{1/2,z}$ and CL/F |
| | than that of healthy subjects (at 60- and 90-mg doses). The | were unchanged across dose groups. Compared to healthy |
| | median volume of distribution following extravascular | subjects, the disposition of tolvaptan is slower with longer $t_{1/2,z}$ |
| | administration of tolvaptan ranged from 1 to 2.5 L/kg and was | (7.8 to 11.1 hours) and smaller CL/F (0.9 to 3.3 mL/min/kg). The |
| | not different from healthy subjects. 16 | C <sub>max</sub> was 2- to 2.5-fold greater than that of healthy subjects (at |
| | Tolvaptan is a weak substrate for cytochrome P450 (CYP) | 60- and 90-mg doses). The median volume of distribution |
| | 3A4 and has no inhibitory activity at CYP3A4. Tolvaptan | following extravascular administration of tolvaptan ranged from 1 |
| | administration does not produce clinically significant changes | to 2.5 L/kg and was not different from healthy subjects. 16 |
| | in amiodarone, warfarin (or its 7-hydroxy and 10-hydroxy | Tolvaptan is a sensitive substrate for cytochrome P450 (CYP) 3A4 |
| | metabolites), lovastatin, furosemide, or hydrochlorothiazide | and has no inhibitory activity at CYP3A4. Tolvaptan |
| | plasma concentrations. Steady state digoxin concentrations | administration does not produce clinically significant changes in |
| | were increased approximately 20% (as determined by | amiodarone, warfarin (or its 7-hydroxy and 10-hydroxy |
| | $AUC_{\tau}$ ). <sup>16</sup> | metabolites), lovastatin, furosemide, or hydrochlorothiazide |
| | When administered with the potent CYP3A4 inhibitor | plasma concentrations. Steady state digoxin concentrations were |
| | ketoconazole, the ketoconazole + tolvaptan/tolvaptan alone | increased approximately 20% (as determined by $AUC_{\tau}$ ). <sup>16</sup> |
| | ratio for tolvaptan mean C <sub>max</sub> and AUC from time zero to | When administered with the potent CYP3A4 inhibitor |
| | infinity values were 3.48 and 5.40, respectively. Therefore, a | ketoconazole, the ketoconazole + tolvaptan/tolvaptan alone ratio |
| | 4-fold reduction in tolvaptan dose is recommended when | for tolvaptan mean $C_{max}$ and AUC from time zero to infinity |
| | initiating tolvaptan therapy in subjects using potent CYP3A4 | values were 3.48 and 5.40, respectively. Therefore, a 4-fold |
| | inhibitors and a 2-fold reduction in tolvaptan dose is | reduction in tolvaptan dose is recommended when initiating |
| | recommended for subjects using moderate CYP3A4 | tolvaptan therapy in subjects using potent CYP3A4 inhibitors and |
| | inhibitors. Lovastatin increases tolvaptan C <sub>max</sub> by | a 2-fold reduction in tolvaptan dose is recommended for subjects |
| | approximately 20% but CL/F is unchanged. Tolvaptan C <sub>max</sub> | using moderate CYP3A4 inhibitors. Lovastatin increases |
| | and AUC calculated to the last observable concentration at | tolvaptan C <sub>max</sub> by approximately 20% but CL/F is unchanged. |
| | time t (AUC <sub>t</sub> ) are increased 1.9- and 1.6-fold, respectively, | Tolvaptan C <sub>max</sub> and AUC calculated to the last observable |
| | when tolvaptan is coadministered with grapefruit juice. | concentration at time t (AUC <sub>t</sub> ) are increased 1.9- and 1.6-fold, |
| | Following coadministration with 600 mg once daily rifampin | respectively, when tolvaptan is coadministered with grapefruit |

| Location | Old Text | Updated Text |
|---|---|---|
| | at steady state, tolvaptan $C_{\text{max}}$ and $AUC_{\text{t}}$ are decreased 83% | juice. Following coadministration with 600 mg once daily |
| | and 87%, respectively. 16 | rifampin at steady state, tolvaptan C <sub>max</sub> and AUC <sub>t</sub> are decreased |
| | When 30- or 60-mg doses were given following a standard | 83% and 87%, respectively. 16 |
| | high-fat, high-calorie meal, no clinically significant | When 30- or 60-mg tablet doses were given following a standard |
| | differences in urine output were observed. <sup>32,33</sup> | high-fat, high-calorie meal, no clinically significant differences in urine output were observed. 32,33 |
| | | Following multiple oral doses, the tolvaptan metabolite DM-4103 was found to accumulate. This metabolite has no pharmacological activity and has shown an acceptable toxicity profile. The metabolite has not been shown to accumulate in nonclinical toxicokinetic studies; however, in a 26-week study in rats, DM-4103 plasma concentrations greater than those expected at the dose used in this trial revealed no evidence of time-dependent toxicological effects. <sup>13</sup> |
| 1.2.2 | Tolvaptan increases urine excretion rate at concentrations | 1.2.2 Pharmacodynamics |
| Pharmacodynamics: | around 20 ng/mL and maximal urine excretion rates are | |
| | reached between 100 and 150 ng/mL. A single oral dose trial | |
| | in healthy subjects using doses from 60 to 240 mg showed | Tolvaptan increases urine excretion rate at concentrations around |
| | that there were 1) no further increases in urine excretion rate | 20 ng/mL and maximal urine excretion rates are reached between |
| | with doses beyond 180 mg; 2) no further increases in zero to | 100 and 150 ng/mL. A single oral dose trial in healthy subjects |
| | 24 hour urine excretion with doses beyond 180 mg; and 3) as | using doses from 60 to 240 mg showed that there were 1) no |
| | dose was increased, increases in urine excretion were | further increases in urine excretion rate with doses beyond 180 |
| | sustained over time. Tolvaptan elevated electrolyte-free water | mg; 2) no further increases in zero to 24 hour urine excretion with |
| | clearance to a positive value, increased serum sodium and | doses beyond 180 mg; and 3) as dose was increased, increases in |
| | serum osmolality, and increased plasma AVP concentrations | urine excretion were sustained over time. Tolvaptan elevated |
| | and renin activity, but no dose-related increases were | electrolyte-free water clearance to a positive value, increased |

| Location | Old Text | Updated Text |
|---|---|---|
| | observed for any other parameter. <sup>16</sup> | serum sodium and serum osmolality, and increased plasma AVP |
| | Following multiple oral doses, the tolvaptan metabolite DM- | concentrations and renin activity, but no dose-related increases |
| | 4103 was found to accumulate. This metabolite has no | were observed for any other parameter. <sup>16</sup> |
| | pharmacological activity and has shown an acceptable toxicity | When compared to a 15-mg spray-dried tablet, the |
| | profile. The metabolite has not been shown to accumulate in | pharmacodynamic profiles of urine excretion rate, cumulative |
| | nonclinical toxicokinetic studies; however, in a 26-week study | urine volume, free water clearance, urine osmolality, and serum |
| | in rats, DM-4103 plasma concentrations greater than those | sodium were not different for 15-mg of the suspension. 16 |
| | expected at the dose used in this trial revealed no evidence of | Details of the currently available PK/PD data for the compound |
| | time-dependent toxicological effects. 16 | are available in the investigator's brochure (IB). <sup>16</sup> |
| | Details of the currently available PK/PD data for the | |
| | compound are available in the investigator's brochure (IB). 16 | |
| 1.3 Known and | As of 31 Mar 2013, 6,794 adult subjects have been exposed to | As of 31 Mar 2013, 6,794 adult subjects have been exposed to oral |
| Potential Risks and Benefits: | oral doses of tolvaptan in 82 completed or terminated | doses of tolvaptan spray-dried tablets in 82 completed or |
| Delicitis: | tolvaptan trials in the US, Europe, South America, and Asia: | terminated tolvaptan trials in the US, Europe, South America, and |
| | 1,047 healthy subjects, 37 subjects with renal impairment | Asia: 1,047 healthy subjects, 37 subjects with renal impairment |
| | (phase 1 trial), 3,115 subjects in trials for CHF, 425 subjects | (phase 1 trial), 3,115 subjects in trials for CHF, 425 subjects in |
| | in trials for hyponatremia, 961 subjects in the pivotal | trials for hyponatremia, 961 subjects in the pivotal long-term |
| | long-term ADPKD trial, 137 subjects in short-term trials for | ADPKD trial, 137 subjects in short-term trials for ADPKD or |
| | ADPKD or renal impairment, 217 subjects with cardiac | renal impairment, 217 subjects with cardiac edema, and |
| | edema, and 855 subjects with hepatic edema. Additionally, | 855 subjects with hepatic edema. Fourteen healthy adult subjects |
| | 14 healthy adult subjects were exposed to a single 1-mg IV | were exposed to a single 1-mg IV dose of tolvaptan in a phase 1 |
| | dose of tolvaptan in a phase 1 bioavailability trial (Trial 156- | bioavailability trial (Trial 156-05-254) in the US.1 <sup>6</sup> As of 31 Mar |
| | 05-254) in the US. <sup>16</sup> | 2014, additionally, 14 healthy adult subjects were also exposed to |
| | The most commonly reported treatment-emergent adverse | the tolvaptan suspension formulation. |
| | events (TEAEs; > 10% and greater than placebo) in healthy | The most commonly reported treatment-emergent adverse events |

| Location | Old Text | Updated Text |
|---|---|---|
| | subjects treated with tolvaptan were thirst, pollakiuria, and | (TEAEs; > 10% and greater than placebo) in healthy subjects |
| | headache. The most commonly reported TEAEs (> 5% | treated with tolvaptan were thirst, pollakiuria, and headache. The |
| | incidence) in hyponatremia trials for subjects treated with | most commonly reported TEAEs (> 5% incidence) in |
| | tolvaptan were thirst, dry mouth, peripheral edema, nausea, | hyponatremia trials for subjects treated with tolvaptan were thirst, |
| | fatigue, dizziness, pollakiuria, diarrhea, headache, | dry mouth, peripheral edema, nausea, fatigue, dizziness, |
| | constipation, and pyrexia. The most commonly reported | pollakiuria, diarrhea, headache, constipation, and pyrexia. The |
| | TEAE (by $>$ 5% incidence) in hyponatremia trials for subjects | most commonly reported TEAE (by > 5% incidence) in |
| | treated with placebo were peripheral edema, diarrhea, | hyponatremia trials for subjects treated with placebo were |
| | dyspnea, vomiting, fatigue, headache, and nausea. The IB | peripheral edema, diarrhea, dyspnea, vomiting, fatigue, headache, |
| | provides a thorough review of the adverse events (AEs) | and nausea. The IB provides a review of the adverse events (AEs) |
| | experienced with this compound during clinical trials. 16 | experienced with the spray-dried tablet and suspension |
| | Analyses of the completed 3-year pivotal Trial 156-04-251 | formulation of tolvaptan during clinical trials. 16 |
| | (double-blind, placebo-controlled trial to determine long-term | There is the potential for osmotic diarrhea due to the sorbitol |
| | safety and efficacy of oral tolvaptan in adult subjects with | content in the suspension. D-Sorbitol is a hexahydric sugar |
| | ADPKD) have revealed new and important safety | alcohol that naturally occurs in fruits and animal tissue. The daily |
| | information. In this trial, a new signal for imbalanced | per capita consumption of sorbitol as a food ingredient is |
| | elevations of liver transaminases in ADPKD subjects | approximately 200mg. The compound is about 35-60% as sweet |
| | receiving tolvaptan compared with placebo was detected and | as sugar, and has been the impetus as a substitute for sugar to |
| | formally adjudicated by an expert panel blinded to treatment. | reduce caloric intake and prophylactic measures against the |
| | | formation of dental caries. Absorption of sorbitol by humans is |
| | | limited by its rate of diffusion from the gastrointestinal tract and |
| | | by laxation that may occur after ingestion of high doses. |
| | | Typically, 25-50 g in adults may cause osmotic diarrhea. The |
| | | corresponding dose in children is thought to be 10 g and higher, |
| | | but is dependent on body weight and types of foods ingested. |
| | | Similar findings are also observed with other sugar alcohols, eg, |
| | | xylitol. <sup>17</sup> |
| | | Following a single 15 mg tolvaptan dose of the suspension, |

| Location | Old Text | Updated Text |
|---|---|---|
| | | containing 8 g of sorbitol, in healthy adults, no diarrhea was reported. <sup>34</sup> |
| | | Therefore, in this trial, suspension dosing is limited to subjects who weigh ≤30 kg; the maximum dose of sorbitol is expected to be approximately 9.6 grams in a 0.6 mg/kg dose for a subject who weighs 30 kg. Subjects will be started on the lowest dose for their weight and titrated to higher doses as appropriate for their clinical condition. Subjects will be in a hospital setting during titration and will be closely monitored for rate of sodium correction and signs of dehydration including diarrhea. |
| | | Analyses of the completed 3-year pivotal Trial 156-04-251 (double-blind, placebo-controlled trial to determine long-term safety and efficacy of oral tolvaptan in adult subjects with ADPKD) have revealed new and important safety information. In this trial, a new signal for imbalanced elevations of liver transaminases in ADPKD subjects receiving tolvaptan compared with placebo was detected and formally adjudicated by an expert panel blinded to treatment. |
| 2.1 Trial Rationale: | The proposed population size of 100 subjects is expected to yield 70 subjects who respond to tolvaptan (henceforth termed "responders"), which has adequate power (> 90%) to test for statistical significance in the primary endpoint. Enrollment is expected to take 3 years using up to 50 sites globally. Additional blood sampling will be included across populations to provide PK information. | The proposed population size of 100 subjects is expected to yield 70 subjects who respond to tolvaptan (henceforth termed "responders"), which has adequate power (> 90%) to test for statistical significance in the primary endpoint. Enrollment is expected to take approximately 3 years using approximately 60 sites globally. Additional blood sampling will be included across populations to provide PK information. |

| Location | Old Text Updated Text | |
|---|---|---|
| | Even with a limited size, recruitment for such a trial is | Even with a limited size, recruitment for such a trial is expected to |
| | expected to be challenging due to the low frequency of AVP- | be challenging due to the low frequency of AVP-mediated |
| | mediated hyponatremia in children. Therefore, the trial will | hyponatremia in children. Therefore, the trial will be organized at |
| | be organized at major pediatric referral centers to access the | major pediatric referral centers to access the largest patient |
| | largest patient population. | population. |
| | | It is recognized that the pediatric population is a vulnerable subgroup and there are risks in conducting a clinical trial in the pediatric population. However, given the possible serious and life-threatening consequences of untreated hyponatremia, it is necessary to study hyponatremia treatment in children. Children have different physiology and metabolisms from adults and, therefore, it is not sufficient to study hyponatremia treatment in the adult population to determine the proper course of treatment for hyponatremia in the pediatric population. A clear understanding of exposure-response in adults that can be applied to pediatrics (or from one pediatric group to another) has not yet been established, furthering the need for this trial. <sup>19</sup> |
| | | Every effort will be made to anticipate and reduce known risks. This trial was designed to minimize the number of participants and the number of procedures, consistent with good study design.2 <sup>0</sup> Children will be continuously monitored for signs of distress during this trial. The risk threshold for subjects will be constantly monitored by the investigator. A detailed list and description of the safety monitoring to be conducted during this trial can be found in Section 3.7.4. |
| 2.1.1 Dosing<br>Rationale: | Enrolled subjects will be dosed based on age, weight, and the use of CYP3A4 inhibitors. Subjects < 2 years of age or < 10 | Enrolled subjects will be dosed based on formulation type, age, weight, and the use of CYP3A4 inhibitors. |

| Location | Old Text | Updated Text |
|---|---|---|
| | or moderate CYP3A4 inhibitors. | Therefore, subjects < 2 years of age or < 10 kg will be |
| | | administered tolvaptan as the suspension formulation with doses |
| | | starting at 0.1 mg/kg. Subjects $\geq$ 2 years of age, weighing $\geq$ 10 to |
| | | < 20 kg and who can swallow a tablet will be administered an oral |
| | | tablet once daily starting at a dose of 3.75-mg. Subjects weighing |
| | | 20 to 50 kg, inclusive, and who can safely swallow a tablet, will |
| | | receive an oral once daily dose of tolvaptan starting as a 7.5-mg |
| | | spray-dried tablet. Subjects $\geq 2$ years of age, weighing $\leq 30$ kg |
| | | and who cannot safely swallow a tablet, will receive an oral, once |
| | | daily dose of tolvaptan suspension staring at 0.15 mg/kg. Subjects |
| | | weighing > 50 kg will receive an oral once daily dose of tolvaptan |
| | | starting as a 15-mg spray-dried tablet. |
| | | Tolvaptan is a sensitive CYP3A4 substrate; plasma concentrations |
| | | increased approximately 4-fold when tolvaptan was administered |
| | | with the potent CYP3A4 inhibitor ketoconazole. 16,24 Where |
| | | appropriate dose reductions are possible, tolvaptan doses may be |
| | | coadministered with potent or moderate CYP3A4 inhibitors. |
| | | Table 2.1.1-2 outlines starting dose adjustments when tolvaptan is |
| | | administered concurrently with potent or moderate CYP3A |
| | | inhibitors. Tolvaptan doses will be reduced 75% and 50% if a |
| | | potent or moderate inhibitor, respectively, is being concurrently |
| | | administered. As the smallest volume of suspension that can be |
| | | administered is 0.3 mL (0.3kg), subjects weighing < 3 kg, < 6 kg |
| | | and taking a moderate CYP3A4 inhibitor or weighing < 10kg and |
| | | taking a potent CYP3A4 inhibitor may not be enrolled. |

New Text: Table 2.1.1-2 Starting Tolvaptan Tablet Doses as mg/kg of Body Weight

| Table 2.1.1-2 Starting Tolvaptan Tablet Doses in the Presence of Potent or<br>Moderate CYP3A Inhibitors | | | |
|---|---|---|---|
| Tolvaptan Dose | Age/Body Weight (as applicable) | Potent Inhibitor | Moderate Inhibitor |
| 0.1 mg/kg<br>suspension | 44 wk to < 2 y or<br>< 10 kg | - | 0.05 mg/kg suspension |
| 0.15 mg/kg<br>suspension | ≥ 2 y, ≤ 30 kg | 0.04 mg/kg suspension | 0.8 mg/kg suspension |
| 3.75 mg tablet | $\geq 10 \text{ kg to} < 20 \text{ kg}$ | 0.94 mL suspension | 0.19 mL suspension |
| 7.5 mg tablet | 20 kg to 50 kg | 1.90 mL suspension | 3.75 mg tablet |
| 15 mg tablet | ≥ 50 kg | 3.75 mg tablet | 7.5 mg tablet |

a The smallest volume of suspension that may be administered is 0.3 mL (0.3 mg), therefore dose reductions for potent inhibitors cannot be accommodated and for moderate inhibitors children weighing < 6 kg cannot be accommodated.

| Location | Old Text | Updated Text |
|---|---|---|
| 3.1 Type of | This is the first clinical trial of tolvaptan in a pediatric | This is the first clinical trial of tolvaptan in a pediatric population, |
| Trial: | population, and the majority of subjects may require only short- | and the majority of subjects may require only short-term treatment |
| | term treatment of hyponatremia, however some subjects may | of hyponatremia, however some subjects may require prolonged |
| | require prolonged treatment and additional follow-up information | treatment and additional follow-up information on their response to |
| | on their response to tolvaptan may be desired to better understand | tolvaptan may be desired to better understand its long-term safety |
| | its long-term safety profile in this pediatric population. Hence, | profile in this pediatric population. Hence, all subjects (responders |
| | all subjects (responders and nonresponders) who complete this | and nonresponders) who participate in this trial will be eligible for |
| | trial will be eligible for enrollment into an extension trial | enrollment into an extension trial (156-11-294) for a 6-month safety |
| | (156-11-294) to continue receiving tolvaptan, as clinically | follow-up, regardless of treatment, and the option to continue |
| | appropriate, until it is approved and available locally. If eligible, | receiving treatment with tolvaptan for hyponatremia based on |
| | subjects could continue therapy with tolvaptan in that trial after | clinical need. |
| | completing the 14 (+2) day Follow-up Visit and completion of | |
| | this trial. (The extension study will also provide long-term post- | |
| | treatment safety follow-up information for a minimum of 6 | |
| | months.) | |
| | The trial will be conducted in two stages. The first stage will be | |
| | conducted using the available tablet formulation of tolvaptan | |
| | whereas the second stage will expand to the use of a suspension | |
| | once that formulation becomes available. | |
| | 0.00 0.00 10.00 0.00 0.00 0.00 0.00 0.0 | |
| Figure 3.1-1<br>Trial Design<br>Schematic: | | Schematic revised to reflect updated text in this section. |
| 3.2.1 Tablet | The maximum starting doses, by weight, for subjects are shown | The maximum starting doses, by weight and age, for subjects are |
| Formulation: | in Table 2.1.1-1 and are within the range previously used in trials | shown in Table 2.1.1-1 and are within the range previously used in |
| | involving adult hyponatremic subjects. | trials involving adult hyponatremic subjects. |
| | The palatability of tolvaptan tablets will be assessed. | The palatability and acceptability of tolvaptan tablets will be |

| Location | Old Text | Updated Text |
|---|---|---|
| 3.2.2 Suspension | Additional information on the proposed suspension formulation | assessed. The investigator has the option of performing a swallow test and providing coaching on swallowing techniques using placebo tablets if it is known or suspected that the subject is unable to swallow tablets. Placebo tablets will be provided for use in performing this test at screening. Tolvaptan suspension, 1 mg/mL (0.1% w/v) will be administered |
| Formulation: | of tolvaptan (currently in development) will be added to the protocol in an amendment when available. Until that time, subjects < 2 years of age or weighing < 10 kg and those unable to swallow tablets, are excluded from the trial. | orally once daily, preferably in the morning hours. The treatment duration will be up to 5 days. Any initiation or titration of tolvaptan must occur in a hospital setting. Subjects < 2 years of age or < 10 kg will be administered tolvaptan as the suspension formulation with doses starting at 0.1 mg/kg. Subjects ≥ 2 to < 4 years of age, weighing ≥ 10 to < 20 kg and who cannot swallow a tablet, can receive tolvaptan as the suspension formulation starting at 0.15 mg/kg. The palatability and acceptability of tolvaptan suspension will be assessed. |
| 3.2.3 Dosing<br>Guidelines: | Subjects will be administered tolvaptan on an age- and weight-based scale. Titration of tolvaptan doses can occur once daily and will be based on serum sodium levels assessed at > 20 hours following initiation of therapy and each subsequent dose; titration may not occur within 20 hours of the previous dose. Up-titration | Subjects will be administered tolvaptan on a formulation, age- and weight-based scale. Titration of tolvaptan doses can occur once daily and will be based on serum sodium levels assessed at > 20 hours following initiation of therapy and each subsequent dose; titration may not occur within 20 hours of the previous dose. |
| | is limited to no more than twice the previous dose. | Up-titration is limited to no more than twice the previous dose. |

| Location | Old Text | Updated Text |
|---|---|---|
| | Subjects < 2 years of age or weighing < 10 kg are excluded until | Subjects < 2 years of age, weighing < 10 kg will receive 0.1 mg/kg |
| | an oral suspension formulation is available. | of the suspension on Day 1 with possible up-titration to 0.2 mg/kg |
| | Subjects $\geq 2$ years of age and weighing $\geq 10$ to $< 20$ kg will | and 0.4 mg/kg doses. |
| | receive a 3.75 mg tablet on Day 1 with possible up-titration to 7.5 | Subjects $\geq 2$ years of age, weighing $\geq 10$ to $\leq 20$ kg and who can |
| | mg and 15 mg tablet doses. | safely swallow a tablet will receive a 3.75 mg tablet on Day 1 with |
| | Subjects weighing 20 to 50 kg, inclusive, will receive a 7.5 mg | possible up-titration to 7.5 mg and 15 mg tablet doses. |
| | tablet on Day 1 with possible up-titration to 15 mg and 30 mg | Subjects weighing 20 to 50 kg, inclusive, and who can safely |
| | tablet doses. | swallow a tablet, will receive a 7.5 mg tablet on Day 1 with |
| | Subjects weighing > 50 kg will receive a 15 mg tablet on Day 1 | possible up-titration to 15 mg and 30 mg doses. |
| | with possible up-titration to 30 mg and 60 mg tablet doses. | Subjects $\geq 2$ years of age, weighing $\leq 30$ kg and who cannot safely |
| | | swallow a tablet, can be given a 0.15 mg/kg dose of the suspension |
| | | on Day 1 with possible up-titration to 0.3 mg/kg and 0.6 mg/kg |
| | For subjects weighing ≥ 20 kg and taking moderate inhibitors | doses. |
| | of CYP3A4, one half of the standard dose will be used (3.75 or | |
| | 7.5 mg, by weight). For subjects weighing > 50 kg and taking | Subjects weighing > 50 kg will be given a 15 mg tablet on Day 1 |
| | potent inhibitors of CYP3A4, a one-quarter dose will be used | with possible up-titration to 30 mg and 60 mg doses. |
| | (3.75 mg). Subjects weighing < 20 kg and who are taking any | |
| | CYP3A4 inhibitors will be excluded until such time that an | For subjects taking medenate inhibitors of CVP2 A A one helf of |
| | alternate dosing formulation is available. | For subjects taking moderate inhibitors of CYP3A4, one half of the standard dose will be used. For subjects taking potent inhibitors |
| | Table in a deciminate of a second and in the second in the second in | · |
| | Following their initial tolvaptan dose in the trial subjects will | of CYP3A4, a one-quarter dose will be used. The suspension |
| | continue dosing according to the titration scheme (see | formulation may be used in dose reductions for the tablet, see Table |
| | Section 3.2.4), targeting a final serum sodium concentration | 2.1.1-2. |
| | between 135 and 140 mEq/L (mmol/L). Titration guidelines are | Following their initial tolvaptan dose in the trial subjects will |
| | designed to achieve a change in serum sodium concentration of at | continue dosing according to the titration scheme (see |
| | least 4 to 8 mEq/L (mmol/L)/24 hours but not exceeding | Section 3.2.4), targeting a final serum sodium concentration |
| | | between 135 and 140 mEq/L (mmol/L). Titration guidelines are |
| | | designed to achieve a change in serum sodium concentration of at |

| Location | Old Text | Updated Text |
|----------|----------|--------------------------------------------------------|
| | | least 4 to 8 mEq/L (mmol/L)/24 hours but not exceeding |
## **Old Text:** Table 3.2.3-1 Dosing Schedule

| Table 3 | .2.3-1 Dosing Sche | dule | |
|---|---|---|---|
| Trial<br>Day | Group | Time | Dose |
| Day 1 | All subjects | Hour 0 | 3.75, 7.5, or 15 mg<br>(as applicable) |
| Day 2 | All subjects | 24 ( $\pm$ 4) h post first dose | 3.75, 7.5, 15, or 30 mg (as applicable) |
| Day 2a | (optional) | 24 (± 4) h post previous dose | 3.75, 7.5, 15, 30 or 60 mg (as applicable) |
| Day 3 | Late Withdrawal<br>and<br>Nonresponders<br>continuing on<br>tolvaptan | 24 (± 4) h post previous dose | 3.75, 7.5, 15, 30, or 60 mg<br>(as applicable) |
| Day 4 | Late Withdrawal<br>and<br>Nonresponders<br>continuing on<br>tolvaptan | 24 (± 4) h post previous dose | 3.75, 7.5, 15, 30, or 60 mg<br>(as applicable) |

# **New Text:** Table 3.2.3-1 Dosing Schedule

| Table 3.2 | Table 3.2.3-1 Dosing Schedule | | |
|---|---|---|---|
| Trial<br>Day | Group | Time | Dose |
| Day 1 | All subjects | Hour 0 | 0.1 or 0.15 mg/kg suspension<br>3.75, 7.5, or 15 mg tablets<br>(as applicable) |
| Day 2 | All subjects | 24 (± 4) h post first dose | 0.1, 0.15, 0.2, or 0.3 mg/kg<br>suspension<br>3.75, 7.5, 15, or 30 mg<br>(as applicable) |
| Day 2a | (optional) | 24 (± 4) h post previous dose | 0.1, 0.15, 0.2, 0.3, 0.4, or 0.6 mg/kg<br>suspension<br>3.75, 7.5, 15, 30 or 60 mg<br>(as applicable) |
| Day 3 | Late Withdrawal<br>and<br>Nonresponders<br>continuing on<br>tolvaptan | 24 (± 4) h post previous dose | 0.1, 0.15, 0.2, 0.3, 0.4, or 0.6 mg/kg<br>suspension3.75, 7.5, 15, 30, or 60<br>mg<br>(as applicable) |
| Day 4 | Late Withdrawal<br>and<br>Nonresponders<br>continuing on<br>tolvaptan | 24 (± 4) h post previous dose | 0.1, 0.15, 0.2, 0.3, 0.4, or 0.6 mg/kg<br>suspension<br>3.75, 7.5, 15, 30, or 60 mg<br>(as applicable) |

| Location | Old Text | New Text |
|---|---|---|
| Figure 3.2.4-1 Titration and Rescue Therapy Scheme: | | Schematic revised to reflect updated text in this section. |
| 3.2.4.2 Rescue<br>Therapy: | <ul> <li>If at any point during the trial serum sodium levels or hyponatremia symptoms worsen or fail to improve adequately and definitive therapy (eg, isotonic or hypertonic saline) is required, the subject will be withdrawn from trial treatment to receive rescue therapy.</li> <li>Additional guidelines for rescue therapy concerning hyponatremia symptoms and decreasing serum sodium level:</li> <li>If a subject has worsening symptoms and/or has a serum sodium level at or below the baseline value, repeat serum sodium [STAT] to confirm level, and begin rescue therapy.</li> <li>If a subject is asymptomatic and serum sodium has decreased by ≥ 4 mEq/L (mmol/L), but is still above the baseline value, consider need for rescue therapy.</li> <li>If a subject is asymptomatic and serum sodium has decreased by ≤ 3 mEq/L (mmol/L), but is still above the baseline value, no action is required.</li> </ul> | <ul> <li>If at any point during the trial serum sodium levels or hyponatremia symptoms worsen or fail to improve adequately and definitive therapy (eg, isotonic or hypertonic saline) is required, the subject will be withdrawn from trial treatment to receive rescue therapy Please see Section 4.2 for further details.</li> <li>Additional guidelines for rescue therapy concerning hyponatremia symptoms and decreasing serum sodium level:</li> <li>If a subject has worsening symptoms and/or has a serum sodium level to robelow the baseline value, repeat serum sodium [STAT] to confirm level, and begin rescue therapy.</li> <li>If a subject is asymptomatic and serum sodium has decreased by ≥ 4 mEq/L (mmol/L), but is still above the baseline value, consider need for rescue therapy according to local standard of care.</li> <li>If a subject is asymptomatic and serum sodium has decreased by ≤ 3 mEq/L (mmol/L), but is still above the baseline value, no action is required.</li> </ul> |
| | Subjects who are randomized to the Early Withdrawal group will initially be observed to determine whether additional intervention is required to maintain appropriate serum sodium levels. Those subjects whose serum sodium declines by $\geq 4$ mEq/L (mmol/L) or whose overall clinical condition requires further treatment to increase serum sodium will be treated per standard of care. Any | Subjects who are randomized to the Early Withdrawal group will initially be observed to determine whether additional intervention is required to maintain appropriate serum sodium levels. For those subjects whose serum sodium declines by $\geq 4$ mEq/L (mmol/L) or whose overall clinical condition requires further treatment to |

| Location | Old Text | New Text |
|---|---|---|
| | intervention intended to raise serum sodium level during the first 48 hours in the responder Early Withdrawal group (including fluid restriction) will be defined as rescue therapy. These subjects will be considered to have reached their clinical endpoint, and their data will be censored from that time forward. | increase serum sodium, the investigator may consider rescue therapy per local standard of care. Any intervention intended to raise serum sodium level during the first 48 hours in the responder Early Withdrawal group (including fluid restriction) will be defined as rescue therapy. These subjects will be considered to have reached their clinical endpoint, and their data will be censored from that time forward. |
| 3.3 Trial<br>Population: | This trial will include up to 100 male and female subjects aged $\geq 4$ weeks (or $\geq 44$ weeks adjusted gestational age) to < 18 years who have been diagnosed with euvolemic or hypervolemic hyponatremia (< 130 mEq/L [mmol/L]) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). Age groups will be enrolled such that 50% of these subjects will be < 10 years old and at least 25% of subjects < 6 years old. Subjects who are defined as responders will be further stratified by the magnitude of serum sodium response to tolvaptan ( $\leq 7$ and $\geq 7$ mEq/L [mmol/L]), and underlying etiology of hyponatremia. | This trial will include approximately 100 male and female subjects aged $\geq 4$ weeks (or $\geq 44$ weeks adjusted gestational age) to < 18 years who have been diagnosed with euvolemic or hypervolemic hyponatremia (< 130 mEq/L [mmol/L]) that persists despite initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist). Age groups will be enrolled such that at least 50% of these subjects will be < 10 years old and at least 25% of subjects < 6 years old. Subjects who are defined as responders will be further stratified by the magnitude of serum sodium response to tolvaptan ( $\leq 7$ and $\geq 7$ mEq/L [mmol/L]), age, and underlying etiology of hyponatremia. |
| | Subjects with euvolemic or hypervolemic hyponatremia eligible to be screened for participation in this trial include, but are not limited to, those diagnosed and admitted to a hospital for treatment of HF, hepatocellular disease (including cirrhosis), or SIADH/other. Subjects with acute hyponatremia or hyponatremia expected to resolve spontaneously will be excluded from the trial. Children with an impaired ability to sense or communicate their thirst will either be required per protocol to undergo closer in-hospital observation, laboratory and urine | Subjects with euvolemic or hypervolemic hyponatremia eligible to be screened for participation in this trial include, but are not limited to, those diagnosed and admitted to a hospital for treatment of HF, hepatocellular disease (including cirrhosis), or SIADH/other. Subjects with acute hyponatremia or hyponatremia expected to resolve spontaneously will be excluded from the trial. Children with an impaired ability to sense or communicate their thirst will either be required to undergo closer in-hospital observation, laboratory and urine output monitoring, or will be excluded from |

| Location | Old Text | New Text |
|---|---|---|
| | output monitoring, or will be excluded from the trial if this is not possible. Children with hypovolemic hyponatremia or those who are at risk of such, secondary to any underlying conditions that cause volume depletion, are excluded from this trial. | the trial if this is not possible. Children with hypovolemic hyponatremia or those who are at risk of such, secondary to any underlying conditions that cause volume depletion, are excluded from this trial. |
| | All potential subjects must have chronic (≥ 48 hours) dilutional hyponatremia (euvolemic or hypervolemic) associated with HF, hepatocellular disease (including cirrhosis), or SIADH/other and be deemed by the investigator as likely to benefit from a therapy that raises serum sodium levels. The etiology of hyponatremia (presumed cause) must be documented and evaluated per Section 3.3.1. Those subjects who have acute or transient hyponatremia, have overt symptoms of hyponatremia requiring immediate intervention, or who are at increased risk for developing hyponatremic encephalopathy or osmotic demyelination are excluded from this trial. | All potential subjects must have chronic (≥ 48 hours) dilutional hyponatremia (euvolemic or hypervolemic) associated with HF, hepatocellular disease (including cirrhosis), or SIADH/other and be deemed by the investigator as likely to benefit from a therapy that raises serum sodium levels. The etiology of hyponatremia (presumed cause) must be documented and evaluated per Section 3.3.1. Those subjects who have acute or transient hyponatremia, have overt symptoms of hyponatremia requiring immediate intervention, or who are at increased risk for developing hyponatremic encephalopathy or osmotic demyelination are excluded from this trial. |
| | Since hyponatremia in this patient population can often be transient and/or may be secondary to hypovolemic states, potential subjects will be screened for hyponatremic histories as well as clinically evaluated to rule out such cases. For the purpose of this protocol, persistent hyponatremia will be defined as serum sodium level < 130 mEq/L (mmol/L) documented as present for at least 48 hours. Specifically, subjects must have at least 2 serum sodium assessments < 130 mEq/L (mmol/L) drawn at least 12 hours apart. These values can be documented using historical values previously obtained as per standard of care. A third (STAT) serum sodium assessment < 130 mEq/L (mmol/L), which will serve as the baseline value for efficacy endpoints, is to | Since hyponatremia in this patient population can often be transient and/or may be secondary to hypovolemic states, potential subjects will be screened for hyponatremic histories as well as clinically evaluated to rule out such cases. For the purpose of this protocol, persistent hyponatremia will be defined as serum sodium level < 130 mEq/L (mmol/L) documented as present for at least 48 hours. Specifically, subjects must have at least 2 serum sodium assessments < 130 mEq/L (mmol/L) drawn at least 12 hours apart. These values can be documented using historical values previously obtained as per standard of care. A third (STAT) serum sodium assessment < 130 mEq/L (mmol/L), which will serve as the baseline value for final trial qualification and clinical management |

| Location | Old Text | New Text |
|---|---|---|
| | be obtained within 2-4 hours prior to the first dose of trial medication. | strategy, is to be obtained within 2-4 hours prior to the first dose of trial medication. This assessment will also serve as the baseline value for secondary and exploratory endpoints. |
| 3.4 Eligibility<br>Criteria: | Eligible subjects must satisfy all informed consent requirements, as well as meet all inclusion and exclusion criteria. Subjects who do not meet all of these requirements are to be defined as screen failures and may rescreen, if eligible, at a later date. | Eligible subjects must satisfy all informed consent and assent requirements, as well as meet all inclusion and exclusion criteria. Subjects who do not meet all of these requirements are to be defined as screen failures and may rescreen, if eligible, at a later date. |
| 3.4.1 Informed<br>Consent/Assent: | 3.4.1 Informed Consent Written informed consent and assent as appropriate will be obtained from the subject's parent or legal guardian, in accordance with requirements of the trial center's institutional review board/independent ethics committee (IRB/IEC). The subject, as required by the trial center's IRB/IEC, must provide informed assent at Screening and as such must be able to understand that he or she can withdraw from the trial at any time. | 3.4.1 Informed Consent/Assent Written informed consent and assent as appropriate will be freely obtained from the subject's parent or legal guardian, as applicable for local laws, in accordance with requirements of the trial center's institutional review board/independent ethics committee (IRB/IEC). The subject, as required by the trial center's IRB/IEC, must provide informed assent at Screening and as such must be able to understand that he or she can withdraw from the trial at any time. Subjects' parents or legal guardian(s) may be asked to sign additional ICFs if the protocol is amended to significantly add or change procedures. Subjects who are able may be asked to reassent as appropriate if the protocol is amended to significantly add or change procedures. |

## **Old Text:** Table 3.4.2-1 Inclusion Criteria

Subjects are required to meet the following inclusion criteria:

| 1. | Male and female subjects ≥ 4 weeks (or ≥ 44 weeks adjusted gestational age for premature births) to < 18 years old |
|---|---|
| 2. | Subjects hospitalized with euvolemic or hypervolemic hyponatremia resistant to initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist) and who are deemed by the investigator as likely to benefit from a therapy that raises serum sodium levels |
| 3. | Persistent euvolemic or hypervolemic hyponatremia defined as being documented as present for at least 48 hours, evidenced by at least 2 serum sodium assessments < 130 mEq/L (mmol/L) drawn at least 12 hours apart (these values can be documented using historical values previously obtained per standard of care); a third (STAT) serum sodium assessment < 130 mEq/L (mmol/L), which will serve as the baseline value for efficacy endpoints, is to be obtained within 2-4 hours prior to the first dose of tolvaptan |
| 4. | Ability to take oral medication |
| 5. | Ability to maintain adequate fluid intake whether orally or via IV support with adequate monitoring |
| 6. | Ability to comply with all requirements of the trial |
| 7. | Trial-specific written informed consent/assent obtained from a parent/guardian or legally acceptable representative, as applicable per age of subject or local laws, prior to the initiation of any protocol-required procedures. In addition, the subject as required by local laws must provide informed assent at Screening and must be able to understand that he or she can withdraw from the trial at any time. All informed consent/assent procedures must be in accordance with the trial center's IRB/IEC and local regulatory requirements |
| 8. | Ability to commit to remain abstinent or practice double-barrier birth control during the trial and for 14 days following the last dose of IMP for sexually active females of childbearing potential |

IMP = investigational medicinal product.

## **New Text:** Table 3.4.2-1 Inclusion Criteria

Subjects are required to meet the following inclusion criteria:

| Tab | ele 3.4.2-1 Inclusion Criteria |
|---|---|
| 1. | Male and female subjects $\geq$ 4 weeks (or $\geq$ 44 weeks adjusted gestational age for premature births) to $<$ 18 years old |
| 2. | Subjects hospitalized with euvolemic or hypervolemic hyponatremia resistant to initial standard background therapy (including fluid restriction and excluding a vasopressin antagonist) and who are deemed by the investigator as likely to benefit from a therapy that raises serum sodium levels |
| 3. | Persistent euvolemic or hypervolemic hyponatremia defined as being documented as present for at least 48 hours, evidenced by at least 2 serum sodium assessments < 130 mEq/L (mmol/L) drawn at least 12 hours apart (these values can be documented using historical values previously obtained per standard of care); a third (STAT) serum sodium assessment < 130 mEq/L (mmol/L), which will serve as the baseline value for final trial qualification and clinical management strategy, is to be obtained within 2-4 hours prior to the first dose of tolvaptan |
| 4. | Ability to take oral medication |
| 5. | Ability to maintain adequate fluid intake whether orally or via IV support with adequate monitoring |
| 6. | Ability to comply with all requirements of the trial |
| 7. | Trial-specific written informed consent/assent obtained from a parent/guardian or legally acceptable representative, as applicable per age of subject or local laws, prior to the initiation of any protocol-required procedures. In addition, the subject as required by local laws must provide informed assent at Screening and must be able to understand that he or she can withdraw from the trial at any time. All informed consent/assent procedures must be in accordance with the trial center's IRB/IEC and local regulatory requirements |
| 8. | Ability to commit to remain fully abstinent (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] or withdrawal are not acceptable methods of contraception) or practice double-barrier birth control during the trial and for 30 days following the last dose of IMP for sexually active females of childbearing potential |

IMP = investigational medicinal product.

#### **Old Text:** Table 3.4.3-1 Exclusion Criteria

Subjects will be excluded if they meet any of the following exclusion criteria prior to trial entry.

| Table 3 | 3.4.3-1 Exclusion Criteria |
|---|---|
| 3. | Use of potent CYP3A4 inhibitors in subjects ≤ 50 kg or moderate CYP3A4 inhibitors in subjects < 20 kg |
| 25. | Subjects <2 years of age, weight <10 kg, or who cannot swallow an oral tablet are excluded until an oral suspension formulation becomes available |

#### **New Text:** Table 3.4.3-1 Exclusion Criteria

Subjects will be excluded if they meet any of the following exclusion criteria prior to trial entry.

| Table | 23.4.3-1 Exclusion Criteria |
|---|---|
| 3. | Current use or expected use during the trial of a potent CYP3A4 inhibitor in subjects weighing < 10 kg or a moderate CYP3A4 inhibitor in subjects weighing < 6 kg |
| 25. | Subjects who weigh < 3 kg |
| 26. | Unable to swallow tablets if the suspension formulation is unavailable |

Use of the suspension formulation is at the discretion of the local regulatory authorities and IRB/IECs. In such cases, subjects who require use of suspension for either standard dosing or adjusted dosing (eg, concomitant use of CYP3A4 inhibitors) cannot be enrolled.

| Location | Old Text | Updated Text |
|---|---|---|
| 3.7 Trial | In Treatment Phase A, subjects who meet the inclusion and | In Treatment Phase A, subjects who meet the inclusion and |
| Procedures: | exclusion criteria will be enrolled and will be administered a | exclusion criteria will be enrolled and will be administered |
| | 3.75-, 7.5-, or 15-mg dose tablet based on age, weight, and the | tolvaptan doses based on age, weight, ability to swallow a tablet, |
| | use of CYP3A4 inhibitors. At the end of Day 2 (or 2a) in | and the use of CYP3A4 inhibitors. At the end of Day 2 (or 2a) in |
| | Treatment Phase A, subjects who are responders will be | Treatment Phase A, subjects who are responders will be |
| | randomized to either continue treatment with tolvaptan for | randomized to either continue treatment with tolvaptan for |
| | 2 additional days (Late Withdrawal) or to discontinue tolvaptan | 2 additional days (Late Withdrawal) or to discontinue tolvaptan |
| | treatment (Early Withdrawal). | treatment (Early Withdrawal). |
| | In Treatment Phase B, subjects who are nonresponders may | In Treatment Phase B, subjects who are nonresponders may |
| | continue on tolvaptan therapy for 2 additional days or may be | continue on tolvaptan therapy for 2 additional days or may be |
| | withdrawn from tolvaptan to be treated per the investigator's | withdrawn from tolvaptan to be treated per the investigator's |
| | preferred standard of care. During Treatment Phase B, subjects | preferred standard of care. During Treatment Phase B, subjects in |
| | in the Late Withdrawal group and nonresponders continuing | the Late Withdrawal group and nonresponders continuing treatment |
| | treatment will continue to receive tolvaptan for 2 additional days | will continue to receive tolvaptan for 2 additional days and all |
| | and all subjects will have serum sodium levels measured at 12 (± | subjects will have serum sodium levels measured at 12 ( $\pm$ 4) hours |
| | 4) hours post-dose and at trough each day. Subjects in the Early | postdose and at trough each day. Subjects in the Early Withdrawal |
| | Withdrawal group should be monitored for the first 48 hours | group should be monitored for the first 48 hours post-last dose. |
| | post-last dose. | |

## **Old Text: Table 3.7-1 Schedule of Assessments**

| Table 3.7-1 Schedule of Assessments | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening | Treatment Phase A | | Treatment Phase B | | | Follow-up Phase C | | | | |
| | Day -2<br>and -1 | Day 1 | Day 2 | Day 2a<br>(optional) | Day 3 | Day 4 | Day 5 | 72 (±4) h<br>post last<br>dose | 7 (±1)<br>days post-<br>last dose | 14 (+2)<br>days post-<br>last dose | Early<br>Termin-<br>ation (ET) |
| Informed Consent/Assent | X | | | | | | | | | | |
| Inclusion/exclusion criteria a | X | X | | | | | | | | | |
| Demographic information | X | | | | | | | | | | |
| Medical and hyponatremia history | X | | | | | | | | | | |
| Vital signs b | X | X | X | X | X | X | X | X | X | | X |
| 12-lead ECG | X | | | | | | | | | | |
| Height | X<br>X | | | | | | | | | | |
| Body weight <sup>c</sup> | X | X | X | X | X | X | X | X | X | | X |
| Directed physical examination | X | X | X | X | X | X | | X | X | | X |
| Tanner staging | X | | | | | | | | | | |
| Neurological examination | X | X | X | | X | X | | X | X | | X |
| Neurocognitive assessment | X | X | X | X | X | X | X | X | X | | X |
| Quality of life assessment | X | | | | | X | | | X | | |
| Clinical status<br>assessment e | X | X | X | X | X | X | | X | X | | X |
| Alcohol/drug screen | X | | | | | | | | | | |
| Pregnancy test (if applicable) f | X | | | | | | | | | | |
| Fluid intake <sup>g</sup> | | X | X | | | | | | | | |
| Urine volume <sup>g</sup> | | X | X | | | | | | | | |

| Table 3.7-1 Schedul | le of Assess | ments | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening | Tre | eatment 1 | Phase A | Treatment Phase B | | Follow-up Phase C | | | | |
| | Day -2<br>and -1 | Day 1 | Day 2 | Day 2a<br>(optional) | Day 3 | Day 4 | Day 5 | 72 (±4) h<br>post last<br>dose | 7 (±1)<br>days post-<br>last dose | 14 (+2)<br>days post-<br>last dose | Early<br>Termin-<br>ation (ET) |
| Urinalysis | X | | | | | | | X | | | X |
| Urine chemistry <sup>g,h</sup> | X | X | X | | | | | | | | |
| Serum sodium <sup>i</sup> | X | X | X | X | X | X | X | X | X | | X |
| Hematology, coagulation, and serum chemistry | X | | | | | | | X | | | X |
| Serum osmolality, FENa, and FE urate | X | | | | | | | | | | |
| TSH and cortisol <sup>k</sup> | X | | | | | | | | | | |
| PK plasma samples | | X | X | | X | X | X | | | | X |
| Tolvaptan dosing m | | X | X | X | X | X | | | | | |
| Assessment for response to tolvaptan | | | X | X | | | | | | | |
| Palatability assessment | | | X | | | | | | | | |
| Randomization | | | | | X | | | | | | |
| Follow-up phone call or visit | | | | | | | | | | X | |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X |

ECG = electrocardiogram; TSH = thyroid-stimulating hormone.

<sup>&</sup>lt;sup>a</sup>Inclusion/exclusion criteria will be checked at screening and predose on Day 1.

<sup>&</sup>lt;sup>b</sup>Vital signs to be assessed include supine blood pressure, heart rate, respiratory rate, and temperature. Vital signs should be assessed prior to any blood draws.

<sup>&</sup>lt;sup>c</sup>Weight will be taken predose as possible.

dNeurocognitive assessments are closely tied to serum sodium assessments and should be done within 1 hour of sodium blood draws.

- Screening: 2 assessments should be taken, at least 12 hours apart (may be part of medical history). 1 assessment can be combined with the serum chemistry panel.
- Treatment Phase A: Baseline [STAT] assessment will be at 2-4 hours prior to first dose. Post-first dose assessments: 8 and 24 (trough) hours. Then every 12 hours thereafter (alternating 12 hours post-dose and at trough)
- Treatment Phase B: Assessments to be taken every 12 hours (alternating 12 hours post-dose and at trough)
- Treatment Phase C: Assessments to be taken at 72 (± 4) hours post-last dose (can be combined with the serum chemistry panel) and at the 7 day post-last dose visit.

- In Treatment Phase A PK samples should be collected at 2 and 8 hours and at trough post-first dose.
- In Treatment Phase B PK will be assessed in subjects continuing treatment with tolvaptan (Late Withdrawal group and nonresponders continuing on tolvaptan) at trough on Days 3, 4 and 5.

<sup>&</sup>lt;sup>e</sup>Clinical status assessments will be performed per inpatient standard of care, ie, review patient chart entries (including hyponatremia assessment notes and laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate overall subject eligibility in terms of hyponatremia state.

Urine pregnancy tests will be performed on female subjects  $\geq 12$  years of age and all female subjects  $\leq 12$  years of age if menstruation has started.

<sup>&</sup>lt;sup>g</sup>Intervals starting immediately after dosing at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours).

<sup>&</sup>lt;sup>h</sup>Samples within a collection interval are to be refrigerated and pooled. An aliquot for urine chemistry tests will be taken for each collection interval. Uric acid is to be measured at screening only.

Serum sodium assessments are closely tied to neurocognitive assessments, dosing time points and PK blood draws.

<sup>&</sup>lt;sup>J</sup>Serum chemisty panel includes serum sodium and assessments can be combined for visits where both assessments are indicated.

Results of these tests will further characterize hyponatremia etiology for the Hyponatremia History CRF and are not required to determine eligibility. Subjects who have clinically relevant TSH or cortisol levels may not respond properly to tolvaptan and will be withdrawn from the trial.

PK samples are closely tied to dosing time points and serum sodium assessments. An ET sample will be collected only if ET is before the last scheduled PK assessment.

<sup>&</sup>lt;sup>m</sup>The tolvaptan dose will be titrated based on serum sodium levels as described in Section 3.2.4.

## **NewText: Table 3.7-1 Schedule of Assessments**

| Procedures Screening Treatment Phase A Treatment Phase B Follow-up Phase C | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Trocedures | Day -2<br>and -1 | Day 1 | Day 2 | Day 2a<br>(optional) | Day 3 | Day 4 | Day 5 | 72 (±4) h<br>post last<br>dose | 7 (±1) days post- last dose | 14 (+2)<br>days post-<br>last dose | Early<br>Termin-<br>ation (ET) |
| Informed Consent/Assent | X | | | | | | | | | | |
| Inclusion/exclusion criteria <sup>a</sup> | X | X | | | | | | | | | |
| Demographic information | X | | | | | | | | | | |
| Medical and hyponatremia history | X | | | | | | | | | | |
| Vital signs b | X | X | X | X | X | X | X | X | X | | X |
| 12-lead ECG | X | | | | | | | | | | |
| Height | X | | | | | | | | | | |
| Body weight <sup>c</sup> | X | X | X | X | X | X | X | X | X | | X |
| Physical examination | x <sup>d</sup> | X | X | X | X | X | | X | X | | X |
| Tanner staging | X | | | | | | | | | | |
| Neurological examination | X | X | X | | X | X | | X | X | | X |
| Neurocognitive assessment e | X | X | X | X | X | X | X | X | X | | X |
| Quality of life assessment | X | | | | | X | | | X | | |
| Clinical status assessment f | X | X | X | X | X | X | | X | X | | X |
| Alcohol/drug screen | X | | | | | | | | | | |
| Pregnancy test (if applicable) <sup>g</sup> | X | | | | | | | | X | | |
| Fluid intake h | | X | X | | | | | | | | |
| Urine volume h | | X | X | | | | | | | | |
| Urinalysis | X | | | | | | | X | | | X |

| Table 3.7-1 Schedul | le of Assess | sments | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedures | Screening | Tre | eatment 1 | Phase A | Trea | Treatment Phase B | | Follow-up Phase C | | | |
| | Day -2<br>and -1 | Day 1 | | Day 2a<br>(optional) | Day 3 | Day 4 | Day 5 | 72 (±4) h<br>post last<br>dose | 7 (±1)<br>days post-<br>last dose | 14 (+2)<br>days post-<br>last dose | Early<br>Termin-<br>ation (ET) |
| Urine chemistry h,i | X | X | X | | | | | | | | |
| Serum sodium <sup>j</sup> | X | X | X | X | X | X | X | X | X | | X |
| Hematology, coagulation, and serum chemistry | X | | | | | | | X | | | X |
| Serum osmolality, FENa, and FE urate | X | | | | | | | | | | |
| TSH and cortisol <sup>1</sup> | X | | | | | | | | | | |
| PK plasma samples m | | X | X | | X | X | X | | | | X |
| Tolvaptan dosing <sup>n</sup> | | X | X | X | X | X | | | | | |
| Swallow test | X <sup>o</sup> | | | | | | | | | | |
| Assessment for response to tolvaptan | | | X | X | | | | | | | |
| Palatability and acceptability assessment | | | X | | | | | | | | |
| Randomization | | | | | X | | | | | | |
| Follow-up phone call or visit | | | | | | | | | | X | |
| Concomitant medications | X | X | X | X | X | X | X | X | X | X | X |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X |

ECG = electrocardiogram; TSH = thyroid-stimulating hormone.

<sup>&</sup>lt;sup>a</sup>Inclusion/exclusion criteria will be checked at screening and predose on Day 1.

bVital signs to be assessed include supine blood pressure, heart rate, respiratory rate, and temperature. Vital signs should be assessed prior to any blood draws.

<sup>&</sup>lt;sup>c</sup>Weight will be taken predose as possible.

- Screening: 2 assessments should be taken, at least 12 hours apart (may be part of medical history). One assessment can be combined with the serum chemistry panel.
- Treatment Phase A: Baseline [STAT] assessment will be at 2-4 hours prior to first dose. Post-first dose assessments: 8 and 24 (trough) hours. Then every 12 hours thereafter (alternating 12 hours postdose and at trough)
- Treatment Phase B: Assessments to be taken every 12 hours (alternating 12 hours postdose and at trough)
- Treatment Phase C: Assessments to be taken at 72 (± 4) hours post-last dose (can be combined with the serum chemistry panel) and at the 7 day post-last dose visit.

In addition to serum sodium samples obtained for trial qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, on Day 1 at 4 to 6 hours postdose and at 18 hours postdose, and on Day 2 (and Day 2a, if applicable) at 6 hours postdose as well as at 18 hours postdose. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if they can be combined with standard of care labs).

- In Treatment Phase A PK samples should be collected at 2 and 8 hours and at trough post-first dose.
- In Treatment Phase B PK will be assessed in subjects continuing treatment with tolvaptan (Late Withdrawal group and nonresponders continuing on tolvaptan) at trough (24 hours post last dose, immediately prior to next dose) on Days 3, 4 and 5.

<sup>&</sup>lt;sup>d</sup>The initial physical examination should be a full physical. Subsequent physical examinations can be directed physical examinations that are focused on hyponatremia-related signs and symptoms as well as any major changes from baseline.

<sup>&</sup>lt;sup>e</sup>Neurocognitive assessments are closely tied to serum sodium assessments and should be done within 1 hour of sodium blood draws.

<sup>&</sup>lt;sup>f</sup>Clinical status assessments will be performed per inpatient standard of care, ie, review patient chart entries (including hyponatremia assessment notes and laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate overall subject eligibility in terms of hyponatremia state. Volume status will be assessed every 6 hours prior to trial entry and every 6 hours during Treatment Phase A.

<sup>&</sup>lt;sup>g</sup>Pregnancy tests will be performed on female subjects  $\geq$  12 years of age and all female subjects  $\leq$  12 years of age if menstruation has started.

hIntervals starting immediately after dosing at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours).

Samples within a collection interval are to be refrigerated and pooled. An aliquot for urine chemistry tests will be taken for each collection interval. Uric acid is to be measured at screening only.

<sup>&</sup>lt;sup>J</sup>Serum sodium assessments are closely tied to neurocognitive assessments, dosing time points and PK blood draws.

<sup>&</sup>lt;sup>k</sup>Serum chemisty panel includes serum sodium and assessments can be combined for visits where both assessments are indicated.

Results of these tests will further characterize hyponatremia etiology for the Hyponatremia History CRF and are not required to determine eligibility. Subjects who have clinically relevant TSH or cortisol levels may not respond properly to tolvaptan and will be withdrawn from the trial.

<sup>&</sup>lt;sup>m</sup>PK samples are closely tied to dosing time points and serum sodium assessments. An ET sample will be collected only if ET is before the last scheduled PK assessment.

<sup>&</sup>lt;sup>n</sup>The tolvaptan dose will be titrated based on serum sodium levels as described in Section 3.2.4. <sup>o</sup>Optional swallow test for subjects who are known or suspected to be unable to swallow tablets, at the investigator's discretion.

| Location | Old Text | Updated Text |
|---|---|---|
| 3.7.1.1 | A directed physical examination will be performed. | A full physical examination will be performed. The initial physical |
| Screening: | Tanner staging will be performed. | examination should be a full physical. Subsequent physical examinations can be directed physical examinations that are |
| | A neurocognitive assessment will be performed, as appropriate by age and where available. | focused on hyponatremia-related signs and symptoms as well as any major changes from baseline. |
| | Quality-of-life (QoL) assessment will be performed, as appropriate by age and where available. | Tanner staging will be performed. |
| | Clinical status assessments will be performed per inpatient standard of care. | A neurocognitive assessment will be performed, as appropriate by age and where available and should be done within 1 hour of serum sodium blood draw. |
| | Alcohol and drug screens will be performed, as age appropriate. A urine pregnancy test will be performed on all female subjects | Quality-of-life (QoL) assessment will be performed, as appropriate by age and where available. |
| | ≥ 12 years of age and all female subjects < 12 years of age if menstruation has started. | Clinical status assessments will be performed per inpatient standard of care. |
| | Urinalysis and urine chemistry laboratory samples will be collected for analysis. | Alcohol and drug screens will be performed, as age appropriate. A pregnancy test will be performed on all female subjects |
| | Two blood samples for serum sodium testing will be collected at | ≥ 12 years of age and all female subjects < 12 years of age if menstruation has started. |
| | to document chronic hyponatremia. (One of these blood draws can be combined with the serum chemistry panel as appropriate to minimize blood draws.) | Urinalysis and urine chemistry laboratory samples will be collected for analysis. |
| | Hematology, coagulation, and serum chemistry laboratory samples will be collected for analysis. | Two blood samples for serum sodium testing will be collected at least 12 hours apart and can be part of the recent medical history to document chronic hyponatremia. (One of these blood draws can be |

| Location | Old Text | Updated Text |
|---|---|---|
| | Serum osmolality, FENa, and FE urate will be determined. | combined with the serum chemistry panel as appropriate to |
| | Thyroid-stimulating hormone (TSH) and cortisol blood samples | minimize blood draws.) |
| | will be collected to determine possible need for alternate mode of | Hematology, coagulation, and serum chemistry laboratory samples |
| | therapy. | will be collected for analysis. |
| | Concomitant medications will be recorded. | Serum osmolality, FENa, and FE urate will be determined. |
| | Adverse events will be recorded. | Thyroid-stimulating hormone (TSH) and cortisol blood samples will be collected to determine possible need for alternate mode of therapy. |
| | | Concomitant medications will be recorded. |
| | | Adverse events will be recorded. |
| | | Optional swallow test for subjects who are known or suspected to be unable to swallow tablets, at the investigator's discretion. Placebo tablets will be provided for use in performing this test at screening. |
| 3.7.1.2.1 Day 1: | 16) A neurological examination will be performed at 8 hours post-first dose. | A neurological examination will be performed at 8 hours post-first dose. |
| | | In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, on Day 1 at 4 to 6 hours postdose and at 18 hours postdose. This sodium safety assessment will be repeated at 6 and 18 hours postdose each day for the remainder of titration. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if |

| Location | Old Text | Updated Text |
|---|---|---|
| | | they can be combined with standard of care labs). |
| 3.7.1.2.2 Day 2: | Postdose | Postdose |
| | Assess palatability of tolvaptan tablets for subjects. | Assess palatability and acceptability of tolvaptan dose for subjects. |
| | Fluid intake will be recorded at 6-hour intervals starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours). | Fluid intake will be recorded at 6-hour intervals starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours). |
| | Urine will be collected at 6-hour intervals starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours). Subjects should be asked to void just prior to the end time of each collection interval, as possible. | Urine will be collected at 6-hour intervals starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours). Subjects should be asked to void just prior to the end time of each collection interval, as possible. |
| | Urine volume will be determined from urine voids made during the 6-hour collection intervals which will be pooled prior to determination of final volume. | Urine volume will be determined from urine voids made during the 6-hour collection intervals which will be pooled prior to determination of final volume. |
| | A urine chemistry sample will be collected and assessed from each 6-hour volume interval starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours). | A urine chemistry sample will be collected and assessed from each 6-hour volume interval starting at Hour 0 (0-6, 6-12, 12-18, and 18-24 hours). |
| | Clinical status assessments will be performed per inpatient standard of care, ie, patient chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state. | Clinical status assessments will be performed per inpatient standard of care, ie, patient chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state. |
| | A blood sample will be collected for serum sodium testing at 12 hours post-dose. | A blood sample will be collected for serum sodium testing at 12 hours postdose. |
| | | In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point |

| Location | Old Text | Updated Text |
|---|---|---|
| | | of care sodium assessment unit, where available, at 6 and 18 hours postdose. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if they can be combined with standard of care labs). |
| 3.7.1.2.3 Day 2a (optional): | Postdose 7) Clinical status assessments will be performed per inpatient standard of care, ie, patient chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state. 8) A blood sample will be collected for serum sodium testing at 12 hours postdose. | Postdose Clinical status assessments will be performed per inpatient standard of care, ie, patient chart entries will be reviewed (including hyponatremia assessment notes, including laboratory results [trial and nontrial specific], any examination findings, medical problem list changes, and fluid intake and output) to evaluate the subject's hyponatremia state. A blood sample will be collected for serum sodium testing at 12 hours postdose. In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, at 6 and 18 hours postdose. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if they can be combined with standard of care labs). |
| 3.7.1.4.2 7 Days<br>Post-last Dose: | <ol> <li>Vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be performed prior to blood draws.</li> <li>A blood sample for serum sodium testing will be collected.</li> </ol> | <ul> <li>11) Vital signs (blood pressure, heart rate, respiratory rate, and temperature) will be assessed after the subject has been supine for ≥ 3 minutes. Vital signs should be performed prior to blood draws.</li> <li>12) A blood sample for serum sodium testing will be collected.</li> <li>13) A pregnancy test will be performed on all female subjects</li> </ul> |

| Location | Old Text | Updated Text |
|---|---|---|
| | 3) A neurocognitive assessment will be performed within 1 hour of the serum sodium sample. | ≥ 12 years of age and all female subjects < 12 years of age if menstruation has started. |
| | | 14) A neurocognitive assessment will be performed within 1 hour of the serum sodium sample. |
| 3.7.2.1 Serum Sodium Concentrations: | Monitoring frequency of serum sodium is at the discretion of the clinical investigator; however, the minimum sample collection required for all subjects is described in Section 3.7.1. In order to qualify for this trial, subjects must have documentation of chronic dilutional hyponatremia (serum sodium < 130 mEq/L [mmol/L]) that is present for ≥ 48 hours. Specifically, each subject must have 2 blood samples collected at least 12 hours apart over a minimum of 48 hours for assessment of baseline serum sodium level to determine subject eligibility. These can be either part of the recent medical history concerning the current hospital stay or prospectively collected as part of this trial. On Day 1, a third (STAT) serum sodium sample should be drawn within 2-4 hours prior to dosing; the results must be verified to be < 130 mmol/L prior to the first dose. Serum sodium assessments should be performed at 8 hours post-first dose and at trough 24 hours post-first dose (this assessment will fall on Day 2 predose). On Day 2 (or 2a), Day 3, and Day 4 (through the following morning on Day 5): For all subjects receiving tolvaptan (Late Withdrawal and Nonresponders continuing on tolvaptan) serum sodium assessments will be performed at trough and 12 hours post-dose | Monitoring frequency of serum sodium is at the discretion of the clinical investigator; however, the minimum sample collection required for all subjects is described in Section 3.7.1 and Section 3.7.4.2.1. In addition to serum sodium samples obtained for treatment qualification and efficacy endpoints, supplemental samples for the purposes of safety assessment only can be obtained using a point of care sodium assessment unit, where available, on Day 1 at 4 to 6 hours postdose and at 18 hours postdose. This sodium safety assessment will be repeated at 6 and 18 hours postdose each day for the remainder of titration. A point of care assessment unit is preferred; however, regular blood draws may be used (especially if they can be combined with standard of care labs). In order to qualify for this trial, subjects must have documentation of chronic dilutional hyponatremia (serum sodium < 130 mEq/L [mmol/L]) that is present for ≥ 48 hours. Specifically, each subject must have 2 blood samples collected at least 12 hours apart over a minimum of 48 hours for assessment of baseline serum sodium level to determine subject eligibility. These can be either part of the recent medical history concerning the current hospital stay or prospectively collected as part of this trial. On Day 1, a third (STAT) serum sodium sample should be drawn |
| | each day during Treatment Phase A and Treatment Phase B. | within 2-4 hours prior to dosing; the results must be verified to be < 130 mmol/L prior to the first dose. Serum sodium assessments |

| Location | Old Text | Updated Text |
|---|---|---|
| | For all subjects not receiving tolvaptan (Early Withdrawal and Nonresponders on standard of care) serum sodium assessments | should be performed at 8 hours post-first dose and at trough 24 hours post-first dose (this assessment will fall on Day 2 predose). |
| | will be performed every 12 hours throughout Treatment Phase A and Treatment Phase B. | On Day 2 (or 2a), Day 3, and Day 4 (through the following morning on Day 5): |
| | For all subjects final serum sodium assessments will be taken at 24 ( $\pm$ 4) and 72 ( $\pm$ 4) hours post-last dose as well as at 7 days post-last dose. | <ul> <li>For all subjects receiving tolvaptan (Late Withdrawal and Nonresponders continuing on tolvaptan) serum sodium assessments will be performed at trough and 12 hours postdose each day during Treatment Phase A and Treatment Phase B.</li> </ul> |
| | Additional unscheduled serum sodium assessments may be performed at the discretion of the clinical investigator and other physicians of record, depending on the local standards and subject's clinical condition. All serum sodium concentrations collected as part of standard of care will be reported as | For all subjects not receiving tolvaptan (Early Withdrawal and Nonresponders on standard of care) serum sodium assessments will be performed every 12 hours throughout Treatment Phase A and Treatment Phase B. |
| | unscheduled sodium assessments in the electronic CRF through the follow-up sodium assessments. | For all subjects final serum sodium assessments will be taken at 24 $(\pm 4)$ and 72 $(\pm 4)$ hours post-last dose as well as at 7 days post-last dose. |
| 3.7.3.1.1 Blood<br>Collection<br>Times: | Blood samples will be taken so that tolvaptan and metabolite concentrations can be determined. Samples will be taken on Day 1 at 2 hours (± 5 minutes) and 8 hours (concurrent with 8 h serum | Blood samples will be taken so that tolvaptan and metabolite concentrations can be determined. Samples will be taken at the following times: |
| | sodium sample) post-first dose. On Days 2, 3, 4 and 5 samples will be taken at trough (24 hours post previous dose but prior to the subsequent dose), concurrent with serum sodium samples, | On Day 1 at 2 hours (± 5 minutes) and 8 hours (concurrent with 8 h serum sodium sample) post-first dose. |
| | for subjects dosed with tolvaptan on Days 1, 2, 3, and/or 4, respectively, regardless of status as responder/non-responder. An early termination (ET) sample will be taken if ET occurs prior to the last planned PK sample. No ET sample is required if ET | On Days 2, 3, 4 and 5 samples will be taken at trough (prior to the subsequent dose), concurrent with serum sodium samples, for subjects dosed with tolvaptan on Days 1, 2, 3, and/or 4, respectively, regardless of status as responder/non-responder. |

| Location | Old Text | Updated Text |
|---|---|---|
| | occurs at the same visit where a PK sample has already been | An early termination (ET) sample will be taken if ET occurs prior |
| | obtained. | to the last planned PK sample. No ET sample is required if ET |
| | For each PK blood sample collected volumes are not expected to exceed 1.2 mL. Total volume per sample may be lower | occurs at the same visit where a PK sample has already been obtained. |
| | depending on finalization of blood collection supplies. | For each PK blood sample collected volumes are not expected to |
| | Serum sodium assessments and other clinically necessary blood samples take priority, therefore, due to restrictions in allowable | exceed 1.2 mL. Total volume per sample may be lower depending on finalization of blood collection supplies. |
| | total daily blood volumes based on local guidelines and subject age, it may not be possible to take more than one PK sample per day. If so, the PK sampling should be changed to: Day 1: 2 hours post dose (± 5 minutes) | Serum sodium assessments and other clinically necessary blood samples take priority, therefore, due to restrictions in allowable total daily blood volumes based on local guidelines and subject age, it may not be possible to take more than one PK sample per day. If so, the PK sampling should be changed to: |
| | Day 2: 8 ( $\pm$ 2) hours post dose (may be concurrent with serum sodium or other blood sampling) | Day 1: 2 hours postdose (± 5 minutes) |
| | Day 3 at trough, ie, pre-dose/24 hours post prior dose (concurrent with serum sodium sample) | Day 2: 8 ( $\pm$ 2) hours postdose (may be concurrent with serum sodium or other blood sampling) |
| | | Day 3 at trough, ie, predose/24 hours post prior dose (concurrent with serum sodium sample) |
| 3.7.3.2.4 Palatability and Acceptability Assessment: | New section for this amendment | A questionnaire will be administered once to assess palatability to rate flavor/taste, smell, sweetnees, and overall liking of the study medication immediately after dosing. Subjects will also be asked about the ease of swallowing the study medication. Between 15 to 20 minutes after dosing, subjects will be asked again about overall liking of the study medication. This assessment will only be done in subjects aged 3 years to 18 years. |
| 3.7.4 Safety<br>Assessments: | The monitoring frequency of safety assessments is at the | The monitoring frequency of safety assessments is at the discretion |

| Location | Old Text | Updated Text |
|---|---|---|
| | discretion of the clinical investigator; however, the trial requires | of the clinical investigator; however, the trial requires the minimum |
| | the minimum sample collection for all subjects noted in Section | sample collection for all subjects noted in Section 3.7.1 and Section |
| | 3.7.1. | 3.7.4.2.1. |
| 3.7.4.2.1 Serum | New section for this amendment | In addition to serum sodium samples obtained for trial qualification |
| Sodium: | | and efficacy endpoints, supplemental samples for the purposes of |
| | | safety assessment only can be obtained using a point of care |
| | | sodium assessment unit, where available, on Day 1 at 4 to 6 hours |
| | | postdose and at 18 hours postdose. This sodium safety assessment |
| | | will be repeated at 6 and 18 hours postdose each day for the |
| | | remainder of Treatment Phase A. A point of care assessment unit is |
| | | preferred since it is expected to reduce overall daily blood volume |
| | | needed for assessments (expected 0.5 mL for regular blood draws |
| | | versus up to several drops for a point of care assessment, depending |
| | | on the device used); however, regular blood draws may be used |
| | | (especially if they can be combined with standard of care labs). |
| | | Additional unscheduled serum sodium assessments may be |
| | | performed at the discretion of the clinical investigator and other |
| | | physicians of record, depending on the local standards and subject's |
| | | clinical condition. All unscheduled serum sodium concentrations |
| | | collected as part of standard of care will be reported as unscheduled |
| | | sodium assessments in the electronic CRF through the follow-up |
| | | sodium assessments. |
| 3.7.4.2.3 Clinical | Table 3.7.4.2-1 presents required clinical laboratory assessments | Table 3.7.4.2-1 presents required clinical laboratory assessments |
| Lab Tests: | (serum chemistry, hematology, coagulation, urinalysis, and urine | (serum chemistry, hematology, coagulation, urinalysis, and urine |
| | chemistry). All clinical laboratory tests will be performed by | chemistry). All clinical laboratory tests will be performed by local |
| | local laboratories. Serum cortisol and TSH will be measured | laboratories. Serum cortisol and TSH will be measured during |
| | during screening using the remaining blood sample obtained for | screening using the remaining blood sample obtained for serum |

| Location | Old Text | Updated Text |
|---|---|---|
| | serum chemistry. If these results are obtained as part of the | chemistry. If these results are obtained as part of the standard of |
| | standard of care for the subject, a trial-specific sample should be | care for the subject, a trial-specific sample should be obtained and |
| | obtained and sent to the local laboratory for analysis per the | sent to the local laboratory for analysis per the schedule of |
| | schedule of assessments (Section 3.7.1). Uric acid will be | assessments (Section 3.7.1). Uric acid will be measured during |
| | measured during screening for calculation of FENa and FE urate. | screening for calculation of FENa and FE urate. |
| | | It is recognized that there may be limitations based on age and weight of children for the amount of blood that can be drawn at a single time point, per day, and the overall conduct of the trial. Wherever possible, it is encouraged to combine standard of care samples that would be taken regardless of trial participation with those samples required for the trial. |
| | | In case of limited blood or urine volume availability, the bolded assessments in Table 3.7.4.2.3-1 take priority. Serum sodium and liver function tests are essential to the conduct of the trial. |
| Table 3.7.4.2.3-1<br>Clinical | Urobilinogen | Urobilinogen |
| Laboratory Tests | Additional Test: | Additional Test: |
| to be Performed<br>Locally: | Urine pregnancy (if applicable) | Serum or urine pregnancy test (if applicable) |
| 3.7.4.3 Physical | Directed physical examinations will be performed and | Directed physical examinations will be performed and documented |
| Examination: | documented according to the schedule of assessments | according to the schedule of assessments (Section 3.7.1). The |
| | (Section 3.7.1). | initial physical examination should be a full physical. Subsequent |
| | The principal investigator or his/her appointed designee is primarily responsible to perform the physical examination. If the appointed designee is to perform the physical examination, | physical examinations can be directed physical examinations that are focused on hyponatremia-related signs and symptoms as well as any major changes from baseline. |
| | he/she must be permitted by local regulations. Whenever | The principal investigator or his/her appointed designee is primarily |

| Location | Old Text | Updated Text |
|---|---|---|
| | possible, the same individual should perform all physical | responsible to perform the physical examination. If the appointed |
| | examinations for a given subject. Any condition present at the | designee is to perform the physical examination, he/she must be |
| | post-treatment directed physical examination that was not present | permitted by local regulations. Whenever possible, the same |
| | at Screening should be documented as an AE and followed to a | individual should perform all physical examinations for a given |
| | satisfactory conclusion. | subject. Any condition present at the post-treatment directed |
| | All physical examination assessments should include assessments of all major body systems, including but not limited to, ears, | physical examination that was not present at Screening should be documented as an AE and followed to a satisfactory conclusion. |
| | nose, and throat, the thorax area, abdomen, urogenital, | All full physical examination assessments should include |
| | extremities, and skin and mucosae. Neurological examinations | assessments of all major body systems, including but not limited to, |
| | will be performed in an age-appropriate manner per | ears, nose, and throat, the thorax area, abdomen, urogenital, |
| | Section 3.7.4.3.1. | extremities, and skin and mucosae. Neurological examinations will |
| | | be performed in an age-appropriate manner per Section 3.7.4.3.1. |
| 3.7.4.8 Volume | New section for this amendment | Volume status will be assessed every 6 hours prior to trial entry and |
| Status | | every 6 hours during Treatment Phase A. |
| Assessment: | | |
| 3.9 Screen | Subjects who are deemed screen failures may be rescreened for | Subjects who are deemed screen failures may be rescreened for |
| Failures: | possible participation at a later date if no randomization number has been assigned. Subjects who receive a randomization | possible participation if they have not taken a dose of IMP. |
| | number may not be rescreened regardless of whether they receive | |
| | trial medication. | |
| 4.1 Prohibited | Continuous or short term use of other medications, while not | Continuous or short term use of other medications, while not |
| Medications: | prohibited, may be restricted by the investigator because of their | prohibited, may be restricted by the investigator because of their |
| | potential for interference with tolvaptan metabolism. Since | potential for interference with tolvaptan metabolism. Tolvaptan is a |
| | tolvaptan is a sensitive CYP3A4 substrate, subjects weighing ≥ | sensitive CYP3A4 substrate; plasma concentrations increased |
| | 20 kg and taking moderate inhibitors of CYP3A4 will be | approximately 4-fold when tolvaptan was administered with the |
| | administered half of their regular dose of tolvaptan. For subjects | potent CYP3A4 inhibitor ketoconazole. 16,24 Where appropriate |
| | weighing > 50 kg and taking potent CYP3A4 inhibitors, with the | dose reductions are possible, tolvaptan doses may be |

| Location | Old Text | Updated Text |
|---|---|---|
| | exception of amiodarone, which was previously found to have no | coadministered with potent or moderate CYP3A4 inhibitors (see |
| | effect on tolvaptan, a one-quarter dose will be used (3.75 mg). | Section 2.1.1 and Table 2.2.2-1). |
| | Moderate and potent CYP3A4 inhibitors are not allowed for | A partial list of CYP3A4 inhibitors is provided in Table 4.1-1. |
| | subjects weighing $< 20$ and $\le 50$ kg, respectively. <sup>16,24</sup> A partial | 71 partial list of C113711 minorous is provided in Tubic 1.1 1. |
| | list of CYP3A4 inhibitors is provided in Table 4.1-1. | |
| 4.2 Other | The use of saline in this population should be closely monitored. | The use of saline in this population should be closely monitored. |
| Restrictions: | The use of hypertonic saline (3%), including normal saline | The use of hypertonic saline (3%), including normal saline |
| | challenge) within 8 hours of the qualifying screening serum sodium laboratory assessment is prohibited. | challenge within 8 hours of the qualifying screening serum sodium laboratory assessment is prohibited. The use of hypertonic saline (3% or greater) is prohibited during tolvaptan treatment. Routine use of hypertonic saline, while prohibited, may be considered only if used emergently (ie, with a severe symptomatic episode) and with the understanding that free water clearance may be stimulated if tolvaptan had been administered in the prior 24 hours, based on the medical judgment of the investigator. |
| 5.5 Pregnancy: | Female subjects of childbearing potential who are sexually active must use an effective method of birth control during the course of the trial and for 14 days after the last dose of IMP in a manner such that risk of failure is minimized. Unless the subject or her partner(s) is sterile (ie, female subjects who have had an oophorectomy and/or hysterectomy; or male partners who have had orchiectomy) or remain abstinent, two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, birth control pills, birth control depot injection, birth control implant, condom, or sponge with spermicide. Any single method of birth control, including | Women of childbearing potential (WOCBP) are defined as female subjects for whom menstruation has started and who are not documented as sterile (ie, have had a bilateral oopherectomy and/or hysterectomy or who have been postmenopausal for at least 12 months). For WOCBP who are sexually active, there must be a documented agreement that the subject and/or their partner will take effective measures (ie, double-barrier method) to prevent pregnancy during the course of the trial and for 30 days after the last dose of IMP. Unless the subject is sterile (ie, women who have had a bilateral oophorectomy and/or hysterectomy or who have been |

| Location | Old Text | Updated Text |
|---|---|---|
| | vasectomy and tubal ligation, may fail, leading to pregnancy. | postmenopausal for at least 12 consecutive months) or remains |
| | Before enrolling female subjects of childbearing potential in this clinical trial, investigators must review guidelines about trial | fully abstinent (periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] or withdrawal are not |
| | participation for female subjects of childbearing potential. The topics should generally include: | acceptable methods of contraception), two of the following precautions must be used: vasectomy, tubal ligation, vaginal diaphragm, intrauterine device, condom with spermicide, or sponge |
| | General information | with spermicide. The following 3 contraceptive methods are not |
| | ICF/assent form, as applicable | allowed in this trial: birth control pills, birth control depot injection, and birth control implant. Any single method of birth |
| | Pregnancy prevention information | control, including vasectomy and tubal ligation, may fail, leading to |
| | Drug interactions with hormonal contraceptives | pregnancy. The contraceptive method will be documented at each trial visit. |
| | Contraceptives in current use | |
| | Guidelines for the follow-up of a reported pregnancy | Before enrolling WOCBP in this clinical trial, investigators must review the below guidelines about trial participation with all WOCBP. The topics should generally include: |
| | Prior to trial enrollment, female subjects of childbearing potential | General information |
| | must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an | ICF/assent form, as applicable |
| | unintentional pregnancy. The subject's parent or legal guardian | Pregnancy prevention information |
| | must sign an ICF stating that the above-mentioned risk factors and the consequences were discussed with the subject and | Drug interactions with hormonal contraceptives |
| | parent/guardian. | Contraceptives in current use |
| | During the trial, all female subjects of childbearing potential should be instructed to contact the investigator immediately if | Guidelines for the follow-up of a reported pregnancy |
| | they suspect they might be pregnant (eg, missed or late menstrual cycle). | Before trial enrollment, WOCBP must be advised of the importance of avoiding pregnancy during trial participation and the potential |
| | If a subject or investigator suspects that the subject may be | risk factors for an unintentional pregnancy. The subject or the |

| Location | Old Text | Updated Text |
|---|---|---|
| | pregnant prior to IMP administration, the IMP administration | subject's parent or legal guardian must sign an ICF stating that the |
| | must be withheld until the results of serum pregnancy tests are | above-mentioned risk factors and the consequences were discussed |
| | available. If the pregnancy is confirmed, the subject must be | with the subject and/or the parent/guardian. |
| | withdrawn from the trial. If pregnancy is suspected while the subject is taking IMP, the IMP must be withheld immediately (if reasonable, taking into consideration any potential withdrawal risks) until the result of the pregnancy is known. If pregnancy is confirmed, the IMP will be permanently discontinued in an appropriate manner (eg, dose tapering if necessary for subject safety) and the subject will be withdrawn from the trial. | A urine and/or serum pregnancy test for human chorionic gonadotropin (hCG) will be performed at screening on all WOCBP and female subjects ≥12 years of age and all female subjects < 12 years of age, if menstruation has started. If a urine test is performed and is positive, the investigator will follow up with a confirmatory serum test. |
| | (Exceptions to trial discontinuation may be considered for life-threatening conditions only after consultations with the trial medical monitor.) | During the trial, all WOCBP should be instructed to contact the investigator immediately if they suspect they might be pregnant (eg, missed or late menstrual cycle). |
| | The investigator must immediately notify INC Research of any pregnancy associated with IMP exposure, including 14 days after the last dose of IMP and record the event on the IRE form and forward it to INC Research. INC Research will forward Pregnancy Surveillance Form(s) for monitoring the outcome of the pregnancy. Protocol-required procedures for trial discontinuation and follow-up must be performed on the subject unless contraindicated by pregnancy (eg, x-ray trials). Other appropriate pregnancy follow-up procedures should be considered if indicated. In addition, the investigator must report to INC Research, on appropriate Pregnancy Surveillance form(s), follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome. Infants will be followed for a minimum of 6 months. | If a subject is suspected to be pregnant before she receives IMP, the IMP administration must be withheld until the results of serum pregnancy tests are available. If the pregnancy is confirmed, the subject must not receive the IMP and must not be enrolled in the trial. If pregnancy is suspected while the subject is taking IMP, the IMP must be withheld immediately (if reasonable, taking into consideration any potential withdrawal risks) until the result of the pregnancy is known. If pregnancy is confirmed, the IMP will be permanently discontinued in an appropriate manner (eg, dose tapering if necessary for subject safety) and the subject will be withdrawn from the trial. (Exceptions to trial discontinuation may be considered for life-threatening conditions only after consultations with the Clinical Safety and Pharmacovigilance department [see Appendix 1 for contact information]) The investigator must immediately notify the sponsor of any |

| Location | Old Text | Updated Text |
|---|---|---|
| | | pregnancy associated with IMP exposure during the trial and for |
| | | 30 days after the last dose of IMP, and record the event on the IRE |
| | | form and forward it to the sponsor. The sponsor will forward |
| | | Pregnancy Surveillance Form(s) for monitoring the outcome of the pregnancy. |
| | | Protocol-required procedures for trial discontinuation and follow- |
| | | up must be performed on the subject unless contraindicated by |
| | | pregnancy (eg, x-ray trials). Other appropriate pregnancy follow-<br>up procedures should be considered, if indicated. In addition, the |
| | | investigator must report to the sponsor, on appropriate Pregnancy |
| | | Surveillance form(s), follow-up information regarding the course of |
| | | the pregnancy, including perinatal and neonatal outcome. Infants |
| | | will be followed for a minimum of 6 months from the date of birth. |
| 7.1.1 Sample Size | Sample size re-estimation will be conducted when 90% of the | Sample size re-estimation will be conducted when 90% of the |
| for Efficacy: | subjects finish (complete or discontinue) the trial. | subjects finish (complete or discontinue) the trial. The trial must |
| | | include no fewer than 60 subjects on IMP for the assessment of |
| | | safety based on regulatory feedback. |
| 8.1 Packaging | The IMP will be provided to the investigator(s) by the sponsor | The IMP will be provided to the investigator(s) by the sponsor (or |
| and Labeling: | (or designated agent). The IMP will be supplied as 3.75-, 7.5-, | designated agent). The IMP will be supplied as 3.75-, 7.5-, 15-, |
| | 15-, and 30-mg spray-dried tablets in blister packs. Each blister | and 30-mg spray-dried tablets in blister packs or as 60 mL bottles |
| | pack used in the dosing period will be labeled to clearly disclose | containing 1 mg/mL (0.1% w/v) tolvaptan suspension. Each blister |
| | the, compound ID, trial number, the sponsor's name and address, | pack and suspension bottle used in the dosing period will be |
| | instructions for use, route of administration, appropriate | labeled to clearly disclose the compound ID, trial number, the |
| | precautionary statements, and other information required by local | sponsor's name and address, instructions for use, route of |
| | regulatory authorities. | administration, appropriate precautionary statements, and other |
| | | information required by local regulatory authorities. Each site will |

| Location | Old Text | Updated Text |
|---|---|---|
| | The current tolvaptan tablet formulation intended for use in this | be supplied with bottle(s) containing placebo tablets to use for |
| | trial is limited to administration to those who can easily swallow | subject screening purposes. Each placebo bottle will be labeled to |
| | a 3.75-mg tablet (6 mm) and weigh $\geq$ 10 kg. A suspension | clearly disclose the compound ID, trial number, instruction for use, |
| | formulation is in development that will be suitable for children | route of administration, appropriate precautionary statement, and |
| | who cannot swallow tablets (eg, < 4 years) and will also allow | other information required by the local regulatory authorities. For |
| | dosage adjustment for children with body weight < 20 or ≤ 50 kg | dosing suspension, syringes and bottle adaptors will be made |
| | who are taking moderate or potent inhibitors of CYP3A4, | available to the sites. |
| | respectively. Once available, the protocol will be amended to | |
| | include the details of this formulation and will include | |
| | information on the packaging and labeling for that formulation | |
| 8.2 Storage: | The IMP will be stored at 25°C (77°F) or below, with excursions | The IMP blister packs will be stored at 25°C (77°F) or below, with |
| | allowed from 15 to 30°C (59 to 86°F). The clinical site staff or | excursions allowed from 15 to 30°C (59 to 86°F). The IMP |
| | designated personnel will maintain a temperature log in the drug | suspension bottles will be stored at 2 to 8°C (35.6 to 46.4°F) and |
| | storage area recording the temperature at least once each working | protected from light. The clinical site staff or designated personnel |
| | day. | will maintain a temperature log in the drug storage area recording |
| | | the temperature at least once each working day. |
| 9.1 Source | Investigator(s)/institution(s) will permit trial-related | Investigator(s)/institution(s) will permit trial-related monitoring, |
| <b>Documents:</b> | monitoring, audits, IRB/IEC review, and regulatory inspection(s) | audits, IRB/IEC review, and regulatory inspection(s) by providing |
| | by providing direct access to source data/documents by | direct access to source data/documents by authorized persons as |
| | authorized persons as defined in the ICF. | defined in the ICF. In all cases, subject confidentiality must be |
| | | maintained in accordance with local regulatory requirements. |
| 0.2 D-4- | | |
| 9.2 Data Collection: | <ul> <li>Documentation of the informed consent process,<br/>including any revised consents;</li> </ul> | <ul> <li>Documentation of the informed consent process, including<br/>any revised consents;</li> </ul> |
| | <ul> <li>The date of the visit and the corresponding visit or day<br/>in the trial schedule;</li> </ul> | Documentation of the investigator's decision to enroll the subject into the trial, the review of all inclusion/exclusion |
| | General subject status remarks, including any <i>significant</i> medical findings. The severity, frequency, and duration | criteria prior to IMP administration, and confirmation of the subject's actual participation in the trial; |

| Location | Old Text | Updated Text |
|---|---|---|
| | of any AEs and the investigator's assessment of relationship to the IMP must also be recorded; | The date of the visit and the corresponding Visit or Day in the trial schedule; |
| | <ul> <li>Any changes in concomitant medications or dosages;</li> <li>A general reference to the procedures completed;</li> <li>The signature (or initials) and date of all clinicians who made an entry in the progress notes.</li> </ul> | <ul> <li>General subject status remarks, including any significant<br/>medical findings. The severity, frequency, duration,<br/>action taken, and outcome of any AEs and the<br/>investigator's assessment of relationship to IMP must also<br/>be recorded;</li> </ul> |
| | Changes will be made by striking a single line through erroneous data, and clearly entering the correct data (eg, wrong data-right data). If the reason for the change is not apparent, a brief explanation for the change will be written in the source | <ul> <li>Any changes in concomitant medications or dosages;</li> <li>A general reference to the procedures completed;</li> <li>The signature (or initials) and date of each clinician (or designee) who made an entry in the progress notes.</li> </ul> |
| | documentation by the clinician. | Changes will be made by striking a single line through erroneous data (so as not to obliterate the original data), and clearly entering the correct data (eg, wrong data right data). If the reason for the change is not apparent, a brief explanation for the change will be written in the source documentation by the clinician. If electronic data systems are being utilized, a full audit trail of changes must be maintained. |
| 9.3 File<br>Management at<br>the Trial Site: | The investigator will ensure that the trial center file is maintained in accordance with Section 8 of the ICH Guideline for GCP <sup>29</sup> and as required by applicable local regulations | The investigator will ensure that the trial site file is maintained in accordance with Section 8 of the ICH GCP Guideline E6 <sup>29</sup> and as required by applicable local regulations |
| 9.4 Records<br>Retention at the<br>Trial Site: | A period of at least 2 years following the date on which approval to market the drug is obtained (or if IMP development is discontinued, the date of discontinuation); OR | A period of at least 2 years following the date on which approval to market the drug is obtained (or if IMP development is discontinued, the date regulatory authorities were notified of discontinuation); OR |
| | The investigator will be responsible to maintain adequate and | The investigator will be responsible to maintain adequate and |

| Location | Old Text | Updated Text |
|---|---|---|
| | accurate electronic or hard copy source documents of all | accurate electronic or hard copy source documents of all |
| | observations and data generated during this trial. | observations and data generated during this trial including any data |
| | | clarification forms received from the sponsor. |
| 10.1 Monitoring: | The sponsor has ethical, legal, and scientific obligations to follow | The sponsor has ethical, legal, and scientific obligations to follow |
| 10.1 Monitoring. | this trial in a detailed and orderly manner in accordance with | this trial in accordance with established research principles, the ICH |
| | • | * * * |
| | established research principles, the ICH GCP Guideline, and | E6 GCP: Consolidated Guidance, and applicable regulatory |
| | applicable regulatory requirements and local laws. As part of a | requirements and local laws. As part of a concerted effort to fulfill |
| | concerted effort to fulfill these obligations (maintain current | these obligations (maintain current personal knowledge of the |
| | personal knowledge of the progress of the trial), the sponsor's | progress of the trial), the sponsor's monitors will visit the site |
| | monitors will visit the site during the trial, as well as | during the trial, as well as communicate frequently via telephone, e- |
| | communicate frequently via telephone and written | mail, and written communications. In addition, all investigators |
| | communications. | and clinical site personnel will undergo initial and ongoing training |
| | | for this particular trial, and this training will be clearly documented. |
| 10.2 Auditing: | The sponsor's Quality Management Unit (or representative) may | The sponsor's Quality Assurance Unit (or representative) may |
| | conduct trial site audits. Audits will include, but are not be | conduct trial site audits. Audits will include, but are not be limited |
| | limited to, drug supply, presence of required documents, the | to, IMP supply, presence of required documents, the informed |
| | informed consent process, and comparison of CRFs with source | consent process, and comparison of CRFs with source documents. |
| | documents. | |
| 11 Ethics and | This trial must be conducted in compliance with the protocol, the | This trial must be conducted in compliance with the protocol, ICH |
| Responsibility: | ICH GCP Guideline, and applicable local laws and regulatory | GCP Guideline (E6), international ethical principles derived from |
| | requirements. Each trial site will seek approval by an IRB or IEC | the Declaration of Helsinki and Council for International |
| | according to regional requirements. | Organizations of Medical Science (CIOMS) guidelines, and |
| | | applicable local laws and regulations. Each trial site will seek |
| | | approval/favorable opinion by an IRB or IEC according to regional |
| | | requirements, and the investigator will provide that documentation |
| | | to the sponsor. |
| | | to the sponsor. |

| Location | Old Text | Updated Text |
|---|---|---|
| 12 | However, authorized regulatory officials and sponsor personnel | However, authorized regulatory officials and sponsor personnel |
| Confidentiality: | (or their representatives) will be allowed full access to inspect | (or their representatives) may be allowed full access to inspect and |
| | and copy the records. All IMPs, subject bodily fluids, and/or | copy the records, consistent with local requirements. All IMPs, |
| | other materials collected shall be used solely in accordance with | subject bodily fluids, and/or other materials collected shall be used |
| | this protocol, unless otherwise agreed to in writing by the | solely in accordance with this protocol, unless otherwise agreed to |
| | sponsor. | in writing by the sponsor. |
| | Subjects will be identified only by initials and unique subject | Subjects will be identified only by unique subject numbers in |
| | numbers in CRFs. Their full names may, however, be made | CRFs. If further subject identification is required, subjects' full |
| | known to a regulatory agency or other authorized officials if | names may be made known to a regulatory agency or other |
| | necessary. | authorized officials if necessary, subject to local regulations. |
| 13 Amendment | The investigator will not make any changes to this protocol | The investigator will not make any changes to this protocol without |
| Policy: | without the sponsor's prior written consent and subsequent | the sponsor's prior written consent and subsequent |
| | approval by the IRB/IEC. Any permanent change to the | approval/favorable opinion by the IRB/IEC. Any permanent |
| | protocol, whether it be an overall change or a change for specific | change to the protocol, whether an overall change or a change for |
| | trial site(s), must be handled as a protocol amendment. Any | specific trial site(s), must be handled as a protocol amendment. |
| | amendment will be written by the sponsor. Each amendment will | Any amendment will be written by the sponsor. Each amendment |
| | be submitted to the IRB/IEC. Except for "administrative" or | will be submitted to the IRB/IEC, as required by local regulations. |
| | "non-substantial" amendments, investigators will wait for | Except for "administrative" or "non-substantial" amendments, |
| | IRB/IEC approval of the amended protocol before implementing | investigators will wait for IRB/IEC approval/favorable opinion of |
| | the change(s). Administrative amendments are defined as having | the amended protocol before implementing the change(s). |
| | no effect on the safety of subjects, conduct or management of the | Administrative amendments are defined as having no effect on the |
| | trial, trial design, or the quality or safety of IMP(s) used in the | safety of subjects, conduct or management of the trial, trial design, |
| | trial. A protocol change intended to eliminate an apparent | or the quality or safety of IMP(s) used in the trial. A protocol |
| | immediate hazard to subjects should be implemented | change intended to eliminate an apparent immediate hazard to |
| | immediately, followed by IRB/IEC notification within 5 working | subjects should be implemented immediately after agreement by the |
| | days. The sponsor will submit protocol amendments to the | sponsor and investigator, followed by IRB/IEC notification within |
| | applicable regulatory agencies. | local applicable timelines. The sponsor will submit protocol |
| | | amendments to the applicable regulatory agencies within local |

| Location | Old Text | Updated Text |
|---|---|---|
| | When the IRB/IEC, investigators, and/or the sponsor conclude that the protocol amendment substantially alters the trial design and/or increases the potential risk to the subject, the currently approved written ICF will require similar modification. In such cases, repeat informed consent will be obtained from subjects enrolled in the trial before expecting continued participation. | applicable timelines. When the IRB/IEC, investigators, and/or the sponsor conclude that the protocol amendment substantially alters the trial design and/or increases the potential risk to the subject, the currently approved written ICF will require similar modification. In such cases, after approval/favorable opinion of the new ICF by the IRB/IEC, repeat written informed consent will be obtained from subjects enrolled in the trial before expecting continued participation and before the amendment-specified changes in the trial are implemented. |
| 14 Publication<br>Authorship<br>Requirements: | New section for this amendment | |
| Appendix 2: | Phone Mobile E-Mail Study Communications & Patient/Site Support Phone: | Phone ; Mobile Fax: E-Mail: Study Communications & Patient/Site Support Phone: IDMC Support Phone: Fax: |

| Location | Old Text | Updated Text |
|---|---|---|
| Agreement: | and in the sponsor's (or designee's) Clinical Research | and in the sponsor's (or designee's) Clinical Trial Agreement. |
| | Agreement. | I am aware that this protocol must be approved by the |
| | I am aware that this protocol must be approved by the | Institutional Review Board (IRB) or receive a favorable opinion by |
| | Institutional Review Board (IRB) or Independent Ethics | the Independent Ethics Committee (IEC) responsible for such |
| | Committee (IEC) responsible for such matters in the clinical trial | matters in the clinical trial facility where tolvaptan will be tested |
| | facility where tolvaptan will be tested prior to commencement of | prior to commencement of this trial. I agree to adhere strictly to the |
| | this trial. I agree to adhere strictly to the attached protocol | attached protocol (unless amended in the manner set forth in the |
| | (unless amended in the manner set forth in Paragraph I of the | sponsor's Clinical Trial Agreement, at which time I agree to adhere |
| | sponsor's Clinical Research Agreement, at which time I agree to | strictly to the protocol as amended). |
| | adhere strictly to the protocol as amended). | I agree to await IRB/IEC approval before implementation of any |
| | I agree to await IRB/IEC approval before implementation of | substantial amendments to this protocol. If, however, there is an |
| | any protocol amendments to this protocol. If, however, there is | immediate hazard to subjects, I will implement the amendment |
| | an immediate hazard to subjects, I will implement the | immediately, and provide the information to the IRB/IEC within |
| | amendment immediately, and provide the information to the | the required local applicable timelines. Administrative changes to |
| | IRB/IEC within 5 working days. Administrative changes to the | the protocol will be transmitted to the IRB/IEC for informational |
| | protocol will be transmitted to the IRB/IEC for informational | purposes only, if required by local regulations. |
| | purposes only. | I agree to report to the sponsor any adverse experiences in |
| | I agree to report to the sponsor any adverse experiences in | accordance with the terms of the sponsor's Clinical Trial Agreement |
| | accordance with the terms of the sponsor's Clinical Research | and the relevant regional regulation(s) and guideline(s). I further |
| | Agreement and the relevant regional regulation(s) and | agree to provide all required information regarding financial |
| | guideline(s). I further agree to provide all required information | certification or disclosure to the sponsor for all investigators and |
| | regarding financial certification or disclosure to the sponsor for | sub-investigators in accordance with the terms of the relevant |
| | all investigators and sub-investigators in accordance with the | regional regulation(s). I understand that participation in the |
| | terms of the relevant regional regulation(s). I understand that | protocol involves a commitment to publish the data from this trial |
| | participation in the protocol involves a commitment to publish | in a cooperative publication before publication of efficacy and |
| | the data from this trial in a cooperative publication prior to | safety results on an individual basis may occur, and I consent to be |
| | publication of efficacy and safety results on an individual basis. | acknowledged in any such cooperative publications that result. |

| Location | Old Text | Updated Text |
|---|---|---|
| | Principal or Coordinating Investigator Signature and Date | Principal Investigator |
| | Sponsor Representative Signature and Date | Print Name |
| | | Signature |
| | | Date |

**ADDITIONAL RISK TO THE SUBJECT:** There is no additional risk to the subjects.

Protocol 156-08-276

Amendment Number: 4

**Issue Date:** 07 May 2015

#### **PURPOSE:**

• Correction of typographical errors in the dosing table (Table 2.1.1-2) for the suspension for subjects taking a CYP3A inhibitor.

- Removed the word "Tablet" from the title of Table 2.1.1-2 as the table includes dosing information for tolvaptan tablets and for the suspension formulation of tolvaptan.
- Updated the Clinical Management contact information on the title page and in Appendix 1.
- Correction of typographical error in Section 2.1.1 Dosing Rationale.

#### **BACKGROUND:**

Table 2.1.1-2 was added to this protocol with Amendment Number 3. Subsequent to the approval of Amendment Number 3, typographical errors were discovered in Table 2.1.1-2. The errors are being corrected with this protocol amendment (Amendment Number 4).

The Clinical Management contact information has been updated.

A typographical error in Section 2.1.1 Dosing Rationale has been corrected. The word "staring" has been corrected to "starting".

#### MODIFICATIONS TO PROTOCOL:

**Sectional Revisions:** changes made to specific sections of the protocol are listed in the table below.

| Location | Old Text | | Updated Text | |
|---|---|---|---|---|
| Title Page: | Clinical Management | | Clinical Management | |
| | Pho | one ; | P | thone; |
| | Fax | | Fax | |
| | E-mail: | | E-mail: | |
| | Issue Date: 03 | 03 Jul 2013 | Issue Date: | 03 Jul 2013 |
| | Date of Amendment 1: 04 | 04 Nov 201 | Date of Amendment 1: | 04 Nov 201 |
| | Date of Amendment 2: | 9 May 2014 | Date of Amendment 2: | 19 May 2014 |
| | Date of Amendment 3: 20 | 26 February 2015 | Date of Amendment 3: | 26 February 2015 |
| | | • | Date of Amendment 4: | 07 May 2015 |
| 2.1.1 | | | | |
| Dosing | Subjects $\geq 2$ years of age, weighing $\leq 30$ kg and who cannot safely | | | weighing ≤30 kg and who cannot safely |
| Rationale: | swallow a tablet, will receive | re an oral, once daily dose of tolvaptan | swallow a tablet, will receive an oral, once daily dose of tolvaptan | |
| | suspension staring at 0.15 m | ng/kg. | suspension starting at 0.1: | 5 mg/kg. |

Old Text: Table 2.1.1-2

| Table 2.1.1-2 Starting Tolvaptan Tablet Doses in the Presence of Potent or Moderate CYP3A Inhibitors | | | |
|---|---|---|---|
| Tolvaptan Dose | Age/Body Weight (as applicable) | Potent Inhibitor | Moderate Inhibitor |
| 0.1 mg/kg<br>suspension <sup>a</sup> | 44 wk to < 2 y or<br>< 10 kg | - | 0.05 mg/kg suspension |
| 0.15 mg/kg<br>suspension | ≥ 2 y, ≤ 30 kg | 0.04 mg/kg suspension | 0.8 mg/kg suspension |
| 3.75 mg tablet | $\geq$ 10 kg to $\leq$ 20 kg | 0.94 mL suspension | 0.19 mL suspension |
| 7.5 mg tablet | 20 kg to 50 kg | 1.90 mL suspension | 3.75 mg tablet |
| 15 mg tablet | ≥ 50 kg | 3.75 mg tablet | 7.5 mg tablet |

<sup>&</sup>lt;sup>a</sup>The smallest volume of suspension that may be administered is 0.3 mL (0.3 mg), therefore dose reductions for potent inhibitors cannot be accommodated and for moderate inhibitors children weighing < 6 kg cannot be accommodated.

**Updated Text: Table 2.1.1-2** 

| Table 2.1.1-2 Starting Tolvaptan Doses in the Presence of Potent or Moderate CYP3A Inhibitors | | | |
|---|---|---|---|
| Tolvaptan Dose | Age/Body Weight (as applicable) | Potent Inhibitor | Moderate Inhibitor |
| 0.1 mg/kg<br>suspension | 44 wk to < 2 y or<br>< 10 kg | _ | 0.05 mg/kg suspension |
| 0.15 mg/kg<br>suspension | ≥ 2 y, ≤ 30 kg | 0.04 mg/kg suspension | 0.08 mg/kg suspension |
| 3.75 mg tablet | $\geq 10 \text{ kg to} < 20 \text{ kg}$ | 0.94 mL suspension | 1.90 mL suspension |
| 7.5 mg tablet | 20 kg to 50 kg | 1.90 mL suspension | 3.75 mg tablet |
| 15 mg tablet | ≥ 50 kg | 3.75 mg tablet | 7.5 mg tablet |

<sup>&</sup>lt;sup>a</sup>The smallest volume of suspension that may be administered is 0.3 mL (0.3 mg), therefore dose reductions for potent inhibitors cannot be accommodated and for moderate inhibitors children weighing < 6 kg cannot be accommodated.



**ADDITIONAL RISK TO THE SUBJECT:** There is no additional risk to the subjects.

Protocol 156-08-276

Amendment Number: 5

**Issue Date:** 17 Nov 2015

**PURPOSE:** 

The main intent of the Amendment is to clarify administrative sections, align with current protocol templates, and incorporate recent requests from Regulatory Authorities (Food and Drug Administration [FDA]).

#### **BACKGROUND:**

This protocol serves as the single trial for the Pediatric Written Request with the FDA and the Pediatric Research Equity Act (PREA) requirement for the US. The FDA has agreed to the current version of the protocol and updates have been made to address further comments from the FDA, and other regulatory agencies.

#### **MODIFICATIONS TO PROTOCOL:**

#### **General Revisions:**

- Removed the neurocognition test battery. This was an exploratory endpoint and the removal of the neurocognition test battery has no impact on the safety aspects of the trial.
- Clarified dosing as dual formulations are employed: tablet and suspension.
- Alignment within the protocol descriptor sections of time points for pharmacokinetic assessments and serum sodium assessments; no change to requirement of time points or assessments.
- Clarification of Exclusion Criteria and added an exclusion criterion to reflect the suspension use and protocol template update.
- Removed reference to the extension study, 156-11-294.
- Standard Protocol template updates made to reflect Investigator's Brochure (IB) Edition 21 issuance.
- Clarified requirements for a full versus directed physical examination and neurological examination. Added a fontanelle assessment as age appropriate.
- Clarified urine vs. serum pregnancy test requirements.
- FE urate changed to FE urea throughout the protocol.
- Urine uric acid changed to urine urea throughout the protocol.
- Provided additional information related to the Tanner Staging Assessment, including an Appendix for classification reference.
- Updated the protocol template to make consistent with changes in the Phase 3 global protocol template (ie. revised definition of AE, SAE definition related to hospitalization, IRE definition, including potential DILI, Clinical lab test value changes, IMP Causality, Eliciting and Reporting AEs).
- Clarified pregnancies to be reported to INC Research instead of the sponsor.

#### Protocol 156-08-276

- Clarified the time points in which nonserious and serious AEs will be followed.
- Updated list of abbreviations and references.

## ADDITIONAL RISK TO THE SUBJECT: There is no additional risk to the subjects.

A complete redline version of this amendment showing all changes from the previous version will be produced and available upon final approval of this amendment.

#### Agreement

I, the undersigned principal investigator, have read and understand the protocol (including the Investigator's Brochure) and agree that it contains all the ethical, legal, and scientific information necessary to conduct this trial in accordance with the principles of Good Clinical Practices and as described herein and in the sponsor's (or designee's) Clinical Trial Agreement.

I will provide copies of the protocol to all physicians, nurses, and other professional personnel to whom I delegate trial responsibilities. I will discuss the protocol with them to ensure that they are sufficiently informed regarding the investigational new drug, tolvaptan, the concurrent medications, the efficacy and safety parameters and the conduct of the trial in general. I am aware that this protocol must be approved by the Institutional Review Board (IRB) or receive a favorable opinion by the Independent Ethics Committee (IEC) responsible for such matters in the clinical trial facility where tolvaptan will be tested prior to commencement of this trial. I agree to adhere strictly to the attached protocol (unless amended in the manner set forth in the sponsor's Clinical Trial Agreement, at which time I agree to adhere strictly to the protocol as amended).

I understand that this IRB- or IEC-approved protocol will be submitted to the appropriate regulatory authority/ies by the sponsor. I agree that clinical data entered on case report forms by me and my staff will be utilized by the sponsor in various ways such as for submission to governmental regulatory authorities and/or in combination with clinical data gathered from other research sites, whenever applicable. I agree to allow sponsor monitors and auditors full access to all medical records at the research facility for subjects screened or enrolled in the trial.

I agree to await IRB/IEC approval before implementation of any substantial amendments to this protocol. If, however, there is an immediate hazard to subjects, I will implement the amendment immediately, and provide the information to the IRB/IEC within the required local applicable timelines. Administrative changes to the protocol will be transmitted to the IRB/IEC for informational purposes only, if required by local regulations.

I agree to provide all subjects with informed consent forms, as required by the applicable regulations and by ICH guidelines. I agree to report to the sponsor any adverse experiences in accordance with the terms of the sponsor's Clinical Trial Agreement and the relevant regional regulation(s) and guideline(s). I further agree to provide all required information regarding financial certification or disclosure to the sponsor for all investigators and sub-investigators in accordance with the terms of the relevant regional regulation(s). I understand that participation in the protocol involves a commitment to publish the data from this trial in a cooperative publication before publication of efficacy and safety results on an individual basis may occur, and I consent to be acknowledged in any such cooperative publications that result.

| Principal Investigator Print Name | Signature | Date |
|-----------------------------------|-----------|------|

# Otsuka Pharmaceutical Development & Commercialization, Inc. This page is a manifestation of an electronically captured signature

OPC-41061

SIGNATURE PAGE

**Document Name: 156-08-276 Protocol Amendment 5** 

Document Number: 0001027730

**Document Version: 9.0** 

| Signed by | Meaning of Signature | Server Date (dd-MMM-yyyy HH:mm 'GMT'Z) |
|-----------|------------------------|----------------------------------------|
| | Biostatistics Approval | 17-Nov-2015 21:03 GMT+00 |
| | Clinical Pharmacology | 17-Nov-2015 21:46 GMT+00 |
| | Clinical Approval | 18-Nov-2015 03:34 GMT+00 |